

# 16.1.9 Documentation of Statistical Codes



# **Statistical Analysis Plan**

| Sponsor: | BioDelivery Sciences International, Inc. |
|---|---|
| Protocol No: | BUP-401 |
| Protocol Title: | A RANDOMIZED, DOUBLE-BLIND, DOUBLE-DUMMY, 6-PERIOD, PLACEBO-CONTROLLED, CROSSOVER STUDY TO EXPLORE AND COMPARE THE VENTILATORY RESPONSE TO HYPERCAPNIA (VRH), OF BELBUCA, OXYCODONE HYDROCHLORIDE, AND PLACEBO IN RECREATIONAL OPIOID USERS |
| PRA Project ID: | BDL673SL-186739 |
| Version Date: | 07-Oct-2019 (SAP) |

# 1.0 Approvals

The undersigned have approved this Statistical Analysis Plan for use in this study.

| Name of Sponsor<br>Representative /<br>Title: |
|------------------------------------------------------|
| Signature of<br>Sponsor<br>Representative /<br>Date: |
| Name of Author /<br>Title: |
| Signature of Author / Date: |

EDSREP 009 T 01 G 




# 2.0 Table of Contents

| 1.0 Approvals | 1 |
|-------------------------------------------------------|------|
| 2.0 Table of Contents | 2 |
| 3.0 Introduction | 4 |
| 4.0 Changes from Previous Version of Approved SAP | 4 |
| 5.0 Study Objectives | 4 |
| 5.1 Primary | |
| 5.1.1 Primary Endpoints | 4 |
| 5.2 Secondary | |
| 5.2.1 Secondary Endpoints | |
| 5.3 Exploratory | |
| 5.4 Study Hypothesis | |
| 6.0 Study Design | |
| 6.1 Sample Size Considerations | |
| 6.2 Randomization | |
| 7.0 Overview of Planned Analysis | |
| 7.1 Changes from Protocol | |
| 7.2 Interim Analysis and Key Results | |
| 7.3 Final Analysis | |
| 8.0 Data Review | |
| 8.1 Data Management | |
| 8.2 Acceptance of Data for Summarization | |
| 9.0 Definitions and General Analysis Methods | |
| 9.1 Analysis Data Presentation | |
| 9.1.1 Rounding | |
| 9.1.2 Imputation | |
| 9.1.3 Daylight Savings Time Adjustments | |
| 9.1.4 Descriptive Statistics | |
| 9.1.5 Pooling | |
| 9.1.6 Unscheduled Measurements | |
| 9.2 Analysis Data Definitions | 8 |
| 9.2.1 Baseline Definition | |
| 9.2.2 Treatment/Subject Grouping | |
| 9.2.3 Common Variable Derivations | 9 |
| 9.2.4 QC | |
| 9.2.5 ADaM Datasets and Metadata | |
| 9.3 Software | |
| 9.4 Statistical Methods | |
| 9.4.1 Statistical Outlier Determination | |
| 9.4.2 Predetermined Covariates and Prognostic Factors | |
| 9.4.3 Hypothesis Testing | . 10 |
| 9.5 TFL Layout | |
| 10.0 Analysis Sets | .11 |
| 10.1 Randomized Set | |
| 10.2 Safety Set | |
| 10.3 Pharmacokinetic Set | |
| 10.4 Completers Set | |
| 10.5 Partial Completers Set | |
| 11.0 Subject Disposition | |
| 12.0 Protocol Deviations | |
| 13.0 Demographic and Baseline Characteristics | |
| 13.1 Demographics | |
| 13.2 Medical History | 12 |



| 13.3 Recreational Drug, Alcohol and Tobacco History | 12 |
|---------------------------------------------------------------|----|
| 14.0 Concomitant Medications | 12 |
| 15.0 Treatment Compliance and Exposure | 12 |
| 16.0 Pharmacokinetic Analyses | 12 |
| 16.1 Pharmacokinetic Variables | 12 |
| 16.2 Plasma Pharmacokinetic Summaries | 13 |
| 16.2.1 Plasma Concentrations | |
| 16.2.2 Plasma Pharmacokinetic Parameters | 13 |
| 17.0 Pharmacodynamic Analysis | 14 |
| 17.1 Pharmacodynamic Measurements | 14 |
| 17.2 Pharmacodynamic Parameters | |
| 17.3 Pharmacodynamic Statistical Analyses | 16 |
| 18.0 Secondary Endpoints | 17 |
| 19.0 Safety Analyses | 17 |
| 19.1 Safety Variables | |
| 19.1.1 Adverse Events | |
| 19.1.2 Deaths and Serious Adverse Events | |
| 19.1.3 Laboratory Data | 19 |
| 19.1.4 Vital Signs | |
| 19.1.5 Electrocardiograms | |
| 19.1.6 Continuous Pulse Oximetry | |
| 19.1.7 Physical Examinations | |
| 19.1.8 Cardiac Telemetry | |
| 19.1.9 Columbia-Suicide Severity Rating Scale | |
| 19.1.10 Clinical Opiate Withdrawal Scale | |
| 20.0 References | |
| Appendix 1: Glossary of Abbreviations | |
| Appendix 2: Schedule of Assessments | |
| Appendix 3: List of End of Text Outputs | |
| Appendix 4: Shells for Post-Text Tables, Figures and Listings | 27 |
| 21.0 Document History | 27 |

Statistical Analysis Plan BDL673SL-186739 Protocol: BUP-401

Version Date: 07-Oct-2019

# 3.0 Introduction

This Statistical Analysis Plan (SAP) describes the statistical methods that will be used during the analysis and reporting of data collected under BioDelivery Sciences International, Inc. Protocol BUP-401.

This SAP should be read in conjunction with the study protocol and electronic case report form (eCRF). This version of the plan has been developed using the protocol dated 24-May-201912 (including all amendments up to this protocol date) and the final eCRF(s) dated 24-Aug-2019.

An approved and signed SAP is a requirement for database lock. An approved SAP is also required for unblinding of the study treatments.

This SAP only covers the results that will be processed by the PRA Early Development Services (EDS) Biostatistics Department.

PRA EDS will perform the pharmacokinetic (PK), pharmacodynamic (PD), and safety and tolerability evaluation.

This SAP supersedes the statistical considerations identified in the protocol; where considerations are substantially different, they will be so identified. Any post-hoc or unplanned analyses, or significant changes from the planned analysis in this SAP performed to provide results for inclusion in the clinical study report (CSR) but not included in this SAP, will be clearly identified in the CSR. Changes to planned analyses do not require an updated SAP but should be included in the CSR if significant.

# 4.0 Changes from Previous Version of Approved SAP

This is the first version of the SAP.

# 5.0 Study Objectives

# 5.1 Primary

Respiratory drive will be evaluated by measuring the ventilatory response to hypercapnia (VRH) by maximum decrease in minute ventilation after administration of Belbuca, oxycodone hydrochloride, and placebo.

# 5.1.1 Primary Endpoints

- Ventilatory response to hypercapnia
  - Minute ventilation (expired minute volume, V<sub>E</sub>; L/min)
  - Respiratory rate (breaths/min)
  - Flow rates (peak expired flow, PEF; L/min)
  - Tidal volume (expired tidal volume, V<sub>T</sub>; mL)
  - o End-tidal CO<sub>2</sub> (ET<sub>CO2</sub>, mmHg)
  - Hypercapnic Ventilatory Response, expressed in L/min per mm Hg
  - Ratio of V<sub>E</sub> / ET<sub>CO2</sub>, expressed in L/min per mm Hg

# 5.2 Secondary

- · Pupil diameter will be assessed by pupillometry predose and at multiple timepoints after completion of Belbuca, oxycodone hydrochloride, and placebo dosing.
- Change in ratio of minute ventilation over end-tidal CO2 predose and at multiple timepoints after oral administration of Belbuca, oxycodone hydrochloride, and placebo.

EDSREP 009 T 01 G 


Clinical safety data from adverse event (AE) reporting, clinical observations, 12-lead
electrocardiograms (ECGs), vital signs (blood pressure [BP], heart rate [HR], respiratory rate, and
oral temperature), oxygen saturation, and safety laboratory tests following administration of
Belbuca, oxycodone hydrochloride, and placebo will be summarized, and any clinically significant
abnormalities will be described.

# 5.2.1 Secondary Endpoints

- Pupil diameter (for each measurement during pupillometry, a single pupil diameter will be recorded)
- · Safety endpoints including:
  - o AFs
  - Safety laboratory (hematology, blood chemistry, urinalysis, serology, alcohol breath test, pregnancy & FSH)
  - Vital signs (BP, RR, oral temperature)
  - o ECG (HR, PR-interval, QRS-duration, QT-interval, QTc-interval (Fridericia's))
  - Pulse Oximetry (continuous oxygen saturation monitoring of peripheral capillary oxygen saturation (SpO<sub>2</sub>))
  - o Columbia-Suicide Severity Rating Scale
  - Cardiac Telemetry (continuous measurement during VHR testing)
  - o Physical Exam
  - o COWS (assessments of opiate withdrawal symptoms during Naloxone Challenge)

# 5.3 Exploratory

• Blood samples will be collected to evaluate pharmacokinetic (PK) and blood levels of Belbuca and oxycodone hydrochloride at important pharmacodynamic (PD) endpoints.

# 5.4 Study Hypothesis

Although there is no formal study hypothesis, the rationale for this study is to compare the effects of increasing dose and respiratory depression between a Schedule II opioid (oxycodone hydrochloride) and Schedule III opioid (Belbuca). In this study, the effect of 300 µg, 600 µg, and 900 µg doses of Belbuca (Schedule III), 30 mg and 60 mg of oxycodone hydrochloride (Schedule II), and placebo, on the respiratory drive will be evaluated by measuring the ventilatory response to hypercapnia (VRH).

# 6.0 Study Design

This is a double-blind, double-dummy, oral/buccal, 6-treatment, 6-period, placebo-controlled, randomized, crossover study with the following treatments (given in the sequences specified in Table 1 below), each separated by an approximate 7-day washout period, in up to 18 male or female subjects self-identifying as recreational drug users. The study will consist of a Screening Phase, a Treatment Phase (which includes the Naloxone Challenge Test), and a Follow-Up Phase.

- Belbuca 300 µg and oral placebo
- Belbuca 600 µg and oral placebo
- Belbuca 900 µg and oral placebo
- Oxycodone 30 mg and buccal placebo
- Oxycodone 60 mg and buccal placebo
- Oral placebo and buccal placebo

EDSREP 009 T 01 G 


Statistical Analysis Plan BDL673SL-186739 Protocol: BUP-401

Version Date: 07-Oct-2019

## **Screening Phase**

Study-specific screening procedures will include: a physical examination (PE), including measurement of height, weight, and vital signs; blood and urine laboratory testing; review of medical and medication history; and a 12-lead ECG. The subjects will also undergo the VRH procedure to determine tolerability of the procedure and demonstrate adequate VRH.

#### **Treatment Phase**

All subjects with a negative urine drug screen on Day -1 will undergo the Naloxone Challenge Test. Subjects will receive an initial dose of naloxone hydrochloride 0.2 mg by intravenous bolus, followed by an assessment of signs of withdrawal. The subject will be assessed by a medical provider for signs or symptoms of withdrawal through assessments of the COWS scores. If no evidence of withdrawal occurs within 30 seconds, an additional 0.6 mg naloxone will be administered by intravenous bolus. A second COWS assessment will be done 5 minutes after the 0.6 mg naloxone dose administration. A COWS score of >5 will result in a failed naloxone challenge. Subject safety will be monitored for 60 minutes after the administration of naloxone.

After completing and passing the Naloxone Challenge Test, subjects will be randomized to 1 of 6 treatment sequences in a 1:1:1:1:1 ratio on Day 1. Subjects will receive all six treatments in the order specified by a Williams design sequence where every treatment follows every other treatment at least once (Table 1). Treatment will be double-blind, double-dummy whereby subjects will receive both buccal film (active or placebo) and a capsule (active or placebo).

Table 1 Assignment of Subjects to Treatments

| Sequence | Period 1 | Period 2 | Period 3 | Period 4 | Period 5 | Period 6 |
|---|---|---|---|---|---|---|
| 1 | Treatment C | Treatment A | Treatment D | Treatment B | Treatment F | Treatment E |
| 2 | Treatment D | Treatment C | Treatment F | Treatment A | Treatment E | Treatment B |
| 3 | Treatment F | Treatment D | Treatment E | Treatment C | Treatment B | Treatment A |
| 4 | Treatment E | Treatment F | Treatment B | Treatment D | Treatment A | Treatment C |
| 5 | Treatment B | Treatment E | Treatment A | Treatment F | Treatment C | Treatment D |
| 6 | Treatment A | Treatment B | Treatment C | Treatment E | Treatment D | Treatment F |

Treatment A: Belbuca 300 µg and oral placebo

Treatment B: Belbuca 600 µg and oral placebo

Treatment C: Belbuca 900 µg and oral placebo

Treatment D: Oxycodone 30 mg and buccal placebo

Treatment E: Oxycodone 60 mg and buccal placebo

Treatment F: Oral placebo and buccal placebo

Primary assessments include ventilatory responses to hypercapnia, and secondary assessments include pupillometry and safety measurements.

# 6.1 Sample Size Considerations

No formal sample size calculation was made. Based on similar studies, the number of subjects is considered appropriate for this Phase 1 study.

EDSREP 009 T 01 G 


# 6.2 Randomization

Subjects will be randomized to 1 of 6 treatment sequences (Table 1) according to the randomization code generated by the Biostatistics Department of PRA. The subject number will ensure identification throughout the study. Randomization numbers will range from 1001 to 1018. Replacement subjects will receive the number of the subject to be replaced, increased by 1000 (e.g., 2001 replacement number for subject number 1001), and will be administered the same (or remaining) treatments in the same order.

# 7.0 Overview of Planned Analysis

# 7.1 Changes from Protocol

There are no changes from the protocol.

# 7.2 Interim Analysis and Key Results

There will be no interim analyses or summaries of data provided prior to the delivery of the full set of post-lock tables, figures and listings (TFLs).

# 7.3 Final Analysis

Draft TFLs will be provided after database lock. After Sponsor comments have been incorporated, the TFLs will be finalized and incorporated in the first draft CSR.

#### 8.0 Data Review

# 8.1 Data Management

Data handling and transfer will take place under the PRA Data Management Plan for the study.

# 8.2 Acceptance of Data for Summarization

Programming of analysis datasets and TFLs may be ongoing during the data management of the study. However, programming of analysis datasets and TFLs will be completed and quality controlled (QC'd) after database lock. Only quality assured (QA'd) results released by the Safety Laboratory, Bioanalytical Laboratory, or other external data source will be used for the programming of analysis datasets and TFLs for the final report. Any data values requiring investigation or corrections that are identified while programming the analysis datasets and TFLs will be sent to the project Data Manager. If the issue affects the TFLs the Programmer or Statistician who identified the issue will follow it to resolution.

# 9.0 Definitions and General Analysis Methods

# 9.1 Analysis Data Presentation

# 9.1.1 Rounding

In listings all data will be presented with the same precision as the original data. Derived data will be rounded for presentation purposes.

For summaries, the minimum and maximum will be presented to the same number of decimal places as the original data, the mean, median, and quartiles (Q1 and Q3) will be presented to 1 decimal greater than the original data, and the standard deviation (SD) and standard error (SE) to 2 decimals greater than the original data. Frequency percentages and coefficient of variation (%CV) will be presented with 1 decimal.

EDSREP 009 T 01 G 




The above rule can be applied directly to collected data. For derived data rounding will occur prior to summarization so a specific number of decimal places will have to be assumed to apply the above rounding rules for summary statistics.

PK parameters will be rounded in the derived dataset as determined by the pharmacokineticist. Each parameter will have a fixed number of decimals. The pharmacokineticist will follow this rule when deciding the number of decimals for each parameter: no decimal if data for a parameter are generally greater than or equal to 100; 1 decimal if data are generally between 10 and 100; 2 decimals if data are generally between 1 and 10; 3 decimals if data are generally below 1.

PD parameters will be rounded in the derived dataset as guided by the statistician and presented as is in the listings. Each parameter will have a fixed number of decimals. The statistician will use discretion when deciding the number of decimals for each parameter.

P-values are descriptive only as there is no formal hypothesis test. P-values will be reported to four decimal places; p-values less than 0.0001 will be reported as p <0.0001.

## 9.1.2 Imputation

Unless otherwise noted, data will not be imputed.

# 9.1.3 Daylight Savings Time Adjustments

This study is not expected to fall over Daylight Savings Time and no adjustments for time change are planned.

#### 9.1.4 Descriptive Statistics

Unless otherwise indicated, continuous variables will be summarized with the following descriptive statistics: n (number of observations), (arithmetic) mean, standard deviation (SD), minimum (min) value, median, and maximum (max) value.

Categorical data will be summarized with frequencies and percentages. Percentages by categories will be based on the number of subjects exposed within a treatment.

For categorical data the categories will be presented in the tables exactly as they appear in the CRF / Database.

# 9.1.5 Pooling

Summary statistics will be calculated by treatment and timepoint, if applicable.

#### 9.1.6 Unscheduled Measurements

Unscheduled and early termination measurements will be included in the listings. With the exception of unscheduled measurements used for baseline, unscheduled measurements will be excluded from the descriptive statistics and statistical analysis.

# 9.2 Analysis Data Definitions

#### 9.2.1 Baseline Definition

Unless otherwise stated, baseline for all post-dose evaluations is defined as the last observation recorded before the first study drug administration, predose is defined as the last observation recorded before the first study drug administration in each period. The last observation can be an unscheduled / repeated measurement. If a pre-treatment observation is missing in a given period then the screening value may be used.

# 9.2.2 Treatment/Subject Grouping

EDSREP 009 T 01 G 


| Label | Grouping |
|---|---|
| Study Drug | Belbuca 300 μg, Belbuca 600 μg, Belbuca 900 μg, Oxycodone 30 mg,<br>Oxycodone 60 mg, oral placebo, buccal placebo |
| Treatment | Treatment A: Belbuca 300 µg and oral placebo Treatment B: Belbuca 600 µg and oral placebo Treatment C: Belbuca 900 µg and oral placebo Treatment D: Oxycodone 30 mg and buccal placebo Treatment E: Oxycodone 60 mg and buccal placebo Treatment F: Oral placebo and buccal placebo |
| Dose Level | Belbuca 300 μg, Belbuca 600 μg, Belbuca 900 μg, Oxycodone 30 mg, and Oxycodone 60 mg |

#### 9.2.3 Common Variable Derivations

| Variable | Data<br>Type | Definition/Calculation |
|---|---|---|
| Change from<br>Baseline/Predose | All | Post-dose Observation minus Baseline/Predose Observation |
| Analysis Study Day (Prior to Dose) | All | Date of Measurement minus Dose Date |
| Analysis Study Day (Post Dose) | All | Date of Measurement minus Dose Date +1 |
| Period | All | Interval of time during which treatment is constant. Treatment Phase only. |
| TEAE | ADAE | AE is a TEAE if the AE Date/Time is greater than or equal to the first dose Date/Time |

#### 9.2.4 QC

The analysis datasets and the TFLs will be QC'd according to the PRA EDS QC plan.

# 9.2.4.1 Critical Data

The QC plan requires datasets be classified as critical or non-critical. The datasets considered critical are subject level, pharmacokinetic, pharmacodynamic, and adverse events (ADSL, ADPC, ADPP, ADPD, ADAE). As these are related to the primary objectives these datasets will be double programmed per the QC Plan.

#### 9.2.5 ADaM Datasets and Metadata

The analysis datasets will be generated in accordance with Clinical Data Interchange Standard Consortium (CDISC) Analysis Data Model (ADaM) Version 2.1.

ADaM compliant datasets will be delivered to the sponsor. A define.xml file version 2 with the corresponding metadata will be included. Analysis results metadata are excluded.

EDSREP 009 T 01 G 




# 9.3 Software

The statistical analysis and reporting will be done using SAS® for Windows™ Version 9.4 or higher (SAS Institute, Inc.).

PK parameter calculations will primarily be done using Phoenix® WinNonlin® version 8.1 or higher (Certara, L.P.). Additional PK computations may be performed in SAS®.

# 9.4 Statistical Methods

#### 9.4.1 Statistical Outlier Determination

No statistical outlier analysis is planned.

# 9.4.2 Predetermined Covariates and Prognostic Factors

There are no predetermined covariates or prognostic factors.

# 9.4.3 Hypothesis Testing

Although no formal hypothesis testing will be done, the pairwise comparisons outlined in section 17.3 will be performed.

# 9.5 TFL Layout

Report layout will be according to the PRA EDS – ICH E3 compliant – CSR Template. The layout of TFLs will be according to the PRA EDS standards.

Table shells are provided with and approved as part of this SAP. Small changes to shell layout due to the nature of the data may be required after lock at the discretion of the PRA project statistician. Other changes to the shells may be out of scope. The TFLs will be provided as a single document in Adobe PDF format (in Letter format), and as individual files for each table, figure or listing in Rich Text Format (.rtf).

EDSREP 009 T 01 G 


# 10.0 Analysis Sets

| Analyses | Randomized<br>Set | Safety Set | PK Set | Completers | Partial<br>Completers |
|---|---|---|---|---|---|
| Disposition<br>Summaries | ✓ | ✓ | ✓ | ✓ | <b>✓</b> |
| Baseline<br>Characteristics | ✓ | ✓ | ✓ | ✓ | <b>✓</b> |
| Safety<br>Assessments | | <b>√</b> | | | |
| PK<br>Concentrations | | ✓ | | | |
| PK Parameters | | | ✓ | | |
| Primary PD<br>Analysis | | | | <b>✓</b> | <b>✓</b> |

#### 10.1 Randomized Set

The Randomized Set will consist of subjects who are assigned a randomization number in the study. This set will be used for disposition summaries. This set will be analyzed as randomized.

# 10.2 Safety Set

The Safety Set will consist of subjects who receive at least one dose of any study drug in the Treatment Phase. This set will be used for the safety data summaries, baseline characteristic summaries, and PK concentration summaries. This set will be analyzed as treated.

#### 10.3 Pharmacokinetic Set

The PK Set will consist of all subjects who receive at least 1 dose of any study drug during Treatment Phase and have sufficient concentration-time data to calculate at least one of the primary PK parameters  $(T_{max}, C_{max}, or AUC_{last})$ . Subjects or individual PK parameters may be excluded at the discretion of the pharmacokineticist (i.e. in the case of a protocol deviation). This set will be used for the PK parameters and will be analyzed as treated.

# 10.4 Completers Set

The Completer Set will consist of all randomized subjects who complete all 6 treatment periods in the Treatment Phase with a valid VRH  $V_E$   $E_{max}$  measurement in each completed treatment period. Subjects with any major protocol deviations may be excluded. This set will be used for all PD analyses and will be analyzed as treated.

#### 10.5 Partial Completers Set

The Partial Completer Set will consist of all randomized subjects who complete at least 2 treatment periods in the Treatment Phase with a valid VRH  $V_E$   $E_{max}$  measurement in each completed treatment period. Note that the mixed model used for this analysis (section 16.3) can accommodate subjects who may not complete all 6 treatment periods. Subjects with any major protocol deviations may be excluded. This set will be used for PD sensitivity analyses and will be analyzed as treated.

EDSREP 009 T 01 G 


# 11.0 Subject Disposition

The number and percentage of subjects randomized, dosed, and members of each analysis set will be presented. The number and percentage of subjects who withdrew from the study prematurely and a breakdown of the corresponding reasons for withdrawal will also be presented.

### 12.0 Protocol Deviations

Protocol deviations will be collected and entered into the Clinical Trial Management System (CTMS) per clinical monitoring Standard Operating Procedures. Important protocol deviation data will be listed by subject.

# 13.0 Demographic and Baseline Characteristics

# 13.1 Demographics

Subject demographics will be summarized overall for each analysis set. The summary will include the subjects' age (years), sex, race, ethnicity, weight (kg), height (cm), and BMI (kg/m²).

All demographic data as collected during the screening visit will be listed by subject.

# 13.2 Medical History

Medical history, categorized by preferred term according to MedDRA, will be summarized. The number and percentage of subjects in each preferred term will be displayed.

Medical history will be listed by subject.

# 13.3 Recreational Drug, Alcohol and Tobacco History

Recreational drug, alcohol and tobacco history will be summarized and listed by subject.

# 14.0 Concomitant Medications

Concomitant medications, categorized by medication group and subgroup according to WHO Drug Dictionary, will be summarized. The number and percentage of subjects using each medication will be displayed with the number and percentage of subjects using at least one medication within each medication group and subgroup, by treatment.

Concomitant medication will be listed by subject. Medications with an end date prior to the first dose of study drug will be considered prior medications and will be noted in the listing. If a partial date allows a medication to be considered concomitant it will be categorized as such.

# 15.0 Treatment Compliance and Exposure

The number of subjects receiving each dose of study drug will be summarized by treatment and listed.

# 16.0 Pharmacokinetic Analyses

# 16.1 Pharmacokinetic Variables

Concentrations and PK parameters of buprenorphine, nor-buprenorphine, and oxycodone will be collected in plasma, and the set of PK variables are considered exploratory endpoints.

EDSREP 009 T 01 G 


# 16.2 Plasma Pharmacokinetic Summaries

#### 16.2.1 Plasma Concentrations

Plasma concentrations for buprenorphine, nor-buprenorphine, and oxycodone below the quantifiable limit (BQL) will be set to 0 in the computation of mean concentration values. Descriptive statistics (number of subjects, arithmetic mean, geometric mean, SD, coefficient of variation, median, min, and max) will be used to summarize the plasma concentrations by treatment at each scheduled timepoint. If the mean at a given timepoint is BQL then the descriptive statistics will not be presented and will instead display as BQL for the mean and minimum. With the exception of n and max, all other statistics will be missing.

Linear and semi-logarithmic plots of the arithmetic mean plasma concentration by scheduled sampling time will be provided by treatment. These plots will show time in hours. The plots will show all calculated means and will show a reference line for LLOQ.

Linear and semi-logarithmic plots of the individual plasma concentration by actual sampling time will be provided by subject (one subject per page). These plots will show time in hours. Individual plots will use the BQL handling procedure described below for "Pharmacokinetic Parameters".

All individual subject plasma concentration data will be listed by subject.

#### 16.2.2 Plasma Pharmacokinetic Parameters

| Parameter | Description | Analyte | SAS Programming Notes |
|---|---|---|---|
| Cmax | Maximum plasma concentration. Observed peak analyte concentration obtained directly from the experimental data without interpolation, expressed in concentration units | All | Cmax from WNL |
| Tmax | Time to maximum plasma concentration. First observed time to reach peak analyte concentration obtained directly from the experimental data without interpolation, expressed in time units. | All | Tmax from WNL |
| AUClast | Area under the concentration-<br>time curve (time 0 to time of last<br>quantifiable concentration). | All | AUClast from WNL |
| AQ | Abuse quotient | All | Cmax/Tmax |
| Lz | Terminal phase rate constant calculated by linear regression of the terminal log-linear portion of the concentration vs. time curve. Linear regression of at least three points occurring after Cmax and an r <sup>2</sup> greater than 0.80 are | All | Lambda_z from WNL If Rsq ≤ .80 then parameter is not included |

EDSREP 009 T 01 G 


| | required to obtain a reliable λz. | | |
|---|---|---|---|
| t1/2 | Terminal phase half-life expressed in time units. Percent extrapolation less than or equal to 20% and r <sup>2</sup> greater than 0.80 is required to obtain a reliable t <sub>1/2</sub> . | All | HL_Lambda_z from WNL If AUC_%Extrap_obs >20% or Rsq ≤ .80 then parameter is not included |

Plasma PK parameters for buprenorphine, nor-buprenorphine, and oxycodone will be estimated using non-compartmental methods with WinNonlin®. The plasma PK parameters will be estimated from the concentration-time profiles, and AUCs will be calculated using linear up / log down. In estimating the PK parameters, BQL values will be set to zero. Actual sampling times, rather than scheduled sampling times, will be used in all computations involving sampling times. If the actual time is missing, the scheduled time may be substituted and flagged.

Determination of points to be included in λz range will follow the Guideline for Defining, Calculating and Summarizing Pharmacokinetic / Pharmacodynamic Parameters (EDSREP 009 R 01).

Descriptive statistics (number of subjects, mean, geometric mean, SD, coefficient of variation (%CV), median, min, and max) will be used to summarize the calculated PK parameters by treatment. For Tmax, only median, min and max will be presented.

# 17.0 Pharmacodynamic Analysis

All VRH summaries will be performed using the Completer Set. The selected measures will assess VRH associated with Belbuca relative to oxycodone and placebo, and oxycodone relative to placebo.

# 17.1 Pharmacodynamic Measurements

The PD measurements:  $V_E$ , RR, PEF,  $V_T$ , and ET<sub>CO2</sub> will be collected at each of the planned VRH timepoints listed in the Schedule of Assessments (See Appendix 2). Numerous observations will be recorded for each PD measurement at each of these timepoints; however, not all observations are considered clinically valid. Due to the sensitivity of the pneumotachometer machines, small adjustments in posture may be picked up by the machines resulting in false, or "artifact", breaths. For this reason, the following VRH output will be excluded:

- Where ET<sub>CO2</sub> is missing or marked as ".p" or ".u" by clinic staff
- Where V<sub>E</sub> is < 3 L/min or is > 60 L/min
- Where RR is < 4 breaths/min or is > 30 breaths/min

For each of these cases, the entire observation (all VRH measurements) will be excluded. Additionally, any observations recorded during the first 30 seconds of each timepoint ("filetimestamp <= 30" from file) will be excluded as the gas is not considered to have fully infiltrated the breathing machine and residual amounts of oxygen will still be present.

After the above exclusions have been made, one value will be derived for each PD measurement, per subject, per treatment, per timepoint (See table below for calculation of derived PD measurements).

| Pharmacodynamic Measurements | |
|---|---|
| Measurement | Description |
| VE | Minute ventilation. Volume of gas exhaled per minute from the lungs, expressed in L/min. Calculated as the mean $V_E$ measurement ("MV" from file) per subject, per treatment, per timepoint. |
| RR | Respiratory rate, expressed in breaths/min. |

EDSREP 009 T 01 G 




| Pharmacodynamic Measurements | |
|---|---|
| Measurement | Description |
| | Calculated as the mean RR measurement ["RR (spont)" from file] per subject, per treatment, per timepoint, excluding zeros. |
| | Peak expiratory flow rate. Maximum speed of expiration, expressed in L/min. |
| PEF | Calculated as the mean PEF measurement per subject, per treatment, per timepoint, excluding zeros. |
| V | Tidal volume. Volume of gas displaced between normal inhalation and exhalation when extra effort is not applied, expressed in mL. |
| VT | Calculated as the mean [sum of inspiratory and expiratory tidal volumes ("Tvi" + "Tve" from file)] per subject, per treatment, per timepoint, excluding zeros. |
| - | End tidal CO <sub>2</sub> . Partial pressure of carbon dioxide at the end of an exhaled breath, expressed in mm Hg. |
| ET <sub>CO2</sub> | Calculated as the mean ET <sub>CO2</sub> measurement per subject, per treatment, per timepoint, excluding zeros. |
| | Hypercapnic Ventilatory Response, expressed in L/min per mm Hg. |
| S | Calculated as the slope of the linear regression line created by plotting $V_E$ values versus $ET_{CO2}$ values for each subject per treatment per timepoint. This calculation will use all valid $V_E$ and $ET_{CO2}$ values prior to the calculation of mean $V_E$ and $ET_{CO2}$ values. See SAS code below. |
| | Ratio of V <sub>E</sub> / ET <sub>CO2</sub> , expressed in L/min per mm Hg. |
| R | Calculated as the mean of the ratios of $V_E$ / $ET_{CO2}$ for each subject per treatment per timepoint. This calculation will use all valid $V_E$ and $ET_{CO2}$ values prior to the calculation of mean $V_E$ and $ET_{CO2}$ values. |

The SAS PROC REG code for the calculation of S is as follows:

proc reg data= VRH; by subject treatment timepoint; model V<sub>E</sub> = ET<sub>CO2</sub>; ods output ParameterEstimates = Estimates; run:

PD measurements and derived changes from baseline will be summarized by treatment and scheduled timepoint using descriptive statistics (n, mean, SD, SE, %CV, median, Q1, Q3, min, and max).

Linear plots of the mean ( $\pm$ SD) PD measurements over time will be provided for V<sub>E</sub>, RR, PEF, V<sub>T</sub>, and ET<sub>CO2</sub> by treatment. These plots will show time in hours. Box plots of PD Emax parameters by treatment will also be presented.

Individual plots of V<sub>E</sub> versus ET<sub>CO2</sub> will be provided by treatment and timepoint, with a regression line and corresponding regression equation displayed for each treatment.

All valid PD measurements will be listed by subject.

# 17.2 Pharmacodynamic Parameters

The primary endpoint of interest is the PD parameter of maximum effect ( $E_{max}$ ) of minute ventilation:  $V_E$   $E_{max}$ .

Secondary endpoints of interest include the  $E_{max}$  values for the PD measurements: RR, PEF,  $V_T$ , and  $ET_{CO2}$ .

EDSREP 009 T 01 G 


| Pharmacodynamic Parameters | |
|---|---|
| Parameter | Description |
| E <sub>max</sub> | Maximum effect, obtained directly from the post-dose mean PD measurements: $V_E$ , RR, PEF, $V_T$ , and ET <sub>CO2</sub> , and from the postdose derived PD measurements: S and R, per subject and treatment. |

The PD measurement E<sub>max</sub> values will be summarized by treatment using descriptive statistics (n, mean, SD, SE, %CV, median, Q1, Q3, min, and max).

Box plots of the  $E_{max}$  of all PD measurements by treatment will be provided. The box plots will include the individual subject  $E_{max}$  values.

All PD parameters will be listed by subject.

# 17.3 Pharmacodynamic Statistical Analyses

The primary endpoint of interest for the analysis is the PD parameter: VE Emax.

The statistical analyses will be performed using the Completer population. The analyses will be repeated with the Partial Completer population for a sensitivity analysis (if not all subjects complete the 6 treatments). The treatment comparisons to assess the respiratory drive of Belbuca relative to oxycodone and placebo will include the following:

- Study Validity (Active Comparator vs. Placebo)
  - Oxycodone 30 mg vs placebo
  - Oxycodone 60 mg vs placebo
- Relative Respiratory Drive (Test vs. Active Comparator)
  - o Belbuca 300 ug vs Oxycodone 30 mg
  - o Belbuca 300 ug vs Oxycodone 60 mg
  - o Belbuca 600 ug vs Oxycodone 30 mg
  - o Belbuca 600 ug vs Oxycodone 60 mg
  - o Belbuca 900 ug vs Oxycodone 30 mg
  - o Belbuca 900 ug vs Oxycodone 60 mg
- Absolute Respiratory Drive (Test vs. Placebo)
  - o Belbuca 300 ug vs Placebo
  - o Belbuca 600 ug vs Placebo
  - o Belbuca 900 ug vs Placebo

As this is a pilot study which is not statistically powered to detect treatment differences, the results of the validity comparison will not affect the reporting of further comparisons.

The SAS mixed effects linear model procedure (PROC MIXED) will be used to construct analysis of variance (ANOVA) models. For each PD measurement:  $V_E$ , RR, PEF,  $V_T$ ,  $ET_{CO2}$ , S, and R, an analysis of the  $E_{max}$  values will be performed. The models will include terms for treatment, period, and sequence as fixed effects, with subject nested within sequence as a random effect.

The SAS PROC MIXED code for the  $E_{max}$  analyses is as follows:

proc mixed data= VRH\_Emax; by measurement; class subject treatment period sequence; model aval= treatment period sequence; random subject(sequence);

EDSREP 009 T 01 G 


```
Ismeans treatment;
***** Study Validity;
estimate 'Oxy 30 vs Placebo' treatment 0 0 0 1 0 -1 / e cl alpha=0.05;
estimate 'Oxy 60 vs Placebo' treatment 0 0 0 0 1 -1 / e cl alpha=0.05;
***** Relative Respiratory Drive;
estimate 'Bel 300 vs Oxy 30' treatment 1 0 0 -1 0 0 / e cl alpha=0.05;
estimate 'Bel 300 vs Oxy 60' treatment 1 0 0 0 -1 0 / e cl alpha=0.05;
estimate 'Bel 600 vs Oxy 30' treatment 0 1 0 -1 0 0 / e cl alpha=0.05;
estimate 'Bel 600 vs Oxy 60' treatment 0 1 0 0 -1 0 / e cl alpha=0.05;
estimate 'Bel 900 vs Oxy 30' treatment 0 0 1 -1 0 0 / e cl alpha=0.05;
estimate 'Bel 900 vs Oxy 60' treatment 0 0 1 0 -1 0 / e cl alpha=0.05;
***** Absolute Respiratory Drive;
estimate 'Bel 300 vs Placebo' treatment 1 0 0 0 0 0 -1/e cl alpha=0.05;
estimate 'Bel 600 vs Placebo' treatment 0 1 0 0 0 0 -1/e cl alpha=0.05;
estimate 'Bel 900 vs Placebo' treatment 0 0 1 0 0 0 -1/e cl alpha=0.05;
run;
```

A summary table will include the least squares (LS) mean for the test and reference  $E_{\text{max}}$  value for each parameter, as well as the LS mean difference (test-reference) and 95% confidence interval (CI) and p-value.

# 18.0 Secondary Endpoints

- Pupillometry
- Change in ratio of minute ventilation over end-tidal CO2

Pupillometry measurements and changes from predose at each post baseline timepoint will be summarized by treatment using descriptive statistics (n, mean, SD, SE, %CV, median, Q1, Q3, min, and max). Pupillometry data will also be listed for each subject by treatment and timepoint.

The change in ratio of minute ventilation over end-tidal CO2 will be presented in a graph, plotting each individual subject's minute ventilation (V<sub>E</sub>) versus end tidal CO2 (ET<sub>CO2</sub>), and also including the regression equations and regression lines for all treatments at each planned timepoint.

# 19.0 Safety Analyses

# 19.1 Safety Variables

- Adverse Events (AEs)
- Clinical Laboratory Evaluations
  - Clinical chemistry
  - Hematology
  - o Urinalysis
  - Serology
  - Pregnancy test and FSH
  - o Urine drug screen
  - Alcohol breath test
- Vital Signs
  - Supine Blood Pressure
    - Systolic blood pressure
    - Diastolic blood pressure
  - o Pulse rate
  - Oral body temperature
  - o Respiratory Rate

EDSREP 009 T 01 G 


- Oxygen Saturation
- Electrocardiograms (ECG)
  - o Heart rate
  - o PR interval
  - o QRS-Duration
  - o QT interval
  - o QTc (Frederica) interval
- Continuous pulse oximetry
- Physical examinations
- Columbia-Suicide Severity Rating Scale (C-SSRS)
- Cardiac Telemetry (continuous measurement during VHR testing)
- COWS (assessments of opiate withdrawal symptoms during Naloxone Challenge)

#### 19.1.1 Adverse Events

Treatment emergence will be evaluated for all AEs. Treatment-emergent adverse events (TEAE) are those which occur after the first dose of study drug.

TEAEs occurring following dosing in a specific period but before dosing in the next period will be attributed to the treatment in that period. If the time is missing for an AE on a dosing day then the AE will be attributed to the treatment given on that day.

The following missing data will be imputed as defined (for calculations only / will not be presented):

- Missing AE start and / or end times for the calculation of onset and duration will be assumed to be at 00:01 for a start time and 23:59 for end times
- Missing AE severity or relationship will be assumed to be severe or related, respectively
- Missing AE start times for the determination of treatment emergence will be assumed to occur
  after treatment unless partial date documents the AE as happening prior to treatment
- Missing AE start times for the determination of treatment assignment will be assumed to occur after treatment on the recorded date one minute after dosing
- Missing AE start date will be assumed to be after treatment for the determination of TEAE but will not be attributed to a specific treatment.

A summary of number and percentage of subjects reporting TEAEs, TEAEs by severity and relationship, serious AEs (SAEs), and subjects who discontinued study drug due to an AE will be provided.

A summary of the number and percentage of subjects reporting each TEAE, categorized by system organ class and preferred term coded according to the Medical Dictionary for Regulatory Activities (MedDRA), will be presented by treatment, and overall. Counting will be done by subject only, not by event; subjects will only be counted once within each body system or preferred term.

A summary of the number and percentage of subjects reporting each TEAE will be presented according to relationship to study drug (as recorded on the eCRF), by treatment and overall. Subjects with multiple events within a system organ class or preferred term will be counted under the category of their most drug-related event within that system organ class or preferred term.

A summary of the number and percentage of subjects reporting each TEAE will be presented according to severity (as recorded on eCRF), by treatment and overall. Subjects with multiple events within a system organ class or preferred term will be counted under the category of their most severe event within that system organ class or preferred term.

All AEs (including non-treatment-emergent events) recorded on the eCRF will be listed by subject.

A separate listing of AEs leading to study drug discontinuation will be provided.

#### 19.1.2 Deaths and Serious Adverse Events

A listing of deaths and other SAEs will be provided by subject.

EDSREP 009 T 01 G 


# 19.1.3 Laboratory Data

Clinical laboratory data will be presented using units from the study data tabulation model (SDTM) Controlled Terminology.

Descriptive statistics summarizing continuous laboratory results of clinical chemistry, hematology, and urinalysis (and changes from baseline) by visit will be provided. A summary table of shifts from baseline will also be provided.

All laboratory data will be listed by subject, including laboratory variables not listed in the protocol. A separate listing of out-of-range values will also be provided. Normal ranges will be used directly from the clinical laboratory and will be included in the listings for reference.

# 19.1.4 Vital Signs

Descriptive statistics summarizing vital signs (and changes from predose) by treatment and scheduled time will be provided.

All vital signs will be listed by subject.

# 19.1.5 Electrocardiograms

Descriptive statistics summarizing ECG parameters (and changes from predose) by treatment and visit (Day -1 and Day 2 for each treatment period) will be provided. A summary table of shifts from predose will also be provided.

All ECG parameters and the corresponding abnormalities will be listed by subject.

# 19.1.6 Continuous Pulse Oximetry

Continuous pulse oximetry will be performed throughout the study during the VRH tests, from at least 15 minutes predose until 8 hours postdose. Data will not be recorded in the database but will be used for real-time safety monitoring. Oxygen saturation data will be presented in a descriptive statistics summary table by treatment and timepoint. Individual subject data will be presented in a listing. Observations of abnormal data that lead to medical treatment, non-scheduled procedures and/or discontinuation from the study will be recorded as AEs.

#### 19.1.7 Physical Examinations

Physical examination result shifts from Baseline (screening visit) to Day 2 of each treatment period will be summarized by treatment. All physical examination data will also be listed by subject.

# 19.1.8 Cardiac Telemetry

A listing of the start and stop times for cardiac telemetry will be provided. Any clinically significant abnormal objective test findings will be recorded as AEs..

#### 19.1.9 Columbia-Suicide Severity Rating Scale

The C-SSRS data will be listed by subject and timepoint.

### 19.1.10 Clinical Opiate Withdrawal Scale

COWS results will be listed by subject.

# 20.0 References

SAS Institute, Inc., SAS® Version 9.4 software, Cary, NC.

EDSREP 009 T 01 G 




**Appendix 1: Glossary of Abbreviations** 

| Glossary of Abbre | eviations: |
|---|---|
| AE | Adverse event |
| ADaM | Analysis data model |
| AUC | Area under the curve |
| ANOVA | Analysis of variance |
| ВМІ | Body mass index |
| BP | Blood pressure |
| BQL | Below the quantifiable limit |
| CDISC | Clinical Data Interchange Standard Consortium |
| CI | Confidence interval |
| cows | Clinical Opiate Withdrawal Scale |
| CO2 | Carbon dioxide |
| CSR | Clinical study report |
| C-SSRS | Columbia Suicide Severity Rating Scale |
| CTMS | Clinical Trial Management System |
| CV | Coefficient of variation |
| ECG | Electrocardiogram |
| eCRF | Electronic case report form |
| E <sub>MAX</sub> | Maximum effect |
| EDS | Early Development Services |
| FSH | Follicle stimulating hormone |
| HR | Heart rate |
| ICH | The International Conference on Harmonization of Technical Requirements for Registration of Pharmaceuticals for Human Use |
| LLOQ | Lower limit of quantification |
| LOCF | Last observation carried forward |
| MedDRA | Medical Dictionary for Regulatory Activities |
| PD | Pharmacodynamic |
| PEF | Peak expiratory flow |
| PK | Pharmacokinetic |
| QA'd | Quality assured |
| QC'd | Quality controlled |

EDSREP 009 T 01 G Page 20 of 21






| Version Date: 07-Oct-2019 |
|---------------------------|

| QTc | Corrected QT interval |
|----------------|------------------------------------------------------|
| RR | Respiration rate |
| SAP | Statistical analysis plan |
| SAE | Serious adverse event |
| SDTM | Study data tabulation model |
| SPO2 | Peripheral capillary oxygen saturation |
| TEAE | Treatment-emergent adverse event |
| TFL(s) | Tables, figures and listings |
| VE | Minute ventilation |
| VRH | Ventilatory response to hypercapnia |
| V <sub>T</sub> | Tidal volume |
| WHO-DDE | World Health Organization – Drug Dictionary Enhanced |
| WNL | WinNonlin |

EDSREP 009 T 01 G Page 21 of 22




# **Appendix 2: Schedule of Assessments**

| | Screening | Inj | oatient Visi | t | Early Termination | Follow-Up Call |
|---|---|---|---|---|---|---|
| Visit ID | V1 | V2-V7 <sup>a</sup> | | | ET | V9 |
| Study Day(s) Procedures | -28 to -2 | -1 | 1 | 2 | | 7 days from final<br>IMP<br>(+/- 2 days) |
| Informed consent | X | | | | | |
| Eligibility criteria | Х | confirm | | | | |
| Demographics | Х | | | | | |
| Medical history, including recreational drug use history | Х | update | | | | |
| Physical examination | Х | | | Х | Xp | |
| Oral mucosa examination | Х | Х | | | | |
| Pregnancy test <sup>c</sup> | Х | Х | | | | |
| Follicle stimulating hormone and estradiol leveld | Х | | | | | |
| Height, weight, BMI | Х | | | | | |
| Blood pressure, heart rate, and respiration rate | Х | Х | Xe | Х | Х | |
| Temperature | Х | Х | Xe | Х | Х | |
| O <sub>2</sub> saturation | Х | | Xe | Х | Х | |
| Continuous pulse oximetry | | | X <sup>f</sup> | | | |
| 12-lead ECG | Х | Х | | Х | Х | |
| Continuous cardiac telemetry | | | Xg | | | |
| Chemistry and hematology labs <sup>h</sup> | X | Х | | | Х | |
| Viral serology (HBsAG, anti-HCV, HIV) | X | | | | | |
| Urinalysis | Х | Х | | | Х | |
| Alcohol breathalyzer/urine drug screen | Х | Х | | | | |
| Naloxone Challenge <sup>i</sup> | | Х | | | | |
| Randomization (first treatment period only) | | | Х | | | |

EDSREP 009 T 01 G 



Statistical Analysis Plan BDL673SL-186739 Protocol: BUP-401

Version Date: 07-Oct-2019

| IMP administration | | | Х | | | |
|-------------------------------------|---|---|----|---|---|---|
| Pupillometry | | | Xe | | | |
| Ventilatory Response to Hypercapnia | Х | | Xj | | | |
| PK <sup>k</sup> | | | Х | | | |
| C-SSRS <sup>I</sup> | X | Х | | | X | |
| Adverse events | | | Х | Х | X | X |
| Prior/Concomitant medications | X | Х | Х | Х | X | X |
| Discharge from clinic | | | | Х | | |

BMI=body mass index; C-SSRS=Columbia-Suicide Severity Rating Scale; ECG=electrocardiogram; ET=early termination; HBsAg=hepatitis B surface antigen; HCV=hepatitis C virus; HIV=human immunodeficiency virus; ID=identification; IMP=investigational medicinal product; PK=pharmacokinetics

EDSREP 009 T 01 G 

<sup>&</sup>lt;sup>a</sup> Each treatment period will be separated by at least 7 days.

<sup>&</sup>lt;sup>b</sup> Physical examination to be completed at ET at discretion of investigator. Unscheduled symptom-directed PEs may be conducted at any time per the investigator's discretion.

<sup>&</sup>lt;sup>c</sup> Serum pregnancy test will be done for all female subjects at screening. Urine pregnancy test will be done for all female subjects at check-in to each period.

<sup>&</sup>lt;sup>d</sup> Postmenopausal female subjects only to confirm postmenopausal status.

e Vital signs, and pupillometry collected at predose and 0.5, 1, 1.5, 2, 2.5, 3, and 4 hours postdose. Body temperature collected once predose each treatment period.

<sup>&</sup>lt;sup>f</sup> Continuous pulse oximetry from at least 15 minutes predose through 8 hours postdose, and recorded at 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, and 8 hours postdose.

<sup>&</sup>lt;sup>9</sup> Continuous cardiac telemetry during VRH procedures from at least 15 minutes predose until at least 4 hours postdose.

<sup>&</sup>lt;sup>h</sup> Creatinine clearance and thyroid stimulating hormone (TSH) will be measured at screening only.

<sup>&</sup>lt;sup>1</sup> Naloxone challenge will be done during Treatment Period 1 and will consist of vital signs (BP, HR, RR and O<sub>2</sub> Saturation) at least 30 minutes before naloxone administration and at 5 minutes, 30 minutes and 60 minutes after administration. Clinical Opiate Withdrawal Scale (COWS) associated with the naloxone challenge will occur immediately predose and within 1 minute and 5 minutes after administration of naloxone.

<sup>&</sup>lt;sup>j</sup> VRH at predose and 0.5, 1, 2, 3, and 4 hours postdose.

<sup>&</sup>lt;sup>k</sup> PK at predose, 0.5, 1, 2, 3, 4, and 6 hours postdose.

<sup>&</sup>lt;sup>1</sup> C-SSRS Baseline version will be used at screening. At the subsequent visits, C-SSRS Since Last Visit version will be used.



# **Appendix 3: List of End of Text Outputs**

| End of Text Tabl | es and Figures: | |
|---|---|---|
| Output | Title | Analysis Set |
| | Demographic Data | |
| Table 14.1.1 | Summary of Analysis Sets | All Analysis<br>Sets |
| Table 14.1.2 | Summary of Subject Disposition | All Analysis<br>Sets |
| Table 14.1.3 | Summary of Dosing | Safety |
| Table 14.1.4 | Summary of Demographics | All Analysis<br>Sets |
| Table 14.1.5 | Summary of Recreational Drug Use History | Safety |
| | PD and PK Summaries | |
| Table 14.2.1.1 | Summary of VRH Measurements and Changes from Baseline | Completer |
| Table 14.2.1.2 | Summary of VRH Parameters | Completer |
| Table 14.2.2 | Statistical Analysis of Respiratory Drive of Belbuca | Completer |
| Table 14.2.3 | Statistical Analysis of Respiratory Drive of Belbuca | Partial<br>Completer |
| Figure 14.2.4.1 | Plot of Mean (±SD) Minute Ventilation over Time | Completer |
| Figure 14.2.4.2 | Box Plot of Minute Ventilation E <sub>max</sub> by Treatment | Completer |
| Figure 14.2.5.1 | Plot of Mean (±SD) Respiratory Rate over Time | Completer |
| Figure 14.2.5.2 | Box Plot of Respiratory Rate E <sub>max</sub> by Treatment | Completer |
| Figure 14.2.6.1 | Plot of Mean (±SD) Peak Expiratory Flow Rate over Time | Completer |
| Figure 14.2.6.2 | Box Plot of Respiratory Rate E <sub>max</sub> by Treatment | Completer |
| Figure 14.2.7.1 | Plot of Mean (±SD) Tidal Volume over Time | Completer |
| Figure 14.2.7.2 | Box Plot of Tidal Volume E <sub>max</sub> by Treatment | Completer |
| Figure 14.2.8.1 | Plot of Mean (±SD) End Tidal CO <sub>2</sub> over Time | Completer |
| Figure 14.2.8.2 | Box Plot of End Tidal CO <sub>2</sub> E <sub>max</sub> by Treatment | Completer |
| Figure 14.2.9.1 | Plot of Individual Minute Ventilation versus End Tidal CO <sub>2</sub> | Completer |
| Figure 14.2.9.2 | Box Plot of Slope E <sub>max</sub> by Treatment | Completer |
| Figure 14.2.9.3 | Box Plot of Ratio E <sub>max</sub> by Treatment | Completer |
| Table 14.2.10 | Summary of Pupillometry and Changes from Predose | Completer |
| Table 14.2.11.1 | Summary of Plasma Concentrations of Belbuca | Safety |
| Table 14.2.11.2 | Summary of Plasma Concentrations of Oxycodone | Safety |
| Table 14.2.12.1 | Summary of Plasma Pharmacokinetic Parameters of Belbuca | PK |
| Table 14.2.12.2 | Summary of Plasma Pharmacokinetic Parameters of Oxycodone | PK |
| Figure 14.2.13.1 | Plot of Mean (±SD) Plasma Concentrations Versus Time on a Linear Scale - Belbuca | PK |
| Figure 14.2.13.2 | Plot of Mean (±SD) Plasma Concentrations Versus Time on a | PK |

EDSREP 009 T 01 G 


| | Linear Scale - Oxycodone | |
|---|---|---|
| Figure 14.2.13.3 | Plot of Mean (±SD) Plasma Concentrations Versus Time on a Semi-Log Scale - Belbuca | PK |
| Figure 14.2.13.4 | Plot of Mean (±SD) Plasma Concentrations Versus Time on a Semi-Log Scale - Oxycodone | PK |
| Figure 14.2.13.5 | Plot of Individual Plasma Concentrations Versus Time on a Linear Scale - Belbuca | PK |
| Figure 14.2.13.6 | Plot of Individual Plasma Concentrations Versus Time on a Linear Scale - Oxycodone | PK |
| Figure 14.2.13.7 | Plot of Individual Plasma Concentrations Versus Time on a Semi-<br>Log Scale - Belbuca | PK |
| Figure 14.2.13.8 | Plot of Individual Plasma Concentrations Versus Time on a Semi-<br>Log Scale - Oxycodone | PK |
| | Safety Data | |
| Table 14.3.1.1 | Summary of Adverse Events | Safety |
| Table 14.3.1.2 | Summary of Treatment Emergent Adverse Events by System Organ Class and Preferred Term | Safety |
| Table 14.3.1.3 | Summary of Treatment Emergent Adverse Events by Relationship to Study Drug | Safety |
| Table 14.3.1.4 | Summary of Treatment Emergent Adverse Events by Severity | Safety |
| Table 14.3.2 | Listing of Deaths and Other Serious Adverse Events | All Subjects |
| Table 14.3.3 | Not part of the TFLs – Reserved for narratives in the CSR | |
| Table 14.3.4 | Listing of Abnormal Laboratory Values | All Subjects |
| Table 14.3.5.1 | Summary of Laboratory Results | Safety |
| Table 14.3.5.2 | Summary of Laboratory Shifts from Baseline | Safety |
| Table 14.3.6 | Summary of Vital Signs | Safety |
| Table 14.3.7 | Summary of Continuous Oxygen Saturation Monitoring | Safety |
| Table 14.3.8.1 | Summary of 12-Lead Electrocardiograms | Safety |
| Table 14.3.8.2 | Summary of 12-Lead Electrocardiograms Shifts from Predose | Safety |
| Table 14.3.9 | Summary of Physical Exam Shifts from Baseline | Safety |

| End of Text Listings: | |
|---|---|
| Output | Title |
| Listing 16.2.1.1 | Subject Disposition |
| Listing 16.2.1.2 | Medical History |
| Listing 16.2.1.3 | Prior and Concomitant Medications |
| Listing 16.2.2 | Not part of the TFLs – Reserved for protocol deviations in the CSR |
| Listing 16.2.3 | Analysis Populations |
| Listing 16.2.4.1 | Subject Demographics |

EDSREP 009 T 01 G 


| Listing 16.2.4.2 | Recreational Drug History |
|---|---|
| Listing 16.2.5.1 | Naloxone Challenge Dosing |
| Listing 16.2.5.2 | Clinical Opiate Withdrawal Scale Results |
| Listing 16.2.5.3 | Study Drug Administration |
| Listing 16.2.6.1 | VRH Measurements |
| Listing 16.2.6.2 | VRH Parameters |
| Listing 16.2.6.3.1 | Listing of Plasma Concentrations of Belbuca |
| Listing 16.2.6.3.2 | Listing of Plasma Concentrations of Oxycodone |
| Listing 16.2.6.4.1 | Listing of Plasma Pharmacokinetic Parameters of Belbuca |
| Listing 16.2.6.4.2 | Listing of Plasma Pharmacokinetic Parameters of Oxycodone |
| Listing 16.2.6.5 | Listing of Pupillometry |
| Listing 16.2.7.1 | Adverse Events |
| Listing 16.2.7.2 | Adverse Events Resulting in Discontinuation |
| Listing 16.2.8.1 | Clinical Laboratory Results – Hematology |
| Listing 16.2.8.2 | Clinical Laboratory Results – Chemistry |
| Listing 16.2.8.3 | Clinical Laboratory Results – Urinalysis |
| Listing 16.2.8.4 | Clinical Laboratory Results – Additional |
| Listing 16.2.8.5 | Clinical Laboratory Results – Urine Drug Screen and Alcohol Breath |
| Listing 16.2.9 | Vital Signs |
| Listing 16.2.10 | 12-Lead Electrocardiograms |
| Listing 16.2.11 | Physical Examinations |
| Listing 16.2.12 | Columbia-Suicide Severity Rating Scale Results |
| Listing 16.2.13 | SPO2 Monitoring |
| Listing 16.2.14 | Cardiac Telemetry |

| Other Appendix Outputs: | |
|-------------------------|------------------------|
| Output | Title |
| Appendix 16.1.9.2 | Statistical Appendices |

EDSREP 009 T 01 G 



# Appendix 4: Shells for Post-Text Tables, Figures and Listings Shells are provided in a separate document.

chene are previous in a coparate accumen

# 21.0 Document History

| Version Date | Modified/Reviewed<br>By | Brief Summary of Changes (if created from a template, include template code) |
|---|---|---|
| 23-Sep-2019 | Jacqueline Cater<br>Reilly Reis<br>Thomas Thompson | |

| Effective Date | | Brief Summary of Changes (if created from a template, include template code) |
|---|---|---|
| | Dy | template, include template code |

EDSREP 009 T 01 G 


BioDelivery Sciences, Inc. Protocol: BUP-401

# Appendix 16.1.9.2.1 Statistical Methods and Analysis Output Supporting Table 14.2.2 Supporting Table 14.2.2

#### The Mixed Procedure

#### Parameter Code=ETCOEMAX

#### Model Information

| Data Set | WORK.ADXV |
|---------------------------|---------------------|
| Dependent Variable | AVAL |
| Covariance Structure | Variance Components |
| Estimation Method | REML |
| Residual Variance Method | Profile |
| Fixed Effects SE Method | Model-Based |
| Degrees of Freedom Method | Containment |

#### Class Level Information

| Class | LevelsValues |
|---|---|
| SUBJID | 151001 1002 1003 1004 1005 1006 1007 1008 1010 1012 1013 1014 1015 1016 1017 |
| TRTPN | 61 2 3 4 5 6 |
| APERIOD | 6P1 P2 P3 P4 P5 P6 |
| ARMCD | 6ABCEDF BEAFCD CADBFE DCFAEB EFBDAC FDECBA |

| Dimensions | | |
|-------------|------------|----|
| Covariance | Parameters | 2 |
| Columns in | X | 19 |
| Columns in | Z | 15 |
| Subjects | | 1 |
| Max Obs per | Subject | 90 |

BioDelivery Sciences, Inc. Protocol: BUP-401

#### Appendix 16.1.9.2.1 Statistical Methods and Analysis Output Supporting Table 14.2.2 Supporting Table 14.2.2

The Mixed Procedure

#### Parameter Code=ETCOEMAX

| Number | of | Observations | Read | 90 |
|--------|----|--------------|----------|----|
| Number | of | Observations | Used | 90 |
| Number | of | Observations | Not Used | 0 |

# Iteration History Iteration Evaluations -2 Res Log Like Criterion 0 1 425.16851375 1 1 403.50606077 0.00000000

Convergence criteria met.

# Estimates Cov Parm Estimate SUBJID(ARMCD) 5.9883 Residual 6.3569

Covariance Parameter

| Fit Statistics | |
|--------------------------|-------|
| -2 Res Log Likelihood | 403.5 |
| AIC (Smaller is Better) | 407.5 |
| AICC (Smaller is Better) | 407.7 |
| BIC (Smaller is Better) | 408.9 |

Program: A Biol.sas Created: 02APR2020 7:35 POSTLOCK 

The Mixed Procedure

Parameter Code=ETCOEMAX

Type 3 Tests of Fixed Effects
Num Den

| | Nulli | Jen | |
|---------|-------|------|--------------|
| Effect | DF | DF F | Value Pr > F |
| TRTPN | 5 | 65 | 2.920.0193 |
| APERIOD | 5 | 65 | 0.490.7801 |
| ARMCD | 5 | 9 | 0.770.5916 |

Coefficients for Oxy 30 vs Placebo
Planned Planned

| | Arm | Treatm | nent |
|----------|--------------|--------|------|
| Effect | APERIOD Code | (N) | Row1 |
| Intorgor | + | | |

| Filect | APERIOD | loae (N | I) KOWI |
|----------|---------|---------|---------|
| Intercep | t | | _ |
| TRTPN | | 1 | |
| TRTPN | | 2 | |
| TRTPN | | 3 | |
| TRTPN | | 4 | 1 |
| TRTPN | | 5 | |
| TRTPN | | 6 | -1 |
| APERIOD | P1 | | |
| APERIOD | P2 | | |
| APERIOD | Р3 | | |
| APERIOD | P4 | | |
| APERIOD | P5 | | |
| APERIOD | P6 | | |
| ARMCD | I | ABCEDF | |
| ARMCD | E | BEAFCD | |
| ARMCD | C | CADBFE | |
| ARMCD | Ι | CFAEB | |

#### The Mixed Procedure

#### Parameter Code=ETCOEMAX

#### Coefficients for Oxy 30 vs Placebo

Planned Planned

 Arm
 Treatment

 Effect
 APERIOD Code
 (N)
 Row1

 ARMCD
 EFBDAC

 ARMCD
 FDECBA

#### Coefficients for Oxy 60 vs Placebo

Planned Planned Arm Treatment

| | | Z 3 11 111 | I I Ca chich c | |
|-----------|---------|------------|----------------|------|
| Effect | APERIOD | Code | (N) | Row1 |
| Intercept | | | | |
| TRTPN | | | 1 | |
| TRTPN | | | 2 | |
| TRTPN | | | 3 | |
| TRTPN | | | 4 | |
| TRTPN | | | 5 | 1 |
| TRTPN | | | 6 | -1 |
| APERIOD | P1 | | | |
| APERIOD | P2 | | | |
| APERIOD | P3 | | | |
| APERIOD | P4 | | | |
| APERIOD | P5 | | | |
| APERIOD | P6 | | | |
| ARMCD | | ABCEDF | | |
| ARMCD | | BEAFCD | | |
| ARMCD | | CADBFE | | |
| ARMCD | | DCFAEB | | |

Program: A\_Biol.sas Created: 02APR2020 7:35 POSTLOCK 

The Mixed Procedure

#### Parameter Code=ETCOEMAX

Coefficients for Oxy 60 vs Placebo

Planned Planned

 Arm
 Treatment

 Effect
 APERIOD Code
 (N)
 Row1

 ARMCD
 EFBDAC

 ARMCD
 FDECBA

Coefficients for Bel 300 vs Oxy 30

Planned Planned
Arm Treatment

| | | Arm | Treatment | |
|-----------|---------|--------|-----------|------|
| Effect | APERIOD | Code | (N) | Row1 |
| Intercept | | | | |
| TRTPN | | | 1 | 1 |
| TRTPN | | | 2 | |
| TRTPN | | | 3 | |
| TRTPN | | | 4 | -1 |
| TRTPN | | | 5 | |
| TRTPN | | | 6 | |
| APERIOD | P1 | | | |
| APERIOD | P2 | | | |
| APERIOD | P3 | | | |
| APERIOD | P4 | | | |
| APERIOD | P5 | | | |
| APERIOD | P6 | | | |
| ARMCD | | ABCEDF | | |
| ARMCD | | BEAFCD | | |
| ARMCD | | CADBFE | | |
| ARMCD | | DCFAEB | | |

Program: A\_Bio1.sas Created: 02APR2020 7:35 POSTLOCK


#### The Mixed Procedure

#### Parameter Code=ETCOEMAX

Coefficients for Bel 300 vs Oxy 30

Planned Planned

 Arm
 Treatment

 Effect
 APERIOD Code
 (N)
 Row1

 ARMCD
 EFBDAC

 ARMCD
 FDECBA

Coefficients for Bel 300 vs Oxy 60 Planned Planned

| | | Arm | Treatment | |
|-----------|---------|--------|-----------|------|
| Effect | APERIOD | Code | (N) | Row1 |
| Intercept | | | | |
| TRTPN | | | 1 | 1 |
| TRTPN | | | 2 | |
| TRTPN | | | 3 | |
| TRTPN | | | 4 | |
| TRTPN | | | 5 | -1 |
| TRTPN | | | 6 | |
| APERIOD | P1 | | | |
| APERIOD | P2 | | | |
| APERIOD | P3 | | | |
| APERIOD | P4 | | | |
| APERIOD | P5 | | | |
| APERIOD | P6 | | | |
| ARMCD | | ABCEDF | | |
| ARMCD | | BEAFCD | | |
| ARMCD | | CADBFE | | |
| ARMCD | | DCFAEB | | |

#### The Mixed Procedure

#### Parameter Code=ETCOEMAX

Coefficients for Bel 300 vs Oxy 60

Planned Planned

Treatment

Arm Treatment Effect APERIOD Code Row1 ARMCD EFBDAC ARMCD **FDECBA** 

Coefficients for Bel 600 vs Oxy 30 Planned Planned Arm

Effect APERIOD Code (N) Row1 Intercept TRTPN 1 1 3 -1

TRTPN TRTPN TRTPN TRTPN TRTPN APERIOD P1 APERIOD P2 APERIOD P3 APERIOD P4 APERIOD P5 APERIOD P6 ARMCD ABCEDF ARMCD BEAFCD ARMCD CADBFE ARMCD DCFAEB

Program: A Biol.sas Created: 02APR2020 7:35 POSTLOCK

#### The Mixed Procedure

#### Parameter Code=ETCOEMAX

Coefficients for Bel 600 vs Oxy 30

Planned Planned

 Arm
 Treatment

 Effect
 APERIOD Code
 (N)
 Row1

 ARMCD
 EFBDAC

 ARMCD
 FDECBA

Coefficients for Bel 600 vs 0xy 60
Planned Planned

Arm Treatment

| | | 7 1 T 111 | II Ca chichi c | • |
|----------|---------|-----------|----------------|------|
| Effect | APERIOD | Code | (N) | Row1 |
| Intercep | t | | | |
| TRTPN | | | 1 | |
| TRTPN | | | 2 | 1 |
| TRTPN | | | 3 | |
| TRTPN | | | 4 | |
| TRTPN | | | 5 | -1 |
| TRTPN | | | 6 | |
| APERIOD | P1 | | | |
| APERIOD | P2 | | | |
| APERIOD | Р3 | | | |
| APERIOD | P4 | | | |
| APERIOD | P5 | | | |
| APERIOD | P6 | | | |
| ARMCD | | ABCEDF | | |
| ARMCD | | BEAFCD | | |
| ARMCD | | CADBFE | | |
| ARMCD | | DCFAEB | | |
The Mixed Procedure

### Parameter Code=ETCOEMAX

Coefficients for Bel 600 vs Oxy 60

Planned Planned

 Arm
 Treatment

 Effect
 APERIOD Code
 (N)
 Row1

 ARMCD
 EFBDAC

 ARMCD
 FDECBA

Coefficients for Bel 900 vs Oxy 30 Planned Planned

Arm Treatment

| | | 2 2 2 111 | I I Ca chichi c | |
|-----------|--------|-----------|-----------------|------|
| Effect | APERIO | ) Code | (N) | Row1 |
| Intercept | 5 | | | |
| TRTPN | | | 1 | |
| TRTPN | | | 2 | |
| TRTPN | | | 3 | 1 |
| TRTPN | | | 4 | -1 |
| TRTPN | | | 5 | |
| TRTPN | | | 6 | |
| APERIOD | P1 | | | |
| APERIOD | P2 | | | |
| APERIOD | Р3 | | | |
| APERIOD | P4 | | | |
| APERIOD | P5 | | | |
| APERIOD | P6 | | | |
| ARMCD | | ABCEDF | | |
| ARMCD | | BEAFCD | | |
| ARMCD | | CADBFE | | |
| ARMCD | | DCFAEB | | |

Program: A Biol.sas Created: 02APR2020 7:35 POSTLOCK 

The Mixed Procedure

### Parameter Code=ETCOEMAX

Coefficients for Bel 900 vs Oxy 30

Planned Planned

 Effect
 APERIOD Code
 (N)
 Row1

 ARMCD
 EFBDAC

 ARMCD
 FDECBA

Coefficients for Bel 900 vs Oxy 60
Planned Planned

| | | Arm | Treatment | |
|-----------|---------|--------|-----------|------|
| Effect | APERIOD | Code | (N) | Row1 |
| Intercept | | | | |
| TRTPN | | | 1 | |
| TRTPN | | | 2 | |
| TRTPN | | | 3 | 1 |
| TRTPN | | | 4 | |
| TRTPN | | | 5 | -1 |
| TRTPN | | | 6 | |
| APERIOD | P1 | | | |
| APERIOD | P2 | | | |
| APERIOD | P3 | | | |
| APERIOD | P4 | | | |
| APERIOD | P5 | | | |
| APERIOD | P6 | | | |
| ARMCD | | ABCEDF | | |
| ARMCD | | BEAFCD | | |
| ARMCD | | CADBFE | | |
| ARMCD | | DCFAEB | | |

Program: A Biol.sas Created: 02APR2020 7:35 POSTLOCK 

### The Mixed Procedure

### Parameter Code=ETCOEMAX

Coefficients for Bel 900 vs Oxy 60

Planned Planned

 Arm
 Treatment

 Effect
 APERIOD Code
 (N)
 Row1

 ARMCD
 EFBDAC

 ARMCD
 FDECBA

Coefficients for Bel 300 vs Placebo
Planned Planned

| | | 1 1 aiiii Ca | TTammed | |
|-----------|---------|--------------|-----------|------|
| | | Arm | Treatment | |
| Effect | APERIOD | Code | (N) | Row1 |
| Intercept | | | | |
| TRTPN | | | 1 | 1 |
| TRTPN | | | 2 | |
| TRTPN | | | 3 | |
| TRTPN | | | 4 | |
| TRTPN | | | 5 | |
| TRTPN | | | 6 | -1 |
| APERIOD | P1 | | | |
| APERIOD | P2 | | | |
| APERIOD | Р3 | | | |
| APERIOD | P4 | | | |
| APERIOD | P5 | | | |
| APERIOD | P6 | | | |
| ARMCD | | ABCEDF | | |
| ARMCD | | BEAFCD | | |
| ARMCD | | CADBFE | | |
| ARMCD | | DCFAEB | | |

Program: A\_Biol.sas Created: 02APR2020 7:35 POSTLOCK

### The Mixed Procedure

### Parameter Code=ETCOEMAX

### Coefficients for Bel 300 vs Placebo

Planned Planned

| Arm | Treatment | Effect | APERIOD Code | (N) | Row1 | ARMCD | EFBDAC | ARMCD | FDECBA |

### Coefficients for Bel 600 vs Placebo

Planned Planned
Arm Treatment

| | | ALIII | TIEatment | |
|-----------|---------|--------|-----------|------|
| Effect | APERIOD | Code | (N) | Row1 |
| Intercept | • | | | |
| TRTPN | | | 1 | |
| TRTPN | | | 2 | 1 |
| TRTPN | | | 3 | |
| TRTPN | | | 4 | |
| TRTPN | | | 5 | |
| TRTPN | | | 6 | -1 |
| APERIOD | P1 | | | |
| APERIOD | P2 | | | |
| APERIOD | P3 | | | |
| APERIOD | P4 | | | |
| APERIOD | P5 | | | |
| APERIOD | P6 | | | |
| ARMCD | | ABCEDF | | |
| ARMCD | | BEAFCD | | |
| ARMCD | | CADBFE | | |
| ARMCD | | DCFAEB | | |

### The Mixed Procedure

### Parameter Code=ETCOEMAX

### Coefficients for Bel 600 vs Placebo

Planned Planned

 Arm
 Treatment

 Effect
 APERIOD Code
 (N)
 Row1

 ARMCD
 EFBDAC

 ARMCD
 FDECBA

### Coefficients for Bel 900 vs Placebo

Planned Planned Arm Treatment

| | | ATIII | TTEatment | |
|-----------|---------|--------|-----------|------|
| Effect | APERIOD | Code | (N) | Row1 |
| Intercept | | | | |
| TRTPN | | | 1 | |
| TRTPN | | | 2 | |
| TRTPN | | | 3 | 1 |
| TRTPN | | | 4 | |
| TRTPN | | | 5 | |
| TRTPN | | | 6 | -1 |
| APERIOD | P1 | | | |
| APERIOD | P2 | | | |
| APERIOD | P3 | | | |
| APERIOD | P4 | | | |
| APERIOD | P5 | | | |
| APERIOD | P6 | | | |
| ARMCD | | ABCEDF | | |
| ARMCD | | BEAFCD | | |
| ARMCD | | CADBFE | | |
| ARMCD | | DCFAEB | | |

## Appendix 16.1.9.2.1 Statistical Methods and Analysis Output Supporting Table 14.2.2 Supporting Table 14.2.2

### The Mixed Procedure

### Parameter Code=ETCOEMAX

Coefficients for Bel 900 vs Placebo

Planned Planned

Arm Treatment

Effect APERIOD Code (N) Row1

ARMCD EFBDAC

ARMCD FDECBA

#### Estimates

### Standard

| Label | Estimate | Error DF t | Value F | r > t | Alpha Lower | Upper |
|---|---|---|---|---|---|---|
| Oxy 30 vs Placebo | 1.2467 | 0.924865 | 1.35 | 0.1823 | 0.05-0.6002 | 3.0936 |
| Oxy 60 vs Placebo | 2.1371 | 0.924865 | 2.31 | 0.0240 | 0.05 0.2901 | 3.9840 |
| Bel 300 vs Oxy 30 | -2.3279 | 0.924865 | -2.52 | 0.0143 | 0.05-4.1748 | -0.4810 |
| Bel 300 vs Oxy 60 | -3.2183 | 0.924865 | -3.48 | 0.0009 | 0.05-5.0652 | -1.3714 |
| Bel 600 vs Oxy 30 | -0.09483 | 0.922765 | -0.10 | 0.9185 | 0.05-1.9376 | 1.7479 |
| Bel 600 vs Oxy 60 | -0.9852 | 0.924865 | -1.07 | 0.2907 | 0.05-2.8321 | 0.8617 |
| Bel 900 vs Oxy 30 | -0.3557 | 0.924865 | -0.38 | 0.7018 | 0.05-2.2026 | 1.4912 |
| Bel 900 vs Oxy 60 | -1.2461 | 0.922765 | -1.35 | 0.1816 | 0.05-3.0888 | 0.5967 |
| Bel 300 vs Placebo | -1.0812 | 0.922765 | -1.17 | 0.2455 | 0.05-2.9240 | 0.7615 |
| Bel 600 vs Placebo | 1.1519 | 0.924865 | 1.25 | 0.2174 | 0.05-0.6950 | 2.9988 |
| Bel 900 vs Placebo | 0.8910 | 0.924865 | 0.96 | 0.3389 | 0.05-0.9559 | 2.7379 |

Program: A Biol.sas Created: 02APR2020 7:35 POSTLOCK 

## Appendix 16.1.9.2.1 Statistical Methods and Analysis Output Supporting Table 14.2.2 Supporting Table 14.2.2

The Mixed Procedure

### Parameter Code=ETCOEMAX

### Least Squares Means

| | Planned | | _ | | | | | |
|---|---|---|---|---|---|---|---|---|
| | Treatment | | Standard | | | | | |
| Effect | (N) | Estimate | Error DF t | Value | Pr > t | Alpha | Lower | Upper |
| TRTPN | 1 | 40.6766 | 0.919565 | 44.24 | <.0001 | 0.05 | 38.8402 | 42.5129 |
| TRTPN | 2 | 42.9097 | 0.919565 | 46.67 | <.0001 | 0.05 | 41.0733 | 44.7460 |
| TRTPN | 3 | 42.6488 | 0.919565 | 46.38 | <.0001 | 0.05 | 40.8124 | 44.4851 |
| TRTPN | 4 | 43.0045 | 0.919565 | 46.77 | <.0001 | 0.05 | 41.1682 | 44.8408 |
| TRTPN | 5 | 43.8948 | 0.919565 | 47.74 | <.0001 | 0.05 | 42.0585 | 45.7312 |
| TRTPN | 6 | 41.7578 | 0.919565 | 45.41 | <.0001 | 0.05 | 39.9215 | 43.5941 |

### Differences of Least Squares Means

| | | | | _ | | | | |
|---|---|---|---|---|---|---|---|---|
| | Planned | Planned | | | | | | |
| | Treatment | Treatment | | Standard | | | | |
| Effect | (N) | (N) | Estimate | Error DF t | Value | Pr > t | Alpha Lower | Upper |
| TRTPN | 1 | 2 | -2.2331 | 0.924865 | -2.41 | 0.0186 | 0.05-4.0800 | -0.3862 |
| TRTPN | 1 | 3 | -1.9722 | 0.924865 | -2.13 | 0.0367 | 0.05-3.8191 | -0.1253 |
| TRTPN | 1 | 4 | -2.3279 | 0.924865 | -2.52 | 0.0143 | 0.05-4.1748 | -0.4810 |
| TRTPN | 1 | 5 | -3.2183 | 0.924865 | -3.48 | 0.0009 | 0.05-5.0652 | -1.3714 |
| TRTPN | 1 | 6 | -1.0812 | 0.922765 | -1.17 | 0.2455 | 0.05-2.9240 | 0.7615 |
| TRTPN | 2 | 3 | 0.2609 | 0.924865 | 0.28 | 0.7788 | 0.05-1.5860 | 2.1078 |
| TRTPN | 2 | 4 | -0.09483 | 0.922765 | -0.10 | 0.9185 | 0.05-1.9376 | 1.7479 |
| TRTPN | 2 | 5 | -0.9852 | 0.924865 | -1.07 | 0.2907 | 0.05-2.8321 | 0.8617 |
| TRTPN | 2 | 6 | 1.1519 | 0.924865 | 1.25 | 0.2174 | 0.05-0.6950 | 2.9988 |
| TRTPN | 3 | 4 | -0.3557 | 0.924865 | -0.38 | 0.7018 | 0.05-2.2026 | 1.4912 |
| TRTPN | 3 | 5 | -1.2461 | 0.922765 | -1.35 | 0.1816 | 0.05-3.0888 | 0.5967 |
| TRTPN | 3 | 6 | 0.8910 | 0.924865 | 0.96 | 0.3389 | 0.05-0.9559 | 2.7379 |
| TRTPN | 4 | 5 | -0.8903 | 0.924865 | -0.96 | 0.3392 | 0.05-2.7372 | 0.9566 |

Program: A Biol.sas Created: 02APR2020 7:35 POSTLOCK 

## Appendix 16.1.9.2.1 Statistical Methods and Analysis Output Supporting Table 14.2.2 Supporting Table 14.2.2

The Mixed Procedure

### Parameter Code=ETCOEMAX

### Differences of Least Squares Means

| | Planned | Planned | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| | Treatment | Treatment | S | tandard | | | | | |
| Effect | (N) | (N) | Estimate | Error DF t | Value Pr | > t | Alpha | Lower | Upper |
| TRTPN | 4 | 6 | 1.2467 | 0.924865 | 1.35 | 0.1823 | 0.05 | -0.6002 | 3.0936 |
| TRTPN | 5 | 6 | 2.1371 | 0.924865 | 2.31 | 0.0240 | 0.05 | 0.2901 | 3.9840 |

Program: A\_Biol.sas Created: 02APR2020 7:35 POSTLOCK 

## Appendix 16.1.9.2.1 Statistical Methods and Analysis Output Supporting Table 14.2.2 Supporting Table 14.2.2

### The Mixed Procedure

### Parameter Code=MVMIEMAX

### Model Information

| Data Set | WORK.ADXV |
|---------------------------|---------------------|
| Dependent Variable | AVAL |
| Covariance Structure | Variance Components |
| Estimation Method | REML |
| Residual Variance Method | Profile |
| Fixed Effects SE Method | Model-Based |
| Degrees of Freedom Method | Containment |

### Class Level Information

| Class | LevelsValues |
|---|---|
| SUBJID | 151001 1002 1003 1004 1005 1006 1007 1008 1010 1012 1013 1014 1015 1016 1017 |
| TRTPN | 61 2 3 4 5 6 |
| APERIOD | 6P1 P2 P3 P4 P5 P6 |
| ARMCD | 6ABCEDF BEAFCD CADBFE DCFAEB EFBDAC FDECBA |

| Dimensions | | |
|-------------|------------|----|
| Covariance | Parameters | 2 |
| Columns in | X | 19 |
| Columns in | Z | 15 |
| Subjects | | |
| Max Obs per | Subject | 90 |

Program: A\_Biol.sas Created: 02APR2020 7:35 POSTLOCK 

### Appendix 16.1.9.2.1 Statistical Methods and Analysis Output Supporting Table 14.2.2 Supporting Table 14.2.2

The Mixed Procedure

### Parameter Code=MVMIEMAX

| | Numbe | r of Obse | rvations | |
|--------|--------|-----------|----------|----|
| Number | of Obs | ervations | Read | 90 |
| Number | of Obs | ervations | Used | 90 |
| Number | of Obs | ervations | Not Used | 0 |

# Iteration History Iteration Evaluations -2 Res Log Like Criterion 0 1 1541.87045175 1 1532.27894557 0.00000000

Convergence criteria met.

# Estimates Cov Parm Estimate SUBJID(ARMCD) 13297907 Residual 28686215

Covariance Parameter

| Fit Statistics | |
|--------------------------|--------|
| -2 Res Log Likelihood | 1532.3 |
| AIC (Smaller is Better) | 1536.3 |
| AICC (Smaller is Better) | 1536.4 |
| BIC (Smaller is Better) | 1537 7 |

Program: A Biol.sas Created: 02APR2020 7:35 POSTLOCK 

The Mixed Procedure

Parameter Code=MVMIEMAX

Type 3 Tests of Fixed Effects

| | NumI | Den | |
|---------|------|------|--------------|
| Effect | DF | DF F | Value Pr > F |
| TRTPN | 5 | 65 | 2.930.0190 |
| APERIOD | 5 | 65 | 2.160.0699 |
| ARMCD | 5 | 9 | 0.680.6506 |

Coefficients for Oxy 30 vs Placebo
Planned Planned

| | | Arm | Treatment | |
|-----------|---------|--------|-----------|------|
| Effect | APERIOD | ) Code | (N) | Row1 |
| Intercept | ; | | | |
| TRTPN | | | 1 | |
| TRTPN | | | 2 | |
| TRTPN | | | 3 | |
| TRTPN | | | 4 | 1 |
| TRTPN | | | 5 | |
| TRTPN | | | 6 | -1 |
| APERIOD | P1 | | | |
| APERIOD | P2 | | | |
| APERIOD | P3 | | | |
| APERIOD | P4 | | | |
| APERIOD | P5 | | | |
| APERIOD | P6 | | | |
| ARMCD | | ABCEDF | | |
| ARMCD | | BEAFCD | | |
| ARMCD | | CADBFE | | |
| ARMCD | | DCFAEB | | |

Program: A\_Biol.sas Created: 02APR2020 7:35 POSTLOCK

### The Mixed Procedure

### Parameter Code=MVMIEMAX

### Coefficients for Oxy 30 vs Placebo

Planned Planned

 Arm
 Treatment

 Effect
 APERIOD Code
 (N)
 Row1

 ARMCD
 EFBDAC

 ARMCD
 FDECBA

### Coefficients for Oxy 60 vs Placebo

Planned Planned Arm Treatment

| | | ATIII | Treatment | |
|-----------|---------|--------|-----------|------|
| Effect | APERIOD | Code | (N) | Row1 |
| Intercept | | | | |
| TRTPN | | | 1 | |
| TRTPN | | | 2 | |
| TRTPN | | | 3 | |
| TRTPN | | | 4 | |
| TRTPN | | | 5 | 1 |
| TRTPN | | | 6 | -1 |
| APERIOD | P1 | | | |
| APERIOD | P2 | | | |
| APERIOD | P3 | | | |
| APERIOD | P4 | | | |
| APERIOD | P5 | | | |
| APERIOD | P6 | | | |
| ARMCD | | ABCEDF | | |
| ARMCD | | BEAFCD | | |
| ARMCD | | CADBFE | | |
| ARMCD | | DCFAEB | | |

Program: A Biol.sas Created: 02APR2020 7:35 POSTLOCK 

### The Mixed Procedure

### Parameter Code=MVMIEMAX

### Coefficients for Oxy 60 vs Placebo

Planned Planned

 Arm
 Treatment

 Effect
 APERIOD Code
 (N)
 Row1

 ARMCD
 EFBDAC

 ARMCD
 FDECBA

### Coefficients for Bel 300 vs Oxy 30

Planned Planned

| | | Arm | Treatment | |
|---|---|---|---|---|
| Effect | APERIOD | Code | (N) | Row1 |
| Intercept | | | | |
| TRTPN | | | 1 | 1 |
| TRTPN | | | 2 | |
| TRTPN | | | 3 | |
| TRTPN | | | 4 | -1 |
| TRTPN | | | 5 | |
| TRTPN | | | 6 | |
| APERIOD | P1 | | | |
| APERIOD | P2 | | | |
| APERIOD | P3 | | | |
| APERIOD | P4 | | | |
| APERIOD | P5 | | | |
| APERIOD | P6 | | | |
| ARMCD | | ABCEDF | | |
| ARMCD | | BEAFCD | | |
| ARMCD | | CADBFE | | |
| ARMCD | | DCFAEB | | |
| | Intercept TRTPN TRTPN TRTPN TRTPN TRTPN TRTPN TRTPN APERIOD ARMCD ARMCD ARMCD ARMCD | Intercept TRTPN APERIOD P1 APERIOD P2 APERIOD P3 APERIOD P4 APERIOD P5 APERIOD P6 ARMCD ARMCD ARMCD ARMCD | Effect APERIOD Code Intercept TRTPN APERIOD P1 APERIOD P2 APERIOD P3 APERIOD P4 APERIOD P5 APERIOD P6 ARMCD ABCEDF ARMCD ABCEDF ARMCD CADBFE | ### Effect APERIOD Code (N) Intercept TRTPN |

### The Mixed Procedure

### Parameter Code=MVMIEMAX

Coefficients for Bel 300 vs Oxy 30

Planned Planned

 Arm
 Treatment

 Effect
 APERIOD Code
 (N)
 Row1

 ARMCD
 EFBDAC

**FDECBA** 

ARMCD

Coefficients for Bel 300 vs 0xy 60
Planned Planned

Arm Treatment Effect APERIOD Code (N) Row1 Intercept 1 TRTPN 1 TRTPN TRTPN 3 TRTPN -1 TRTPN TRTPN APERIOD P1 APERIOD P2 APERIOD P3 APERIOD P4 APERIOD P5 APERIOD P6 ARMCD ABCEDF ARMCD BEAFCD ARMCD CADBFE ARMCD DCFAEB

Program: A Biol.sas Created: 02APR2020 7:35 POSTLOCK 

### The Mixed Procedure

### Parameter Code=MVMIEMAX

Coefficients for Bel 300 vs Oxy 60

Planned Planned

 Arm
 Treatment

 Effect
 APERIOD Code
 (N)
 Row1

 ARMCD
 EFBDAC

 ARMCD
 FDECBA

Coefficients for Bel 600 vs 0xy 30 Planned Planned

Arm Treatment

| | | 211111 | I I Ca chich | • |
|-----------|--------|--------|--------------|------|
| Effect | APERIO | ) Code | (N) | Row1 |
| Intercept | ; | | | |
| TRTPN | | | 1 | |
| TRTPN | | | 2 | 1 |
| TRTPN | | | 3 | |
| TRTPN | | | 4 | -1 |
| TRTPN | | | 5 | |
| TRTPN | | | 6 | |
| APERIOD | P1 | | | |
| APERIOD | P2 | | | |
| APERIOD | Р3 | | | |
| APERIOD | P4 | | | |
| APERIOD | P5 | | | |
| APERIOD | P6 | | | |
| ARMCD | | ABCEDF | | |
| ARMCD | | BEAFCD | | |
| ARMCD | | CADBFE | | |
| ARMCD | | DCFAEB | | |

Program: A\_Biol.sas Created: 02APR2020 7:35 POSTLOCK


The Mixed Procedure

### Parameter Code=MVMIEMAX

Coefficients for Bel 600 vs Oxy 30

Planned Planned

 Arm
 Treatment

 Effect
 APERIOD Code
 (N)
 Row1

 ARMCD
 EFBDAC

 ARMCD
 FDECBA

Coefficients for Bel 600 vs Oxy 60 Planned Planned

| | | Arm | Treatment | |
|-----------|---------|--------|-----------|------|
| Effect | APERIOD | Code | (N) | Row1 |
| Intercept | | | | |
| TRTPN | | | 1 | |
| TRTPN | | | 2 | 1 |
| TRTPN | | | 3 | |
| TRTPN | | | 4 | |
| TRTPN | | | 5 | -1 |
| TRTPN | | | 6 | |
| APERIOD | P1 | | | |
| APERIOD | P2 | | | |
| APERIOD | Р3 | | | |
| APERIOD | P4 | | | |
| APERIOD | P5 | | | |
| APERIOD | P6 | | | |
| ARMCD | | ABCEDF | | |
| ARMCD | | BEAFCD | | |
| ARMCD | | CADBFE | | |
| ARMCD | | DCFAEB | | |
| ARMCD | | DCFAEB | | |

Program: A Biol.sas Created: 02APR2020 7:35 POSTLOCK 

### The Mixed Procedure

### Parameter Code=MVMIEMAX

Coefficients for Bel 600 vs Oxy 60

Planned Planned

 Arm
 Treatment

 Effect
 APERIOD Code
 (N)
 Row1

 ARMCD
 EFBDAC

 ARMCD
 FDECBA

Coefficients for Bel 900 vs Oxy 30

Planned Planned
Arm Treatment

| | | 2 2 2 111 | I I Ca chichi c | |
|-----------|--------|-----------|-----------------|------|
| Effect | APERIO | ) Code | (N) | Row1 |
| Intercept | | | | |
| TRTPN | | | 1 | |
| TRTPN | | | 2 | |
| TRTPN | | | 3 | 1 |
| TRTPN | | | 4 | -1 |
| TRTPN | | | 5 | |
| TRTPN | | | 6 | |
| APERIOD | P1 | | | |
| APERIOD | P2 | | | |
| APERIOD | Р3 | | | |
| APERIOD | P4 | | | |
| APERIOD | P5 | | | |
| APERIOD | P6 | | | |
| ARMCD | | ABCEDF | | |
| ARMCD | | BEAFCD | | |
| ARMCD | | CADBFE | | |
| ARMCD | | DCFAEB | | |

Program: A\_Bio1.sas Created: 02APR2020 7:35 POSTLOCK

### The Mixed Procedure

### Parameter Code=MVMIEMAX

Coefficients for Bel 900 vs Oxy 30

Planned Planned

 Arm
 Treatment

 Effect
 APERIOD Code
 (N)
 Row1

 ARMCD
 EFBDAC

 ARMCD
 FDECBA

Coefficients for Bel 900 vs Oxy 60 Planned Planned

| | | Arm | Treatment | |
|-----------|---------|--------|-----------|------|
| Effect | APERIOD | Code | (N) | Row1 |
| Intercept | | | | |
| TRTPN | | | 1 | |
| TRTPN | | | 2 | |
| TRTPN | | | 3 | 1 |
| TRTPN | | | 4 | |
| TRTPN | | | 5 | -1 |
| TRTPN | | | 6 | |
| APERIOD | P1 | | | |
| APERIOD | P2 | | | |
| APERIOD | P3 | | | |
| APERIOD | P4 | | | |
| APERIOD | P5 | | | |
| APERIOD | P6 | | | |
| ARMCD | | ABCEDF | | |
| ARMCD | | BEAFCD | | |
| ARMCD | | CADBFE | | |
| ARMCD | | DCFAEB | | |

### The Mixed Procedure

### Parameter Code=MVMIEMAX

Coefficients for Bel 900 vs Oxy 60

Planned Planned

 Arm
 Treatment

 Effect
 APERIOD Code
 (N)
 Row1

 ARMCD
 EFBDAC

 ARMCD
 FDECBA

Coefficients for Bel 300 vs Placebo
Planned Planned

| | | Arm | Treatment | |
|-----------|--------|--------|-----------|------|
| Effect | APERIO | O Code | (N) | Row1 |
| Intercept | | | | |
| TRTPN | | | 1 | 1 |
| TRTPN | | | 2 | |
| TRTPN | | | 3 | |
| TRTPN | | | 4 | |
| TRTPN | | | 5 | |
| TRTPN | | | 6 | -1 |
| APERIOD | P1 | | | |
| APERIOD | P2 | | | |
| APERIOD | Р3 | | | |
| APERIOD | P4 | | | |
| APERIOD | P5 | | | |
| APERIOD | P6 | | | |
| ARMCD | | ABCEDF | | |
| ARMCD | | BEAFCD | | |
| ARMCD | | CADBFE | | |
| ARMCD | | DCFAEB | | |

### The Mixed Procedure

### Parameter Code=MVMIEMAX

Coefficients for Bel 300 vs Placebo

Planned Planned

 Arm
 Treatment

 Effect
 APERIOD Code
 (N)
 Row1

 ARMCD
 EFBDAC

 ARMCD
 FDECBA

Coefficients for Bel 600 vs Placebo
Planned Planned

Arm Treatment Effect APERIOD Code (N) Row1 Intercept TRTPN 1 TRTPN 1 TRTPN 3 TRTPN TRTPN TRTPN -1 APERIOD P1 APERIOD P2 APERIOD P3 APERIOD P4 APERIOD P5 APERIOD P6 ARMCD ABCEDF ARMCD BEAFCD ARMCD CADBFE

Program: A Biol.sas Created: 02APR2020 7:35 POSTLOCK 

DCFAEB

ARMCD

### The Mixed Procedure

### Parameter Code=MVMIEMAX

### Coefficients for Bel 600 vs Placebo

Planned Planned

 Arm
 Treatment

 Effect
 APERIOD Code
 (N)
 Row1

 ARMCD
 EFBDAC

 ARMCD
 FDECBA

### Coefficients for Bel 900 vs Placebo

Planned Planned

| | | Arm | Treatment | |
|-----------|---------|--------|-----------|------|
| Effect | APERIOD | Code | (N) | Row1 |
| Intercept | | | | |
| TRTPN | | | 1 | |
| TRTPN | | | 2 | |
| TRTPN | | | 3 | 1 |
| TRTPN | | | 4 | |
| TRTPN | | | 5 | |
| TRTPN | | | 6 | -1 |
| APERIOD | P1 | | | |
| APERIOD | P2 | | | |
| APERIOD | P3 | | | |
| APERIOD | P4 | | | |
| APERIOD | P5 | | | |
| APERIOD | P6 | | | |
| ARMCD | | ABCEDF | | |
| ARMCD | | BEAFCD | | |
| ARMCD | | CADBFE | | |
| ARMCD | | DCFAEB | | |

### Appendix 16.1.9.2.1 Statistical Methods and Analysis Output Supporting Table 14.2.2 Supporting Table 14.2.2

### The Mixed Procedure

### Parameter Code=MVMIEMAX

Coefficients for Bel 900 vs Placebo

Planned Planned

Arm Treatment

Effect APERIOD Code (N) Row1

ARMCD EFBDAC

ARMCD FDECBA

### Estimates

### Standard

| Label | Estimate | Error DF t | Value H | ?r > t <i>i</i> | Alpha | Lower | Upper |
|---|---|---|---|---|---|---|---|
| Oxy 30 vs Placebo | -794.77 | 1964.4965 | -0.40 | 0.6871 | 0.05- | -4718.12 | 3128.58 |
| Oxy 60 vs Placebo | -5228.92 | 1964.4965 | -2.66 | 0.0098 | 0.05- | -9152.27 - | -1305.57 |
| Bel 300 vs Oxy 30 | 2034.61 | 1964.4965 | 1.04 | 0.3042 | 0.05- | -1888.74 | 5957.96 |
| Bel 300 vs Oxy 60 | 6468.76 | 1964.4965 | 3.29 | 0.0016 | 0.05 | 2545.41 | 10392 |
| Bel 600 vs Oxy 30 | 1022.24 | 1960.0865 | 0.52 | 0.6038 | 0.05- | -2892.31 | 4936.78 |
| Bel 600 vs Oxy 60 | 5456.39 | 1964.4965 | 2.78 | 0.0072 | 0.05 | 1533.04 | 9379.74 |
| Bel 900 vs Oxy 30 | 1726.13 | 1964.4965 | 0.88 | 0.3828 | 0.05- | -2197.22 | 5649.48 |
| Bel 900 vs Oxy 60 | 6160.28 | 1960.0865 | 3.14 | 0.0025 | 0.05 | 2245.73 | 10075 |
| Bel 300 vs Placebo | 1239.84 | 1960.0865 | 0.63 | 0.5292 | 0.05- | -2674.70 | 5154.39 |
| Bel 600 vs Placebo | 227.47 | 1964.4965 | 0.12 | 0.9082 | 0.05- | -3695.88 | 4150.82 |
| Bel 900 vs Placebo | 931.36 | 1964.4965 | 0.47 | 0.6370 | 0.05- | -2991.99 | 4854.71 |

Program: A Biol.sas Created: 02APR2020 7:35 POSTLOCK 

## Appendix 16.1.9.2.1 Statistical Methods and Analysis Output Supporting Table 14.2.2 Supporting Table 14.2.2

The Mixed Procedure

### Parameter Code=MVMIEMAX

### Least Squares Means

| | | | _ | | | |
|---|---|---|---|---|---|---|
| | Planned | | | | | |
| | Treatment | | Standard | | | |
| Effect | (N) | ${\tt Estimate}$ | Error DF t | Value Pr | > t . | Alpha Lower Upper |
| TRTPN | 1 | 23741 | 1691.7665 | 14.03 | <.0001 | 0.052036227120 |
| TRTPN | 2 | 22729 | 1691.7665 | 13.43 | <.0001 | 0.051935026107 |
| TRTPN | 3 | 23433 | 1691.7665 | 13.85 | <.0001 | 0.052005426811 |
| TRTPN | 4 | 21706 | 1691.7665 | 12.83 | <.0001 | 0.051832825085 |
| TRTPN | 5 | 17272 | 1691.7665 | 10.21 | <.0001 | 0.051389420651 |
| TRTPN | 6 | 22501 | 1691.7665 | 13.30 | <.0001 | 0.051912325880 |

### Differences of Least Squares Means

| | Planned | Planned | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| | Treatment | Treatment | | Standard | | | | | |
| Effect | (N) | (N) | Estimate | Error DF t | Value F | ?r > t | Alpha | Lower | Upper |
| TRTPN | 1 | 2 | 1012.37 | 1964.4965 | 0.52 | 0.6081 | 0.05 | -2910.98 | 4935.72 |
| TRTPN | 1 | 3 | 308.48 | 1964.4965 | 0.16 | 0.8757 | 0.05 | -3614.87 | 4231.83 |
| TRTPN | 1 | 4 | 2034.61 | 1964.4965 | 1.04 | 0.3042 | 0.05 | -1888.74 | 5957.96 |
| TRTPN | 1 | 5 | 6468.76 | 1964.4965 | 3.29 | 0.0016 | 0.05 | 2545.41 | 10392 |
| TRTPN | 1 | 6 | 1239.84 | 1960.0865 | 0.63 | 0.5292 | 0.05 | -2674.70 | 5154.39 |
| TRTPN | 2 | 3 | -703.89 | 1964.4965 | -0.36 | 0.7213 | 0.05 | -4627.24 | 3219.46 |
| TRTPN | 2 | 4 | 1022.24 | 1960.0865 | 0.52 | 0.6038 | 0.05 | -2892.31 | 4936.78 |
| TRTPN | 2 | 5 | 5456.39 | 1964.4965 | 2.78 | 0.0072 | 0.05 | 1533.04 | 9379.74 |
| TRTPN | 2 | 6 | 227.47 | 1964.4965 | 0.12 | 0.9082 | 0.05 | -3695.88 | 4150.82 |
| TRTPN | 3 | 4 | 1726.13 | 1964.4965 | 0.88 | 0.3828 | 0.05 | -2197.22 | 5649.48 |
| TRTPN | 3 | 5 | 6160.28 | 1960.0865 | 3.14 | 0.0025 | 0.05 | 2245.73 | 10075 |
| TRTPN | 3 | 6 | 931.36 | 1964.4965 | 0.47 | 0.6370 | 0.05 | -2991.99 | 4854.71 |
| TRTPN | 4 | 5 | 4434.15 | 1964.4965 | 2.26 | 0.0274 | 0.05 | 510.80 | 8357.50 |

Program: A\_Biol.sas Created: 02APR2020 7:35 POSTLOCK 

## Appendix 16.1.9.2.1 Statistical Methods and Analysis Output Supporting Table 14.2.2 Supporting Table 14.2.2

### The Mixed Procedure

### Parameter Code=MVMIEMAX

### Differences of Least Squares Means

Planned Planned Treatment

| | Treatment | Treatment | 5 | Standard | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| Effect | (N) | (N) | Estimate | Error DF t | Value Pr | c > t A | Alpha | Lower | Upper |
| TRTPN | 4 | 6 | -794.77 | 1964.4965 | -0.40 | 0.6871 | 0.05-47 | 718.12 | 3128.58 |
| TRTPN | 5 | 6 | -5228.92 | 1964.4965 | -2.66 | 0.0098 | 0.05-93 | 152.27 - | -1305.57 |

Program: A Biol.sas Created: 02APR2020 7:35 POSTLOCK 

## Appendix 16.1.9.2.1 Statistical Methods and Analysis Output Supporting Table 14.2.2 Supporting Table 14.2.2

### The Mixed Procedure

### Parameter Code=PEFMEMAX

### Model Information

| Data Set | WORK.ADXV |
|---------------------------|---------------------|
| Dependent Variable | AVAL |
| Covariance Structure | Variance Components |
| Estimation Method | REML |
| Residual Variance Method | Profile |
| Fixed Effects SE Method | Model-Based |
| Degrees of Freedom Method | Containment |

### Class Level Information

| Class | LevelsValues |
|---|---|
| SUBJID | 151001 1002 1003 1004 1005 1006 1007 1008 1010 1012 1013 1014 1015 1016 1017 |
| TRTPN | 61 2 3 4 5 6 |
| APERIOD | 6P1 P2 P3 P4 P5 P6 |
| ARMCD | 6ABCEDF BEAFCD CADBFE DCFAEB EFBDAC FDECBA |

| Dimensions | | | |
|------------|-------------|------------|----|
| | Covariance | Parameters | 2 |
| | Columns in | X | 19 |
| | Columns in | Z | 15 |
| | Subjects | | 1 |
| | Max Obs per | Subject | 90 |

Program: A\_Biol.sas Created: 02APR2020 7:35 POSTLOCK 

### Appendix 16.1.9.2.1 Statistical Methods and Analysis Output Supporting Table 14.2.2 Supporting Table 14.2.2

The Mixed Procedure

### Parameter Code=PEFMEMAX

| | Nι | umber of Obse | rvations | |
|--------|----|---------------|----------|----|
| Number | of | Observations | Read | 90 |
| Number | of | Observations | Used | 90 |
| Number | of | Observations | Not Used | 0 |

#### Iteration History Iteration Evaluations -2 Res Log Like Criterion 0 1 668.81167810 1 1 659.346344790.00000000

Convergence criteria met.

### Covariance Parameter Estimates

| Cov Parm | Estimate |
|----------------|----------|
| SUBJID (ARMCD) | 99.2034 |
| Residual | 216.26 |

| Fit Statistics | |
|--------------------------|-------|
| -2 Res Log Likelihood | 659.3 |
| AIC (Smaller is Better) | 663.3 |
| AICC (Smaller is Better) | 663.5 |
| BIC (Smaller is Better) | 664.8 |

 Program: A Biol.sas Created: 02APR2020 7:35 POSTLOCK

The Mixed Procedure

Parameter Code=PEFMEMAX

Type 3 Tests of Fixed Effects

| 1 | Num I | | |
|---------|-------|------|----------------------|
| Effect | DF | DF F | ${\tt Value Pr > F}$ |
| TRTPN | 5 | 65 | 2.640.0313 |
| APERIOD | 5 | 65 | 2.530.0374 |
| ARMCD | 5 | 9 | 0.580.7181 |

### Coefficients for Oxy 30 vs Placebo Planned Planned

| | | Arm | Treatment | ; |
|----------|---------|--------|-----------|----------|
| Effect | APERIOD | ) Code | (N) | Row1 |
| Intercep | t | | | <u>.</u> |
| TRTPN | | | 1 | |
| TRTPN | | | 2 | |
| TRTPN | | | 3 | |
| TRTPN | | | 4 | 1 |
| TRTPN | | | 5 | |
| TRTPN | | | 6 | -1 |
| APERIOD | P1 | | | |
| APERIOD | P2 | | | |
| APERIOD | P3 | | | |
| APERIOD | P4 | | | |
| APERIOD | P5 | | | |
| APERIOD | P6 | | | |
| ARMCD | | ABCEDF | | |
| ARMCD | | BEAFCD | | |

CADBFE

DCFAEB

Program: A\_Bio1.sas Created: 02APR2020 7:35 POSTLOCK

ARMCD

ARMCD

### The Mixed Procedure

### Parameter Code=PEFMEMAX

### Coefficients for Oxy 30 vs Placebo

Planned Planned

 Arm
 Treatment

 Effect
 APERIOD Code
 (N)
 Row1

 ARMCD
 EFBDAC

 ARMCD
 FDECBA

### Coefficients for Oxy 60 vs Placebo

Planned Planned
Arm Treatment

| | | ATIII | Treatment | |
|-----------|---------|--------|-----------|------|
| Effect | APERIOD | Code | (N) | Row1 |
| Intercept | | | | |
| TRTPN | | | 1 | |
| TRTPN | | | 2 | |
| TRTPN | | | 3 | |
| TRTPN | | | 4 | |
| TRTPN | | | 5 | 1 |
| TRTPN | | | 6 | -1 |
| APERIOD | P1 | | | |
| APERIOD | P2 | | | |
| APERIOD | Р3 | | | |
| APERIOD | P4 | | | |
| APERIOD | P5 | | | |
| APERIOD | P6 | | | |
| ARMCD | | ABCEDF | | |
| ARMCD | | BEAFCD | | |
| ARMCD | | CADBFE | | |
| ARMCD | | DCFAEB | | |

The Mixed Procedure

### Parameter Code=PEFMEMAX

Coefficients for Oxy 60 vs Placebo

Planned Planned

 Arm
 Treatment

 Effect
 APERIOD Code
 (N)
 Row1

 ARMCD
 EFBDAC

 ARMCD
 FDECBA

Coefficients for Bel 300 vs Oxy 30

Planned Planned
Arm Treatment

| | | Arm | Treatment | |
|-----------|---------|--------|-----------|------|
| Effect | APERIOD | Code | (N) | Row1 |
| Intercept | | | | |
| TRTPN | | | 1 | 1 |
| TRTPN | | | 2 | |
| TRTPN | | | 3 | |
| TRTPN | | | 4 | -1 |
| TRTPN | | | 5 | |
| TRTPN | | | 6 | |
| APERIOD | P1 | | | |
| APERIOD | P2 | | | |
| APERIOD | P3 | | | |
| APERIOD | P4 | | | |
| APERIOD | P5 | | | |
| APERIOD | P6 | | | |
| ARMCD | | ABCEDF | | |
| ARMCD | | BEAFCD | | |
| ARMCD | | CADBFE | | |
| ARMCD | | DCFAEB | | |

### The Mixed Procedure

### Parameter Code=PEFMEMAX

Coefficients for Bel 300 vs Oxy 30

Planned Planned

 Arm
 Treatment

 Effect
 APERIOD Code
 (N)
 Row1

 ARMCD
 EFBDAC

 ARMCD
 FDECBA

Coefficients for Bel 300 vs Oxy 60

Planned Planned

| | | Arm | Treatment | |
|-----------|---------|--------|-----------|------|
| Effect | APERIOD | Code | (N) | Row1 |
| Intercept | | | | |
| TRTPN | | | 1 | 1 |
| TRTPN | | | 2 | |
| TRTPN | | | 3 | |
| TRTPN | | | 4 | |
| TRTPN | | | 5 | -1 |
| TRTPN | | | 6 | |
| APERIOD | P1 | | | |
| APERIOD | P2 | | | |
| APERIOD | P3 | | | |
| APERIOD | P4 | | | |
| APERIOD | P5 | | | |
| APERIOD | P6 | | | |
| ARMCD | | ABCEDF | | |
| ARMCD | | BEAFCD | | |
| ARMCD | | CADBFE | | |
| ARMCD | | DCFAEB | | |

### The Mixed Procedure

### Parameter Code=PEFMEMAX

Coefficients for Bel 300 vs Oxy 60

Planned Planned

 Arm
 Treatment

 Effect
 APERIOD Code
 (N)
 Row1

 ARMCD
 EFBDAC

 ARMCD
 FDECBA

Coefficients for Bel 600 vs Oxy 30
Planned Planned

Arm Treatment

| | | 2 1 L 111 | I I Ca cincii c | • |
|-----------|--------|-----------|-----------------|------|
| Effect | APERIO | ) Code | (N) | Row1 |
| Intercept | | | | |
| TRTPN | | | 1 | |
| TRTPN | | | 2 | 1 |
| TRTPN | | | 3 | |
| TRTPN | | | 4 | -1 |
| TRTPN | | | 5 | |
| TRTPN | | | 6 | |
| APERIOD | P1 | | | |
| APERIOD | P2 | | | |
| APERIOD | Р3 | | | |
| APERIOD | P4 | | | |
| APERIOD | P5 | | | |
| APERIOD | P6 | | | |
| ARMCD | | ABCEDF | | |
| ARMCD | | BEAFCD | | |
| ARMCD | | CADBFE | | |
| ARMCD | | DCFAEB | | |

Program: A\_Biol.sas Created: 02APR2020 7:35 POSTLOCK 

### The Mixed Procedure

### Parameter Code=PEFMEMAX

Coefficients for Bel 600 vs Oxy 30

Planned Planned

 Arm
 Treatment

 Effect
 APERIOD Code
 (N)
 Row1

 ARMCD
 EFBDAC

 ARMCD
 FDECBA

Coefficients for Bel 600 vs 0xy 60
Planned Planned

| | | Arm | Treatment | |
|-----------|---------|--------|-----------|------|
| Effect | APERIOD | Code | (N) | Row1 |
| Intercept | | | | |
| TRTPN | | | 1 | |
| TRTPN | | | 2 | 1 |
| TRTPN | | | 3 | |
| TRTPN | | | 4 | |
| TRTPN | | | 5 | -1 |
| TRTPN | | | 6 | |
| APERIOD | P1 | | | |
| APERIOD | P2 | | | |
| APERIOD | P3 | | | |
| APERIOD | P4 | | | |
| APERIOD | P5 | | | |
| APERIOD | P6 | | | |
| ARMCD | | ABCEDF | | |
| ARMCD | | BEAFCD | | |
| ARMCD | | CADBFE | | |
| ARMCD | | DCFAEB | | |

Program: A Biol.sas Created: 02APR2020 7:35 POSTLOCK 

### The Mixed Procedure

### Parameter Code=PEFMEMAX

Coefficients for Bel 600 vs Oxy 60

Planned Planned

 Arm
 Treatment

 Effect
 APERIOD Code
 (N)
 Row1

 ARMCD
 EFBDAC

 ARMCD
 FDECBA

Coefficients for Bel 900 vs Oxy 30
Planned Planned

Arm Treatment

| | | | | - |
|----------|---------|--------|-----|------|
| Effect | APERIOD | Code | (N) | Row1 |
| Intercep | t | | | |
| TRTPN | | | 1 | |
| TRTPN | | | 2 | |
| TRTPN | | | 3 | 1 |
| TRTPN | | | 4 | -1 |
| TRTPN | | | 5 | |
| TRTPN | | | 6 | |
| APERIOD | P1 | | | |
| APERIOD | P2 | | | |
| APERIOD | Р3 | | | |
| APERIOD | P4 | | | |
| APERIOD | P5 | | | |
| APERIOD | P6 | | | |
| ARMCD | | ABCEDF | | |
| ARMCD | | BEAFCD | | |
| ARMCD | | CADBFE | | |
| ARMCD | | DCFAEB | | |

### The Mixed Procedure

### Parameter Code=PEFMEMAX

Coefficients for Bel 900 vs Oxy 30

Planned Planned

 Arm
 Treatment

 Effect
 APERIOD Code
 (N)
 Row1

 ARMCD
 EFBDAC

 ARMCD
 FDECBA

Coefficients for Bel 900 vs 0xy 60
Planned Planned
Arm Treatment

| | | Arm | Treatment | |
|-----------|--------|--------|-----------|------|
| Effect | APERIO | O Code | (N) | Row1 |
| Intercept | ; | | | |
| TRTPN | | | 1 | |
| TRTPN | | | 2 | |
| TRTPN | | | 3 | 1 |
| TRTPN | | | 4 | |
| TRTPN | | | 5 | -1 |
| TRTPN | | | 6 | |
| APERIOD | P1 | | | |
| APERIOD | P2 | | | |
| APERIOD | Р3 | | | |
| APERIOD | P4 | | | |
| APERIOD | P5 | | | |
| APERIOD | P6 | | | |
| ARMCD | | ABCEDF | | |
| ARMCD | | BEAFCD | | |
| ARMCD | | CADBFE | | |
| ARMCD | | DCFAEB | | |

### The Mixed Procedure

### Parameter Code=PEFMEMAX

Coefficients for Bel 900 vs Oxy 60

Planned Planned

 Arm
 Treatment

 Effect
 APERIOD Code
 (N)
 Row1

 ARMCD
 EFBDAC

FDECBA

ARMCD

Coefficients for Bel 300 vs Placebo
Planned Planned

| | | Arm | Treatment | |
|-----------|---------|--------|-----------|------|
| Effect | APERIOD | Code | (N) | Row1 |
| Intercept | | | | |
| TRTPN | | | 1 | 1 |
| TRTPN | | | 2 | |
| TRTPN | | | 3 | |
| TRTPN | | | 4 | |
| TRTPN | | | 5 | |
| TRTPN | | | 6 | -1 |
| APERIOD | P1 | | | |
| APERIOD | P2 | | | |
| APERIOD | Р3 | | | |
| APERIOD | P4 | | | |
| APERIOD | P5 | | | |
| APERIOD | P6 | | | |
| ARMCD | | ABCEDF | | |
| ARMCD | | BEAFCD | | |
| ARMCD | | CADBFE | | |
| ARMCD | | DCFAEB | | |

Program: A\_Biol.sas Created: 02APR2020 7:35 POSTLOCK

The Mixed Procedure

### Parameter Code=PEFMEMAX

Coefficients for Bel 300 vs Placebo

Planned Planned

 $\begin{array}{c|cccc} & & Arm & Treatment \\ \hline Effect & APERIOD\,Code & (N) & Row1 \\ \hline ARMCD & EFBDAC \end{array}$ 

ARMCD FDECBA

### Coefficients for Bel 600 vs Placebo Planned Planned

Arm Treatment

| | | Arm | Treatment | |
|-----------|---------|--------|-----------|------|
| Effect | APERIOD | Code | (N) | Row1 |
| Intercept | | | | |
| TRTPN | | | 1 | |
| TRTPN | | | 2 | 1 |
| TRTPN | | | 3 | |
| TRTPN | | | 4 | |
| TRTPN | | | 5 | |
| TRTPN | | | 6 | -1 |
| APERIOD | P1 | | | |
| APERIOD | P2 | | | |
| APERIOD | P3 | | | |
| APERIOD | P4 | | | |
| APERIOD | P5 | | | |
| APERIOD | P6 | | | |
| ARMCD | | ABCEDF | | |
| ARMCD | | BEAFCD | | |
| ARMCD | | CADBFE | | |
| ARMCD | | DCFAEB | | |
The Mixed Procedure

### Parameter Code=PEFMEMAX

Coefficients for Bel 600 vs Placebo

Planned Planned

 Arm
 Treatment

 Effect
 APERIOD Code
 (N)
 Row1

 ARMCD
 EFBDAC

 ARMCD
 FDECBA

Coefficients for Bel 900 vs Placebo
Planned Planned

| | | Arm | Treatment | |
|-----------|---------|--------|-----------|------|
| Effect | APERIOD | ) Code | (N) | Row1 |
| Intercept | | | | |
| TRTPN | | | 1 | |
| TRTPN | | | 2 | |
| TRTPN | | | 3 | 1 |
| TRTPN | | | 4 | |
| TRTPN | | | 5 | |
| TRTPN | | | 6 | -1 |
| APERIOD | P1 | | | |
| APERIOD | P2 | | | |
| APERIOD | P3 | | | |
| APERIOD | P4 | | | |
| APERIOD | P5 | | | |
| APERIOD | P6 | | | |
| ARMCD | | ABCEDF | | |
| ARMCD | | BEAFCD | | |
| ARMCD | | CADBFE | | |
| ARMCD | | DCFAEB | | |

# Appendix 16.1.9.2.1 Statistical Methods and Analysis Output Supporting Table 14.2.2 Supporting Table 14.2.2

### The Mixed Procedure

### Parameter Code=PEFMEMAX

Coefficients for Bel 900 vs Placebo

Planned Planned

Arm Treatment

Effect APERIOD Code (N) Row1
ARMCD EFBDAC
ARMCD FDECBA

### Estimates

### Standard

| Label | Estimate | Error DF t | Value P | r > t . | Alpha | Lower | Upper |
|---|---|---|---|---|---|---|---|
| Oxy 30 vs Placebo | 0.01627 | 5.393965 | 0.00 | 0.9976 | 0.05 | -10.7560 | 10.7886 |
| Oxy 60 vs Placebo | -13.6055 | 5.393965 | -2.52 | 0.0141 | 0.05 | -24.3778 | -2.8332 |
| Bel 300 vs Oxy 30 | 2.8228 | 5.393965 | 0.52 | 0.6025 | 0.05 | -7.9495 | 13.5951 |
| Bel 300 vs Oxy 60 | 16.4446 | 5.393965 | 3.05 | 0.0033 | 0.05 | 5.6723 | 27.2169 |
| Bel 600 vs Oxy 30 | 1.6470 | 5.381865 | 0.31 | 0.7606 | 0.05 | -9.1012 | 12.3951 |
| Bel 600 vs Oxy 60 | 15.2687 | 5.393965 | 2.83 | 0.0062 | 0.05 | 4.4964 | 26.0410 |
| Bel 900 vs Oxy 30 | 1.9547 | 5.393965 | 0.36 | 0.7182 | 0.05 | -8.8176 | 12.7270 |
| Bel 900 vs Oxy 60 | 15.5765 | 5.381865 | 2.89 | 0.0052 | 0.05 | 4.8283 | 26.3246 |
| Bel 300 vs Placebo | 2.8391 | 5.381865 | 0.53 | 0.5996 | 0.05 | -7.9090 | 13.5872 |
| Bel 600 vs Placebo | 1.6632 | 5.393965 | 0.31 | 0.7588 | 0.05 | -9.1091 | 12.4355 |
| Bel 900 vs Placebo | 1.9710 | 5.393965 | 0.37 | 0.7160 | 0.05 | -8.8013 | 12.7433 |

Program: A Biol.sas Created: 02APR2020 7:35 POSTLOCK 

# Appendix 16.1.9.2.1 Statistical Methods and Analysis Output Supporting Table 14.2.2 Supporting Table 14.2.2

The Mixed Procedure

### Parameter Code=PEFMEMAX

## Least Squares Means

| | Planned | | | | | | | |
|---|---|---|---|---|---|---|---|---|
| | Treatment | | Standard | | | | | |
| Effect | (N) | Estimate | Error DF t | Value | Pr > t | Alpha | Lower | Upper |
| TRTPN | 1 | 62.0303 | 4.637265 | 13.38 | <.0001 | 0.05 | 52.7692 | 71.2915 |
| TRTPN | 2 | 60.8544 | 4.637265 | 13.12 | <.0001 | 0.05 | 51.5933 | 70.1156 |
| TRTPN | 3 | 61.1622 | 4.637265 | 13.19 | <.0001 | 0.05 | 51.9011 | 70.4233 |
| TRTPN | 4 | 59.2075 | 4.637265 | 12.77 | <.0001 | 0.05 | 49.9464 | 68.4686 |
| TRTPN | 5 | 45.5857 | 4.637265 | 9.83 | <.0001 | 0.05 | 36.3246 | 54.8469 |
| TRTPN | 6 | 59.1912 | 4.637265 | 12.76 | <.0001 | 0.05 | 49.9301 | 68.4524 |

# Differences of Least Squares Means

| | Planned | Planned | | | - | | | | |
|---|---|---|---|---|---|---|---|---|---|
| | | t Treatment | - | Standard | | | | | |
| Effect | (N) | (N) | Estimate | Error DF t | Value E | ?r > t . | Alpha | Lower | Upper |
| TRTPN | 1 | 2 | 1.1759 | 5.393965 | 0.22 | 0.8281 | 0.05 | -9.5964 | 11.9482 |
| TRTPN | 1 | 3 | 0.8681 | 5.393965 | 0.16 | 0.8726 | 0.05 | -9.9042 | 11.6404 |
| TRTPN | 1 | 4 | 2.8228 | 5.393965 | 0.52 | 0.6025 | 0.05 | -7.9495 | 13.5951 |
| TRTPN | 1 | 5 | 16.4446 | 5.393965 | 3.05 | 0.0033 | 0.05 | 5.6723 | 27.2169 |
| TRTPN | 1 | 6 | 2.8391 | 5.381865 | 0.53 | 0.5996 | 0.05 | -7.9090 | 13.5872 |
| TRTPN | 2 | 3 | -0.3078 | 5.393965 | -0.06 | 0.9547 | 0.05 | -11.0800 | 10.4645 |
| TRTPN | 2 | 4 | 1.6470 | 5.381865 | 0.31 | 0.7606 | 0.05 | -9.1012 | 12.3951 |
| TRTPN | 2 | 5 | 15.2687 | 5.393965 | 2.83 | 0.0062 | 0.05 | 4.4964 | 26.0410 |
| TRTPN | 2 | 6 | 1.6632 | 5.393965 | 0.31 | 0.7588 | 0.05 | -9.1091 | 12.4355 |
| TRTPN | 3 | 4 | 1.9547 | 5.393965 | 0.36 | 0.7182 | 0.05 | -8.8176 | 12.7270 |
| TRTPN | 3 | 5 | 15.5765 | 5.381865 | 2.89 | 0.0052 | 0.05 | 4.8283 | 26.3246 |
| TRTPN | 3 | 6 | 1.9710 | 5.393965 | 0.37 | 0.7160 | 0.05 | -8.8013 | 12.7433 |
| TRTPN | 4 | 5 | 13.6217 | 5.393965 | 2.53 | 0.0140 | 0.05 | 2.8495 | 24.3940 |

Program: A Biol.sas Created: 02APR2020 7:35 POSTLOCK 

# Appendix 16.1.9.2.1 Statistical Methods and Analysis Output Supporting Table 14.2.2 Supporting Table 14.2.2

### The Mixed Procedure

### Parameter Code=PEFMEMAX

# Differences of Least Squares Means

| | Planned | Planned | | | - | | | | |
|---|---|---|---|---|---|---|---|---|---|
| | Treatment | Treatment | | Standard | | | | | |
| Effect | (N) | (N) | Estimate | Error DF t | Value Pr | : > t | Alpha | Lower | Upper |
| TRTPN | 4 | 6 | 0.01627 | 5.393965 | 0.00 | 0.9976 | 0.05 | -10.7560 | 10.7886 |
| TRTPN | 5 | 6 | -13.6055 | 5.393965 | -2.52 | 0.0141 | 0.05 | -24.3778 | -2.8332 |

Program: A\_Biol.sas Created: 02APR2020 7:35 POSTLOCK 

# Appendix 16.1.9.2.1 Statistical Methods and Analysis Output Supporting Table 14.2.2 Supporting Table 14.2.2

### The Mixed Procedure

### Parameter Code=REMAX

### Model Information

| Data Set | WORK.ADXV |
|---------------------------|---------------------|
| Dependent Variable | AVAL |
| Covariance Structure | Variance Components |
| Estimation Method | REML |
| Residual Variance Method | Profile |
| Fixed Effects SE Method | Model-Based |
| Degrees of Freedom Method | Containment |

### Class Level Information

| Class | LevelsValues |
|---|---|
| SUBJID | 151001 1002 1003 1004 1005 1006 1007 1008 1010 1012 1013 1014 1015 1016 1017 |
| TRTPN | 61 2 3 4 5 6 |
| APERIOD | 6P1 P2 P3 P4 P5 P6 |
| ARMCD | 6ABCEDF BEAFCD CADBFE DCFAEB EFBDAC FDECBA |

| Dimensions | | | |
|------------|-------------|------------|----|
| | Covariance | Parameters | 2 |
| | Columns in | X | 19 |
| | Columns in | Z | 15 |
| | Subjects | | 1 |
| | Max Obs per | Subject | 90 |

Program: A\_Biol.sas Created: 02APR2020 7:35 POSTLOCK 

# Appendix 16.1.9.2.1 Statistical Methods and Analysis Output Supporting Table 14.2.2 Supporting Table 14.2.2

The Mixed Procedure

### Parameter Code=REMAX

| | Nι | umber of Obse | rvations | |
|--------|----|---------------|----------|----|
| Number | of | Observations | Read | 90 |
| Number | of | Observations | Used | 90 |
| Number | οf | Observations | Not Used | 0 |

# Iteration History Iteration Evaluations -2 Res Log Like Criterion 0 1 983.84438280 1 1 974.534388150.00000000

Convergence criteria met.

# Estimates Cov Parm Estimate SUBJID(ARMCD) 6936.53 Residual 15320

Covariance Parameter

| Fit Statistics | |
|--------------------------|-------|
| -2 Res Log Likelihood | 974.5 |
| AIC (Smaller is Better) | 978.5 |
| AICC (Smaller is Better) | 978.7 |
| BIC (Smaller is Better) | 980.0 |

Program: A Biol.sas Created: 02APR2020 7:35 POSTLOCK 

The Mixed Procedure

Parameter Code=REMAX

Type 3 Tests of Fixed Effects

| | Num I | Den | |
|---------|-------|------|--------------|
| Effect | DF | DF F | Value Pr > F |
| TRTPN | 5 | 65 | 3.720.0051 |
| APERIOD | 5 | 65 | 2.320.0528 |
| ARMCD | 5 | 9 | 0.890.5270 |

# Coefficients for Oxy 30 vs Placebo Planned Planned

| | | Arm | Treatment | |
|-----------|---------|--------|-----------|------|
| Effect | APERIOD | Code | (N) | Row1 |
| Intercept | | | | |
| TRTPN | | | 1 | |
| TRTPN | | | 2 | |
| TRTPN | | | 3 | |
| TRTPN | | | 4 | 1 |
| TRTPN | | | 5 | |
| TRTPN | | | 6 | -1 |
| APERIOD | P1 | | | |
| APERIOD | P2 | | | |
| APERIOD | Р3 | | | |
| APERIOD | P4 | | | |
| APERIOD | P5 | | | |
| APERIOD | P6 | | | |
| ARMCD | | ABCEDF | | |
| ARMCD | | BEAFCD | | |
| ARMCD | | CADBFE | | |
| ARMCD | | DCFAEB | | |

The Mixed Procedure

Parameter Code=REMAX

Coefficients for Oxy 30 vs Placebo

Planned Planned

 $\begin{array}{c|cccc} & & Arm & Treatment \\ \hline Effect & APERIOD\,Code & (N) & Row1 \\ \hline ARMCD & EFBDAC \end{array}$ 

ARMCD EFBDAC FDECBA

Coefficients for Oxy 60 vs Placebo

Planned Planned
Arm Treatment

Effect APERIOD Code (N) Row1 Intercept TRTPN 1 TRTPN TRTPN 3 TRTPN 1 TRTPN -1 TRTPN APERIOD P1 APERIOD P2 APERIOD P3 APERIOD P4 APERIOD P5 APERIOD P6 ARMCD ABCEDF ARMCD BEAFCD ARMCD CADBFE ARMCD DCFAEB

The Mixed Procedure

### Parameter Code=REMAX

Coefficients for Oxy 60 vs Placebo

Planned Planned

Arm Treatment
Effect APERIOD Code (N) Row1
ARMCD EFBDAC
ARMCD FDECBA

Coefficients for Bel 300 vs Oxy 30

Planned Planned Arm Treatment

| | | 211111 | I I Ca chichi c | |
|-----------|---------|--------|-----------------|------|
| Effect | APERIOD | ) Code | (N) | Row1 |
| Intercept | ; | | | |
| TRTPN | | | 1 | 1 |
| TRTPN | | | 2 | |
| TRTPN | | | 3 | |
| TRTPN | | | 4 | -1 |
| TRTPN | | | 5 | |
| TRTPN | | | 6 | |
| APERIOD | P1 | | | |
| APERIOD | P2 | | | |
| APERIOD | Р3 | | | |
| APERIOD | P4 | | | |
| APERIOD | P5 | | | |
| APERIOD | P6 | | | |
| ARMCD | | ABCEDF | | |
| ARMCD | | BEAFCD | | |
| ARMCD | | CADBFE | | |
| ARMCD | | DCFAEB | | |

Program: A\_Biol.sas Created: 02APR2020 7:35 POSTLOCK

The Mixed Procedure

Parameter Code=REMAX

Coefficients for Bel 300 vs Oxy 30

Planned Planned

Arm Treatment Effect APERIOD Code (N) Row1

ARMCD EFBDAC ARMCD FDECBA

Coefficients for Bel 300 vs Oxy 60

Planned Planned

| | | Arm | Treatment | |
|-----------|---------|--------|-----------|------|
| Effect | APERIOD | Code | (N) | Row1 |
| Intercept | | | | |
| TRTPN | | | 1 | 1 |
| TRTPN | | | 2 | |
| TRTPN | | | 3 | |
| TRTPN | | | 4 | |
| TRTPN | | | 5 | -1 |
| TRTPN | | | 6 | |
| APERIOD | P1 | | | |
| APERIOD | P2 | | | |
| APERIOD | P3 | | | |
| APERIOD | P4 | | | |
| APERIOD | P5 | | | |
| APERIOD | P6 | | | |
| ARMCD | | ABCEDF | | |
| ARMCD | | BEAFCD | | |
| ARMCD | | CADBFE | | |
| ARMCD | | DCFAEB | | |

The Mixed Procedure

Parameter Code=REMAX

Coefficients for Bel 300 vs Oxy 60

Planned Planned

 Arm
 Treatment

 Effect
 APERIOD Code
 (N)
 Row1

 ARMCD
 EFBDAC

 ARMCD
 FDECBA

Coefficients for Bel 600 vs Oxy 30
Planned Planned

Arm Treatment

| | | 211111 | I I Ca chich | • |
|-----------|--------|--------|--------------|------|
| Effect | APERIO | ) Code | (N) | Row1 |
| Intercept | ; | | | |
| TRTPN | | | 1 | |
| TRTPN | | | 2 | 1 |
| TRTPN | | | 3 | |
| TRTPN | | | 4 | -1 |
| TRTPN | | | 5 | |
| TRTPN | | | 6 | |
| APERIOD | P1 | | | |
| APERIOD | P2 | | | |
| APERIOD | Р3 | | | |
| APERIOD | P4 | | | |
| APERIOD | P5 | | | |
| APERIOD | P6 | | | |
| ARMCD | | ABCEDF | | |
| ARMCD | | BEAFCD | | |
| ARMCD | | CADBFE | | |
| ARMCD | | DCFAEB | | |

Program: A\_Biol.sas Created: 02APR2020 7:35 POSTLOCK 

The Mixed Procedure

Parameter Code=REMAX

Coefficients for Bel 600 vs Oxy 30

Planned Planned

Arm Treatment Effect APERIOD Code (N) Row1

ARMCD EFBDAC ARMCD FDECBA

Coefficients for Bel 600 vs Oxy 60

Planned Planned

Arm Treatment Effect APERIOD Code (N) Row1 Intercept TRTPN 1 TRTPN 1 TRTPN 3 TRTPN -1 TRTPN TRTPN APERIOD P1 APERIOD P2 APERIOD P3 APERIOD P4 APERIOD P5 APERIOD P6 ARMCD ABCEDF ARMCD BEAFCD ARMCD CADBFE

DCFAEB

Program: A\_Biol.sas Created: 02APR2020 7:35 POSTLOCK

ARMCD


The Mixed Procedure

Parameter Code=REMAX

Coefficients for Bel 600 vs Oxy 60

Planned Planned

Arm Treatment fect APERIOD Code (N) Row1

Effect APERIOD Code (N)

ARMCD EFBDAC

ARMCD FDECBA

Coefficients for Bel 900 vs Oxy 30

Planned Planned

Arm Treatment Effect APERIOD Code (N) Row1 Intercept 1 TRTPN TRTPN 3 TRTPN 1 TRTPN -1 TRTPN TRTPN APERIOD P1 APERIOD P2 APERIOD P3 APERIOD P4 APERIOD P5 APERIOD P6 ARMCD ABCEDF ARMCD BEAFCD ARMCD CADBFE ARMCD DCFAEB

Program: A\_Biol.sas Created: 02APR2020 7:35 POSTLOCK


The Mixed Procedure

Parameter Code=REMAX

Coefficients for Bel 900 vs Oxy 30

Planned Planned

 $\begin{array}{ccc} & & \text{Arm} & & \text{Treatment} \\ \text{Effect} & & \text{APERIOD\,Code} & & \text{(N)} & & \text{Row1} \\ \end{array}$ 

ARMCD EFBDAC ARMCD FDECBA

Coefficients for Bel 900 vs Oxy 60

Planned Planned

Arm Treatment fect APERIOD Code (N)

| Effect | APERIOD C | Code | (N) | Row1 |
|----------|-----------|--------|-----|------|
| Intercep | t | | | |
| TRTPN | | | 1 | |
| TRTPN | | | 2 | |
| TRTPN | | | 3 | 1 |
| TRTPN | | | 4 | |
| TRTPN | | | 5 | -1 |
| TRTPN | | | 6 | |
| APERIOD | P1 | | | |
| APERIOD | P2 | | | |
| APERIOD | Р3 | | | |
| APERIOD | P4 | | | |
| APERIOD | P5 | | | |
| APERIOD | P6 | | | |
| ARMCD | A | ABCEDF | | |
| ARMCD | E | BEAFCD | | |
| ARMCD | C | CADBFE | | |
| ARMCD | Ε | CFAEB | | |

The Mixed Procedure

### Parameter Code=REMAX

Coefficients for Bel 900 vs Oxy 60

Planned Planned

 Arm
 Treatment

 Effect
 APERIOD Code
 (N)
 Row1

 ARMCD
 EFBDAC

 ARMCD
 FDECBA

Coefficients for Bel 300 vs Placebo
Planned Planned

| | | Arm | Treatment | |
|-----------|--------|--------|-----------|------|
| Effect | APERIO | ) Code | (N) | Row1 |
| Intercept | ; | | | |
| TRTPN | | | 1 | 1 |
| TRTPN | | | 2 | |
| TRTPN | | | 3 | |
| TRTPN | | | 4 | |
| TRTPN | | | 5 | |
| TRTPN | | | 6 | -1 |
| APERIOD | P1 | | | |
| APERIOD | P2 | | | |
| APERIOD | Р3 | | | |
| APERIOD | P4 | | | |
| APERIOD | P5 | | | |
| APERIOD | P6 | | | |
| ARMCD | | ABCEDF | | |
| ARMCD | | BEAFCD | | |
| ARMCD | | CADBFE | | |
| ARMCD | | DCFAEB | | |

### The Mixed Procedure

### Parameter Code=REMAX

Coefficients for Bel 300 vs Placebo

Planned Planned

Arm Treatment
Effect APERIOD Code (N) Row1

| LITCCC | THE BILLIOD COUC | ( + 4 ) |
|--------|------------------|---------|
| ARMCD | EFBDAC | |
| ARMCD | FDECBA | |

# Coefficients for Bel 600 vs Placebo

Planned Planned

| | | Arm | Treatment | |
|-----------|---------|--------|-----------|------|
| Effect | APERIOD | Code | (N) | Row1 |
| Intercept | | | | |
| TRTPN | | | 1 | |
| TRTPN | | | 2 | 1 |
| TRTPN | | | 3 | |
| TRTPN | | | 4 | |
| TRTPN | | | 5 | |
| TRTPN | | | 6 | -1 |
| APERIOD | P1 | | | |
| APERIOD | P2 | | | |
| APERIOD | Р3 | | | |
| APERIOD | P4 | | | |
| APERIOD | P5 | | | |
| APERIOD | P6 | | | |
| ARMCD | | ABCEDF | | |
| ARMCD | | BEAFCD | | |
| ARMCD | | CADBFE | | |
| ARMCD | | DCFAEB | | |

Program: A Biol.sas Created: 02APR2020 7:35 POSTLOCK 

The Mixed Procedure

Parameter Code=REMAX

Coefficients for Bel 600 vs Placebo

Planned Planned

 $\begin{array}{c|cccc} & & Arm & Treatment \\ \hline Effect & APERIOD\,Code & (N) & Row1 \\ \hline ARMCD & EFBDAC \end{array}$ 

ARMCD FDECBA

Coefficients for Bel 900 vs Placebo

Planned Planned Arm Treatment

Effect APERIOD Code (N) Row1 Intercept 1 TRTPN TRTPN 3 TRTPN 1 TRTPN TRTPN TRTPN -1 APERIOD P1 APERIOD P2 APERIOD P3 APERIOD P4 APERIOD P5 APERIOD P6 ARMCD ABCEDF ARMCD BEAFCD ARMCD CADBFE ARMCD DCFAEB

# Appendix 16.1.9.2.1 Statistical Methods and Analysis Output Supporting Table 14.2.2 Supporting Table 14.2.2

The Mixed Procedure

### Parameter Code=REMAX

Coefficients for Bel 900 vs Placebo

Planned Planned

Arm Treatment

Effect APERIOD Code (N) Row1
ARMCD EFBDAC
ARMCD FDECBA

### Estimates

### Standard

| Label | Estimate | Error DF t | Value E | r > t | Alpha | Lower | Upper |
|---|---|---|---|---|---|---|---|
| Oxy 30 vs Placebo | -20.2097 | 45.399165 | -0.45 | 0.6577 | 0.05 | -110.88 | 70.4586 |
| Oxy 60 vs Placebo | -129.70 | 45.399165 | -2.86 | 0.0057 | 0.05 | -220.37 | -39.0311 |
| Bel 300 vs Oxy 30 | 64.5958 | 45.399165 | 1.42 | 0.1596 | 0.05 | -26.0726 | 155.26 |
| Bel 300 vs Oxy 60 | 174.09 | 45.399165 | 3.83 | 0.0003 | 0.05 | 83.4171 | 264.75 |
| Bel 600 vs Oxy 30 | 20.6471 | 45.297265 | 0.46 | 0.6500 | 0.05 | -69.8177 | 111.11 |
| Bel 600 vs Oxy 60 | 130.14 | 45.399165 | 2.87 | 0.0056 | 0.05 | 39.4684 | 220.81 |
| Bel 900 vs Oxy 30 | 49.7034 | 45.399165 | 1.09 | 0.2776 | 0.05 | -40.9650 | 140.37 |
| Bel 900 vs Oxy 60 | 159.19 | 45.297265 | 3.51 | 0.0008 | 0.05 | 68.7282 | 249.66 |
| Bel 300 vs Placebo | 44.3861 | 45.297265 | 0.98 | 0.3308 | 0.05 | -46.0788 | 134.85 |
| Bel 600 vs Placebo | 0.4374 | 45.399165 | 0.01 | 0.9923 | 0.05 | -90.2310 | 91.1057 |
| Bel 900 vs Placebo | 29.4936 | 45.399165 | 0.65 | 0.5182 | 0.05 | -61.1747 | 120.16 |

Program: A Biol.sas Created: 02APR2020 7:35 POSTLOCK 

# Appendix 16.1.9.2.1 Statistical Methods and Analysis Output Supporting Table 14.2.2 Supporting Table 14.2.2

The Mixed Procedure

Parameter Code=REMAX

Least Squares Means

| | | | _ | | | | | |
|---|---|---|---|---|---|---|---|---|
| | Planned | | | | | | | |
| | Treatment | | Standard | | | | | |
| Effect | (N) | Estimate | Error DF t | Value P | r > t | Alpha | Lower | Upper |
| TRTPN | 1 | 586.67 | 38.949265 | 15.06 | <.0001 | 0.05 | 508.88 | 664.46 |
| TRTPN | 2 | 542.72 | 38.949265 | 13.93 | <.0001 | 0.05 | 464.93 | 620.51 |
| TRTPN | 3 | 571.78 | 38.949265 | 14.68 | <.0001 | 0.05 | 493.99 | 649.56 |
| TRTPN | 4 | 522.07 | 38.949265 | 13.40 | <.0001 | 0.05 | 444.29 | 599.86 |
| TRTPN | 5 | 412.58 | 38.949265 | 10.59 | <.0001 | 0.05 | 334.80 | 490.37 |
| TRTPN | 6 | 542.28 | 38.949265 | 13.92 | <.0001 | 0.05 | 464.50 | 620.07 |

Differences of Least Squares Means

| | | | | | 1 | | | |
|---|---|---|---|---|---|---|---|---|
| | Planned | Planned | | | | | | |
| | Treatment | Treatment | 9 | Standard | | | | |
| Effect | (N) | (N) | Estimate | Error DF t | Value P | r > t | Alpha Lower | Upper |
| TRTPN | 1 | 2 | 43.9487 | 45.399165 | 0.97 | 0.3366 | 0.05-46.7197 | 134.62 |
| TRTPN | 1 | 3 | 14.8924 | 45.399165 | 0.33 | 0.7439 | 0.05-75.7759 | 105.56 |
| TRTPN | 1 | 4 | 64.5958 | 45.399165 | 1.42 | 0.1596 | 0.05-26.0726 | 155.26 |
| TRTPN | 1 | 5 | 174.09 | 45.399165 | 3.83 | 0.0003 | 0.05 83.4171 | 264.75 |
| TRTPN | 1 | 6 | 44.3861 | 45.297265 | 0.98 | 0.3308 | 0.05-46.0788 | 134.85 |
| TRTPN | 2 | 3 | -29.0563 | 45.399165 | -0.64 | 0.5244 | 0.05 -119.72 | 61.6121 |
| TRTPN | 2 | 4 | 20.6471 | 45.297265 | 0.46 | 0.6500 | 0.05-69.8177 | 111.11 |
| TRTPN | 2 | 5 | 130.14 | 45.399165 | 2.87 | 0.0056 | 0.05 39.4684 | 220.81 |
| TRTPN | 2 | 6 | 0.4374 | 45.399165 | 0.01 | 0.9923 | 0.05-90.2310 | 91.1057 |
| TRTPN | 3 | 4 | 49.7034 | 45.399165 | 1.09 | 0.2776 | 0.05-40.9650 | 140.37 |
| TRTPN | 3 | 5 | 159.19 | 45.297265 | 3.51 | 0.0008 | 0.05 68.7282 | 249.66 |
| TRTPN | 3 | 6 | 29.4936 | 45.399165 | 0.65 | 0.5182 | 0.05-61.1747 | 120.16 |
| TRTPN | 4 | 5 | 109.49 | 45.399165 | 2.41 | 0.0187 | 0.05 18.8213 | 200.16 |

Program: A Biol.sas Created: 02APR2020 7:35 POSTLOCK 

# Appendix 16.1.9.2.1 Statistical Methods and Analysis Output Supporting Table 14.2.2Supporting Table 14.2.2

The Mixed Procedure

Parameter Code=REMAX

Differences of Least Squares Means

Planned Planned Treatment Treatment

| Treatment Treatment | | Standard | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| | Effect | (N) | (N) | Estimate | Error DF t | Value P | r > t P | Alpha | Lower | Upper |
| | TRTPN | 4 | 6 | -20.2097 | 45.399165 | -0.45 | 0.6577 | 0.05 | -110.88 | 70.4586 |
| | TRTPN | 5 | 6 | -129.70 | 45.399165 | -2.86 | 0.0057 | 0.05 | -220.37 | -39.0311 |

 Program: A Biol.sas Created: 02APR2020 7:35 POSTLOCK

# Appendix 16.1.9.2.1 Statistical Methods and Analysis Output Supporting Table 14.2.2 Supporting Table 14.2.2

### The Mixed Procedure

### Parameter Code=RRSPEMAX

### Model Information

| Data Set | WORK.ADXV |
|---------------------------|---------------------|
| Dependent Variable | AVAL |
| Covariance Structure | Variance Components |
| Estimation Method | REML |
| Residual Variance Method | Profile |
| Fixed Effects SE Method | Model-Based |
| Degrees of Freedom Method | Containment |

### Class Level Information

| Class | LevelsValues |
|---|---|
| SUBJID | 151001 1002 1003 1004 1005 1006 1007 1008 1010 1012 1013 1014 1015 1016 1017 |
| TRTPN | 61 2 3 4 5 6 |
| APERIOD | 6P1 P2 P3 P4 P5 P6 |
| ARMCD | 6ABCEDF BEAFCD CADBFE DCFAEB EFBDAC FDECBA |

| Dimensions | |
|----------------|-----------|
| Covariance Par | ameters 2 |
| Columns in X | 19 |
| Columns in Z | 15 |
| Subjects | 1 |
| Max Obs per Su | bject 90 |

Program: A\_Biol.sas Created: 02APR2020 7:35 POSTLOCK 

# Appendix 16.1.9.2.1 Statistical Methods and Analysis Output Supporting Table 14.2.2 Supporting Table 14.2.2

The Mixed Procedure

### Parameter Code=RRSPEMAX

| | Nι | umber of Obse | rvations | |
|--------|----|---------------|----------|----|
| Number | of | Observations | Read | 90 |
| Number | of | Observations | Used | 90 |
| Number | of | Observations | Not Used | 0 |

# Iteration History Iteration Evaluations -2 Res Log Like Criterion 0 1 447.68859180 1 1 419.425315020.00000000

Convergence criteria met.

# Estimates Cov Parm Estimate SUBJID(ARMCD) 9.4252 Residual 7.6646

Covariance Parameter

| Fit Statistics | |
|--------------------------|-------|
| -2 Res Log Likelihood | 419.4 |
| AIC (Smaller is Better) | 423.4 |
| AICC (Smaller is Better) | 423.6 |
| BIC (Smaller is Better) | 424.8 |

Program: A Biol.sas Created: 02APR2020 7:35 POSTLOCK 

The Mixed Procedure

Parameter Code=RRSPEMAX

Type 3 Tests of Fixed Effects

| 1 | NumI | Den | |
|---------|------|------|--------------|
| Effect | DF | DF F | Value Pr > F |
| TRTPN | 5 | 65 | 0.800.5523 |
| APERIOD | 5 | 65 | 1.020.4119 |
| ARMCD | 5 | 9 | 0.610.6987 |

# Coefficients for Oxy 30 vs Placebo Planned Planned

| - | | <br>- | | | | ~ | |
|----|----|-------|----|-------|---|-----|---|
| 7\ | rm | T | 20 | · > + | m | ont | + |

| | | Arm | Treatment | |
|-----------|---------|--------|-----------|------|
| Effect | APERIOD | Code | (N) | Row1 |
| Intercept | ; | | | |
| TRTPN | | | 1 | |
| TRTPN | | | 2 | |
| TRTPN | | | 3 | |
| TRTPN | | | 4 | 1 |
| TRTPN | | | 5 | |
| TRTPN | | | 6 | -1 |
| APERIOD | P1 | | | |
| APERIOD | P2 | | | |
| APERIOD | Р3 | | | |
| APERIOD | P4 | | | |
| APERIOD | P5 | | | |
| APERIOD | P6 | | | |
| ARMCD | | ABCEDF | | |
| ARMCD | | BEAFCD | | |
| ARMCD | | CADBFE | | |
| ARMCD | | DCFAEB | | |

Program: A\_Biol.sas Created: 02APR2020 7:35 POSTLOCK

The Mixed Procedure

### Parameter Code=RRSPEMAX

Coefficients for Oxy 30 vs Placebo

Planned Planned

 Arm
 Treatment

 Effect
 APERIOD Code
 (N)
 Row1

 ARMCD
 EFBDAC

 ARMCD
 FDECBA

Coefficients for Oxy 60 vs Placebo

Planned Planned
Arm Treatment

| | | ATIII | Treatment | |
|-----------|---------|--------|-----------|------|
| Effect | APERIOD | Code | (N) | Row1 |
| Intercept | | | | |
| TRTPN | | | 1 | |
| TRTPN | | | 2 | |
| TRTPN | | | 3 | |
| TRTPN | | | 4 | |
| TRTPN | | | 5 | 1 |
| TRTPN | | | 6 | -1 |
| APERIOD | P1 | | | |
| APERIOD | P2 | | | |
| APERIOD | Р3 | | | |
| APERIOD | P4 | | | |
| APERIOD | P5 | | | |
| APERIOD | P6 | | | |
| ARMCD | | ABCEDF | | |
| ARMCD | | BEAFCD | | |
| ARMCD | | CADBFE | | |
| ARMCD | | DCFAEB | | |

### The Mixed Procedure

### Parameter Code=RRSPEMAX

# Coefficients for Oxy 60 vs Placebo

Planned Planned

 Arm
 Treatment

 Effect
 APERIOD Code
 (N)
 Row1

 ARMCD
 EFBDAC

 ARMCD
 FDECBA

# Coefficients for Bel 300 vs Oxy 30

Planned Planned Arm Treatment

| | | 212111 | I I Ca chich c | |
|-----------|---------|--------|----------------|------|
| Effect | APERIOD | Code | (N) | Row1 |
| Intercept | | | | |
| TRTPN | | | 1 | 1 |
| TRTPN | | | 2 | |
| TRTPN | | | 3 | |
| TRTPN | | | 4 | -1 |
| TRTPN | | | 5 | |
| TRTPN | | | 6 | |
| APERIOD | P1 | | | |
| APERIOD | P2 | | | |
| APERIOD | P3 | | | |
| APERIOD | P4 | | | |
| APERIOD | P5 | | | |
| APERIOD | P6 | | | |
| ARMCD | | ABCEDF | | |
| ARMCD | | BEAFCD | | |
| ARMCD | | CADBFE | | |
| ARMCD | | DCFAEB | | |

Program: A\_Biol.sas Created: 02APR2020 7:35 POSTLOCK 

### The Mixed Procedure

### Parameter Code=RRSPEMAX

Coefficients for Bel 300 vs Oxy 30

Planned Planned

 Arm
 Treatment

 Effect
 APERIOD Code
 (N)
 Row1

 ARMCD
 EFBDAC

 ARMCD
 FDECBA

Coefficients for Bel 300 vs Oxy 60
Planned Planned

Arm Treatment Effect APERIOD Code (N) Row1 Intercept 1 TRTPN 1 TRTPN TRTPN 3 TRTPN -1 TRTPN TRTPN APERIOD P1 APERIOD P2 APERIOD P3 APERIOD P4 APERIOD P5 APERIOD P6 ARMCD ABCEDF ARMCD BEAFCD ARMCD CADBFE ARMCD DCFAEB

Program: A\_Bio1.sas Created: 02APR2020 7:35 POSTLOCK


### The Mixed Procedure

### Parameter Code=RRSPEMAX

Coefficients for Bel 300 vs Oxy 60

Planned Planned

 $\begin{array}{c|cccc} & Arm & Treatment \\ \hline Effect & APERIOD\,Code & (N) & Row1 \\ \hline ARMCD & EFBDAC \\ \end{array}$ 

ARMCD EFBDAC
ARMCD FDECBA

Coefficients for Bel 600 vs Oxy 30

Planned Planned
Arm Treatment

| | | Arm | Treatment | |
|-----------|---------|--------|-----------|------|
| Effect | APERIOD | Code | (N) | Row1 |
| Intercept | | | | |
| TRTPN | | | 1 | |
| TRTPN | | | 2 | 1 |
| TRTPN | | | 3 | |
| TRTPN | | | 4 | -1 |
| TRTPN | | | 5 | |
| TRTPN | | | 6 | |
| APERIOD | P1 | | | |
| APERIOD | P2 | | | |
| APERIOD | P3 | | | |
| APERIOD | P4 | | | |
| APERIOD | P5 | | | |
| APERIOD | P6 | | | |
| ARMCD | | ABCEDF | | |
| ARMCD | | BEAFCD | | |
| ARMCD | | CADBFE | | |
| ARMCD | | DCFAEB | | |

Program: A\_Biol.sas Created: 02APR2020 7:35 POSTLOCK

### The Mixed Procedure

### Parameter Code=RRSPEMAX

Coefficients for Bel 600 vs Oxy 30

Planned Planned

 Arm
 Treatment

 Effect
 APERIOD Code
 (N)
 Row1

 ARMCD
 EFBDAC

 ARMCD
 FDECBA

Coefficients for Bel 600 vs Oxy 60 Planned Planned

| | | Arm | Treatment | |
|-----------|---------|--------|-----------|------|
| Effect | APERIOD | Code | (N) | Row1 |
| Intercept | | | | |
| TRTPN | | | 1 | |
| TRTPN | | | 2 | 1 |
| TRTPN | | | 3 | |
| TRTPN | | | 4 | |
| TRTPN | | | 5 | -1 |
| TRTPN | | | 6 | |
| APERIOD | P1 | | | |
| APERIOD | P2 | | | |
| APERIOD | P3 | | | |
| APERIOD | P4 | | | |
| APERIOD | P5 | | | |
| APERIOD | P6 | | | |
| ARMCD | | ABCEDF | | |
| ARMCD | | BEAFCD | | |
| ARMCD | | CADBFE | | |
| ARMCD | | DCFAEB | | |

### The Mixed Procedure

### Parameter Code=RRSPEMAX

Coefficients for Bel 600 vs Oxy 60

Planned Planned

 Arm
 Treatment

 Effect
 APERIOD Code
 (N)
 Row1

 ARMCD
 EFBDAC

 ARMCD
 FDECBA

Coefficients for Bel 900 vs Oxy 30
Planned Planned

Arm Treatment

| | | 2 2 2 111 | I I Ca chichi c | |
|-----------|--------|-----------|-----------------|------|
| Effect | APERIO | ) Code | (N) | Row1 |
| Intercept | | | | |
| TRTPN | | | 1 | |
| TRTPN | | | 2 | |
| TRTPN | | | 3 | 1 |
| TRTPN | | | 4 | -1 |
| TRTPN | | | 5 | |
| TRTPN | | | 6 | |
| APERIOD | P1 | | | |
| APERIOD | P2 | | | |
| APERIOD | Р3 | | | |
| APERIOD | P4 | | | |
| APERIOD | P5 | | | |
| APERIOD | P6 | | | |
| ARMCD | | ABCEDF | | |
| ARMCD | | BEAFCD | | |
| ARMCD | | CADBFE | | |
| ARMCD | | DCFAEB | | |

Program: A Biol.sas Created: 02APR2020 7:35 POSTLOCK 

### The Mixed Procedure

### Parameter Code=RRSPEMAX

Coefficients for Bel 900 vs Oxy 30

Planned Planned

 Arm
 Treatment

 Effect
 APERIOD Code
 (N)
 Row1

 ARMCD
 EFBDAC

 ARMCD
 FDECBA

Coefficients for Bel 900 vs 0xy 60
Planned Planned

Arm Treatment

| | | 2 1 L 111 | I I Ca cincii c | • |
|-----------|--------|-----------|-----------------|------|
| Effect | APERIO | ) Code | (N) | Row1 |
| Intercept | ; | | | |
| TRTPN | | | 1 | |
| TRTPN | | | 2 | |
| TRTPN | | | 3 | 1 |
| TRTPN | | | 4 | |
| TRTPN | | | 5 | -1 |
| TRTPN | | | 6 | |
| APERIOD | P1 | | | |
| APERIOD | P2 | | | |
| APERIOD | Р3 | | | |
| APERIOD | P4 | | | |
| APERIOD | P5 | | | |
| APERIOD | P6 | | | |
| ARMCD | | ABCEDF | | |
| ARMCD | | BEAFCD | | |
| ARMCD | | CADBFE | | |
| ARMCD | | DCFAEB | | |

Program: A Biol.sas Created: 02APR2020 7:35 POSTLOCK 

### The Mixed Procedure

### Parameter Code=RRSPEMAX

Coefficients for Bel 900 vs Oxy 60

Planned Planned

 Arm
 Treatment

 Effect
 APERIOD Code
 (N)
 Row1

 ARMCD
 EFBDAC

 ARMCD
 FDECBA

Coefficients for Bel 300 vs Placebo
Planned Planned

Arm Treatment

| | | ALIII | TIEacment | |
|-----------|---------|--------|-----------|------|
| Effect | APERIOD | Code | (N) | Row1 |
| Intercept | | | | |
| TRTPN | | | 1 | 1 |
| TRTPN | | | 2 | |
| TRTPN | | | 3 | |
| TRTPN | | | 4 | |
| TRTPN | | | 5 | |
| TRTPN | | | 6 | -1 |
| APERIOD | P1 | | | |
| APERIOD | P2 | | | |
| APERIOD | Р3 | | | |
| APERIOD | P4 | | | |
| APERIOD | P5 | | | |
| APERIOD | P6 | | | |
| ARMCD | | ABCEDF | | |
| ARMCD | | BEAFCD | | |
| ARMCD | | CADBFE | | |
| ARMCD | | DCFAEB | | |


### The Mixed Procedure

### Parameter Code=RRSPEMAX

# Coefficients for Bel 300 vs Placebo

Planned Planned

 Arm
 Treatment

 Effect
 APERIOD Code
 (N)
 Row1

 ARMCD
 EFBDAC

 ARMCD
 FDECBA

# Coefficients for Bel 600 vs Placebo

Planned Planned
Arm Treatment

| | | Arm | Treatment | |
|-----------|---------|--------|-----------|------|
| Effect | APERIOD | Code | (N) | Row1 |
| Intercept | | | | |
| TRTPN | | | 1 | |
| TRTPN | | | 2 | 1 |
| TRTPN | | | 3 | |
| TRTPN | | | 4 | |
| TRTPN | | | 5 | |
| TRTPN | | | 6 | -1 |
| APERIOD | P1 | | | |
| APERIOD | P2 | | | |
| APERIOD | P3 | | | |
| APERIOD | P4 | | | |
| APERIOD | P5 | | | |
| APERIOD | P6 | | | |
| ARMCD | | ABCEDF | | |
| ARMCD | | BEAFCD | | |
| ARMCD | | CADBFE | | |
| ARMCD | | DCFAEB | | |

### The Mixed Procedure

### Parameter Code=RRSPEMAX

# Coefficients for Bel 600 vs Placebo

Planned Planned

# Coefficients for Bel 900 vs Placebo

Planned Planned

| | | Arm | Treatment | |
|-----------|---------|--------|-----------|------|
| Effect | APERIOD | Code | (N) | Row1 |
| Intercept | | | | |
| TRTPN | | | 1 | |
| TRTPN | | | 2 | |
| TRTPN | | | 3 | 1 |
| TRTPN | | | 4 | |
| TRTPN | | | 5 | |
| TRTPN | | | 6 | -1 |
| APERIOD | P1 | | | |
| APERIOD | P2 | | | |
| APERIOD | P3 | | | |
| APERIOD | P4 | | | |
| APERIOD | P5 | | | |
| APERIOD | P6 | | | |
| ARMCD | | ABCEDF | | |
| ARMCD | | BEAFCD | | |
| ARMCD | | CADBFE | | |
| ARMCD | | DCFAEB | | |

# Appendix 16.1.9.2.1 Statistical Methods and Analysis Output Supporting Table 14.2.2 Supporting Table 14.2.2

### The Mixed Procedure

### Parameter Code=RRSPEMAX

Coefficients for Bel 900 vs Placebo

Planned Planned

Arm Treatment

| Effect | APERIOD Code | (N) | Row1 |
|--------|--------------|-----|------|
| ARMCD | EFBDAC | | |
| ARMCD | FDECBA | | |

### Estimates

### Standard

| Label | Estimate | Error DF t | Value F | r > t | Alpha | Lower Upper |
|---|---|---|---|---|---|---|
| Oxy 30 vs Placebo | -1.5420 | 1.015465 | -1.52 | 0.1337 | 0.05 | -3.57000.4860 |
| Oxy 60 vs Placebo | -1.8452 | 1.015465 | -1.82 | 0.0738 | 0.05 | -3.87320.1827 |
| Bel 300 vs Oxy 30 | 0.4076 | 1.015465 | 0.40 | 0.6894 | 0.05 | -1.62042.4356 |
| Bel 300 vs Oxy 60 | 0.7109 | 1.015465 | 0.70 | 0.4864 | 0.05 | -1.31712.7388 |
| Bel 600 vs Oxy 30 | 0.4711 | 1.013265 | 0.46 | 0.6435 | 0.05 | -1.55242.4945 |
| Bel 600 vs Oxy 60 | 0.7743 | 1.015465 | 0.76 | 0.4485 | 0.05 | -1.25372.8023 |
| Bel 900 vs Oxy 30 | 0.06312 | 1.015465 | 0.06 | 0.9506 | 0.05 | -1.96492.0911 |
| Bel 900 vs Oxy 60 | 0.3664 | 1.013265 | 0.36 | 0.7188 | 0.05 | -1.65712.3898 |
| Bel 300 vs Placebo | -1.1344 | 1.013265 | -1.12 | 0.2670 | 0.05 | -3.15780.8890 |
| Bel 600 vs Placebo | -1.0710 | 1.015465 | -1.05 | 0.2955 | 0.05 | -3.09890.9570 |
| Bel 900 vs Placebo | -1.4789 | 1.015465 | -1.46 | 0.1501 | 0.05 | -3.50690.5491 |

Program: A Biol.sas Created: 02APR2020 7:35 POSTLOCK 

# Appendix 16.1.9.2.1 Statistical Methods and Analysis Output Supporting Table 14.2.2 Supporting Table 14.2.2

### The Mixed Procedure

### Parameter Code=RRSPEMAX

## Least Squares Means

Planned

| | I I a i i i c a | | | | | | | |
|---|---|---|---|---|---|---|---|---|
| | Treatment | | Standard | | | | | |
| Effect | (N) | Estimate | Error DF t | Value | Pr > t | Alpha | Lower | Upper |
| TRTPN | 1 | 15.5293 | 1.082865 | 14.34 | <.0001 | 0.05 | 13.3667 | 17.6918 |
| TRTPN | 2 | 15.5927 | 1.082865 | 14.40 | <.0001 | 0.05 | 13.4302 | 17.7552 |
| TRTPN | 3 | 15.1848 | 1.082865 | 14.02 | <.0001 | 0.05 | 13.0222 | 17.3473 |
| TRTPN | 4 | 15.1217 | 1.082865 | 13.97 | <.0001 | 0.05 | 12.9591 | 17.2842 |
| TRTPN | 5 | 14.8184 | 1.082865 | 13.69 | <.0001 | 0.05 | 12.6559 | 16.9809 |
| TRTPN | 6 | 16.6637 | 1.082865 | 15.39 | <.0001 | 0.05 | 14.5011 | 18.8262 |

# Differences of Least Squares Means

| | | | | 1 | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| | Planned | Planned | | | | | | | |
| | Treatment | Treatment | | Standard | | | | | |
| Effect | (N) | (N) | ${\tt Estimate}$ | Error DF t | Value Pr | > t | Alpha | Lower | Upper |
| TRTPN | 1 | 2 | -0.06343 | 1.015465 | -0.06 | 0.9504 | 0.05- | -2.0914 | 1.9645 |
| TRTPN | 1 | 3 | 0.3445 | 1.015465 | 0.34 | 0.7355 | 0.05- | -1.6835 | 2.3725 |
| TRTPN | 1 | 4 | 0.4076 | 1.015465 | 0.40 | 0.6894 | 0.05- | -1.6204 | 2.4356 |
| TRTPN | 1 | 5 | 0.7109 | 1.015465 | 0.70 | 0.4864 | 0.05- | -1.3171 | 2.7388 |
| TRTPN | 1 | 6 | -1.1344 | 1.013265 | -1.12 | 0.2670 | 0.05- | -3.1578 | 0.8890 |
| TRTPN | 2 | 3 | 0.4079 | 1.015465 | 0.40 | 0.6892 | 0.05- | -1.6201 | 2.4359 |
| TRTPN | 2 | 4 | 0.4711 | 1.013265 | 0.46 | 0.6435 | 0.05- | -1.5524 | 2.4945 |
| TRTPN | 2 | 5 | 0.7743 | 1.015465 | 0.76 | 0.4485 | 0.05- | -1.2537 | 2.8023 |
| TRTPN | 2 | 6 | -1.0710 | 1.015465 | -1.05 | 0.2955 | 0.05- | -3.0989 | 0.9570 |
| TRTPN | 3 | 4 | 0.06312 | 1.015465 | 0.06 | 0.9506 | 0.05- | -1.9649 | 2.0911 |
| TRTPN | 3 | 5 | 0.3664 | 1.013265 | 0.36 | 0.7188 | 0.05- | -1.6571 | 2.3898 |
| TRTPN | 3 | 6 | -1.4789 | 1.015465 | -1.46 | 0.1501 | 0.05- | -3.5069 | 0.5491 |
| TRTPN | 4 | 5 | 0.3032 | 1.015465 | 0.30 | 0.7662 | 0.05- | -1.7247 | 2.3312 |

Program: A Biol.sas Created: 02APR2020 7:35 POSTLOCK 

# Appendix 16.1.9.2.1 Statistical Methods and Analysis Output Supporting Table 14.2.2 Supporting Table 14.2.2

The Mixed Procedure

### Parameter Code=RRSPEMAX

# Differences of Least Squares Means

Planned Planned

| | Treatment | Treatment | | Standard | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| Effect | (N) | (N) | Estimate | Error DF t | Value Pr | > t | Alpha | Lower | Upper |
| TRTPN | 4 | 6 | -1.5420 | 1.015465 | -1.52 | 0.1337 | 0.05-3 | 3.5700 | 0.4860 |
| TRTPN | 5 | 6 | -1.8452 | 1.015465 | -1.82 | 0.0738 | 0.05 - | 3.8732 | 0.1827 |

 Program: A\_Biol.sas Created: 02APR2020 7:35 POSTLOCK
## Appendix 16.1.9.2.1 Statistical Methods and Analysis Output Supporting Table 14.2.2 Supporting Table 14.2.2

### The Mixed Procedure

### Parameter Code=SEMAX

### Model Information

| Data Set | WORK.ADXV |
|---------------------------|---------------------|
| Dependent Variable | AVAL |
| Covariance Structure | Variance Components |
| Estimation Method | REML |
| Residual Variance Method | Profile |
| Fixed Effects SE Method | Model-Based |
| Degrees of Freedom Method | Containment |

### Class Level Information

| Class | LevelsValues |
|---|---|
| SUBJID | 151001 1002 1003 1004 1005 1006 1007 1008 1010 1012 1013 1014 1015 1016 1017 |
| TRTPN | 61 2 3 4 5 6 |
| APERIOD | 6P1 P2 P3 P4 P5 P6 |
| ARMCD | 6ABCEDF BEAFCD CADBFE DCFAEB EFBDAC FDECBA |

| Dimensions | | |
|-------------|------------|----|
| Covariance | Parameters | 2 |
| Columns in | X | 19 |
| Columns in | Z | 15 |
| Subjects | | 1 |
| Max Obs per | Subject | 90 |

Program: A\_Biol.sas Created: 02APR2020 7:35 POSTLOCK 

## Appendix 16.1.9.2.1 Statistical Methods and Analysis Output Supporting Table 14.2.2 Supporting Table 14.2.2

The Mixed Procedure

### Parameter Code=SEMAX

| | Nι | umber of Obse | rvations | |
|--------|----|---------------|----------|----|
| Number | of | Observations | Read | 90 |
| Number | of | Observations | Used | 90 |
| Number | of | Observations | Not Used | 0 |

# Iteration History Iteration Evaluations -2 Res Log Like Criterion 0 1 1156.00805775 1 1151.832259990.00000000

Convergence criteria met.

### Covariance Parameter Estimates

| Cov Parm | Estimate |
|----------------|----------|
| SUBJID (ARMCD) | 44274 |
| Residual | 176454 |

### Fit Statistics

| -2 Res Log Likelihood | 1151.8 |
|--------------------------|--------|
| AIC (Smaller is Better) | 1155.8 |
| AICC (Smaller is Better) | 1156.0 |
| BIC (Smaller is Better) | 1157.2 |

Program: A Biol.sas Created: 02APR2020 7:35 POSTLOCK 

The Mixed Procedure

Parameter Code=SEMAX

Type 3 Tests of Fixed Effects
Num Den

| | Nulli | Jen | |
|---------|-------|------|--------------|
| Effect | DF | DF F | Value Pr > F |
| TRTPN | 5 | 65 | 2.660.0299 |
| APERIOD | 5 | 65 | 3.330.0096 |
| ARMCD | 5 | 9 | 1.240.3681 |

Coefficients for Oxy 30 vs Placebo
Planned Planned

| | | Arm | Treatment | : |
|-----------|--------|--------|-----------|------|
| Effect | APERIO | ) Code | (N) | Row1 |
| Intercept | ; | | | |
| TRTPN | | | 1 | |
| TRTPN | | | 2 | |
| TRTPN | | | 3 | |
| TRTPN | | | 4 | 1 |
| TRTPN | | | 5 | |
| TRTPN | | | 6 | -1 |
| APERIOD | P1 | | | |
| APERIOD | P2 | | | |
| APERIOD | Р3 | | | |
| APERIOD | P4 | | | |
| APERIOD | P5 | | | |
| APERIOD | P6 | | | |
| ARMCD | | ABCEDF | | |
| ARMCD | | BEAFCD | | |
| ARMCD | | CADBFE | | |
| ARMCD | | DCFAEB | | |

Program: A\_Bio1.sas Created: 02APR2020 7:35 POSTLOCK

The Mixed Procedure

Parameter Code=SEMAX

Coefficients for Oxy 30 vs Placebo

Planned Planned

Arm Treatment Effect APERIOD Code (N) Row1

ARMCD EFBDAC ARMCD FDECBA

Coefficients for Oxy 60 vs Placebo

Planned Planned

Arm Treatment Effect APERIOD Code (N) Row1 Intercept TRTPN 1 TRTPN TRTPN 3 TRTPN 1 TRTPN -1 TRTPN APERIOD P1 APERIOD P2 APERIOD P3 APERIOD P4 APERIOD P5 APERIOD P6 ARMCD ABCEDF ARMCD BEAFCD ARMCD CADBFE ARMCD DCFAEB

Program: A\_Biol.sas Created: 02APR2020 7:35 POSTLOCK

The Mixed Procedure

Parameter Code=SEMAX

Coefficients for Oxy 60 vs Placebo

Planned Planned

 Arm
 Treatment

 Effect
 APERIOD Code
 (N)
 Row1

 ARMCD
 EFBDAC

 ARMCD
 FDECBA

Coefficients for Bel 300 vs Oxy 30

Planned Planned

Arm Treatment Effect APERIOD Code (N) Row1 Intercept 1 TRTPN 1 TRTPN TRTPN 3 TRTPN -1 TRTPN TRTPN APERIOD P1 APERIOD P2 APERIOD P3 APERIOD P4 APERIOD P5 APERIOD P6 ARMCD ABCEDF ARMCD BEAFCD ARMCD CADBFE ARMCD DCFAEB

The Mixed Procedure

Parameter Code=SEMAX

Coefficients for Bel 300 vs Oxy 30

Planned Planned

 Arm
 Treatment

 Effect
 APERIOD Code
 (N)
 Row1

 ARMCD
 EFBDAC

 ARMCD
 FDECBA

Coefficients for Bel 300 vs Oxy 60 Planned Planned

| | | Arm | Treatment | |
|-----------|---------|--------|-----------|------|
| Effect | APERIOD | Code | (N) | Row1 |
| Intercept | | | | |
| TRTPN | | | 1 | 1 |
| TRTPN | | | 2 | |
| TRTPN | | | 3 | |
| TRTPN | | | 4 | |
| TRTPN | | | 5 | -1 |
| TRTPN | | | 6 | |
| APERIOD | P1 | | | |
| APERIOD | P2 | | | |
| APERIOD | P3 | | | |
| APERIOD | P4 | | | |
| APERIOD | P5 | | | |
| APERIOD | P6 | | | |
| ARMCD | | ABCEDF | | |
| ARMCD | | BEAFCD | | |
| ARMCD | | CADBFE | | |
| ARMCD | | DCFAEB | | |

The Mixed Procedure

Parameter Code=SEMAX

Coefficients for Bel 300 vs Oxy 60

Planned Planned

Arm Treatment
Effect APERIOD Code (N) Row1

ARMCD EFBDAC ARMCD FDECBA

Coefficients for Bel 600 vs Oxy 30

Planned Planned

Arm Treatment Effect APERIOD Code (N) Row1 Intercept TRTPN 1 TRTPN 1 TRTPN 3 TRTPN -1 TRTPN TRTPN APERIOD P1 APERIOD P2 APERIOD P3 APERIOD P4 APERIOD P5 APERIOD P6 ARMCD ABCEDF ARMCD BEAFCD ARMCD CADBFE ARMCD DCFAEB

Program: A\_Biol.sas Created: 02APR2020 7:35 POSTLOCK

The Mixed Procedure

Parameter Code=SEMAX

Coefficients for Bel 600 vs Oxy 30

Planned Planned

Arm Treatment
APERIOD Code (N) Row1

Effect APERIOD Code (N)

ARMCD EFBDAC

ARMCD FDECBA

Coefficients for Bel 600 vs Oxy 60

Planned Planned

Arm Treatment

| | | 21111 | I I Ca chich c | |
|-----------|---------|--------|----------------|------|
| Effect | APERIOD | Code | (N) | Row1 |
| Intercept | | | | |
| TRTPN | | | 1 | |
| TRTPN | | | 2 | 1 |
| TRTPN | | | 3 | |
| TRTPN | | | 4 | |
| TRTPN | | | 5 | -1 |
| TRTPN | | | 6 | |
| APERIOD | P1 | | | |
| APERIOD | P2 | | | |
| APERIOD | P3 | | | |
| APERIOD | P4 | | | |
| APERIOD | P5 | | | |
| APERIOD | P6 | | | |
| ARMCD | | ABCEDF | | |
| ARMCD | | BEAFCD | | |
| ARMCD | | CADBFE | | |
| ARMCD | | DCFAEB | | |

Program: A Biol.sas Created: 02APR2020 7:35 POSTLOCK 

The Mixed Procedure

Parameter Code=SEMAX

Coefficients for Bel 600 vs Oxy 60

Planned Planned

Arm Treatment Effect APERIOD Code (N) Row1

ARMCD EFBDAC ARMCD FDECBA

Coefficients for Bel 900 vs Oxy 30

Planned Planned

Arm Treatment Effect APERIOD Code (N) Row1 Intercept 1 TRTPN TRTPN 3 TRTPN 1 TRTPN -1 TRTPN TRTPN APERIOD P1 APERIOD P2 APERIOD P3 APERIOD P4 APERIOD P5 APERIOD P6 ARMCD ABCEDF ARMCD BEAFCD ARMCD CADBFE ARMCD DCFAEB

Program: A Biol.sas Created: 02APR2020 7:35 POSTLOCK 

The Mixed Procedure

Parameter Code=SEMAX

Coefficients for Bel 900 vs Oxy 30

Planned Planned

Arm Treatment

| Effect | APERIOD Code | (N) | Row1 |
|--------|--------------|-----|------|
| ARMCD | EFBDAC | | |
| ARMCD | FDECBA | | |

Coefficients for Bel 900 vs Oxy 60

Planned Planned

Arm Treatment Effect APERIOD Code (N) Row1 Intercept 1 TRTPN TRTPN 3 TRTPN 1 TRTPN 5 TRTPN -1 TRTPN APERIOD P1 APERIOD P2 APERIOD P3 APERIOD P4 APERIOD P5 APERIOD P6 ARMCD ABCEDF ARMCD BEAFCD ARMCD CADBFE ARMCD DCFAEB

Program: A\_Bio1.sas Created: 02APR2020 7:35 POSTLOCK


The Mixed Procedure

Parameter Code=SEMAX

Coefficients for Bel 900 vs Oxy 60

Planned Planned

 Arm
 Treatment

 Effect
 APERIOD Code
 (N)
 Row1

 ARMCD
 EFBDAC

 ARMCD
 FDECBA

Coefficients for Bel 300 vs Placebo
Planned Planned

| | | Arm | Treatment | |
|-----------|---------|--------|-----------|------|
| Effect | APERIOD | ) Code | (N) | Row1 |
| Intercept | ; | | | |
| TRTPN | | | 1 | 1 |
| TRTPN | | | 2 | |
| TRTPN | | | 3 | |
| TRTPN | | | 4 | |
| TRTPN | | | 5 | |
| TRTPN | | | 6 | -1 |
| APERIOD | P1 | | | |
| APERIOD | P2 | | | |
| APERIOD | P3 | | | |
| APERIOD | P4 | | | |
| APERIOD | P5 | | | |
| APERIOD | P6 | | | |
| ARMCD | | ABCEDF | | |
| ARMCD | | BEAFCD | | |
| ARMCD | | CADBFE | | |
| ARMCD | | DCFAEB | | |

The Mixed Procedure

### Parameter Code=SEMAX

Coefficients for Bel 300 vs Placebo

Planned Planned

 Arm
 Treatment

 Effect
 APERIOD Code
 (N)
 Row1

 ARMCD
 EFBDAC

 ARMCD
 FDECBA

Coefficients for Bel 600 vs Placebo
Planned Planned

| | | Arm | Treatment | |
|-----------|---------|--------|-----------|------|
| Effect | APERIOD | Code | (N) | Row1 |
| Intercept | | | | |
| TRTPN | | | 1 | |
| TRTPN | | | 2 | 1 |
| TRTPN | | | 3 | |
| TRTPN | | | 4 | |
| TRTPN | | | 5 | |
| TRTPN | | | 6 | -1 |
| APERIOD | P1 | | | |
| APERIOD | P2 | | | |
| APERIOD | P3 | | | |
| APERIOD | P4 | | | |
| APERIOD | P5 | | | |
| APERIOD | P6 | | | |
| ARMCD | | ABCEDF | | |
| ARMCD | | BEAFCD | | |
| ARMCD | | CADBFE | | |
| ARMCD | | DCFAEB | | |

The Mixed Procedure

### Parameter Code=SEMAX

Coefficients for Bel 600 vs Placebo

Planned Planned

 Arm
 Treatment

 Effect
 APERIOD Code
 (N)
 Row1

 ARMCD
 EFBDAC

FDECBA

ARMCD

Coefficients for Bel 900 vs Placebo Planned Planned

| | | Arm | Treatment | |
|-----------|---------|--------|-----------|------|
| Effect | APERIOD | Code | (N) | Row1 |
| Intercept | | | | |
| TRTPN | | | 1 | |
| TRTPN | | | 2 | |
| TRTPN | | | 3 | 1 |
| TRTPN | | | 4 | |
| TRTPN | | | 5 | |
| TRTPN | | | 6 | -1 |
| APERIOD | P1 | | | |
| APERIOD | P2 | | | |
| APERIOD | Р3 | | | |
| APERIOD | P4 | | | |
| APERIOD | P5 | | | |
| APERIOD | P6 | | | |
| ARMCD | | ABCEDF | | |
| ARMCD | | BEAFCD | | |
| ARMCD | | CADBFE | | |
| ARMCD | | DCFAEB | | |

## Appendix 16.1.9.2.1 Statistical Methods and Analysis Output Supporting Table 14.2.2 Supporting Table 14.2.2

The Mixed Procedure

### Parameter Code=SEMAX

Coefficients for Bel 900 vs Placebo

Planned Planned

Arm Treatment

Effect APERIOD Code (N) Row1
ARMCD EFBDAC
ARMCD FDECBA

### Estimates

### Standard

| Label | Estimate | ErrorDFt | Value | Pr > t . | Alpha | Lower | Upper |
|---|---|---|---|---|---|---|---|
| Oxy 30 vs Placebo | -72.0201 | 154.0765 | -0.47 | 0.6417 | 0.05 | -379.73 | 235.69 |
| Oxy 60 vs Placebo | -336.37 | 154.0765 | -2.18 | 0.0326 | 0.05 | -644.08 | -28.6636 |
| Bel 300 vs Oxy 30 | 200.18 | 154.0765 | 1.30 | 0.1984 | 0.05 | -107.52 | 507.89 |
| Bel 300 vs Oxy 60 | 464.53 | 154.0765 | 3.01 | 0.0037 | 0.05 | 156.83 | 772.24 |
| Bel 600 vs Oxy 30 | 165.60 | 153.7365 | 1.08 | 0.2854 | 0.05 | -141.42 | 472.62 |
| Bel 600 vs Oxy 60 | 429.95 | 154.0765 | 2.79 | 0.0069 | 0.05 | 122.24 | 737.66 |
| Bel 900 vs Oxy 30 | 193.57 | 154.0765 | 1.26 | 0.2135 | 0.05 | -114.14 | 501.28 |
| Bel 900 vs Oxy 60 | 457.92 | 153.7365 | 2.98 | 0.0041 | 0.05 | 150.90 | 764.94 |
| Bel 300 vs Placebo | 128.16 | 153.7365 | 0.83 | 0.4075 | 0.05 | -178.85 | 435.18 |
| Bel 600 vs Placebo | 93.5803 | 154.0765 | 0.61 | 0.5457 | 0.05 | -214.13 | 401.29 |
| Bel 900 vs Placebo | 121.55 | 154.0765 | 0.79 | 0.4330 | 0.05 | -186.16 | 429.26 |

Program: A Biol.sas Created: 02APR2020 7:35 POSTLOCK 

Appendix 16.1.9.2.1
Statistical Methods and Analysis Output Supporting Table 14.2.2
Supporting Table 14.2.2

The Mixed Procedure

Parameter Code=SEMAX

Least Squares Means

| | Planned | | | | | | | |
|---|---|---|---|---|---|---|---|---|
| | Treatment | | Standard | | | | | |
| Effect | (N) | ${\tt Estimate}$ | Error DF t | Value | Pr > t | Alpha | Lower | Upper |
| TRTPN | 1 | 1272.57 | 122.4765 | 10.39 | <.0001 | 0.05 | 1027.98 | 1517.16 |
| TRTPN | 2 | 1237.99 | 122.4765 | 10.11 | <.0001 | 0.05 | 993.40 | 1482.58 |
| TRTPN | 3 | 1265.96 | 122.4765 | 10.34 | <.0001 | 0.05 | 1021.37 | 1510.55 |
| TRTPN | 4 | 1072.39 | 122.4765 | 8.76 | <.0001 | 0.05 | 827.80 | 1316.98 |
| TRTPN | 5 | 808.04 | 122.4765 | 6.60 | <.0001 | 0.05 | 563.45 | 1052.63 |
| TRTPN | 6 | 1144.41 | 122.4765 | 9.34 | <.0001 | 0.05 | 899.82 | 1389.00 |

Differences of Least Squares Means

| | | | | | 1 | | | | |
|---|---|---|---|---|---|---|---|---|---|
| | Planned | Planned | | | | | | | |
| | Treatment | Treatment | St | tandard | | | | | |
| Effect | (N) | (N) | Estimate | Error DF t | Value Pr | $r > t ^2$ | Alpha | Lower | Upper |
| TRTPN | 1 | 2 | 34.5817 | 154.0765 | 0.22 | 0.8231 | 0.05 | -273.12 | 342.29 |
| TRTPN | 1 | 3 | 6.6126 | 154.0765 | 0.04 | 0.9659 | 0.05 | -301.09 | 314.32 |
| TRTPN | 1 | 4 | 200.18 | 154.0765 | 1.30 | 0.1984 | 0.05 | -107.52 | 507.89 |
| TRTPN | 1 | 5 | 464.53 | 154.0765 | 3.01 | 0.0037 | 0.05 | 156.83 | 772.24 |
| TRTPN | 1 | 6 | 128.16 | 153.7365 | 0.83 | 0.4075 | 0.05 | -178.85 | 435.18 |
| TRTPN | 2 | 3 | -27.9691 | 154.0765 | -0.18 | 0.8565 | 0.05 | -335.68 | 279.74 |
| TRTPN | 2 | 4 | 165.60 | 153.7365 | 1.08 | 0.2854 | 0.05 | -141.42 | 472.62 |
| TRTPN | 2 | 5 | 429.95 | 154.0765 | 2.79 | 0.0069 | 0.05 | 122.24 | 737.66 |
| TRTPN | 2 | 6 | 93.5803 | 154.0765 | 0.61 | 0.5457 | 0.05 | -214.13 | 401.29 |
| TRTPN | 3 | 4 | 193.57 | 154.0765 | 1.26 | 0.2135 | 0.05 | -114.14 | 501.28 |
| TRTPN | 3 | 5 | 457.92 | 153.7365 | 2.98 | 0.0041 | 0.05 | 150.90 | 764.94 |
| TRTPN | 3 | 6 | 121.55 | 154.0765 | 0.79 | 0.4330 | 0.05 | -186.16 | 429.26 |
| TRTPN | 4 | 5 | 264.35 | 154.0765 | 1.72 | 0.0910 | 0.05 | -43.3566 | 572.06 |

Program: A Biol.sas Created: 02APR2020 7:35 POSTLOCK 

### Appendix 16.1.9.2.1 Statistical Methods and Analysis Output Supporting Table 14.2.2Supporting Table 14.2.2

The Mixed Procedure

Parameter Code=SEMAX

Differences of Least Squares Means

Planned Planned Treatment Treatment

| | Treatment | Treatment | : | Standard | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| Effect | (N) | (N) | Estimate | Error DF t | Value Pr | > t . | Alpha | Lower | Upper |
| TRTPN | 4 | 6 | -72.0201 | 154.0765 | -0.47 | 0.6417 | 0.05 | -379.73 | 235.69 |
| TRTPN | 5 | 6 | -336.37 | 154.0765 | -2.18 | 0.0326 | 0.05 | -644.08 | -28.6636 |

 Program: A Biol.sas Created: 02APR2020 7:35 POSTLOCK

## Appendix 16.1.9.2.1 Statistical Methods and Analysis Output Supporting Table 14.2.2 Supporting Table 14.2.2

### The Mixed Procedure

### Parameter Code=TVEMEMAX

### Model Information

| Data Set | WORK.ADXV |
|---------------------------|---------------------|
| Dependent Variable | AVAL |
| Covariance Structure | Variance Components |
| Estimation Method | REML |
| Residual Variance Method | Profile |
| Fixed Effects SE Method | Model-Based |
| Degrees of Freedom Method | Containment |

### Class Level Information

| Class L | evels Values |
|---|---|
| SUBJID | 151001 1002 1003 1004 1005 1006 1007 1008 1010 1012 1013 1014 1015 1016 1017 |
| TRTPN | 61 2 3 4 5 6 |
| APERIOD | 6P1 P2 P3 P4 P5 P6 |
| ARMCD | 6ABCEDF BEAFCD CADBFE DCFAEB EFBDAC FDECBA |

| nensions | | |
|-------------|------------|----|
| Covariance | Parameters | 2 |
| Columns in | X | 19 |
| Columns in | Z | 15 |
| Subjects | | 1 |
| Max Obs per | Subject | 90 |

Program: A Biol.sas Created: 02APR2020 7:35 POSTLOCK 

### Appendix 16.1.9.2.1 Statistical Methods and Analysis Output Supporting Table 14.2.2 Supporting Table 14.2.2

The Mixed Procedure

### Parameter Code=TVEMEMAX

| | Nι | umber of Obse | rvations | |
|--------|----|---------------|----------|----|
| Number | of | Observations | Read | 90 |
| Number | of | Observations | Used | 90 |
| Number | of | Observations | Not Used | 0 |

# Iteration History Iteration Evaluations -2 Res Log Like Criterion 0 1 1214.80530325 1 1149.08926784 0.00000000

Convergence criteria met.

### Covariance Parameter Estimates

| Cov Parm | Estimate |
|----------------|----------|
| SUBJID (ARMCD) | 454187 |
| Residual | 130654 |

### Fit Statistics

| -2 Res Log Likelihood | 1149.1 |
|--------------------------|--------|
| AIC (Smaller is Better) | 1153.1 |
| AICC (Smaller is Better) | 1153.3 |
| BIC (Smaller is Better) | 1154.5 |

Program: A Biol.sas Created: 02APR2020 7:35 POSTLOCK 

The Mixed Procedure

Parameter Code=TVEMEMAX

Type 3 Tests of Fixed Effects
Num Den

| Nulli Dell | | | |
|------------|----|------|--------------|
| Effect | DF | DF F | Value Pr > F |
| TRTPN | 5 | 65 | 3.210.0119 |
| APERIOD | 5 | 65 | 1.990.0923 |
| ARMCD | 5 | 9 | 0.560.7305 |

### Coefficients for Oxy 30 vs Placebo Planned Planned

| | | Arm | Treatment | |
|-----------|---------|--------|-----------|------|
| Effect | APERIOD | Code | (N) | Row1 |
| Intercept | | | | |
| TRTPN | | | 1 | |
| TRTPN | | | 2 | |
| TRTPN | | | 3 | |
| TRTPN | | | 4 | 1 |
| TRTPN | | | 5 | |
| TRTPN | | | 6 | -1 |
| APERIOD | P1 | | | |
| APERIOD | P2 | | | |
| APERIOD | P3 | | | |
| APERIOD | P4 | | | |
| APERIOD | P5 | | | |
| APERIOD | P6 | | | |
| ARMCD | | ABCEDF | | |
| ARMCD | | BEAFCD | | |
| ARMCD | | CADBFE | | |
| ARMCD | | DCFAEB | | |

Program: A Biol.sas Created: 02APR2020 7:35 POSTLOCK 

The Mixed Procedure

### Parameter Code=TVEMEMAX

Coefficients for Oxy 30 vs Placebo

Planned Planned

 Arm
 Treatment

 Effect
 APERIOD Code
 (N)
 Row1

 ARMCD
 EFBDAC

 ARMCD
 FDECBA

Coefficients for Oxy 60 vs Placebo

Planned Planned

| | | Arm | Treatment | |
|-----------|---------|--------|-----------|------|
| Effect | APERIOD | Code | (N) | Row1 |
| Intercept | | | | |
| TRTPN | | | 1 | |
| TRTPN | | | 2 | |
| TRTPN | | | 3 | |
| TRTPN | | | 4 | |
| TRTPN | | | 5 | 1 |
| TRTPN | | | 6 | -1 |
| APERIOD | P1 | | | |
| APERIOD | P2 | | | |
| APERIOD | Р3 | | | |
| APERIOD | P4 | | | |
| APERIOD | P5 | | | |
| APERIOD | P6 | | | |
| ARMCD | | ABCEDF | | |
| ARMCD | | BEAFCD | | |
| ARMCD | | CADBFE | | |
| ARMCD | | DCFAEB | | |

Program: A Biol.sas Created: 02APR2020 7:35 POSTLOCK 

The Mixed Procedure

### Parameter Code=TVEMEMAX

Coefficients for Oxy 60 vs Placebo

Planned Planned

Arm Treatment
Effect APERIOD Code (N) Row1
ARMCD EFBDAC
ARMCD FDECBA

Coefficients for Bel 300 vs Oxy 30

Planned Planned

| | | Arm | Treatment | |
|---|---|---|---|---|
| Effect | APERIOD | Code | (N) | Row1 |
| Intercept | | | | |
| TRTPN | | | 1 | 1 |
| TRTPN | | | 2 | |
| TRTPN | | | 3 | |
| TRTPN | | | 4 | -1 |
| TRTPN | | | 5 | |
| TRTPN | | | 6 | |
| APERIOD | P1 | | | |
| APERIOD | P2 | | | |
| APERIOD | P3 | | | |
| APERIOD | P4 | | | |
| APERIOD | P5 | | | |
| APERIOD | P6 | | | |
| ARMCD | | ABCEDF | | |
| ARMCD | | BEAFCD | | |
| ARMCD | | CADBFE | | |
| ARMCD | | DCFAEB | | |
| | Intercept TRTPN TRTPN TRTPN TRTPN TRTPN TRTPN TRTPN APERIOD ARMCD ARMCD ARMCD ARMCD | Intercept TRTPN APERIOD P1 APERIOD P2 APERIOD P3 APERIOD P4 APERIOD P5 APERIOD P6 ARMCD ARMCD ARMCD ARMCD | Effect APERIOD Code Intercept TRTPN APERIOD P1 APERIOD P2 APERIOD P3 APERIOD P4 APERIOD P5 APERIOD P6 ARMCD ABCEDF ARMCD ABCEDF ARMCD CADBFE | ### Effect APERIOD Code (N) Intercept TRTPN |

### The Mixed Procedure

### Parameter Code=TVEMEMAX

Coefficients for Bel 300 vs Oxy 30

Planned Planned

 Arm
 Treatment

 Effect
 APERIOD Code
 (N)
 Row1

 ARMCD
 EFBDAC

 ARMCD
 FDECBA

Coefficients for Bel 300 vs Oxy 60 Planned Planned

| | | Arm | Treatment | |
|-----------|---------|--------|-----------|------|
| Effect | APERIOD | Code | (N) | Row1 |
| Intercept | | | | |
| TRTPN | | | 1 | 1 |
| TRTPN | | | 2 | |
| TRTPN | | | 3 | |
| TRTPN | | | 4 | |
| TRTPN | | | 5 | -1 |
| TRTPN | | | 6 | |
| APERIOD | P1 | | | |
| APERIOD | P2 | | | |
| APERIOD | P3 | | | |
| APERIOD | P4 | | | |
| APERIOD | P5 | | | |
| APERIOD | P6 | | | |
| ARMCD | | ABCEDF | | |
| ARMCD | | BEAFCD | | |
| ARMCD | | CADBFE | | |
| ARMCD | | DCFAEB | | |

The Mixed Procedure

### Parameter Code=TVEMEMAX

Coefficients for Bel 300 vs Oxy 60

Planned Planned

 Arm
 Treatment

 Effect
 APERIOD Code
 (N)
 Row1

 ARMCD
 EFBDAC

 ARMCD
 FDECBA

Coefficients for Bel 600 vs Oxy 30
Planned Planned

Arm Treatment

| APERIOD Co | de (N | ) Row1 |
|---|---|---|
| : | | |
| | 1 | |
| | 2 | 1 |
| | 3 | |
| | 4 | -1 |
| | 5 | |
| | 6 | |
| P1 | | |
| P2 | | |
| P3 | | |
| P4 | | |
| P5 | | |
| P6 | | |
| AE | CEDF | |
| BE | CAFCD | |
| CA | DBFE | |
| DC | FAEB | |
| | P1<br>P2<br>P3<br>P4<br>P5<br>P6 | 1<br>2<br>3<br>4<br>5<br>6<br>P1<br>P2<br>P3<br>P4<br>P5 |

Program: A Biol.sas Created: 02APR2020 7:35 POSTLOCK 

### The Mixed Procedure

### Parameter Code=TVEMEMAX

Coefficients for Bel 600 vs Oxy 30

Planned Planned

FDECBA

ARMCD

Coefficients for Bel 600 vs Oxy 60 Planned Planned

| | | Arm | Treatment | |
|-----------|---------|--------|-----------|------|
| Effect | APERIOD | Code | (N) | Row1 |
| Intercept | | | | |
| TRTPN | | | 1 | |
| TRTPN | | | 2 | 1 |
| TRTPN | | | 3 | |
| TRTPN | | | 4 | |
| TRTPN | | | 5 | -1 |
| TRTPN | | | 6 | |
| APERIOD | P1 | | | |
| APERIOD | P2 | | | |
| APERIOD | P3 | | | |
| APERIOD | P4 | | | |
| APERIOD | P5 | | | |
| APERIOD | P6 | | | |
| ARMCD | | ABCEDF | | |
| ARMCD | | BEAFCD | | |
| ARMCD | | CADBFE | | |
| ARMCD | | DCFAEB | | |

Program: A Biol.sas Created: 02APR2020 7:35 POSTLOCK 

The Mixed Procedure

### Parameter Code=TVEMEMAX

Coefficients for Bel 600 vs Oxy 60

Planned Planned

| Arm | Treatment | Effect | APERIOD Code | (N) | Row1 | ARMCD | EFBDAC |

FDECBA

ARMCD

Coefficients for Bel 900 vs Oxy 30

Planned Planned

| | | Arm | Treatment | |
|-----------|---------|--------|-----------|------|
| Effect | APERIOD | Code | (N) | Row1 |
| Intercept | | | | |
| TRTPN | | | 1 | |
| TRTPN | | | 2 | |
| TRTPN | | | 3 | 1 |
| TRTPN | | | 4 | -1 |
| TRTPN | | | 5 | |
| TRTPN | | | 6 | |
| APERIOD | P1 | | | |
| APERIOD | P2 | | | |
| APERIOD | Р3 | | | |
| APERIOD | P4 | | | |
| APERIOD | P5 | | | |
| APERIOD | P6 | | | |
| ARMCD | | ABCEDF | | |
| ARMCD | | BEAFCD | | |
| ARMCD | | CADBFE | | |
| ARMCD | | DCFAEB | | |

Program: A Biol.sas Created: 02APR2020 7:35 POSTLOCK 

### The Mixed Procedure

### Parameter Code=TVEMEMAX

Coefficients for Bel 900 vs Oxy 30

Planned Planned

Arm Treatment Effect APERIOD Code (N) Row1

ARMCD EFBDAC ARMCD FDECBA

Coefficients for Bel 900 vs Oxy 60

Planned Planned
Arm Treatment

Effect APERIOD Code (N) Row1 Intercept 1 TRTPN TRTPN 2 3 TRTPN 1 TRTPN 5 -1 TRTPN TRTPN APERIOD P1 APERIOD P2 APERIOD P3 APERIOD P4 APERIOD P5 APERIOD P6 ARMCD ABCEDF ARMCD BEAFCD ARMCD CADBFE ARMCD DCFAEB

Program: A Biol.sas Created: 02APR2020 7:35 POSTLOCK 

### The Mixed Procedure

### Parameter Code=TVEMEMAX

Coefficients for Bel 900 vs Oxy 60

Planned Planned

 Arm
 Treatment

 Effect
 APERIOD Code
 (N)
 Row1

 ARMCD
 EFBDAC

 ARMCD
 FDECBA

Coefficients for Bel 300 vs Placebo
Planned Planned

Arm Treatment Effect APERIOD Code (N) Row1 Intercept 1 TRTPN 1 TRTPN TRTPN 3 TRTPN TRTPN TRTPN -1 APERIOD P1 APERIOD P2 APERIOD P3 APERIOD P4 APERIOD P5 APERIOD P6 ARMCD ABCEDF ARMCD BEAFCD ARMCD CADBFE ARMCD DCFAEB

Program: A Biol.sas Created: 02APR2020 7:35 POSTLOCK 

### The Mixed Procedure

### Parameter Code=TVEMEMAX

Coefficients for Bel 300 vs Placebo

Planned Planned

Arm Treatment

| Effect | APERIOD Code | (N) | Row1 |
|--------|--------------|-----|------|
| ARMCD | EFBDAC | | |
| ARMCD | FDECBA | | |

Coefficients for Bel 600 vs Placebo

Planned Planned

Arm Treatment Effect APERIOD Code (N) Row1 Intercept TRTPN 1 TRTPN 1 TRTPN 3 TRTPN TRTPN TRTPN -1 APERIOD P1 APERIOD P2 APERIOD P3 APERIOD P4 APERIOD P5 APERIOD P6 ARMCD ABCEDF ARMCD BEAFCD ARMCD CADBFE ARMCD DCFAEB

The Mixed Procedure

### Parameter Code=TVEMEMAX

Coefficients for Bel 600 vs Placebo

Planned Planned

 Arm
 Treatment

 Effect
 APERIOD Code
 (N)
 Row1

 ARMCD
 EFBDAC

 ARMCD
 FDECBA

Coefficients for Bel 900 vs Placebo
Planned Planned

| | | Arm | Treatment | |
|-----------|--------|--------|-----------|------|
| Effect | APERIO | ) Code | (N) | Row1 |
| Intercept | | | | |
| TRTPN | | | 1 | |
| TRTPN | | | 2 | |
| TRTPN | | | 3 | 1 |
| TRTPN | | | 4 | |
| TRTPN | | | 5 | |
| TRTPN | | | 6 | -1 |
| APERIOD | P1 | | | |
| APERIOD | P2 | | | |
| APERIOD | P3 | | | |
| APERIOD | P4 | | | |
| APERIOD | P5 | | | |
| APERIOD | P6 | | | |
| ARMCD | | ABCEDF | | |
| ARMCD | | BEAFCD | | |
| ARMCD | | CADBFE | | |
| ARMCD | | DCFAEB | | |

## Appendix 16.1.9.2.1 Statistical Methods and Analysis Output Supporting Table 14.2.2 Supporting Table 14.2.2

### The Mixed Procedure

### Parameter Code=TVEMEMAX

Coefficients for Bel 900 vs Placebo

Planned Planned

Arm Treatment

Effect APERIOD Code (N) Row1
ARMCD EFBDAC
ARMCD FDECBA

#### Estimates

### Standard

| Label | Estimate | Error DF t | Value E | r > t | Alpha | Lower Upper |
|---|---|---|---|---|---|---|
| Oxy 30 vs Placebo | 64.4353 | 132.5865 | 0.49 | 0.6286 | 0.05 | -200.34329.21 |
| Oxy 60 vs Placebo | -258.67 | 132.5865 | -1.95 | 0.0554 | 0.05 | -523.456.1076 |
| Bel 300 vs Oxy 30 | 135.61 | 132.5865 | 1.02 | 0.3102 | 0.05 | -129.17400.39 |
| Bel 300 vs Oxy 60 | 458.72 | 132.5865 | 3.46 | 0.0010 | 0.05 | 193.94723.50 |
| Bel 600 vs Oxy 30 | -12.2582 | 132.2865 | -0.09 | 0.9265 | 0.05 | -276.44251.93 |
| Bel 600 vs Oxy 60 | 310.85 | 132.5865 | 2.34 | 0.0221 | 0.05 | 46.0695575.63 |
| Bel 900 vs Oxy 30 | 128.89 | 132.5865 | 0.97 | 0.3346 | 0.05 | -135.89393.67 |
| Bel 900 vs Oxy 60 | 451.99 | 132.2865 | 3.42 | 0.0011 | 0.05 | 187.81716.18 |
| Bel 300 vs Placebo | 200.05 | 132.2865 | 1.51 | 0.1353 | 0.05 | -64.1373464.23 |
| Bel 600 vs Placebo | 52.1771 | 132.5865 | 0.39 | 0.6952 | 0.05 | -212.60316.96 |
| Bel 900 vs Placebo | 193.32 | 132.5865 | 1.46 | 0.1496 | 0.05 | -71.4549458.10 |

Program: A Biol.sas Created: 02APR2020 7:35 POSTLOCK 

## Appendix 16.1.9.2.1 Statistical Methods and Analysis Output Supporting Table 14.2.2 Supporting Table 14.2.2

### The Mixed Procedure

### Parameter Code=TVEMEMAX

### Least Squares Means

| | Planned | | _ | | | | | |
|---|---|---|---|---|---|---|---|---|
| | Treatment | | Standard | | | | | |
| Effect | (N) | Estimate | Error DF t | Value | Pr > t | Alpha | Lower | Upper |
| TRTPN | 1 | 1959.11 | 200.9265 | 9.75 | <.0001 | 0.05 | 1557.84 | 2360.38 |
| TRTPN | 2 | 1811.24 | 200.9265 | 9.01 | <.0001 | 0.05 | 1409.97 | 2212.51 |
| TRTPN | 3 | 1952.39 | 200.9265 | 9.72 | <.0001 | 0.05 | 1551.12 | 2353.66 |
| TRTPN | 4 | 1823.50 | 200.9265 | 9.08 | <.0001 | 0.05 | 1422.23 | 2224.77 |
| TRTPN | 5 | 1500.39 | 200.9265 | 7.47 | <.0001 | 0.05 | 1099.12 | 1901.66 |
| TRTPN | 6 | 1759.06 | 200.9265 | 8.75 | <.0001 | 0.05 | 1357.79 | 2160.34 |

### Differences of Least Squares Means

| | Planned | Planned | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| | Treatment | Treatment | | Standard | | | | | |
| Effect | (N) | (N) | Estimate | Error DF t | Value I | Pr > t <i>i</i> | Alpha | Lower | Upper |
| TRTPN | 1 | 2 | 147.87 | 132.5865 | 1.12 | 0.2688 | 0.05 | -116.91 | 412.65 |
| TRTPN | 1 | 3 | 6.7232 | 132.5865 | 0.05 | 0.9597 | 0.05 | -258.05 | 271.50 |
| TRTPN | 1 | 4 | 135.61 | 132.5865 | 1.02 | 0.3102 | 0.05 | -129.17 | 400.39 |
| TRTPN | 1 | 5 | 458.72 | 132.5865 | 3.46 | 0.0010 | 0.05 | 193.94 | 723.50 |
| TRTPN | 1 | 6 | 200.05 | 132.2865 | 1.51 | 0.1353 | 0.05 | -64.1373 | 464.23 |
| TRTPN | 2 | 3 | -141.15 | 132.5865 | -1.06 | 0.2910 | 0.05 | -405.92 | 123.63 |
| TRTPN | 2 | 4 | -12.2582 | 132.2865 | -0.09 | 0.9265 | 0.05 | -276.44 | 251.93 |
| TRTPN | 2 | 5 | 310.85 | 132.5865 | 2.34 | 0.0221 | 0.05 | 46.0695 | 575.63 |
| TRTPN | 2 | 6 | 52.1771 | 132.5865 | 0.39 | 0.6952 | 0.05 | -212.60 | 316.96 |
| TRTPN | 3 | 4 | 128.89 | 132.5865 | 0.97 | 0.3346 | 0.05 | -135.89 | 393.67 |
| TRTPN | 3 | 5 | 451.99 | 132.2865 | 3.42 | 0.0011 | 0.05 | 187.81 | 716.18 |
| TRTPN | 3 | 6 | 193.32 | 132.5865 | 1.46 | 0.1496 | 0.05 | -71.4549 | 458.10 |
| TRTPN | 4 | 5 | 323.11 | 132.5865 | 2.44 | 0.0176 | 0.05 | 58.3277 | 587.88 |

Program: A Biol.sas Created: 02APR2020 7:35 POSTLOCK 

## Appendix 16.1.9.2.1 Statistical Methods and Analysis Output Supporting Table 14.2.2 Supporting Table 14.2.2

### The Mixed Procedure

### Parameter Code=TVEMEMAX

### Differences of Least Squares Means

| | Planned | Planned | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| | Treatment | Treatment | | Standard | | | | | |
| Effect | (N) | (N) | Estimate | Error DF t | Value Pr | > t 2 | Alpha | Lower | Upper |
| TRTPN | 4 | 6 | 64.4353 | 132.5865 | 0.49 | 0.6286 | 0.05 | -200.34 | 329.21 |
| TRTPN | 5 | 6 | -258.67 | 132.5865 | -1.95 | 0.0554 | 0.05 | -523.45 | 6.1076 |

Program: A\_Biol.sas Created: 02APR2020 7:35 POSTLOCK 

### Appendix 16.1.9.2.2 Statistical Methods and Analysis Output Supporting Table 14.2.3 Supporting Table 14.2.3

### The Mixed Procedure

### Parameter Code=ETCOEMAX

### Model Information

| Data Set | WORK.ADXV |
|---------------------------|---------------------|
| Dependent Variable | AVAL |
| Covariance Structure | Variance Components |
| Estimation Method | REML |
| Residual Variance Method | Profile |
| Fixed Effects SE Method | Model-Based |
| Degrees of Freedom Method | Containment |

### Class Level Information

| Class | LevelsValues |
|---|---|
| SUBJID | 161001 1002 1003 1004 1005 1006 1007 1008 1010 1012 1013 1014 1015 1016 1017 1018 |
| TRTPN | 61 2 3 4 5 6 |
| APERIOD | O 6P1 P2 P3 P4 P5 P6 |
| ARMCD | 6ABCEDF BEAFCD CADBFE DCFAEB EFBDAC FDECBA |

| Dir | mensions | |
|-------------|------------|----|
| Covariance | Parameters | 2 |
| Columns in | X | 19 |
| Columns in | Z | 16 |
| Subjects | | 1 |
| Max Obs per | Subject | 93 |

Program: A Bio2.sas Created: 02APR2020 7:35 POSTLOCK 

### Appendix 16.1.9.2.2 Statistical Methods and Analysis Output Supporting Table 14.2.3 Supporting Table 14.2.3

The Mixed Procedure

### Parameter Code=ETCOEMAX

| | Nι | umber of Obse | rvations | |
|--------|----|---------------|----------|----|
| Number | of | Observations | Read | 93 |
| Number | of | Observations | Used | 93 |
| Number | οf | Observations | Not Used | 0 |

# Iteration History Iteration Evaluations -2 Res Log Like Criterion 0 1 445.33349796 1 2 425.589813360.00000000

Convergence criteria met.

### Covariance Parameter Estimates

| Cov Parm | Estimate |
|----------------|----------|
| SUBJID (ARMCD) | 5.7636 |
| Residual | 6.9739 |

| Fit Statistics | |
|--------------------------|-------|
| -2 Res Log Likelihood | 425.6 |
| AIC (Smaller is Better) | 429.6 |
| AICC (Smaller is Better) | 429.8 |
| BIC (Smaller is Better) | 431.1 |

Program: A Bio2.sas Created: 02APR2020 7:35 POSTLOCK 

The Mixed Procedure

Parameter Code=ETCOEMAX

Type 3 Tests of Fixed Effects

| 1 | Num I | Den | |
|---------|-------|------|--------------|
| Effect | DF | DF F | Value Pr > F |
| TRTPN | 5 | 67 | 3.460.0077 |
| APERIOD | 5 | 67 | 0.490.7812 |
| ARMCD | 5 | 10 | 0.760.5997 |

### Coefficients for Oxy 30 vs Placebo Planned Planned

| | | Arm | Treatment | |
|-----------|---------|--------|-----------|------|
| Effect | APERIOD | Code | (N) | Row1 |
| Intercept | | | | |
| TRTPN | | | 1 | |
| TRTPN | | | 2 | |
| TRTPN | | | 3 | |
| TRTPN | | | 4 | 1 |
| TRTPN | | | 5 | |
| TRTPN | | | 6 | -1 |
| APERIOD | P1 | | | |
| APERIOD | P2 | | | |
| APERIOD | Р3 | | | |
| APERIOD | P4 | | | |
| APERIOD | P5 | | | |
| APERIOD | P6 | | | |
| ARMCD | | ABCEDF | | |
| ARMCD | | BEAFCD | | |
| ARMCD | | CADBFE | | |
| ARMCD | | DCFAEB | | |

Program: A Bio2.sas Created: 02APR2020 7:35 POSTLOCK 

### The Mixed Procedure

### Parameter Code=ETCOEMAX

### Coefficients for Oxy 30 vs Placebo

Planned Planned

Arm Treatment
Effect APERIOD Code (N) Row1
ARMCD EFBDAC
ARMCD FDECBA

### Coefficients for Oxy 60 vs Placebo

Planned Planned Arm Treatment

| | | ATIII | Treatment | |
|-----------|---------|--------|-----------|------|
| Effect | APERIOD | Code | (N) | Row1 |
| Intercept | | | | |
| TRTPN | | | 1 | |
| TRTPN | | | 2 | |
| TRTPN | | | 3 | |
| TRTPN | | | 4 | |
| TRTPN | | | 5 | 1 |
| TRTPN | | | 6 | -1 |
| APERIOD | P1 | | | |
| APERIOD | P2 | | | |
| APERIOD | P3 | | | |
| APERIOD | P4 | | | |
| APERIOD | P5 | | | |
| APERIOD | P6 | | | |
| ARMCD | | ABCEDF | | |
| ARMCD | | BEAFCD | | |
| ARMCD | | CADBFE | | |
| ARMCD | | DCFAEB | | |
The Mixed Procedure

#### Parameter Code=ETCOEMAX

Coefficients for Oxy 60 vs Placebo

Planned Planned

 Arm
 Treatment

 Effect
 APERIOD Code
 (N)
 Row1

 ARMCD
 EFBDAC

 ARMCD
 FDECBA

Coefficients for Bel 300 vs Oxy 30

Planned Planned
Arm Treatment

| | | Arm | Treatment | |
|-----------|---------|--------|-----------|------|
| Effect | APERIOD | Code | (N) | Row1 |
| Intercept | | | | |
| TRTPN | | | 1 | 1 |
| TRTPN | | | 2 | |
| TRTPN | | | 3 | |
| TRTPN | | | 4 | -1 |
| TRTPN | | | 5 | |
| TRTPN | | | 6 | |
| APERIOD | P1 | | | |
| APERIOD | P2 | | | |
| APERIOD | P3 | | | |
| APERIOD | P4 | | | |
| APERIOD | P5 | | | |
| APERIOD | P6 | | | |
| ARMCD | | ABCEDF | | |
| ARMCD | | BEAFCD | | |
| ARMCD | | CADBFE | | |
| ARMCD | | DCFAEB | | |

Program: A\_Bio2.sas Created: 02APR2020 7:35 POSTLOCK 

The Mixed Procedure

#### Parameter Code=ETCOEMAX

Coefficients for Bel 300 vs Oxy 30

Planned Planned

 $\begin{array}{c|cccc} & & Arm & Treatment \\ \hline Effect & APERIOD\,Code & (N) & Row1 \\ \hline ARMCD & EFBDAC \\ \end{array}$ 

ARMCD FDECBA

Coefficients for Bel 300 vs Oxy 60 Planned Planned

Arm Treatment

| | | Arm | Treatment | |
|-----------|---------|--------|-----------|------|
| Effect | APERIOD | Code | (N) | Row1 |
| Intercept | | | | |
| TRTPN | | | 1 | 1 |
| TRTPN | | | 2 | |
| TRTPN | | | 3 | |
| TRTPN | | | 4 | |
| TRTPN | | | 5 | -1 |
| TRTPN | | | 6 | |
| APERIOD | P1 | | | |
| APERIOD | P2 | | | |
| APERIOD | P3 | | | |
| APERIOD | P4 | | | |
| APERIOD | P5 | | | |
| APERIOD | P6 | | | |
| ARMCD | | ABCEDF | | |
| ARMCD | | BEAFCD | | |
| ARMCD | | CADBFE | | |
| ARMCD | | DCFAEB | | |

The Mixed Procedure

#### Parameter Code=ETCOEMAX

Coefficients for Bel 300 vs Oxy 60

Planned Planned

 Arm
 Treatment

 Effect
 APERIOD Code
 (N)
 Row1

 ARMCD
 EFBDAC

ARMCD EFBDAC ARMCD FDECBA

Coefficients for Bel 600 vs Oxy 30

Planned Planned

| Effect | | | | |
|---|---|---|---|---|
| TITECL | APERIOD | Code | (N) | Row1 |
| Intercept | | | | |
| TRTPN | | | 1 | |
| TRTPN | | | 2 | 1 |
| TRTPN | | | 3 | |
| TRTPN | | | 4 | -1 |
| TRTPN | | | 5 | |
| TRTPN | | | 6 | |
| APERIOD | P1 | | | |
| APERIOD | P2 | | | |
| APERIOD | P3 | | | |
| APERIOD | P4 | | | |
| APERIOD | P5 | | | |
| APERIOD | P6 | | | |
| ARMCD | | ABCEDF | | |
| ARMCD | | BEAFCD | | |
| ARMCD | | CADBFE | | |
| ARMCD | | DCFAEB | | |
| | Intercept TRTPN TRTPN TRTPN TRTPN TRTPN TRTPN TRTPN APERIOD APERIOD APERIOD APERIOD APERIOD APERIOD APERIOD ARMCD ARMCD ARMCD ARMCD | Intercept TRTPN APERIOD P1 APERIOD P2 APERIOD P3 APERIOD P4 APERIOD P5 APERIOD P6 ARMCD ARMCD ARMCD | Intercept TRTPN APERIOD P1 APERIOD P2 APERIOD P3 APERIOD P4 APERIOD P5 APERIOD P6 ARMCD ABCEDF ARMCD ABCEDF ARMCD CADBFE | Intercept TRTPN 1 TRTPN 2 TRTPN 3 TRTPN 4 TRTPN 5 TRTPN 6 APERIOD P1 APERIOD P2 APERIOD P3 APERIOD P4 APERIOD P5 APERIOD P5 APERIOD P6 ARMCD ABCEDF ARMCD BEAFCD ARMCD CADBFE |

Program: A Bio2.sas Created: 02APR2020 7:35 POSTLOCK 

The Mixed Procedure

#### Parameter Code=ETCOEMAX

Coefficients for Bel 600 vs Oxy 30

Planned Planned

 Arm
 Treatment

 Effect
 APERIOD Code
 (N)
 Row1

 ARMCD
 EFBDAC

ARMCD EFBDAC ARMCD FDECBA

Coefficients for Bel 600 vs Oxy 60

Planned Planned Arm Treatment

Effect APERIOD Code (N) Row1 Intercept TRTPN 1 TRTPN 1 TRTPN 3 TRTPN -1 TRTPN TRTPN APERIOD P1 APERIOD P2 APERIOD P3 APERIOD P4 APERIOD P5 APERIOD P6 ARMCD ABCEDF ARMCD BEAFCD ARMCD CADBFE ARMCD DCFAEB

Program: A\_Bio2.sas Created: 02APR2020 7:35 POSTLOCK


The Mixed Procedure

#### Parameter Code=ETCOEMAX

Coefficients for Bel 600 vs Oxy 60

Planned Planned

 Arm
 Treatment

 Effect
 APERIOD Code
 (N)
 Row1

 ARMCD
 EFBDAC

 ARMCD
 FDECBA

Coefficients for Bel 900 vs Oxy 30
Planned Planned

Arm Treatment

| | | 2 1 L 111 | I I Ca chich | • |
|-----------|--------|-----------|--------------|------|
| Effect | APERIO | ) Code | (N) | Row1 |
| Intercept | ; | | | |
| TRTPN | | | 1 | |
| TRTPN | | | 2 | |
| TRTPN | | | 3 | 1 |
| TRTPN | | | 4 | -1 |
| TRTPN | | | 5 | |
| TRTPN | | | 6 | |
| APERIOD | P1 | | | |
| APERIOD | P2 | | | |
| APERIOD | Р3 | | | |
| APERIOD | P4 | | | |
| APERIOD | P5 | | | |
| APERIOD | P6 | | | |
| ARMCD | | ABCEDF | | |
| ARMCD | | BEAFCD | | |
| ARMCD | | CADBFE | | |
| ARMCD | | DCFAEB | | |

Program: A\_Bio2.sas Created: 02APR2020 7:35 POSTLOCK 

The Mixed Procedure

#### Parameter Code=ETCOEMAX

Coefficients for Bel 900 vs Oxy 30

Planned Planned

 Arm
 Treatment

 Effect
 APERIOD Code
 (N)
 Row1

 ARMCD
 EFBDAC

 ARMCD
 FDECBA

Coefficients for Bel 900 vs 0xy 60
Planned Planned

| | | Arm | Treatment | |
|-----------|---------|--------|-----------|------|
| Effect | APERIOD | Code | (N) | Row1 |
| Intercept | | | | |
| TRTPN | | | 1 | |
| TRTPN | | | 2 | |
| TRTPN | | | 3 | 1 |
| TRTPN | | | 4 | |
| TRTPN | | | 5 | -1 |
| TRTPN | | | 6 | |
| APERIOD | P1 | | | |
| APERIOD | P2 | | | |
| APERIOD | P3 | | | |
| APERIOD | P4 | | | |
| APERIOD | P5 | | | |
| APERIOD | P6 | | | |
| ARMCD | | ABCEDF | | |
| ARMCD | | BEAFCD | | |
| ARMCD | | CADBFE | | |
| ARMCD | | DCFAEB | | |

Program: A Bio2.sas Created: 02APR2020 7:35 POSTLOCK 

#### The Mixed Procedure

#### Parameter Code=ETCOEMAX

Coefficients for Bel 900 vs Oxy 60

Planned Planned

 Arm
 Treatment

 Effect
 APERIOD Code
 (N)
 Row1

 ARMCD
 EFBDAC

 ARMCD
 FDECBA

Coefficients for Bel 300 vs Placebo
Planned Planned

| | | Arm | Treatment | |
|-----------|--------|--------|-----------|------|
| Effect | APERIO | ) Code | (N) | Row1 |
| Intercept | ; | | | |
| TRTPN | | | 1 | 1 |
| TRTPN | | | 2 | |
| TRTPN | | | 3 | |
| TRTPN | | | 4 | |
| TRTPN | | | 5 | |
| TRTPN | | | 6 | -1 |
| APERIOD | P1 | | | |
| APERIOD | P2 | | | |
| APERIOD | Р3 | | | |
| APERIOD | P4 | | | |
| APERIOD | P5 | | | |
| APERIOD | P6 | | | |
| ARMCD | | ABCEDF | | |
| ARMCD | | BEAFCD | | |
| ARMCD | | CADBFE | | |
| ARMCD | | DCFAEB | | |

#### The Mixed Procedure

#### Parameter Code=ETCOEMAX

# Coefficients for Bel 300 vs Placebo

Planned Planned

 Arm
 Treatment

 Effect
 APERIOD Code
 (N)
 Row1

 ARMCD
 EFBDAC

ARMCD FDECBA

# Coefficients for Bel 600 vs Placebo

Planned Planned

| | | Arm | Treatment | |
|-----------|--------|--------|-----------|------|
| Effect | APERIO | ) Code | (N) | Row1 |
| Intercept | ; | | | |
| TRTPN | | | 1 | |
| TRTPN | | | 2 | 1 |
| TRTPN | | | 3 | |
| TRTPN | | | 4 | |
| TRTPN | | | 5 | |
| TRTPN | | | 6 | -1 |
| APERIOD | P1 | | | |
| APERIOD | P2 | | | |
| APERIOD | Р3 | | | |
| APERIOD | P4 | | | |
| APERIOD | P5 | | | |
| APERIOD | P6 | | | |
| ARMCD | | ABCEDF | | |
| ARMCD | | BEAFCD | | |
| ARMCD | | CADBFE | | |
| ARMCD | | DCFAEB | | |

The Mixed Procedure

#### Parameter Code=ETCOEMAX

Coefficients for Bel 600 vs Placebo

Planned Planned

Arm Treatment
Effect APERIOD Code (N) Row1
ARMCD EFBDAC
ARMCD FDECBA

Coefficients for Bel 900 vs Placebo Planned Planned

| | | Arm | Treatment | |
|-----------|---------|--------|-----------|------|
| Effect | APERIOD | Code | (N) | Row1 |
| Intercept | | | | |
| TRTPN | | | 1 | |
| TRTPN | | | 2 | |
| TRTPN | | | 3 | 1 |
| TRTPN | | | 4 | |
| TRTPN | | | 5 | |
| TRTPN | | | 6 | -1 |
| APERIOD | P1 | | | |
| APERIOD | P2 | | | |
| APERIOD | P3 | | | |
| APERIOD | P4 | | | |
| APERIOD | P5 | | | |
| APERIOD | P6 | | | |
| ARMCD | | ABCEDF | | |
| ARMCD | | BEAFCD | | |
| ARMCD | | CADBFE | | |
| ARMCD | | DCFAEB | | |

# Appendix 16.1.9.2.2 Statistical Methods and Analysis Output Supporting Table 14.2.3 Supporting Table 14.2.3

#### The Mixed Procedure

#### Parameter Code=ETCOEMAX

Coefficients for Bel 900 vs Placebo

Planned Planned

Arm Treatment

Effect APERIOD Code (N) Row1
ARMCD EFBDAC
ARMCD FDECBA

#### Estimates

#### Standard

| Label | Estimate | Error DF t | Value E | ?r > t . | Alpha | Lower | Upper |
|---|---|---|---|---|---|---|---|
| Oxy 30 vs Placebo | 1.3593 | 0.955967 | 1.42 | 0.1597 | 0.05- | 0.5486 | 3.2672 |
| Oxy 60 vs Placebo | 2.7012 | 0.937567 | 2.88 | 0.0053 | 0.05 | 0.8298 | 4.5725 |
| Bel 300 vs Oxy 30 | -2.3356 | 0.968667 | -2.41 | 0.0186 | 0.05- | 4.2688 | -0.4024 |
| Bel 300 vs Oxy 60 | -3.6775 | 0.955867 | -3.85 | 0.0003 | 0.05- | 5.5853 | -1.7696 |
| Bel 600 vs Oxy 30 | -0.2433 | 0.956367 | -0.25 | 0.7999 | 0.05- | 2.1521 | 1.6655 |
| Bel 600 vs Oxy 60 | -1.5852 | 0.937567 | -1.69 | 0.0955 | 0.05- | 3.4564 | 0.2860 |
| Bel 900 vs Oxy 30 | -0.3133 | 0.968567 | -0.32 | 0.7473 | 0.05- | 2.2464 | 1.6198 |
| Bel 900 vs Oxy 60 | -1.6552 | 0.956367 | -1.73 | 0.0881 | 0.05- | 3.5639 | 0.2535 |
| Bel 300 vs Placebo | -0.9763 | 0.955367 | -1.02 | 0.3105 | 0.05- | 2.8832 | 0.9305 |
| Bel 600 vs Placebo | 1.1159 | 0.935667 | 1.19 | 0.2372 | 0.05- | 0.7515 | 2.9834 |
| Bel 900 vs Placebo | 1.0460 | 0.955967 | 1.09 | 0.2778 | 0.05- | 0.8620 | 2.9539 |

Program: A Bio2.sas Created: 02APR2020 7:35 POSTLOCK 

# Appendix 16.1.9.2.2 Statistical Methods and Analysis Output Supporting Table 14.2.3Supporting Table 14.2.3

The Mixed Procedure

#### Parameter Code=ETCOEMAX

## Least Squares Means

| | Planned | | _ | | | | | |
|---|---|---|---|---|---|---|---|---|
| | Treatment | | Standard | | | | | |
| Effect | (N) | Estimate | Error DF t | Value | Pr > t | Alpha | Lower | Upper |
| TRTPN | 1 | 40.7846 | 0.921867 | 44.24 | <.0001 | 0.1 | 39.2471 | 42.3220 |
| TRTPN | 2 | 42.8768 | 0.902567 | 47.51 | <.0001 | 0.1 | 41.3715 | 44.3822 |
| TRTPN | 3 | 42.8069 | 0.922367 | 46.41 | <.0001 | 0.1 | 41.2686 | 44.3451 |
| TRTPN | 4 | 43.1202 | 0.922367 | 46.75 | <.0001 | 0.1 | 41.5819 | 44.6584 |
| TRTPN | 5 | 44.4621 | 0.902567 | 49.26 | <.0001 | 0.1 | 42.9567 | 45.9674 |
| TRTPN | 6 | 41.7609 | 0.902567 | 46.27 | <.0001 | 0.1 | 40.2556 | 43.2662 |

## Differences of Least Squares Means

| | Planned | Planned | | | | | | |
|---|---|---|---|---|---|---|---|---|
| | Treatment | Treatment | 5 | Standard | | | | |
| Effect | (N) | (N) | Estimate | Error DF t | Value Pr | c > t | Alpha Lower | Upper |
| TRTPN | 1 | 2 | -2.0923 | 0.957867 | -2.18 | 0.0324 | 0.1-3.6898 | -0.4948 |
| TRTPN | 1 | 3 | -2.0223 | 0.968467 | -2.09 | 0.0406 | 0.1-3.6375 | -0.4071 |
| TRTPN | 1 | 4 | -2.3356 | 0.968667 | -2.41 | 0.0186 | 0.1-3.9511 | -0.7201 |
| TRTPN | 1 | 5 | -3.6775 | 0.955867 | -3.85 | 0.0003 | 0.1-5.2717 | -2.0832 |
| TRTPN | 1 | 6 | -0.9763 | 0.955367 | -1.02 | 0.3105 | 0.1-2.5697 | 0.6171 |
| TRTPN | 2 | 3 | 0.06998 | 0.956467 | 0.07 | 0.9419 | 0.1-1.5253 | 1.6652 |
| TRTPN | 2 | 4 | -0.2433 | 0.956367 | -0.25 | 0.7999 | 0.1-1.8384 | 1.3517 |
| TRTPN | 2 | 5 | -1.5852 | 0.937567 | -1.69 | 0.0955 | 0.1-3.1488 | -0.02161 |
| TRTPN | 2 | 6 | 1.1159 | 0.935667 | 1.19 | 0.2372 | 0.1-0.4445 | 2.6764 |
| TRTPN | 3 | 4 | -0.3133 | 0.968567 | -0.32 | 0.7473 | 0.1-1.9286 | 1.3020 |
| TRTPN | 3 | 5 | -1.6552 | 0.956367 | -1.73 | 0.0881 | 0.1-3.2502 | -0.06020 |
| TRTPN | 3 | 6 | 1.0460 | 0.955967 | 1.09 | 0.2778 | 0.1-0.5483 | 2.6403 |

 Program: A Bio2.sas Created: 02APR2020 7:35 POSTLOCK

TRTPN 4 5 -1.3419 0.956367 -1.40 0.1652 0.1-2.9369 0.2531

Appendix 16.1.9.2.2
Statistical Methods and Analysis Output Supporting Table 14.2.3
Supporting Table 14.2.3

#### The Mixed Procedure

#### Parameter Code=ETCOEMAX

# Differences of Least Squares Means

| | Planned | Planned | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| | Treatment | Treatment | S | tandard | | | | | |
| Effect | (N) | (N) | Estimate | Error DF t | Value Pr | : > t | Alpha | Lower | Upper |
| TRTPN | 4 | 6 | 1.3593 | 0.955967 | 1.42 | 0.1597 | 0.1 | -0.2350 | 2.9536 |
| TRTPN | 5 | 6 | 2.7012 | 0.937567 | 2.88 | 0.0053 | 0.1 | 1.1374 | 4.2649 |

Program: A\_Bio2.sas Created: 02APR2020 7:35 POSTLOCK 

# Appendix 16.1.9.2.2 Statistical Methods and Analysis Output Supporting Table 14.2.3 Supporting Table 14.2.3

#### The Mixed Procedure

#### Parameter Code=MVMIEMAX

#### Model Information

| Data Set | WORK.ADXV |
|---------------------------|---------------------|
| Dependent Variable | AVAL |
| Covariance Structure | Variance Components |
| Estimation Method | REML |
| Residual Variance Method | Profile |
| Fixed Effects SE Method | Model-Based |
| Degrees of Freedom Method | Containment |

#### Class Level Information

| Class | LevelsValues |
|---|---|
| SUBJID | 161001 1002 1003 1004 1005 1006 1007 1008 1010 1012 1013 1014 1015 1016 1017 1018 |
| TRTPN | 61 2 3 4 5 6 |
| APERIOD | O 6P1 P2 P3 P4 P5 P6 |
| ARMCD | 6ABCEDF BEAFCD CADBFE DCFAEB EFBDAC FDECBA |

| Dimensions | |
|-----------------------|----|
| Covariance Parameters | 2 |
| Columns in X | 19 |
| Columns in Z | 16 |
| Subjects | 1 |
| Max Obs per Subject | 93 |

Program: A Bio2.sas Created: 02APR2020 7:35 POSTLOCK 

# Appendix 16.1.9.2.2 Statistical Methods and Analysis Output Supporting Table 14.2.3 Supporting Table 14.2.3

The Mixed Procedure

#### Parameter Code=MVMIEMAX

| | Nι | umber of Obse | rvations | |
|--------|----|---------------|----------|----|
| Number | of | Observations | Read | 93 |
| Number | of | Observations | Used | 93 |
| Number | of | Observations | Not Used | 0 |

# Iteration History Iteration Evaluations -2 Res Log Like Criterion 0 1 1601.99363318 1 2 1591.964904820.00000000

Convergence criteria met.

# Covariance Parameter Estimates Cov Parm Estimate

| Cov Parm | Estimate |
|----------------|----------|
| SUBJID (ARMCD) | 12903876 |
| Residual | 28030184 |

| Fit Statistics |
|----------------|
|----------------|

| -2 Res Log Likelihood | 1592.0 |
|--------------------------|--------|
| AIC (Smaller is Better) | 1596.0 |
| AICC (Smaller is Better) | 1596.1 |
| BIC (Smaller is Better) | 1597.5 |

Program: A Bio2.sas Created: 02APR2020 7:35 POSTLOCK 

The Mixed Procedure

#### Parameter Code=MVMIEMAX

Type 3 Tests of Fixed Effects

| | Num I | Den | |
|---------|-------|------|--------------|
| Effect | DF | DF F | Value Pr > F |
| TRTPN | 5 | 67 | 3.060.0152 |
| APERIOD | 5 | 67 | 2.170.0677 |
| ARMCD | 5 | 10 | 0.880.5301 |

# Coefficients for Oxy 30 vs Placebo Planned Planned

| | | Arm | Treatment | |
|-----------|---------|--------|-----------|------|
| Effect | APERIOD | Code | (N) | Row1 |
| Intercept | ; | | | |
| TRTPN | | | 1 | |
| TRTPN | | | 2 | |
| TRTPN | | | 3 | |
| TRTPN | | | 4 | 1 |
| TRTPN | | | 5 | |
| TRTPN | | | 6 | -1 |
| APERIOD | P1 | | | |
| APERIOD | P2 | | | |
| APERIOD | P3 | | | |
| APERIOD | P4 | | | |
| APERIOD | P5 | | | |
| APERIOD | P6 | | | |
| ARMCD | | ABCEDF | | |
| ARMCD | | BEAFCD | | |
| ARMCD | | CADBFE | | |
| ARMCD | | DCFAEB | | |

Program: A Bio2.sas Created: 02APR2020 7:35 POSTLOCK 

#### The Mixed Procedure

#### Parameter Code=MVMIEMAX

# Coefficients for Oxy 30 vs Placebo

Planned Planned

 Effect
 APERIOD Code
 (N)
 Row1

 ARMCD
 EFBDAC

 ARMCD
 FDECBA

#### Coefficients for Oxy 60 vs Placebo

Planned Planned
Arm Treatment

| | | ALIII | Treatment | |
|-----------|---------|--------|-----------|------|
| Effect | APERIOD | Code | (N) | Row1 |
| Intercept | | | | |
| TRTPN | | | 1 | |
| TRTPN | | | 2 | |
| TRTPN | | | 3 | |
| TRTPN | | | 4 | |
| TRTPN | | | 5 | 1 |
| TRTPN | | | 6 | -1 |
| APERIOD | P1 | | | |
| APERIOD | P2 | | | |
| APERIOD | Р3 | | | |
| APERIOD | P4 | | | |
| APERIOD | P5 | | | |
| APERIOD | P6 | | | |
| ARMCD | | ABCEDF | | |
| ARMCD | | BEAFCD | | |
| ARMCD | | CADBFE | | |
| ARMCD | | DCFAEB | | |


#### The Mixed Procedure

#### Parameter Code=MVMIEMAX

Coefficients for Oxy 60 vs Placebo

Planned Planned

Arm Treatment
Effect APERIOD Code (N) Row1
ARMCD EFBDAC
ARMCD FDECBA

Coefficients for Bel 300 vs Oxy 30

Planned Planned

| | | Arm | Treatment | |
|-----------|---------|--------|-----------|------|
| Effect | APERIOD | Code | (N) | Row1 |
| Intercept | | | | |
| TRTPN | | | 1 | 1 |
| TRTPN | | | 2 | |
| TRTPN | | | 3 | |
| TRTPN | | | 4 | -1 |
| TRTPN | | | 5 | |
| TRTPN | | | 6 | |
| APERIOD | P1 | | | |
| APERIOD | P2 | | | |
| APERIOD | P3 | | | |
| APERIOD | P4 | | | |
| APERIOD | P5 | | | |
| APERIOD | P6 | | | |
| ARMCD | | ABCEDF | | |
| ARMCD | | BEAFCD | | |
| ARMCD | | CADBFE | | |
| ARMCD | | DCFAEB | | |

#### The Mixed Procedure

#### Parameter Code=MVMIEMAX

Coefficients for Bel 300 vs Oxy 30

Planned Planned

Coefficients for Bel 300 vs 0xy 60
Planned Planned

Arm Treatment Effect APERIOD Code (N) Row1 Intercept 1 TRTPN 1 TRTPN TRTPN 3 TRTPN -1 TRTPN TRTPN APERIOD P1 APERIOD P2 APERIOD P3 APERIOD P4 APERIOD P5 APERIOD P6 ARMCD ABCEDF ARMCD BEAFCD ARMCD CADBFE ARMCD DCFAEB

Program: A Bio2.sas Created: 02APR2020 7:35 POSTLOCK 

#### The Mixed Procedure

#### Parameter Code=MVMIEMAX

Coefficients for Bel 300 vs Oxy 60

Planned Planned

Arm Treatment Effect APERIOD Code (N) Row1 ARMCD EFBDAC ARMCD FDECBA

Coefficients for Bel 600 vs Oxy 30 Planned Planned

Arm Treatment

| | | Arm | Treatment | |
|-----------|---------|--------|-----------|------|
| Effect | APERIOD | ) Code | (N) | Row1 |
| Intercept | • | | | |
| TRTPN | | | 1 | |
| TRTPN | | | 2 | 1 |
| TRTPN | | | 3 | |
| TRTPN | | | 4 | -1 |
| TRTPN | | | 5 | |
| TRTPN | | | 6 | |
| APERIOD | P1 | | | |
| APERIOD | P2 | | | |
| APERIOD | P3 | | | |
| APERIOD | P4 | | | |
| APERIOD | P5 | | | |
| APERIOD | P6 | | | |
| ARMCD | | ABCEDF | | |
| ARMCD | | BEAFCD | | |
| ARMCD | | CADBFE | | |
| ARMCD | | DCFAEB | | |

The Mixed Procedure

#### Parameter Code=MVMIEMAX

Coefficients for Bel 600 vs Oxy 30

Planned Planned

 Arm
 Treatment

 Effect
 APERIOD Code
 (N)
 Row1

 ARMCD
 EFBDAC

 ARMCD
 FDECBA

Coefficients for Bel 600 vs 0xy 60
Planned Planned
Arm Treatment

| | | Arm | Treatment | |
|-----------|---------|--------|-----------|------|
| Effect | APERIOD | Code | (N) | Row1 |
| Intercept | | | | |
| TRTPN | | | 1 | |
| TRTPN | | | 2 | 1 |
| TRTPN | | | 3 | |
| TRTPN | | | 4 | |
| TRTPN | | | 5 | -1 |
| TRTPN | | | 6 | |
| APERIOD | P1 | | | |
| APERIOD | P2 | | | |
| APERIOD | P3 | | | |
| APERIOD | P4 | | | |
| APERIOD | P5 | | | |
| APERIOD | P6 | | | |
| ARMCD | | ABCEDF | | |
| ARMCD | | BEAFCD | | |
| ARMCD | | CADBFE | | |
| ARMCD | | DCFAEB | | |

#### The Mixed Procedure

#### Parameter Code=MVMIEMAX

Coefficients for Bel 600 vs Oxy 60

Planned Planned

 Arm
 Treatment

 Effect
 APERIOD Code
 (N)
 Row1

 ARMCD
 EFBDAC

 ARMCD
 FDECBA

Coefficients for Bel 900 vs Oxy 30

Planned Planned
Arm Treatment

| | | 2 1 L 111 | I I Ca chich | • |
|-----------|--------|-----------|--------------|------|
| Effect | APERIO | ) Code | (N) | Row1 |
| Intercept | ; | | | |
| TRTPN | | | 1 | |
| TRTPN | | | 2 | |
| TRTPN | | | 3 | 1 |
| TRTPN | | | 4 | -1 |
| TRTPN | | | 5 | |
| TRTPN | | | 6 | |
| APERIOD | P1 | | | |
| APERIOD | P2 | | | |
| APERIOD | Р3 | | | |
| APERIOD | P4 | | | |
| APERIOD | P5 | | | |
| APERIOD | P6 | | | |
| ARMCD | | ABCEDF | | |
| ARMCD | | BEAFCD | | |
| ARMCD | | CADBFE | | |
| ARMCD | | DCFAEB | | |

Program: A Bio2.sas Created: 02APR2020 7:35 POSTLOCK 

#### The Mixed Procedure

#### Parameter Code=MVMIEMAX

Coefficients for Bel 900 vs Oxy 30

Planned Planned

Arm Treatment
Effect APERIOD Code (N) Row1

ARMCD EFBDAC ARMCD FDECBA

Coefficients for Bel 900 vs Oxy 60

Planned Planned

Arm Treatment Effect APERIOD Code (N) Row1 Intercept 1 TRTPN TRTPN 3 TRTPN 1 TRTPN 5 -1 TRTPN TRTPN APERIOD P1 APERIOD P2 APERIOD P3 APERIOD P4 APERIOD P5 APERIOD P6 ARMCD ABCEDF ARMCD BEAFCD ARMCD CADBFE ARMCD DCFAEB

Program: A\_Bio2.sas Created: 02APR2020 7:35 POSTLOCK

#### The Mixed Procedure

#### Parameter Code=MVMIEMAX

Coefficients for Bel 900 vs Oxy 60

Planned Planned

Coefficients for Bel 300 vs Placebo
Planned Planned

Arm Treatment Effect APERIOD Code (N) Row1 Intercept 1 TRTPN 1 TRTPN TRTPN 3 TRTPN TRTPN TRTPN -1 APERIOD P1 APERIOD P2 APERIOD P3 APERIOD P4 APERIOD P5 APERIOD P6 ARMCD ABCEDF ARMCD BEAFCD ARMCD CADBFE ARMCD DCFAEB

Program: A\_Bio2.sas Created: 02APR2020 7:35 POSTLOCK


#### The Mixed Procedure

#### Parameter Code=MVMIEMAX

Coefficients for Bel 300 vs Placebo

Planned Planned

Arm Treatment

Effect APERIOD Code (N) Row1

ARMCD EFBDAC ARMCD FDECBA

Coefficients for Bel 600 vs Placebo
Planned Planned

Arm Treatment

Effect APERIOD Code (N) Row1 Intercept TRTPN 1 TRTPN 1 TRTPN 3 TRTPN TRTPN TRTPN -1 APERIOD P1 APERIOD P2 APERIOD P3 APERIOD P4 APERIOD P5 APERIOD P6 ARMCD ABCEDF ARMCD BEAFCD ARMCD CADBFE ARMCD DCFAEB

#### The Mixed Procedure

#### Parameter Code=MVMIEMAX

# Coefficients for Bel 600 vs Placebo

Planned Planned

| | | Arm | Treatment | |
|--------|---------|--------|-----------|------|
| Effect | APERIOD | Code | (N) | Row1 |
| ARMCD | | EFBDAC | | |
| ARMCD | | FDECBA | | |

# Coefficients for Bel 900 vs Placebo

Planned Planned
Arm Treatment

| | | Arm | Treatment | |
|-----------|---------|--------|-----------|------|
| Effect | APERIOD | Code | (N) | Row1 |
| Intercept | | | | |
| TRTPN | | | 1 | |
| TRTPN | | | 2 | |
| TRTPN | | | 3 | 1 |
| TRTPN | | | 4 | |
| TRTPN | | | 5 | |
| TRTPN | | | 6 | -1 |
| APERIOD | P1 | | | |
| APERIOD | P2 | | | |
| APERIOD | P3 | | | |
| APERIOD | P4 | | | |
| APERIOD | P5 | | | |
| APERIOD | P6 | | | |
| ARMCD | | ABCEDF | | |
| ARMCD | | BEAFCD | | |
| ARMCD | | CADBFE | | |
| ARMCD | | DCFAEB | | |

# Appendix 16.1.9.2.2 Statistical Methods and Analysis Output Supporting Table 14.2.3 Supporting Table 14.2.3

#### The Mixed Procedure

#### Parameter Code=MVMIEMAX

#### Coefficients for Bel 900 vs Placebo

Planned Planned

Arm Treatment

Effect APERIOD Code (N) Row1
ARMCD EFBDAC
ARMCD FDECBA

#### Estimates

#### Standard

| Label | Estimate | Error DF t | Value E | r > t | Alpha | Lower | Upper |
|---|---|---|---|---|---|---|---|
| Oxy 30 vs Placebo | -799.96 | 1915.2867 | -0.42 | 0.6775 | 0.05- | -4622.87 | 3022.94 |
| Oxy 60 vs Placebo | -5189.06 | 1879.6067 | -2.76 | 0.0074 | 0.05 - | -8940.75 - | -1437.38 |
| Bel 300 vs Oxy 30 | 2034.96 | 1941.7867 | 1.05 | 0.2984 | 0.05 - | -1840.84 | 5910.76 |
| Bel 300 vs Oxy 60 | 6424.06 | 1915.2267 | 3.35 | 0.0013 | 0.05 | 2601.26 | 10247 |
| Bel 600 vs Oxy 30 | 736.00 | 1916.0367 | 0.38 | 0.7021 | 0.05 - | -3088.41 | 4560.41 |
| Bel 600 vs Oxy 60 | 5125.10 | 1879.4567 | 2.73 | 0.0082 | 0.05 | 1373.69 | 8876.51 |
| Bel 900 vs Oxy 30 | 1748.48 | 1941.6067 | 0.90 | 0.3711 | 0.05- | -2126.98 | 5623.93 |
| Bel 900 vs Oxy 60 | 6137.58 | 1915.9867 | 3.20 | 0.0021 | 0.05 | 2313.27 | 9961.88 |
| Bel 300 vs Placebo | 1234.99 | 1914.3367 | 0.65 | 0.5210 | 0.05- | -2586.03 | 5056.02 |
| Bel 600 vs Placebo | -63.9639 | 1875.6667 | -0.03 | 0.9729 | 0.05- | -3807.80 | 3679.88 |
| Bel 900 vs Placebo | 948 51 | 1915 2867 | 0.50 | 0 6221 | 0 05- | -2874 40 | 4771 42 |

Program: A Bio2.sas Created: 02APR2020 7:35 POSTLOCK 

# Appendix 16.1.9.2.2 Statistical Methods and Analysis Output Supporting Table 14.2.3 Supporting Table 14.2.3

#### The Mixed Procedure

#### Parameter Code=MVMIEMAX

## Least Squares Means

| | | | _ | | | |
|---|---|---|---|---|---|---|
| | Planned | | | | | |
| | Treatment | : | Standard | | | |
| Effect | (N) | Estimate | Error DF t | Value | Pr > t | Alpha Lower Upper |
| TRTPN | 1 | 23560 | 1657.2867 | 14.22 | <.0001 | 0.12079526324 |
| TRTPN | 2 | 22261 | 1615.1967 | 13.78 | <.0001 | 0.11956724955 |
| TRTPN | 3 | 23273 | 1658.1967 | 14.04 | <.0001 | 0.12050726039 |
| TRTPN | 4 | 21525 | 1658.1967 | 12.98 | <.0001 | 0.11875924290 |
| TRTPN | 5 | 17136 | 1615.1767 | 10.61 | <.0001 | 0.11444219830 |
| TRTPN | 6 | 22325 | 1615.1167 | 13.82 | <.0001 | 0.11963125019 |

# Differences of Least Squares Means

| | Planned | Planned | | | | | | |
|---|---|---|---|---|---|---|---|---|
| | Treatment | Treatment | 6 | Standard | | | | |
| Effect | (N) | (N) | Estimate | Error DF t | Value Pr | > t A | lpha Lower | Upper |
| TRTPN | 1 | 2 | 1298.96 | 1919.1467 | 0.68 | 0.5008 | 0.1-1902.01 | 4499.93 |
| TRTPN | 1 | 3 | 286.48 | 1941.5067 | 0.15 | 0.8831 | 0.1-2951.78 | 3524.74 |
| TRTPN | 1 | 4 | 2034.96 | 1941.7867 | 1.05 | 0.2984 | 0.1-1203.76 | 5273.68 |
| TRTPN | 1 | 5 | 6424.06 | 1915.2267 | 3.35 | 0.0013 | 0.1 3229.63 | 9618.49 |
| TRTPN | 1 | 6 | 1234.99 | 1914.3367 | 0.65 | 0.5210 | 0.1-1957.96 | 4427.94 |
| TRTPN | 2 | 3 | -1012.48 | 1916.2967 | -0.53 | 0.5990 | 0.1-4208.68 | 2183.73 |
| TRTPN | 2 | 4 | 736.00 | 1916.0367 | 0.38 | 0.7021 | 0.1-2459.77 | 3931.77 |
| TRTPN | 2 | 5 | 5125.10 | 1879.4567 | 2.73 | 0.0082 | 0.1 1990.33 | 8259.87 |
| TRTPN | 2 | 6 | -63.9639 | 1875.6667 | -0.03 | 0.9729 | 0.1-3192.41 | 3064.49 |
| TRTPN | 3 | 4 | 1748.48 | 1941.6067 | 0.90 | 0.3711 | 0.1-1489.95 | 4986.91 |
| TRTPN | 3 | 5 | 6137.58 | 1915.9867 | 3.20 | 0.0021 | 0.1 2941.89 | 9333.26 |
| TRTPN | 3 | 6 | 948.51 | 1915.2867 | 0.50 | 0.6221 | 0.1-2246.01 | 4143.04 |
| TRTPN | 4 | 5 | 4389.10 | 1915.9767 | 2.29 | 0.0251 | 0.1 1193.41 | 7584.79 |

Program: A\_Bio2.sas Created: 02APR2020 7:35 POSTLOCK 

# Appendix 16.1.9.2.2 Statistical Methods and Analysis Output Supporting Table 14.2.3 Supporting Table 14.2.3

#### The Mixed Procedure

#### Parameter Code=MVMIEMAX

## Differences of Least Squares Means

Planned Planned Treatment Treatment

| Treatment Treatment | | Standard | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| | Effect | (N) | (N) | Estimate | Error DF t | Value Pr | r > t A | lpha L | ower | Upper |
| | TRTPN | 4 | 6 | -799.96 | 1915.2867 | -0.42 | 0.6775 | 0.1-399 | 4.48 | 2394.55 |
| | TRTPN | 5 | 6 | -5189.06 | 1879.6067 | -2.76 | 0.0074 | 0.1-832 | 4.07 - | -2054.06 |

 Program: A\_Bio2.sas Created: 02APR2020 7:35 POSTLOCK

# Appendix 16.1.9.2.2 Statistical Methods and Analysis Output Supporting Table 14.2.3 Supporting Table 14.2.3

#### The Mixed Procedure

#### Parameter Code=PEFMEMAX

#### Model Information

| Data Set | WORK.ADXV |
|---------------------------|---------------------|
| Dependent Variable | AVAL |
| Covariance Structure | Variance Components |
| Estimation Method | REML |
| Residual Variance Method | Profile |
| Fixed Effects SE Method | Model-Based |
| Degrees of Freedom Method | Containment |

#### Class Level Information

| Class | LevelsValues |
|---|---|
| SUBJID | 161001 1002 1003 1004 1005 1006 1007 1008 1010 1012 1013 1014 1015 1016 1017 1018 |
| TRTPN | 61 2 3 4 5 6 |
| APERIOD | O 6P1 P2 P3 P4 P5 P6 |
| ARMCD | 6ABCEDF BEAFCD CADBFE DCFAEB EFBDAC FDECBA |

| Dimensions | | | |
|------------|-------------|------------|----|
| | Covariance | Parameters | 2 |
| | Columns in | X | 19 |
| | Columns in | Z | 16 |
| | Subjects | | 1 |
| | Max Obs per | Subject | 93 |

Program: A Bio2.sas Created: 02APR2020 7:35 POSTLOCK 

# Appendix 16.1.9.2.2 Statistical Methods and Analysis Output Supporting Table 14.2.3 Supporting Table 14.2.3

The Mixed Procedure

#### Parameter Code=PEFMEMAX

| Number of Observations | | | |
|------------------------|--------------|----------|----|
| Number of | Observations | Read | 93 |
| Number of | Observations | Used | 93 |
| Number of | Observations | Not Used | 0 |

## Iteration History

| Iteration Evaluat | ions -2 | Res | Log | Like | Criterion |
|-------------------|---------|-----|--------|-------|-----------|
| 0 | 1 | 693 | .508 | 73069 | _ |
| 1 | 2 | 683 | .8832 | 29081 | 0.0000004 |
| 2 | 1 | 683 | . 8832 | 7887 | 0.0000000 |

Convergence criteria met.

# Covariance Parameter Estimates

| Cov Parm | Estimate |
|----------------|----------|
| SUBJID (ARMCD) | 94.1104 |
| Residual | 212.55 |

#### Fit Statistics

| -2 Res Log Likelihood | 683.9 |
|--------------------------|-------|
| AIC (Smaller is Better) | 687.9 |
| AICC (Smaller is Better) | 688.0 |
| BIC (Smaller is Better) | 689.4 |

Program: A Bio2.sas Created: 02APR2020 7:35 POSTLOCK 

The Mixed Procedure

#### Parameter Code=PEFMEMAX

Type 3 Tests of Fixed Effects

| | Num I | Den | |
|---------|-------|------|--------------|
| Effect | DF | DF F | Value Pr > F |
| TRTPN | 5 | 67 | 2.580.0339 |
| APERIOD | 5 | 67 | 2.600.0327 |
| ARMCD | 5 | 10 | 0.620.6898 |

# Coefficients for Oxy 30 vs Placebo Planned Planned

| | | Arm | Treatment | ; |
|-----------|---------|--------|-----------|------|
| Effect | APERIOD | ) Code | (N) | Row1 |
| Intercept | 5 | | | |
| TRTPN | | | 1 | |
| TRTPN | | | 2 | |
| TRTPN | | | 3 | |
| TRTPN | | | 4 | 1 |
| TRTPN | | | 5 | |
| TRTPN | | | 6 | -1 |
| APERIOD | P1 | | | |
| APERIOD | P2 | | | |
| APERIOD | P3 | | | |
| APERIOD | P4 | | | |
| APERIOD | P5 | | | |
| APERIOD | P6 | | | |
| ARMCD | | ABCEDF | | |
| ARMCD | | BEAFCD | | |
| ARMCD | | CADBFE | | |
| ARMCD | | DCFAEB | | |

#### The Mixed Procedure

#### Parameter Code=PEFMEMAX

# Coefficients for Oxy 30 vs Placebo

Planned Planned

Arm Treatment
Effect APERIOD Code (N) Row1
ARMCD EFBDAC
ARMCD FDECBA

#### Coefficients for Oxy 60 vs Placebo

Planned Planned Arm Treatment

| | | ATIII | TIEatment | |
|-----------|---------|--------|-----------|------|
| Effect | APERIOD | Code | (N) | Row1 |
| Intercept | | | | |
| TRTPN | | | 1 | |
| TRTPN | | | 2 | |
| TRTPN | | | 3 | |
| TRTPN | | | 4 | |
| TRTPN | | | 5 | 1 |
| TRTPN | | | 6 | -1 |
| APERIOD | P1 | | | |
| APERIOD | P2 | | | |
| APERIOD | P3 | | | |
| APERIOD | P4 | | | |
| APERIOD | P5 | | | |
| APERIOD | P6 | | | |
| ARMCD | | ABCEDF | | |
| ARMCD | | BEAFCD | | |
| ARMCD | | CADBFE | | |
| ARMCD | | DCFAEB | | |

#### The Mixed Procedure

#### Parameter Code=PEFMEMAX

# Coefficients for Oxy 60 vs Placebo

Planned Planned

 Effect
 APERIOD Code
 (N)
 Row1

 ARMCD
 EFBDAC

 ARMCD
 FDECBA

# Coefficients for Bel 300 vs Oxy 30

Planned Planned
Arm Treatment

| | | Arm | Treatment | |
|-----------|---------|--------|-----------|------|
| Effect | APERIOD | Code | (N) | Row1 |
| Intercept | | | | |
| TRTPN | | | 1 | 1 |
| TRTPN | | | 2 | |
| TRTPN | | | 3 | |
| TRTPN | | | 4 | -1 |
| TRTPN | | | 5 | |
| TRTPN | | | 6 | |
| APERIOD | P1 | | | |
| APERIOD | P2 | | | |
| APERIOD | P3 | | | |
| APERIOD | P4 | | | |
| APERIOD | P5 | | | |
| APERIOD | P6 | | | |
| ARMCD | | ABCEDF | | |
| ARMCD | | BEAFCD | | |
| ARMCD | | CADBFE | | |
| ARMCD | | DCFAEB | | |

Program: A\_Bio2.sas Created: 02APR2020 7:35 POSTLOCK


#### The Mixed Procedure

#### Parameter Code=PEFMEMAX

Coefficients for Bel 300 vs Oxy 30

Planned Planned

 Arm
 Treatment

 Effect
 APERIOD Code
 (N)
 Row1

 ARMCD
 EFBDAC

 ARMCD
 FDECBA

Coefficients for Bel 300 vs Oxy 60 Planned Planned

| | | Arm | Treatment | |
|-----------|---------|--------|-----------|------|
| Effect | APERIOD | Code | (N) | Row1 |
| Intercept | | | | |
| TRTPN | | | 1 | 1 |
| TRTPN | | | 2 | |
| TRTPN | | | 3 | |
| TRTPN | | | 4 | |
| TRTPN | | | 5 | -1 |
| TRTPN | | | 6 | |
| APERIOD | P1 | | | |
| APERIOD | P2 | | | |
| APERIOD | P3 | | | |
| APERIOD | P4 | | | |
| APERIOD | P5 | | | |
| APERIOD | P6 | | | |
| ARMCD | | ABCEDF | | |
| ARMCD | | BEAFCD | | |
| ARMCD | | CADBFE | | |
| ARMCD | | DCFAEB | | |

The Mixed Procedure

#### Parameter Code=PEFMEMAX

Coefficients for Bel 300 vs Oxy 60

Planned Planned

 Arm
 Treatment

 Effect
 APERIOD Code
 (N)
 Row1

 ARMCD
 EFBDAC

 ARMCD
 FDECBA

Coefficients for Bel 600 vs Oxy 30 Planned Planned

r Taimed Franced

| | | Arm | Treatment | |
|-----------|---------|--------|-----------|------|
| Effect | APERIOD | Code | (N) | Row1 |
| Intercept | | | | |
| TRTPN | | | 1 | |
| TRTPN | | | 2 | 1 |
| TRTPN | | | 3 | |
| TRTPN | | | 4 | -1 |
| TRTPN | | | 5 | |
| TRTPN | | | 6 | |
| APERIOD | P1 | | | |
| APERIOD | P2 | | | |
| APERIOD | Р3 | | | |
| APERIOD | P4 | | | |
| APERIOD | P5 | | | |
| APERIOD | P6 | | | |
| ARMCD | | ABCEDF | | |
| ARMCD | | BEAFCD | | |
| ARMCD | | CADBFE | | |
| ARMCD | | DCFAEB | | |

#### The Mixed Procedure

#### Parameter Code=PEFMEMAX

Coefficients for Bel 600 vs Oxy 30

Planned Planned

 Arm
 Treatment

 Effect
 APERIOD Code
 (N)
 Row1

 ARMCD
 EFBDAC

 ARMCD
 FDECBA

Coefficients for Bel 600 vs 0xy 60
Planned Planned

Arm Treatment

| | | 21111 | I I Ca chich c | |
|-----------|---------|--------|----------------|------|
| Effect | APERIOD | Code | (N) | Row1 |
| Intercept | | | | |
| TRTPN | | | 1 | |
| TRTPN | | | 2 | 1 |
| TRTPN | | | 3 | |
| TRTPN | | | 4 | |
| TRTPN | | | 5 | -1 |
| TRTPN | | | 6 | |
| APERIOD | P1 | | | |
| APERIOD | P2 | | | |
| APERIOD | P3 | | | |
| APERIOD | P4 | | | |
| APERIOD | P5 | | | |
| APERIOD | P6 | | | |
| ARMCD | | ABCEDF | | |
| ARMCD | | BEAFCD | | |
| ARMCD | | CADBFE | | |
| ARMCD | | DCFAEB | | |

Program: A Bio2.sas Created: 02APR2020 7:35 POSTLOCK 
#### The Mixed Procedure

#### Parameter Code=PEFMEMAX

Coefficients for Bel 600 vs Oxy 60

Planned Planned

 Arm
 Treatment

 Effect
 APERIOD Code
 (N)
 Row1

 ARMCD
 EFBDAC

 ARMCD
 FDECBA

Coefficients for Bel 900 vs 0xy 30

Planned Planned
Arm Treatment

| | | ATIII | Treatment | |
|-----------|---------|--------|-----------|------|
| Effect | APERIOD | Code | (N) | Row1 |
| Intercept | | | | |
| TRTPN | | | 1 | |
| TRTPN | | | 2 | |
| TRTPN | | | 3 | 1 |
| TRTPN | | | 4 | -1 |
| TRTPN | | | 5 | |
| TRTPN | | | 6 | |
| APERIOD | P1 | | | |
| APERIOD | P2 | | | |
| APERIOD | Р3 | | | |
| APERIOD | P4 | | | |
| APERIOD | P5 | | | |
| APERIOD | P6 | | | |
| ARMCD | | ABCEDF | | |
| ARMCD | | BEAFCD | | |
| ARMCD | | CADBFE | | |
| ARMCD | | DCFAEB | | |

#### The Mixed Procedure

#### Parameter Code=PEFMEMAX

Coefficients for Bel 900 vs Oxy 30

Planned Planned

 Arm
 Treatment

 Effect
 APERIOD Code
 (N)
 Row1

 ARMCD
 EFBDAC

 ARMCD
 FDECBA

Coefficients for Bel 900 vs 0xy 60
Planned Planned

| | | Arm | Treatment | |
|-----------|---------|--------|-----------|------|
| Effect | APERIOD | Code | (N) | Row1 |
| Intercept | | | | |
| TRTPN | | | 1 | |
| TRTPN | | | 2 | |
| TRTPN | | | 3 | 1 |
| TRTPN | | | 4 | |
| TRTPN | | | 5 | -1 |
| TRTPN | | | 6 | |
| APERIOD | P1 | | | |
| APERIOD | P2 | | | |
| APERIOD | P3 | | | |
| APERIOD | P4 | | | |
| APERIOD | P5 | | | |
| APERIOD | P6 | | | |
| ARMCD | | ABCEDF | | |
| ARMCD | | BEAFCD | | |
| ARMCD | | CADBFE | | |
| ARMCD | | DCFAEB | | |

Program: A Bio2.sas Created: 02APR2020 7:35 POSTLOCK 

#### The Mixed Procedure

#### Parameter Code=PEFMEMAX

Coefficients for Bel 900 vs Oxy 60

Planned Planned

 Arm
 Treatment

 Effect
 APERIOD Code
 (N)
 Row1

 ARMCD
 EFBDAC

 ARMCD
 FDECBA

Coefficients for Bel 300 vs Placebo Planned Planned

| | | Arm | Treatment | |
|-----------|---------|--------|-----------|------|
| Effect | APERIOD | Code | (N) | Row1 |
| Intercept | | | | |
| TRTPN | | | 1 | 1 |
| TRTPN | | | 2 | |
| TRTPN | | | 3 | |
| TRTPN | | | 4 | |
| TRTPN | | | 5 | |
| TRTPN | | | 6 | -1 |
| APERIOD | P1 | | | |
| APERIOD | P2 | | | |
| APERIOD | P3 | | | |
| APERIOD | P4 | | | |
| APERIOD | P5 | | | |
| APERIOD | P6 | | | |
| ARMCD | | ABCEDF | | |
| ARMCD | | BEAFCD | | |
| ARMCD | | CADBFE | | |
| ARMCD | | DCFAEB | | |

#### The Mixed Procedure

#### Parameter Code=PEFMEMAX

Coefficients for Bel 300 vs Placebo

Planned Planned

Arm Treatment Effect APERIOD Code (N) Row1 ARMCD EFBDAC

FDECBA

ARMCD

Coefficients for Bel 600 vs Placebo Planned Planned

Arm Treatment Effect APERIOD Code (N)

| Effect | APERIOD ( | Code | (N) | Row1 |
|-----------|-----------|--------|-----|------|
| Intercept | | | | |
| TRTPN | | | 1 | |
| TRTPN | | | 2 | 1 |
| TRTPN | | | 3 | |
| TRTPN | | | 4 | |
| TRTPN | | | 5 | |
| TRTPN | | | 6 | -1 |
| APERIOD | P1 | | | |
| APERIOD | P2 | | | |
| APERIOD | P3 | | | |
| APERIOD | P4 | | | |
| APERIOD | P5 | | | |
| APERIOD | P6 | | | |
| ARMCD | Z | ABCEDF | | |
| ARMCD | I | BEAFCD | | |
| ARMCD | ( | CADBFE | | |
| ARMCD | Ī | OCFAEB | | |

The Mixed Procedure

#### Parameter Code=PEFMEMAX

Coefficients for Bel 600 vs Placebo

Planned Planned

 Arm
 Treatment

 Effect
 APERIOD Code
 (N)
 Row1

 ARMCD
 EFBDAC

 ARMCD
 FDECBA

Coefficients for Bel 900 vs Placebo Planned Planned

| | | Arm | Treatment | |
|-----------|---------|--------|-----------|------|
| Effect | APERIOD | Code | (N) | Row1 |
| Intercept | | | | |
| TRTPN | | | 1 | |
| TRTPN | | | 2 | |
| TRTPN | | | 3 | 1 |
| TRTPN | | | 4 | |
| TRTPN | | | 5 | |
| TRTPN | | | 6 | -1 |
| APERIOD | P1 | | | |
| APERIOD | P2 | | | |
| APERIOD | P3 | | | |
| APERIOD | P4 | | | |
| APERIOD | P5 | | | |
| APERIOD | P6 | | | |
| ARMCD | | ABCEDF | | |
| ARMCD | | BEAFCD | | |
| ARMCD | | CADBFE | | |
| ARMCD | | DCFAEB | | |

# Appendix 16.1.9.2.2 Statistical Methods and Analysis Output Supporting Table 14.2.3 Supporting Table 14.2.3

#### The Mixed Procedure

#### Parameter Code=PEFMEMAX

Coefficients for Bel 900 vs Placebo

Planned Planned

Arm Treatment

Effect APERIOD Code (N) Row1
ARMCD EFBDAC
ARMCD FDECBA

#### Estimates

#### Standard

| Label | Estimate | Error DF t | Value H | ?r > t . | Alpha | Lower | Upper |
|---|---|---|---|---|---|---|---|
| Oxy 30 vs Placebo | 0.2197 | 5.273867 | 0.04 | 0.9669 | 0.05 | -10.3069 | 10.7464 |
| Oxy 60 vs Placebo | -12.9112 | 5.175867 | -2.49 | 0.0151 | 0.05 | -23.2422 | -2.5803 |
| Bel 300 vs Oxy 30 | 2.8091 | 5.347067 | 0.53 | 0.6011 | 0.05 | -7.8636 | 13.4818 |
| Bel 300 vs Oxy 60 | 15.9401 | 5.273767 | 3.02 | 0.0035 | 0.05 | 5.4138 | 26.4664 |
| Bel 600 vs Oxy 30 | 0.8329 | 5.275967 | 0.16 | 0.8750 | 0.05 | -9.6978 | 11.3636 |
| Bel 600 vs Oxy 60 | 13.9639 | 5.175467 | 2.70 | 0.0088 | 0.05 | 3.6337 | 24.2941 |
| Bel 900 vs Oxy 30 | 2.0449 | 5.346567 | 0.38 | 0.7033 | 0.05 | -8.6269 | 12.7166 |
| Bel 900 vs Oxy 60 | 15.1758 | 5.275767 | 2.88 | 0.0054 | 0.05 | 4.6454 | 25.7063 |
| Bel 300 vs Placebo | 3.0289 | 5.271367 | 0.57 | 0.5675 | 0.05 | -7.4926 | 13.5504 |
| Bel 600 vs Placebo | 1.0527 | 5.165067 | 0.20 | 0.8391 | 0.05 | -9.2567 | 11.3620 |
| Bel 900 vs Placebo | 2.2646 | 5.273867 | 0.43 | 0.6690 | 0.05 | -8.2620 | 12.7912 |

Program: A Bio2.sas Created: 02APR2020 7:35 POSTLOCK 

# Appendix 16.1.9.2.2 Statistical Methods and Analysis Output Supporting Table 14.2.3 Supporting Table 14.2.3

# The Mixed Procedure

#### Parameter Code=PEFMEMAX

# Least Squares Means

| | Planned | | _ | | | | | |
|---|---|---|---|---|---|---|---|---|
| | Treatment | | Standard | | | | | |
| Effect | (N) | Estimate | Error DF t | Value | Pr > | t Alpha | Lower | Upper |
| TRTPN | 1 | 61.5830 | 4.536867 | 13.57 | <.00 | 01 0.1 | 54.0160 | 69.1499 |
| TRTPN | 2 | 59.6068 | 4.420467 | 13.48 | <.00 | 01 0.1 | 52.2339 | 66.9796 |
| TRTPN | 3 | 60.8187 | 4.539367 | 13.40 | <.00 | 01 0.1 | 53.2476 | 68.3899 |
| TRTPN | 4 | 58.7739 | 4.539367 | 12.95 | <.00 | 01 0.1 | 51.2027 | 66.3450 |
| TRTPN | 5 | 45.6429 | 4.420467 | 10.33 | <.00 | 01 0.1 | 38.2701 | 53.0157 |
| TRTPN | 6 | 58.5541 | 4.420267 | 13.25 | <.00 | 01 0.1 | 51.1816 | 65.9266 |

# Differences of Least Squares Means

| | Planned | Planned | | | - | | | | |
|---|---|---|---|---|---|---|---|---|---|
| | Treatmen | t Treatment | | Standard | | | | | |
| Effect | (N) | (N) | Estimate | Error DF t | Value F | r > t A | Alpha | Lower | Upper |
| TRTPN | 1 | 2 | 1.9762 | 5.284567 | 0.37 | 0.7096 | 0.1 | -6.8379 | 10.7903 |
| TRTPN | 1 | 3 | 0.7643 | 5.346367 | 0.14 | 0.8868 | 0.1 | -8.1529 | 9.6814 |
| TRTPN | 1 | 4 | 2.8091 | 5.347067 | 0.53 | 0.6011 | 0.1 | -6.1093 | 11.7275 |
| TRTPN | 1 | 5 | 15.9401 | 5.273767 | 3.02 | 0.0035 | 0.1 | 7.1440 | 24.7362 |
| TRTPN | 1 | 6 | 3.0289 | 5.271367 | 0.57 | 0.5675 | 0.1 | -5.7632 | 11.8209 |
| TRTPN | 2 | 3 | -1.2120 | 5.276667 | -0.23 | 0.8190 | 0.1 | -10.0129 | 7.5890 |
| TRTPN | 2 | 4 | 0.8329 | 5.275967 | 0.16 | 0.8750 | 0.1 | -7.9668 | 9.6326 |
| TRTPN | 2 | 5 | 13.9639 | 5.175467 | 2.70 | 0.0088 | 0.1 | 5.3317 | 22.5960 |
| TRTPN | 2 | 6 | 1.0527 | 5.165067 | 0.20 | 0.8391 | 0.1 | -7.5621 | 9.6674 |
| TRTPN | 3 | 4 | 2.0449 | 5.346567 | 0.38 | 0.7033 | 0.1 | -6.8727 | 10.9624 |
| TRTPN | 3 | 5 | 15.1758 | 5.275767 | 2.88 | 0.0054 | 0.1 | 6.3764 | 23.9753 |
| TRTPN | 3 | 6 | 2.2646 | 5.273867 | 0.43 | 0.6690 | 0.1 | -6.5317 | 11.0609 |
| TRTPN | 4 | 5 | 13.1310 | 5.275767 | 2.49 | 0.0153 | 0.1 | 4.3315 | 21.9305 |

Program: A Bio2.sas Created: 02APR2020 7:35 POSTLOCK 

# Appendix 16.1.9.2.2 Statistical Methods and Analysis Output Supporting Table 14.2.3 Supporting Table 14.2.3

# The Mixed Procedure

#### Parameter Code=PEFMEMAX

# Differences of Least Squares Means

| | | | | | - | | | | |
|---|---|---|---|---|---|---|---|---|---|
| | Planned | Planned | | | | | | | |
| | Treatment | Treatment | | Standard | | | | | |
| Effect | (N) | (N) | Estimate | Error DF t | Value Pr | > t | Alpha | Lower | Upper |
| TRTPN | 4 | 6 | 0.2197 | 5.273867 | 0.04 | 0.9669 | 0.1 | -8.5766 | 9.0161 |
| TRTPN | 5 | 6 | -12.9112 | 5.175867 | -2.49 | 0.0151 | 0.1 | -21.5440 | -4.2785 |

Program: A\_Bio2.sas Created: 02APR2020 7:35 POSTLOCK 

# Appendix 16.1.9.2.2 Statistical Methods and Analysis Output Supporting Table 14.2.3 Supporting Table 14.2.3

#### The Mixed Procedure

#### Parameter Code=REMAX

#### Model Information

| Data Set | WORK.ADXV |
|---------------------------|---------------------|
| Dependent Variable | AVAL |
| Covariance Structure | Variance Components |
| Estimation Method | REML |
| Residual Variance Method | Profile |
| Fixed Effects SE Method | Model-Based |
| Degrees of Freedom Method | Containment |

# Class Level Information

| Class | LevelsValues |
|---|---|
| SUBJID | 161001 1002 1003 1004 1005 1006 1007 1008 1010 1012 1013 1014 1015 1016 1017 1018 |
| TRTPN | 61 2 3 4 5 6 |
| APERIOD | 6 P1 P2 P3 P4 P5 P6 |
| ARMCD | 6ABCEDF BEAFCD CADBFE DCFAEB EFBDAC FDECBA |

| Dimensions | |
|-----------------------|----|
| Covariance Parameters | 2 |
| Columns in X | 19 |
| Columns in Z | 16 |
| Subjects | 1 |
| Max Obs per Subject | 93 |

Program: A\_Bio2.sas Created: 02APR2020 7:35 POSTLOCK 

# Appendix 16.1.9.2.2 Statistical Methods and Analysis Output Supporting Table 14.2.3 Supporting Table 14.2.3

The Mixed Procedure

#### Parameter Code=REMAX

| | Nι | umber of Obse | rvations | |
|--------|----|---------------|----------|----|
| Number | of | Observations | Read | 93 |
| Number | of | Observations | Used | 93 |
| Number | of | Observations | Not Used | 0 |

# Iteration History Iteration Evaluations -2 Res Log Like Criterion 0 1 1021.29677444 1 2 1011.480179880.00000000

Convergence criteria met.

# Estimates Cov Parm Estimate SUBJID(ARMCD) 6773.79 Residual 14934

Covariance Parameter

| Fit Statistics | |
|------------------------------|--------|
| -2 Res Log Likelihood 1011.5 | |
| AIC (Smaller is Better) | 1015.5 |
| AICC (Smaller is Better) | 1015.6 |
| BIC (Smaller is Better) | 1017.0 |

Program: A Bio2.sas Created: 02APR2020 7:35 POSTLOCK 

The Mixed Procedure

Parameter Code=REMAX

Type 3 Tests of Fixed Effects
Num Den

| | Nulli | | |
|---------|-------|------|--------------|
| Effect | DF | DF F | Value Pr > F |
| TRTPN | 5 | 67 | 4.010.0030 |
| APERIOD | 5 | 67 | 2.310.0537 |
| ARMCD | 5 | 10 | 1.120.4076 |

Coefficients for Oxy 30 vs Placebo Planned Planned

| | | Arm | Treatment | |
|-----------|---------|--------|-----------|------|
| Effect | APERIOD | Code | (N) | Row1 |
| Intercept | : | | | |
| TRTPN | | | 1 | |
| TRTPN | | | 2 | |
| TRTPN | | | 3 | |
| TRTPN | | | 4 | 1 |
| TRTPN | | | 5 | |
| TRTPN | | | 6 | -1 |
| APERIOD | P1 | | | |
| APERIOD | P2 | | | |
| APERIOD | P3 | | | |
| APERIOD | P4 | | | |
| APERIOD | P5 | | | |
| APERIOD | P6 | | | |
| ARMCD | | ABCEDF | | |
| ARMCD | | BEAFCD | | |
| ARMCD | | CADBFE | | |
| ARMCD | | DCFAEB | | |

Program: A\_Bio2.sas Created: 02APR2020 7:35 POSTLOCK

The Mixed Procedure

#### Parameter Code=REMAX

Coefficients for Oxy 30 vs Placebo

Planned Planned

 $\begin{array}{c|cccc} & & Arm & Treatment \\ \hline Effect & APERIOD\,Code & (N) & Row1 \\ \hline ARMCD & EFBDAC \end{array}$ 

ARMCD

Coefficients for Oxy 60 vs Placebo

FDECBA

Planned Planned

| | | Arm | Treatment | |
|-----------|---------|--------|-----------|------|
| Effect | APERIOD | Code | (N) | Row1 |
| Intercept | | | | |
| TRTPN | | | 1 | |
| TRTPN | | | 2 | |
| TRTPN | | | 3 | |
| TRTPN | | | 4 | |
| TRTPN | | | 5 | 1 |
| TRTPN | | | 6 | -1 |
| APERIOD | P1 | | | |
| APERIOD | P2 | | | |
| APERIOD | P3 | | | |
| APERIOD | P4 | | | |
| APERIOD | P5 | | | |
| APERIOD | P6 | | | |
| ARMCD | | ABCEDF | | |
| ARMCD | | BEAFCD | | |
| ARMCD | | CADBFE | | |
| ARMCD | | DCFAEB | | |

The Mixed Procedure

Parameter Code=REMAX

Coefficients for Oxy 60 vs Placebo

Planned Planned

 Arm
 Treatment

 Effect
 APERIOD Code
 (N)
 Row1

 ARMCD
 EFBDAC

 ARMCD
 FDECBA

Coefficients for Bel 300 vs Oxy 30

Planned Planned
Arm Treatment

| | | Arm | Treatment | |
|-----------|---------|--------|-----------|------|
| Effect | APERIOD | Code | (N) | Row1 |
| Intercept | | | | |
| TRTPN | | | 1 | 1 |
| TRTPN | | | 2 | |
| TRTPN | | | 3 | |
| TRTPN | | | 4 | -1 |
| TRTPN | | | 5 | |
| TRTPN | | | 6 | |
| APERIOD | P1 | | | |
| APERIOD | P2 | | | |
| APERIOD | P3 | | | |
| APERIOD | P4 | | | |
| APERIOD | P5 | | | |
| APERIOD | P6 | | | |
| ARMCD | | ABCEDF | | |
| ARMCD | | BEAFCD | | |
| ARMCD | | CADBFE | | |
| ARMCD | | DCFAEB | | |

Program: A\_Bio2.sas Created: 02APR2020 7:35 POSTLOCK 

The Mixed Procedure

Parameter Code=REMAX

Coefficients for Bel 300 vs Oxy 30

Planned Planned

Arm Treatment

| Effect | APERIOD Code | (N) | Row1 |
|--------|--------------|-----|------|
| ARMCD | EFBDAC | | |
| ARMCD | FDECBA | | |

Coefficients for Bel 300 vs Oxy 60 Arm

Planned Planned

Treatment

Effect APERIOD Code (N) Row1 Intercept 1 1 TRTPN TRTPN TRTPN 3 TRTPN TRTPN -1 TRTPN APERIOD P1 APERIOD P2

APERIOD P3 APERIOD P4 APERIOD P5

Program: A Bio2.sas Created: 02APR2020 7:35 POSTLOCK

The Mixed Procedure

Parameter Code=REMAX

Coefficients for Bel 300 vs Oxy 60

Planned Planned

Arm Treatment

| Effect | APERIOD Code | (N) | Row1 |
|--------|--------------|-----|------|
| ARMCD | EFBDAC | | |
| ARMCD | FDECBA | | |

Coefficients for Bel 600 vs Oxy 30

Planned Planned
Arm Treatment

Effect APERIOD Code (N) Row1 Intercept TRTPN 1 TRTPN 1 TRTPN 3 TRTPN -1 TRTPN TRTPN APERIOD P1 APERIOD P2 APERIOD P3 APERIOD P4 APERIOD P5 APERIOD P6 ARMCD ABCEDF ARMCD BEAFCD ARMCD CADBFE ARMCD DCFAEB

Program: A\_Bio2.sas Created: 02APR2020 7:35 POSTLOCK

The Mixed Procedure

Parameter Code=REMAX

Coefficients for Bel 600 vs Oxy 30

Planned Planned

 $\begin{array}{c|cccc} & Arm & Treatment \\ \hline Effect & APERIOD\,Code & (N) & Row1 \\ \hline ARMCD & EFBDAC & & \\ \end{array}$ 

**FDECBA** 

ARMCD

Coefficients for Bel 600 vs 0xy 60
Planned Planned

Arm Treatment Effect APERIOD Code (N) Row1 Intercept TRTPN 1 TRTPN 1 TRTPN 3 TRTPN -1 TRTPN TRTPN APERIOD P1 APERIOD P2 APERIOD P3 APERIOD P4 APERIOD P5 APERIOD P6 ARMCD ABCEDF ARMCD BEAFCD ARMCD CADBFE ARMCD DCFAEB

Program: A\_Bio2.sas Created: 02APR2020 7:35 POSTLOCK


The Mixed Procedure

Parameter Code=REMAX

Coefficients for Bel 600 vs Oxy 60

Planned Planned

Arm Treatment Effect APERIOD Code (N) Row1

ARMCD EFBDAC ARMCD FDECBA

Coefficients for Bel 900 vs Oxy 30

Planned Planned

Arm Treatment Effect APERIOD Code (N) Row1 Intercept 1 TRTPN TRTPN 3 TRTPN 1 TRTPN -1 TRTPN TRTPN APERIOD P1 APERIOD P2 APERIOD P3 APERIOD P4 APERIOD P5 APERIOD P6 ARMCD ABCEDF ARMCD BEAFCD ARMCD CADBFE ARMCD DCFAEB

Program: A\_Bio2.sas Created: 02APR2020 7:35 POSTLOCK

The Mixed Procedure

Parameter Code=REMAX

Coefficients for Bel 900 vs Oxy 30

Planned Planned

Arm Treatment Effect APERIOD Code (N) Row1

ARMCD EFBDAC ARMCD FDECBA

Coefficients for Bel 900 vs Oxy 60

Planned Planned

Arm Treatment Effect APERIOD Code (N) Row1 Intercept 1 TRTPN TRTPN 3 TRTPN 1 TRTPN 5 -1 TRTPN TRTPN APERIOD P1 APERIOD P2 APERIOD P3 APERIOD P4 APERIOD P5 APERIOD P6 ARMCD ABCEDF ARMCD BEAFCD ARMCD CADBFE ARMCD DCFAEB

Program: A Bio2.sas Created: 02APR2020 7:35 POSTLOCK 

The Mixed Procedure

Parameter Code=REMAX

Coefficients for Bel 900 vs Oxy 60

Planned Planned

 Arm
 Treatment

 Effect
 APERIOD Code
 (N)
 Row1

 ARMCD
 EFBDAC

ARMCD FDECBA

Coefficients for Bel 300 vs Placebo

Planned Planned

| | | Arm | Treatment | |
|-----------|---------|--------|-----------|------|
| Effect | APERIOD | Code | (N) | Row1 |
| Intercept | | | | |
| TRTPN | | | 1 | 1 |
| TRTPN | | | 2 | |
| TRTPN | | | 3 | |
| TRTPN | | | 4 | |
| TRTPN | | | 5 | |
| TRTPN | | | 6 | -1 |
| APERIOD | P1 | | | |
| APERIOD | P2 | | | |
| APERIOD | P3 | | | |
| APERIOD | P4 | | | |
| APERIOD | P5 | | | |
| APERIOD | P6 | | | |
| ARMCD | | ABCEDF | | |
| ARMCD | | BEAFCD | | |
| ARMCD | | CADBFE | | |
| ARMCD | | DCFAEB | | |

The Mixed Procedure

Parameter Code=REMAX

Coefficients for Bel 300 vs Placebo

Planned Planned

Arm Treatment

| Effect | APERIOD Code | (N) | Row1 |
|--------|--------------|-----|------|
| ARMCD | EFBDAC | | |
| ARMCD | FDECBA | | |

Coefficients for Bel 600 vs Placebo

Planned Planned

Arm Treatment Effect APERIOD Code (N) Row1 Intercept TRTPN 1 TRTPN 1 TRTPN 3 TRTPN TRTPN TRTPN -1 APERIOD P1 APERIOD P2 APERIOD P3 APERIOD P4 APERIOD P5 APERIOD P6 ARMCD ABCEDF ARMCD BEAFCD ARMCD CADBFE

Program: A Bio2.sas Created: 02APR2020 7:35 POSTLOCK 

DCFAEB

ARMCD

The Mixed Procedure

Parameter Code=REMAX

Coefficients for Bel 600 vs Placebo

Planned Planned

Arm Treatment

Effect APERIOD Code (N) Row1

ARMCD EFBDAC ARMCD FDECBA

Coefficients for Bel 900 vs Placebo

Planned Planned

Arm Treatment Effect APERIOD Code (N) Row1 Intercept 1 TRTPN TRTPN 3 TRTPN 1 TRTPN TRTPN TRTPN -1 APERIOD P1 APERIOD P2 APERIOD P3 APERIOD P4 APERIOD P5 APERIOD P6 ARMCD ABCEDF ARMCD BEAFCD ARMCD CADBFE ARMCD DCFAEB

# Appendix 16.1.9.2.2 Statistical Methods and Analysis Output Supporting Table 14.2.3 Supporting Table 14.2.3

The Mixed Procedure

#### Parameter Code=REMAX

Coefficients for Bel 900 vs Placebo

Planned Planned

Arm Treatment

Effect APERIOD Code (N) Row1
ARMCD EFBDAC
ARMCD FDECBA

#### Estimates

#### Standard

| Label | Estimate | Error DF t | Value H | ?r > t <i>i</i> | Alpha | Lower | Upper |
|---|---|---|---|---|---|---|---|
| Oxy 30 vs Placebo | -21.2343 | 44.208467 | -0.48 | 0.6326 | 0.05 | -109.47 | 67.0060 |
| Oxy 60 vs Placebo | -131.81 | 43.385567 | -3.04 | 0.0034 | 0.05 | -218.41 | -45.2147 |
| Bel 300 vs Oxy 30 | 64.6649 | 44.820767 | 1.44 | 0.1538 | 0.05 | -24.7977 | 154.13 |
| Bel 300 vs Oxy 60 | 175.24 | 44.207267 | 3.96 | 0.0002 | 0.05 | 87.0052 | 263.48 |
| Bel 600 vs Oxy 30 | 14.7699 | 44.225767 | 0.33 | 0.7394 | 0.05 | -73.5049 | 103.04 |
| Bel 600 vs Oxy 60 | 125.35 | 43.382267 | 2.89 | 0.0052 | 0.05 | 38.7567 | 211.94 |
| Bel 900 vs Oxy 30 | 50.0157 | 44.816867 | 1.12 | 0.2684 | 0.05 | -39.4390 | 139.47 |
| Bel 900 vs Oxy 60 | 160.59 | 44.224567 | 3.63 | 0.0005 | 0.05 | 72.3214 | 248.87 |
| Bel 300 vs Placebo | 43.4306 | 44.186867 | 0.98 | 0.3292 | 0.05 | -44.7665 | 131.63 |
| Bel 600 vs Placebo | -6.4645 | 43.294767 | -0.15 | 0.8818 | 0.05 | -92.8811 | 79.9522 |
| Bel 900 vs Placebo | 28.7813 | 44.208567 | 0.65 | 0.5172 | 0.05 | -59.4592 | 117.02 |

Program: A Bio2.sas Created: 02APR2020 7:35 POSTLOCK 

# Appendix 16.1.9.2.2 Statistical Methods and Analysis Output Supporting Table 14.2.3 Supporting Table 14.2.3

The Mixed Procedure

Parameter Code=REMAX

Least Squares Means

| | | | _ | | | | |
|---|---|---|---|---|---|---|---|
| | Planned | | | | | | |
| | Treatment | | Standard | | | | |
| Effect | (N) | Estimate | Error DF t | Value | Pr > t 2 | Alpha Lower | Upper |
| TRTPN | 1 | 582.53 | 38.167267 | 15.26 | <.0001 | 0.1518.87 | 646.19 |
| TRTPN | 2 | 532.64 | 37.194267 | 14.32 | <.0001 | 0.1470.60 | 594.67 |
| TRTPN | 3 | 567.88 | 38.188367 | 14.87 | <.0001 | 0.1504.19 | 631.58 |
| TRTPN | 4 | 517.87 | 38.188267 | 13.56 | <.0001 | 0.1454.17 | 581.56 |
| TRTPN | 5 | 407.29 | 37.193867 | 10.95 | <.0001 | 0.1345.25 | 469.33 |
| TRTPN | 6 | 539.10 | 37.192367 | 14.49 | <.0001 | 0.1477.07 | 601.14 |

Differences of Least Squares Means

Planned Planned

| | rianneu | rianneu | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| | Treatment | Treatment | : | Standard | | | | | |
| Effect | (N) | (N) | Estimate | Error DF t | Value F | ?r > t | Alpha | Lower | Upper |
| TRTPN | 1 | 2 | 49.8950 | 44.297767 | 1.13 | 0.2640 | 0.1-2 | 3.9897 | 123.78 |
| TRTPN | 1 | 3 | 14.6493 | 44.814567 | 0.33 | 0.7448 | 0.1-6 | 0.0975 | 89.3960 |
| TRTPN | 1 | 4 | 64.6649 | 44.820767 | 1.44 | 0.1538 | 0.1-1 | 0.0923 | 139.42 |
| TRTPN | 1 | 5 | 175.24 | 44.207267 | 3.96 | 0.0002 | 0.1 | 101.51 | 248.98 |
| TRTPN | 1 | 6 | 43.4306 | 44.186867 | 0.98 | 0.3292 | 0.1-3 | 0.2692 | 117.13 |
| TRTPN | 2 | 3 | -35.2458 | 44.231767 | -0.80 | 0.4284 | 0.1 - | 109.02 | 38.5290 |
| TRTPN | 2 | 4 | 14.7699 | 44.225767 | 0.33 | 0.7394 | 0.1-5 | 8.9948 | 88.5345 |
| TRTPN | 2 | 5 | 125.35 | 43.382267 | 2.89 | 0.0052 | 0.1 5 | 2.9901 | 197.71 |
| TRTPN | 2 | 6 | -6.4645 | 43.294767 | -0.15 | 0.8818 | 0.1-7 | 8.6764 | 65.7475 |
| TRTPN | 3 | 4 | 50.0157 | 44.816867 | 1.12 | 0.2684 | 0.1-2 | 4.7350 | 124.77 |
| TRTPN | 3 | 5 | 160.59 | 44.224567 | 3.63 | 0.0005 | 0.1 8 | 6.8311 | 234.36 |
| TRTPN | 3 | 6 | 28.7813 | 44.208567 | 0.65 | 0.5172 | 0.1 - 4 | 4.9547 | 102.52 |
| TRTPN | 4 | 5 | 110.58 | 44.224467 | 2.50 | 0.0149 | 0.1 3 | 6.8155 | 184.34 |

Program: A Bio2.sas Created: 02APR2020 7:35 POSTLOCK 

# Appendix 16.1.9.2.2 Statistical Methods and Analysis Output Supporting Table 14.2.3 Supporting Table 14.2.3

# The Mixed Procedure

#### Parameter Code=REMAX

# Differences of Least Squares Means

Planned Planned Treatment Treatment

| | Treatment | Treatment | | Standard | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| Effect | (N) | (N) | Estimate | Error DF t | Value Pr | c > t | Alpha | Lower | Upper |
| TRTPN | 4 | 6 | -21.2343 | 44.208467 | -0.48 | 0.6326 | 0.1- | -94.9702 | 52.5016 |
| TRTPN | 5 | 6 | -131.81 | 43.385567 | -3.04 | 0.0034 | 0.1 | -204.18 | -59.4492 |

 Program: A\_Bio2.sas Created: 02APR2020 7:35 POSTLOCK

# Appendix 16.1.9.2.2 Statistical Methods and Analysis Output Supporting Table 14.2.3 Supporting Table 14.2.3

# The Mixed Procedure

#### Parameter Code=RRSPEMAX

#### Model Information

| Data Set | WORK.ADXV |
|---------------------------|---------------------|
| Dependent Variable | AVAL |
| Covariance Structure | Variance Components |
| Estimation Method | REML |
| Residual Variance Method | Profile |
| Fixed Effects SE Method | Model-Based |
| Degrees of Freedom Method | Containment |

#### Class Level Information

| Class | LevelsValues |
|---|---|
| SUBJID | 161001 1002 1003 1004 1005 1006 1007 1008 1010 1012 1013 1014 1015 1016 1017 1018 |
| TRTPN | 61 2 3 4 5 6 |
| APERIOD | 6P1 P2 P3 P4 P5 P6 |
| ARMCD | 6ABCEDF BEAFCD CADBFE DCFAEB EFBDAC FDECBA |

| Dimensions | | |
|-------------|------------|----|
| Covariance | Parameters | 2 |
| Columns in | X | 19 |
| Columns in | Z | 16 |
| Subjects | | 1 |
| Max Obs per | Subject | 93 |

Program: A Bio2.sas Created: 02APR2020 7:35 POSTLOCK 

# Appendix 16.1.9.2.2 Statistical Methods and Analysis Output Supporting Table 14.2.3 Supporting Table 14.2.3

The Mixed Procedure

#### Parameter Code=RRSPEMAX

| | Nι | umber of Obse | rvations | |
|--------|----|---------------|----------|----|
| Number | of | Observations | Read | 93 |
| Number | of | Observations | Used | 93 |
| Number | of | Observations | Not Used | 0 |

# Iteration History

| Iteration Evaluat | ions -2 | Res | Log | Like | Criterion |
|-------------------|---------|-----|-------|-------|------------|
| 0 | 1 | 462 | .4120 | 08316 | _ |
| 1 | 3 | 434 | .2531 | 16146 | 0.00000768 |
| 2 | 1 | 434 | 2520 | 11500 | 0 0000001 |

Convergence criteria met.

# Covariance Parameter Estimates

| Cov Parm | Estimate |
|----------------|----------|
| SUBJID (ARMCD) | 8.5079 |
| Residual | 7.5427 |

# Fit Statistics

| -2 Res Log Likelihood | 434.3 |
|--------------------------|-------|
| AIC (Smaller is Better) | 438.3 |
| AICC (Smaller is Better) | 438.4 |
| BIC (Smaller is Better) | 439.8 |

Program: A Bio2.sas Created: 02APR2020 7:35 POSTLOCK 

The Mixed Procedure

# Parameter Code=RRSPEMAX

Type 3 Tests of Fixed Effects

| 1 | NumI | | |
|---------|------|------|--------------|
| Effect | DF | DF F | Value Pr > F |
| TRTPN | 5 | 67 | 1.080.3818 |
| APERIOD | 5 | 67 | 1.120.3558 |
| ARMCD | 5 | 10 | 0.810.5698 |

# Coefficients for Oxy 30 vs Placebo Planned Planned

| - | | <br>- | | | | ~ | |
|----|----|-------|----|-------|---|-----|---|
| 7\ | rm | T | 20 | · > + | m | ont | + |

| | | Arm | Treatment | |
|-----------|---------|--------|-----------|------|
| Effect | APERIOD | Code | (N) | Row1 |
| Intercept | | | | |
| TRTPN | | | 1 | |
| TRTPN | | | 2 | |
| TRTPN | | | 3 | |
| TRTPN | | | 4 | 1 |
| TRTPN | | | 5 | |
| TRTPN | | | 6 | -1 |
| APERIOD | P1 | | | |
| APERIOD | P2 | | | |
| APERIOD | P3 | | | |
| APERIOD | P4 | | | |
| APERIOD | P5 | | | |
| APERIOD | P6 | | | |
| ARMCD | | ABCEDF | | |
| ARMCD | | BEAFCD | | |
| ARMCD | | CADBFE | | |
| ARMCD | | DCFAEB | | |

Program: A Bio2.sas Created: 02APR2020 7:35 POSTLOCK 

The Mixed Procedure

#### Parameter Code=RRSPEMAX

Coefficients for Oxy 30 vs Placebo

Planned Planned

Arm Treatment
Effect APERIOD Code (N) Row1
ARMCD EFBDAC
ARMCD FDECBA

Coefficients for Oxy 60 vs Placebo

Planned Planned Arm Treatment

| | | ATIII | Treatment | |
|-----------|---------|--------|-----------|------|
| Effect | APERIOD | Code | (N) | Row1 |
| Intercept | | | | |
| TRTPN | | | 1 | |
| TRTPN | | | 2 | |
| TRTPN | | | 3 | |
| TRTPN | | | 4 | |
| TRTPN | | | 5 | 1 |
| TRTPN | | | 6 | -1 |
| APERIOD | P1 | | | |
| APERIOD | P2 | | | |
| APERIOD | Р3 | | | |
| APERIOD | P4 | | | |
| APERIOD | P5 | | | |
| APERIOD | P6 | | | |
| ARMCD | | ABCEDF | | |
| ARMCD | | BEAFCD | | |
| ARMCD | | CADBFE | | |
| ARMCD | | DCFAEB | | |

#### The Mixed Procedure

#### Parameter Code=RRSPEMAX

# Coefficients for Oxy 60 vs Placebo

Planned Planned

 Arm
 Treatment

 Effect
 APERIOD Code
 (N)
 Row1

 ARMCD
 EFBDAC

 ARMCD
 FDECBA

# Coefficients for Bel 300 vs Oxy 30

Planned Planned
Arm Treatment

| | | 211111 | I I Ca chich | - |
|-----------|---------|--------|--------------|------|
| Effect | APERIOD | Code | (N) | Row1 |
| Intercept | _ | | | |
| TRTPN | | | 1 | 1 |
| TRTPN | | | 2 | |
| TRTPN | | | 3 | |
| TRTPN | | | 4 | -1 |
| TRTPN | | | 5 | |
| TRTPN | | | 6 | |
| APERIOD | P1 | | | |
| APERIOD | P2 | | | |
| APERIOD | Р3 | | | |
| APERIOD | P4 | | | |
| APERIOD | P5 | | | |
| APERIOD | P6 | | | |
| ARMCD | | ABCEDF | | |
| ARMCD | | BEAFCD | | |
| ARMCD | | CADBFE | | |
| ARMCD | | DCFAEB | | |

Program: A Bio2.sas Created: 02APR2020 7:35 POSTLOCK 

#### The Mixed Procedure

#### Parameter Code=RRSPEMAX

Coefficients for Bel 300 vs Oxy 30

Planned Planned

 Arm
 Treatment

 Effect
 APERIOD Code
 (N)
 Row1

 ARMCD
 EFBDAC

 ARMCD
 FDECBA

Coefficients for Bel 300 vs Oxy 60

Planned Planned
Arm Treatment

| | | Arm | Treatment | |
|-----------|--------|--------|-----------|------|
| Effect | APERIO | ) Code | (N) | Row1 |
| Intercept | | | | |
| TRTPN | | | 1 | 1 |
| TRTPN | | | 2 | |
| TRTPN | | | 3 | |
| TRTPN | | | 4 | |
| TRTPN | | | 5 | -1 |
| TRTPN | | | 6 | |
| APERIOD | P1 | | | |
| APERIOD | P2 | | | |
| APERIOD | P3 | | | |
| APERIOD | P4 | | | |
| APERIOD | P5 | | | |
| APERIOD | P6 | | | |
| ARMCD | | ABCEDF | | |
| ARMCD | | BEAFCD | | |
| ARMCD | | CADBFE | | |
| ARMCD | | DCFAEB | | |

#### The Mixed Procedure

#### Parameter Code=RRSPEMAX

Coefficients for Bel 300 vs Oxy 60

Planned Planned

 Arm
 Treatment

 Effect
 APERIOD Code
 (N)
 Row1

 ARMCD
 EFBDAC

 ARMCD
 FDECBA

Coefficients for Bel 600 vs Oxy 30
Planned Planned

Arm Treatment

| | | ATIII | I I E a CIII E II C | |
|-----------|---------|--------|---------------------|------|
| Effect | APERIOD | Code | (N) | Row1 |
| Intercept | | | | |
| TRTPN | | | 1 | |
| TRTPN | | | 2 | 1 |
| TRTPN | | | 3 | |
| TRTPN | | | 4 | -1 |
| TRTPN | | | 5 | |
| TRTPN | | | 6 | |
| APERIOD | P1 | | | |
| APERIOD | P2 | | | |
| APERIOD | P3 | | | |
| APERIOD | P4 | | | |
| APERIOD | P5 | | | |
| APERIOD | P6 | | | |
| ARMCD | | ABCEDF | | |
| ARMCD | | BEAFCD | | |
| ARMCD | | CADBFE | | |
| ARMCD | | DCFAEB | | |

Program: A Bio2.sas Created: 02APR2020 7:35 POSTLOCK 

# The Mixed Procedure

#### Parameter Code=RRSPEMAX

Coefficients for Bel 600 vs Oxy 30

Planned Planned

 Arm
 Treatment

 Effect
 APERIOD Code
 (N)
 Row1

 ARMCD
 EFBDAC

 ARMCD
 FDECBA

Coefficients for Bel 600 vs 0xy 60
Planned Planned

Arm Treatment

| | | ATIII | TTEatment | |
|-----------|---------|--------|-----------|------|
| Effect | APERIOD | Code | (N) | Row1 |
| Intercept | | | | |
| TRTPN | | | 1 | |
| TRTPN | | | 2 | 1 |
| TRTPN | | | 3 | |
| TRTPN | | | 4 | |
| TRTPN | | | 5 | -1 |
| TRTPN | | | 6 | |
| APERIOD | P1 | | | |
| APERIOD | P2 | | | |
| APERIOD | Р3 | | | |
| APERIOD | P4 | | | |
| APERIOD | P5 | | | |
| APERIOD | P6 | | | |
| ARMCD | | ABCEDF | | |
| ARMCD | | BEAFCD | | |
| ARMCD | | CADBFE | | |
| ARMCD | | DCFAEB | | |

Program: A Bio2.sas Created: 02APR2020 7:35 POSTLOCK 

The Mixed Procedure

#### Parameter Code=RRSPEMAX

Coefficients for Bel 600 vs Oxy 60

Planned Planned

 Arm
 Treatment

 Effect
 APERIOD Code
 (N)
 Row1

 ARMCD
 EFBDAC

 ARMCD
 FDECBA

Coefficients for Bel 900 vs Oxy 30
Planned Planned

Arm Treatment

| | | 232111 | IICUC | THCTT C |
|---------|-------|---------|-------|---------|
| Effect | APERI | OD Code | (N) | Row1 |
| Interce | pt | | | |
| TRTPN | | | 1 | |
| TRTPN | | | 2 | |
| TRTPN | | | 3 | 1 |
| TRTPN | | | 4 | -1 |
| TRTPN | | | 5 | |
| TRTPN | | | 6 | |
| APERIOD | P1 | | | |
| APERIOD | P2 | | | |
| APERIOD | P3 | | | |
| APERIOD | P4 | | | |
| APERIOD | P5 | | | |
| APERIOD | P6 | | | |
| ARMCD | | ABCED | F | |
| ARMCD | | BEAFC | D | |
| ARMCD | | CADBF | Ε | |
| ARMCD | | DCFAE | В | |

Program: A Bio2.sas Created: 02APR2020 7:35 POSTLOCK 

# The Mixed Procedure

#### Parameter Code=RRSPEMAX

Coefficients for Bel 900 vs Oxy 30

Planned Planned

| Arm | Treatment | Effect | APERIOD Code | (N) | Row1 | ARMCD | EFBDAC |

**FDECBA** 

ARMCD

Coefficients for Bel 900 vs 0xy 60
Planned Planned

Arm Treatment Effect APERIOD Code (N) Row1 Intercept 1 TRTPN TRTPN 2 3 TRTPN 1 TRTPN 5 -1 TRTPN TRTPN APERIOD P1 APERIOD P2 APERIOD P3 APERIOD P4 APERIOD P5 APERIOD P6 ARMCD ABCEDF ARMCD BEAFCD ARMCD CADBFE ARMCD DCFAEB

Program: A Bio2.sas Created: 02APR2020 7:35 POSTLOCK 

# The Mixed Procedure

#### Parameter Code=RRSPEMAX

Coefficients for Bel 900 vs Oxy 60

Planned Planned

Arm Treatment

Effect APERIOD Code (N) Row1

ARMCD EFBDAC ARMCD FDECBA

Coefficients for Bel 300 vs Placebo

Planned Planned

Arm Treatment Effect APERIOD Code (N) Row1 Intercept 1 TRTPN 1 TRTPN TRTPN 3 TRTPN TRTPN TRTPN -1 APERIOD P1 APERIOD P2 APERIOD P3 APERIOD P4 APERIOD P5 APERIOD P6 ARMCD ABCEDF ARMCD BEAFCD ARMCD CADBFE ARMCD DCFAEB

#### The Mixed Procedure

#### Parameter Code=RRSPEMAX

# Coefficients for Bel 300 vs Placebo

Planned Planned

 Arm
 Treatment

 Effect
 APERIOD Code
 (N)
 Row1

 ARMCD
 EFBDAC

ARMCD EFBDAC ARMCD FDECBA

# Coefficients for Bel 600 vs Placebo

Planned Planned

| | | Arm | Treatment | |
|-----------|--------|--------|-----------|------|
| Effect | APERIO | ) Code | (N) | Row1 |
| Intercept | | | | |
| TRTPN | | | 1 | |
| TRTPN | | | 2 | 1 |
| TRTPN | | | 3 | |
| TRTPN | | | 4 | |
| TRTPN | | | 5 | |
| TRTPN | | | 6 | -1 |
| APERIOD | P1 | | | |
| APERIOD | P2 | | | |
| APERIOD | Р3 | | | |
| APERIOD | P4 | | | |
| APERIOD | P5 | | | |
| APERIOD | P6 | | | |
| ARMCD | | ABCEDF | | |
| ARMCD | | BEAFCD | | |
| ARMCD | | CADBFE | | |
| ARMCD | | DCFAEB | | |
#### The Mixed Procedure

#### Parameter Code=RRSPEMAX

### Coefficients for Bel 600 vs Placebo

Planned Planned

## Coefficients for Bel 900 vs Placebo

Planned Planned

| | | Arm | Treatment | |
|-----------|--------|--------|-----------|------|
| Effect | APERIO | ) Code | (N) | Row1 |
| Intercept | : | | | |
| TRTPN | | | 1 | |
| TRTPN | | | 2 | |
| TRTPN | | | 3 | 1 |
| TRTPN | | | 4 | |
| TRTPN | | | 5 | |
| TRTPN | | | 6 | -1 |
| APERIOD | P1 | | | |
| APERIOD | P2 | | | |
| APERIOD | P3 | | | |
| APERIOD | P4 | | | |
| APERIOD | P5 | | | |
| APERIOD | P6 | | | |
| ARMCD | | ABCEDF | | |
| ARMCD | | BEAFCD | | |
| ARMCD | | CADBFE | | |
| ARMCD | | DCFAEB | | |


## Appendix 16.1.9.2.2 Statistical Methods and Analysis Output Supporting Table 14.2.3 Supporting Table 14.2.3

#### The Mixed Procedure

#### Parameter Code=RRSPEMAX

Coefficients for Bel 900 vs Placebo

Planned Planned

Arm Treatment

Effect APERIOD Code (N) Row1
ARMCD EFBDAC
ARMCD FDECBA

#### Estimates

#### Standard

| Label | Estimate | Error DF t | Value P | r > t 2 | Alpha Lower | Upper |
|---|---|---|---|---|---|---|
| Oxy 30 vs Placebo | -1.6707 | 0.994367 | -1.68 | 0.0976 | 0.05-3.6554 | 0.3140 |
| Oxy 60 vs Placebo | -2.1015 | 0.975067 | -2.16 | 0.0347 | 0.05-4.0476 | -0.1553 |
| Bel 300 vs Oxy 30 | 0.4163 | 1.007367 | 0.41 | 0.6807 | 0.05-1.5943 | 2.4268 |
| Bel 300 vs Oxy 60 | 0.8470 | 0.994367 | 0.85 | 0.3973 | 0.05-1.1376 | 2.8316 |
| Bel 600 vs Oxy 30 | 0.4418 | 0.994867 | 0.44 | 0.6584 | 0.05-1.5438 | 2.4275 |
| Bel 600 vs Oxy 60 | 0.8726 | 0.974967 | 0.89 | 0.3740 | 0.05-1.0734 | 2.8186 |
| Bel 900 vs Oxy 30 | 0.05551 | 1.007267 | 0.06 | 0.9562 | 0.05-1.9548 | 2.0659 |
| Bel 900 vs Oxy 60 | 0.4862 | 0.994867 | 0.49 | 0.6266 | 0.05-1.4993 | 2.4718 |
| Bel 300 vs Placebo | -1.2544 | 0.993767 | -1.26 | 0.2112 | 0.05-3.2379 | 0.7291 |
| Bel 600 vs Placebo | -1.2289 | 0.973067 | -1.26 | 0.2110 | 0.05-3.1710 | 0.7132 |
| Bel 900 vs Placebo | -1.6152 | 0.994367 | -1.62 | 0.1090 | 0.05 - 3.5999 | 0.3695 |

Program: A Bio2.sas Created: 02APR2020 7:35 POSTLOCK 

## Appendix 16.1.9.2.2 Statistical Methods and Analysis Output Supporting Table 14.2.3 Supporting Table 14.2.3

#### The Mixed Procedure

#### Parameter Code=RRSPEMAX

### Least Squares Means

| | Planned | | | | | | | |
|---|---|---|---|---|---|---|---|---|
| | Treatment | | Standard | | | | | |
| Effect | (N) | Estimate | Error DF t | Value | Pr > t | Alpha | Lower | Upper |
| TRTPN | 1 | 15.4944 | 1.032967 | 15.00 | <.0001 | 0.13 | 13.7716 | 17.2171 |
| TRTPN | 2 | 15.5199 | 1.014167 | 15.30 | <.0001 | 0.11 | 13.8285 | 17.2114 |
| TRTPN | 3 | 15.1336 | 1.033467 | 14.64 | <.0001 | 0.11 | 13.4100 | 16.8572 |
| TRTPN | 4 | 15.0781 | 1.033467 | 14.59 | <.0001 | 0.11 | 13.3545 | 16.8017 |
| TRTPN | 5 | 14.6473 | 1.014167 | 14.44 | <.0001 | 0.11 | 12.9559 | 16.3388 |
| TRTPN | 6 | 16.7488 | 1.014167 | 16.52 | <.0001 | 0.11 | 15.0574 | 18.4402 |

## Differences of Least Squares Means

| | | | | | 1 | | | |
|---|---|---|---|---|---|---|---|---|
| | Planned | Planned | | | | | | |
| | Treatment | Treatment | S | tandard | | | | |
| Effect | (N) | (N) | Estimate | Error DF t | Value P | r > t A | lpha Lower | Upper |
| TRTPN | 1 | 2 | -0.02556 | 0.996367 | -0.03 | 0.9796 | 0.1-1.6873 | 1.6362 |
| TRTPN | 1 | 3 | 0.3608 | 1.007167 | 0.36 | 0.7213 | 0.1-1.3191 | 2.0406 |
| TRTPN | 1 | 4 | 0.4163 | 1.007367 | 0.41 | 0.6807 | 0.1-1.2638 | 2.0963 |
| TRTPN | 1 | 5 | 0.8470 | 0.994367 | 0.85 | 0.3973 | 0.1-0.8114 | 2.5054 |
| TRTPN | 1 | 6 | -1.2544 | 0.993767 | -1.26 | 0.2112 | 0.1-2.9119 | 0.4030 |
| TRTPN | 2 | 3 | 0.3863 | 0.995067 | 0.39 | 0.6990 | 0.1-1.2732 | 2.0458 |
| TRTPN | 2 | 4 | 0.4418 | 0.994867 | 0.44 | 0.6584 | 0.1-1.2174 | 2.1011 |
| TRTPN | 2 | 5 | 0.8726 | 0.974967 | 0.89 | 0.3740 | 0.1-0.7536 | 2.4987 |
| TRTPN | 2 | 6 | -1.2289 | 0.973067 | -1.26 | 0.2110 | 0.1-2.8517 | 0.3940 |
| TRTPN | 3 | 4 | 0.05551 | 1.007267 | 0.06 | 0.9562 | 0.1-1.6244 | 1.7354 |
| TRTPN | 3 | 5 | 0.4862 | 0.994867 | 0.49 | 0.6266 | 0.1-1.1730 | 2.1455 |
| TRTPN | 3 | 6 | -1.6152 | 0.994367 | -1.62 | 0.1090 | 0.1-3.2737 | 0.04324 |
| TRTPN | 4 | 5 | 0.4307 | 0.994867 | 0.43 | 0.6664 | 0.1-1.2285 | 2.0900 |

Program: A Bio2.sas Created: 02APR2020 7:35 POSTLOCK 

Appendix 16.1.9.2.2
Statistical Methods and Analysis Output Supporting Table 14.2.3
Supporting Table 14.2.3

#### The Mixed Procedure

#### Parameter Code=RRSPEMAX

## Differences of Least Squares Means

| | Planned | Planned | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| | Treatment | Treatment | S | tandard | | | | | |
| Effect | (N) | (N) | Estimate | Error DF t | Value Pr | r > t | Alpha | Lower | Upper |
| TRTPN | 4 | 6 | -1.6707 | 0.994367 | -1.68 | 0.0976 | 0.1 | -3.3292 - | -0.01227 |
| TRTPN | 5 | 6 | -2.1015 | 0.975067 | -2.16 | 0.0347 | 0.1 | -3.7277 | -0.4752 |

Program: A\_Bio2.sas Created: 02APR2020 7:35 POSTLOCK 

# Appendix 16.1.9.2.2 Statistical Methods and Analysis Output Supporting Table 14.2.3 Supporting Table 14.2.3

#### The Mixed Procedure

#### Parameter Code=SEMAX

#### Model Information

| Data Set | WORK.ADXV |
|---------------------------|---------------------|
| Dependent Variable | AVAL |
| Covariance Structure | Variance Components |
| Estimation Method | REML |
| Residual Variance Method | Profile |
| Fixed Effects SE Method | Model-Based |
| Degrees of Freedom Method | Containment |

#### Class Level Information

| Class | LevelsValues |
|---|---|
| SUBJID | 161001 1002 1003 1004 1005 1006 1007 1008 1010 1012 1013 1014 1015 1016 1017 1018 |
| TRTPN | 61 2 3 4 5 6 |
| APERIOD | O 6P1 P2 P3 P4 P5 P6 |
| ARMCD | 6ABCEDF BEAFCD CADBFE DCFAEB EFBDAC FDECBA |

| Dimensions | | |
|-------------|------------|----|
| Covariance | Parameters | 2 |
| Columns in | X | 19 |
| Columns in | Z | 16 |
| Subjects | | 1 |
| Max Obs per | Subject | 93 |

Program: A Bio2.sas Created: 02APR2020 7:35 POSTLOCK 

## Appendix 16.1.9.2.2 Statistical Methods and Analysis Output Supporting Table 14.2.3 Supporting Table 14.2.3

The Mixed Procedure

#### Parameter Code=SEMAX

| Number of Observations | | |
|------------------------|----------------|------------|
| Number o | f Observations | Read 93 |
| Number o | f Observations | Used 93 |
| Number o | f Observations | Not Used 0 |

### Iteration History

| Iteration Evaluati | ons - | 2 Res | Log | Like | Criterion |
|--------------------|-------|-------|-------|-------|------------|
| 0 | 1 | 1200 | .5512 | 13258 | |
| 1 | 2 | 1196 | .4471 | 10417 | 0.0000001 |
| 2 | 1 | 1196 | .4470 | 9777 | 0.00000000 |

Convergence criteria met.

## Covariance Parameter Estimates

| Cov | Parm | Estimate |
|------|------------|----------|
| SUBJ | JID(ARMCD) | 41275 |
| Resi | idual | 174256 |

#### Fit Statistics

| -2 Res Log Likelihood | 1196.4 |
|--------------------------|--------|
| AIC (Smaller is Better) | 1200.4 |
| AICC (Smaller is Better) | 1200.6 |
| BIC (Smaller is Better) | 1202.0 |

Program: A Bio2.sas Created: 02APR2020 7:35 POSTLOCK 

The Mixed Procedure

Parameter Code=SEMAX

Type 3 Tests of Fixed Effects
Num Den

| Effect | DF | DF F | Value Pr > F |
|---------|----|------|--------------|
| TRTPN | 5 | 67 | 3.070.0149 |
| APERIOD | 5 | 67 | 3.410.0083 |
| ARMCD | 5 | 10 | 1.210.3725 |

Coefficients for Oxy 30 vs Placebo Planned Planned

| | | Arm | Treatment | |
|-----------|---------|--------|-----------|------|
| Effect | APERIOD | Code | (N) | Row1 |
| Intercept | ; | | | |
| TRTPN | | | 1 | |
| TRTPN | | | 2 | |
| TRTPN | | | 3 | |
| TRTPN | | | 4 | 1 |
| TRTPN | | | 5 | |
| TRTPN | | | 6 | -1 |
| APERIOD | P1 | | | |
| APERIOD | P2 | | | |
| APERIOD | Р3 | | | |
| APERIOD | P4 | | | |
| APERIOD | P5 | | | |
| APERIOD | P6 | | | |
| ARMCD | | ABCEDF | | |
| ARMCD | | BEAFCD | | |
| ARMCD | | CADBFE | | |
| ARMCD | | DCFAEB | | |

Program: A Bio2.sas Created: 02APR2020 7:35 POSTLOCK 

The Mixed Procedure

Parameter Code=SEMAX

Coefficients for Oxy 30 vs Placebo

Planned Planned

 $\begin{array}{ccc} & & \text{Arm} & \text{Treatment} \\ \hline \text{Effect} & \text{APERIOD\,Code} & \text{(N)} & \text{Row1} \\ \hline \text{ARMCD} & & \text{EFBDAC} \\ \end{array}$ 

ARMCD

Coefficients for Oxy 60 vs Placebo

FDECBA

Planned Planned

| | | Arm | Treatment | |
|-----------|---------|--------|-----------|------|
| Effect | APERIOD | Code | (N) | Row1 |
| Intercept | | | | |
| TRTPN | | | 1 | |
| TRTPN | | | 2 | |
| TRTPN | | | 3 | |
| TRTPN | | | 4 | |
| TRTPN | | | 5 | 1 |
| TRTPN | | | 6 | -1 |
| APERIOD | P1 | | | |
| APERIOD | P2 | | | |
| APERIOD | P3 | | | |
| APERIOD | P4 | | | |
| APERIOD | P5 | | | |
| APERIOD | P6 | | | |
| ARMCD | | ABCEDF | | |
| ARMCD | | BEAFCD | | |
| ARMCD | | CADBFE | | |
| ARMCD | | DCFAEB | | |

The Mixed Procedure

Parameter Code=SEMAX

Coefficients for Oxy 60 vs Placebo

Planned Planned

 Arm
 Treatment

 Effect
 APERIOD Code
 (N)
 Row1

 ARMCD
 EFBDAC

ARMCD EFBDAC FDECBA

Coefficients for Bel 300 vs Oxy 30

Planned Planned

Arm Treatment Effect APERIOD Code (N) Row1 Intercept 1 TRTPN 1 TRTPN TRTPN 3 TRTPN -1 TRTPN TRTPN APERIOD P1 APERIOD P2 APERIOD P3 APERIOD P4 APERIOD P5 APERIOD P6 ARMCD ABCEDF ARMCD BEAFCD ARMCD CADBFE ARMCD DCFAEB

Program: A\_Bio2.sas Created: 02APR2020 7:35 POSTLOCK

The Mixed Procedure

Parameter Code=SEMAX

Coefficients for Bel 300 vs Oxy 30

Planned Planned

 $\begin{array}{c|cccc} & & Arm & Treatment \\ \hline Effect & APERIOD\,Code & (N) & Row1 \\ \hline ARMCD & EFBDAC \end{array}$ 

ARMCD EFBDAC ARMCD FDECBA

Coefficients for Bel 300 vs Oxy 60

Planned Planned
Arm Treatment

| | | Arm | Treatment | |
|-----------|--------|--------|-----------|------|
| Effect | APERIO | ) Code | (N) | Row1 |
| Intercept | | | | |
| TRTPN | | | 1 | 1 |
| TRTPN | | | 2 | |
| TRTPN | | | 3 | |
| TRTPN | | | 4 | |
| TRTPN | | | 5 | -1 |
| TRTPN | | | 6 | |
| APERIOD | P1 | | | |
| APERIOD | P2 | | | |
| APERIOD | P3 | | | |
| APERIOD | P4 | | | |
| APERIOD | P5 | | | |
| APERIOD | P6 | | | |
| ARMCD | | ABCEDF | | |
| ARMCD | | BEAFCD | | |
| ARMCD | | CADBFE | | |
| ARMCD | | DCFAEB | | |

The Mixed Procedure

Parameter Code=SEMAX

Coefficients for Bel 300 vs Oxy 60

Planned Planned

Coefficients for Bel 600 vs 0xy 30 Planned Planned

Arm Treatment Effect APERIOD Code (N) Row1 Intercept TRTPN 1 TRTPN 1 TRTPN 3 TRTPN -1 TRTPN TRTPN APERIOD P1 APERIOD P2 APERIOD P3 APERIOD P4 APERIOD P5 APERIOD P6 ARMCD ABCEDF ARMCD BEAFCD ARMCD CADBFE

DCFAEB

Program: A\_Bio2.sas Created: 02APR2020 7:35 POSTLOCK

ARMCD

The Mixed Procedure

Parameter Code=SEMAX

Coefficients for Bel 600 vs 0xy 30

Planned Planned

Arm Treatment
Effect APERIOD Code (N) Row1

ARMCD EFBDAC
ARMCD FDECBA

Coefficients for Bel 600 vs Oxy 60

Planned Planned

Arm Treatment

| | | ALIII | Treatment | • |
|-----------|---------|--------|-----------|------|
| Effect | APERIOD | Code | (N) | Row1 |
| Intercept | | | | |
| TRTPN | | | 1 | |
| TRTPN | | | 2 | 1 |
| TRTPN | | | 3 | |
| TRTPN | | | 4 | |
| TRTPN | | | 5 | -1 |
| TRTPN | | | 6 | |
| APERIOD | P1 | | | |
| APERIOD | P2 | | | |
| APERIOD | P3 | | | |
| APERIOD | P4 | | | |
| APERIOD | P5 | | | |
| APERIOD | P6 | | | |
| ARMCD | | ABCEDF | | |
| ARMCD | | BEAFCD | | |
| ARMCD | | CADBFE | | |
| ARMCD | | DCFAEB | | |

Program: A Bio2.sas Created: 02APR2020 7:35 POSTLOCK 

The Mixed Procedure

Parameter Code=SEMAX

Coefficients for Bel 600 vs Oxy 60

Planned Planned

Arm Treatment

Effect APERIOD Code (N) Row1
ARMCD EFBDAC
ARMCD FDECBA

Coefficients for Bel 900 vs Oxy 30

Planned Planned Arm Treatment

Effect APERIOD Code (N) Row1 Intercept 1 TRTPN TRTPN 3 TRTPN 1 TRTPN -1 TRTPN TRTPN APERIOD P1 APERIOD P2 APERIOD P3 APERIOD P4 APERIOD P5 APERIOD P6 ARMCD ABCEDF ARMCD BEAFCD

CADBFE

DCFAEB

Program: A Bio2.sas Created: 02APR2020 7:35 POSTLOCK 

ARMCD

ARMCD

The Mixed Procedure

Parameter Code=SEMAX

Coefficients for Bel 900 vs Oxy 30

Planned Planned

 $\begin{array}{ccc} & \text{Arm} & \text{Treatment} \\ \text{Effect} & \text{APERIOD\,Code} & \text{(N)} & \text{Row1} \\ \end{array}$ 

ARMCD EFBDAC ARMCD FDECBA

Coefficients for Bel 900 vs Oxy 60

Planned Planned

Arm Treatment Effect APERIOD Code (N) Row1 Intercept 1 TRTPN TRTPN 3 TRTPN 1 TRTPN 5 -1 TRTPN TRTPN APERIOD P1 APERIOD P2 APERIOD P3 APERIOD P4 APERIOD P5 APERIOD P6 ARMCD ABCEDF ARMCD BEAFCD ARMCD CADBFE ARMCD DCFAEB

Program: A\_Bio2.sas Created: 02APR2020 7:35 POSTLOCK

#### The Mixed Procedure

#### Parameter Code=SEMAX

## Coefficients for Bel 900 vs Oxy 60

Planned Planned

Arm Treatment
Effect APERIOD Code (N) Row1
ARMCD EFBDAC

FDECBA

ARMCD

## Coefficients for Bel 300 vs Placebo

| | | Planneo | lPianned | |
|-----------|---------|---------|-----------|------|
| | | Arm | Treatment | |
| Effect | APERIOD | Code | (N) | Row1 |
| Intercept | ; | | | |
| TRTPN | | | 1 | 1 |
| TRTPN | | | 2 | |
| TRTPN | | | 3 | |
| TRTPN | | | 4 | |
| TRTPN | | | 5 | |
| TRTPN | | | 6 | -1 |
| APERIOD | P1 | | | |
| APERIOD | P2 | | | |
| APERIOD | Р3 | | | |
| APERIOD | P4 | | | |
| APERIOD | P5 | | | |
| APERIOD | P6 | | | |
| ARMCD | | ABCEDF | | |
| ARMCD | | BEAFCD | | |
| ARMCD | | CADBFE | | |
| ARMCD | | DCFAEB | | |

Program: A\_Bio2.sas Created: 02APR2020 7:35 POSTLOCK

#### The Mixed Procedure

#### Parameter Code=SEMAX

#### Coefficients for Bel 300 vs Placebo

Planned Planned

 Arm
 Treatment

 Effect
 APERIOD Code
 (N)
 Row1

 ARMCD
 EFBDAC

 ARMCD
 FDECBA

## Coefficients for Bel 600 vs Placebo

Planned Planned Arm Treatment

| | | ALIII | IIEau | IICII C |
|-----------|--------|---------|-------|---------|
| Effect | APERIO | DD Code | (N) | Row1 |
| Intercept | t | | | _ |
| TRTPN | | | 1 | |
| TRTPN | | | 2 | 1 |
| TRTPN | | | 3 | |
| TRTPN | | | 4 | |
| TRTPN | | | 5 | |
| TRTPN | | | 6 | -1 |
| APERIOD | P1 | | | |
| APERIOD | P2 | | | |
| APERIOD | Р3 | | | |
| APERIOD | P4 | | | |
| APERIOD | P5 | | | |
| APERIOD | P6 | | | |
| ARMCD | | ABCEDF | | |
| ARMCD | | BEAFCD | | |
| ARMCD | | CADBFE | | |
| ARMCD | | DCFAEB | | |

Program: A Bio2.sas Created: 02APR2020 7:35 POSTLOCK 

The Mixed Procedure

#### Parameter Code=SEMAX

Coefficients for Bel 600 vs Placebo

Planned Planned

Arm Treatment
Effect APERIOD Code (N) Row1
ARMCD EFBDAC
ARMCD FDECBA

Coefficients for Bel 900 vs Placebo Planned Planned

| | | Arm | Treatment | |
|-----------|---------|--------|-----------|------|
| Effect | APERIOD | Code | (N) | Row1 |
| Intercept | | | | |
| TRTPN | | | 1 | |
| TRTPN | | | 2 | |
| TRTPN | | | 3 | 1 |
| TRTPN | | | 4 | |
| TRTPN | | | 5 | |
| TRTPN | | | 6 | -1 |
| APERIOD | P1 | | | |
| APERIOD | P2 | | | |
| APERIOD | Р3 | | | |
| APERIOD | P4 | | | |
| APERIOD | P5 | | | |
| APERIOD | P6 | | | |
| ARMCD | | ABCEDF | | |
| ARMCD | | BEAFCD | | |
| ARMCD | | CADBFE | | |
| ARMCD | | DCFAEB | | |

## Appendix 16.1.9.2.2 Statistical Methods and Analysis Output Supporting Table 14.2.3 Supporting Table 14.2.3

The Mixed Procedure

#### Parameter Code=SEMAX

Coefficients for Bel 900 vs Placebo

Planned Planned

Arm Treatment

Effect APERIOD Code (N) Row1
ARMCD EFBDAC
ARMCD FDECBA

#### Estimates

#### Standard

| Label | Estimate | Error DF t | Value | Pr > t | Alpha Lower | Upper |
|---|---|---|---|---|---|---|
| Oxy 30 vs Placebo | -100.13 | 150.9067 | -0.66 | 0.5093 | 0.05-401.34 | 201.08 |
| Oxy 60 vs Placebo | -379.92 | 148.2067 | -2.56 | 0.0126 | 0.05-675.72 | -84.1134 |
| Bel 300 vs Oxy 30 | 202.07 | 153.1067 | 1.32 | 0.1914 | 0.05-103.52 | 507.66 |
| Bel 300 vs Oxy 60 | 481.86 | 150.9067 | 3.19 | 0.0021 | 0.05 180.66 | 783.06 |
| Bel 600 vs Oxy 30 | 173.86 | 150.9567 | 1.15 | 0.2535 | 0.05-127.43 | 475.16 |
| Bel 600 vs Oxy 60 | 453.65 | 148.1967 | 3.06 | 0.0032 | 0.05 157.87 | 749.44 |
| Bel 900 vs Oxy 30 | 191.81 | 153.0967 | 1.25 | 0.2146 | 0.05-113.76 | 497.37 |
| Bel 900 vs Oxy 60 | 471.60 | 150.9567 | 3.12 | 0.0026 | 0.05 170.31 | 772.89 |
| Bel 300 vs Placebo | 101.94 | 150.8467 | 0.68 | 0.5015 | 0.05-199.15 | 403.03 |
| Bel 600 vs Placebo | 73.7326 | 147.8967 | 0.50 | 0.6197 | 0.05-221.45 | 368.92 |
| Bel 900 vs Placebo | 91.6771 | 150.9067 | 0.61 | 0.5456 | 0.05-209.53 | 392.88 |

Program: A Bio2.sas Created: 02APR2020 7:35 POSTLOCK 

## Appendix 16.1.9.2.2 Statistical Methods and Analysis Output Supporting Table 14.2.3 Supporting Table 14.2.3

The Mixed Procedure

Parameter Code=SEMAX

Least Squares Means

| | Planned | | _ | | | | | |
|---|---|---|---|---|---|---|---|---|
| | Treatment | | Standard | | | | | |
| Effect | (N) | Estimate | Error DF t | Value | Pr > t | Alpha | Lower | Upper |
| TRTPN | 1 | 1281.33 | 120.5167 | 10.63 | <.0001 | 0.1 | 1080.33 | 1482.32 |
| TRTPN | 2 | 1253.12 | 117.0267 | 10.71 | <.0001 | 0.1 | 1057.94 | 1448.30 |
| TRTPN | 3 | 1271.06 | 120.5767 | 10.54 | <.0001 | 0.1 | 1069.97 | 1472.16 |
| TRTPN | 4 | 1079.26 | 120.5767 | 8.95 | <.0001 | 0.1 | 878.16 | 1280.36 |
| TRTPN | 5 | 799.47 | 117.0267 | 6.83 | <.0001 | 0.1 | 604.29 | 994.65 |
| TRTPN | 6 | 1179.39 | 117.0267 | 10.08 | < .0001 | 0.1 | 984.22 | 1374.56 |

Differences of Least Squares Means

| | Planned | Planned | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| | Treatment | Treatment | | Standard | | | | | |
| Effect | (N) | (N) | Estimate | Error DF t | Value H | ?r > t | Alpha | Lower | Upper |
| TRTPN | 1 | 2 | 28.2077 | 151.2167 | 0.19 | 0.8526 | 0.1 | -224.00 | 280.41 |
| TRTPN | 1 | 3 | 10.2632 | 153.0867 | 0.07 | 0.9467 | 0.1 | -245.06 | 265.59 |
| TRTPN | 1 | 4 | 202.07 | 153.1067 | 1.32 | 0.1914 | 0.1 | -53.2914 | 457.43 |
| TRTPN | 1 | 5 | 481.86 | 150.9067 | 3.19 | 0.0021 | 0.1 | 230.17 | 733.55 |
| TRTPN | 1 | 6 | 101.94 | 150.8467 | 0.68 | 0.5015 | 0.1 | -149.66 | 353.54 |
| TRTPN | 2 | 3 | -17.9445 | 150.9767 | -0.12 | 0.9057 | 0.1 | -269.75 | 233.86 |
| TRTPN | 2 | 4 | 173.86 | 150.9567 | 1.15 | 0.2535 | 0.1 | -77.9097 | 425.63 |
| TRTPN | 2 | 5 | 453.65 | 148.1967 | 3.06 | 0.0032 | 0.1 | 206.49 | 700.82 |
| TRTPN | 2 | 6 | 73.7326 | 147.8967 | 0.50 | 0.6197 | 0.1 | -172.93 | 320.40 |
| TRTPN | 3 | 4 | 191.81 | 153.0967 | 1.25 | 0.2146 | 0.1 | -63.5327 | 447.14 |
| TRTPN | 3 | 5 | 471.60 | 150.9567 | 3.12 | 0.0026 | 0.1 | 219.83 | 723.36 |
| TRTPN | 3 | 6 | 91.6771 | 150.9067 | 0.61 | 0.5456 | 0.1 | -160.02 | 343.37 |
| TRTPN | 4 | 5 | 279.79 | 150.9567 | 1.85 | 0.0682 | 0.1 | 28.0255 | 531.56 |

Program: A Bio2.sas Created: 02APR2020 7:35 POSTLOCK 

## Appendix 16.1.9.2.2 Statistical Methods and Analysis Output Supporting Table 14.2.3 Supporting Table 14.2.3

The Mixed Procedure

Parameter Code=SEMAX

## Differences of Least Squares Means

| Planned | Planned | | | | | | | |
|---|---|---|---|---|---|---|---|---|
| Treatmen | t Treatment | : S | tandard | | | | | |
| Effect (N) | (N) | Estimate | Error DF t | Value P | r > t P | lpha | Lower | Upper |
| TRTPN 4 | 6 | -100.13 | 150.9067 | -0.66 | 0.5093 | 0.1 | -351.82 | 151.57 |
| TRTPN 5 | 6 | -379.92 | 148.2067 | -2.56 | 0.0126 | 0.1 | -627.10 | -132.74 |

Program: A\_Bio2.sas Created: 02APR2020 7:35 POSTLOCK 

## Appendix 16.1.9.2.2 Statistical Methods and Analysis Output Supporting Table 14.2.3 Supporting Table 14.2.3

#### The Mixed Procedure

#### Parameter Code=TVEMEMAX

#### Model Information

| Data Set | WORK.ADXV |
|---------------------------|---------------------|
| Dependent Variable | AVAL |
| Covariance Structure | Variance Components |
| Estimation Method | REML |
| Residual Variance Method | Profile |
| Fixed Effects SE Method | Model-Based |
| Degrees of Freedom Method | Containment |

#### Class Level Information

| Class | LevelsValues |
|---|---|
| SUBJID | 161001 1002 1003 1004 1005 1006 1007 1008 1010 1012 1013 1014 1015 1016 1017 1018 |
| TRTPN | 61 2 3 4 5 6 |
| APERIOD | O 6P1 P2 P3 P4 P5 P6 |
| ARMCD | 6ABCEDF BEAFCD CADBFE DCFAEB EFBDAC FDECBA |

| Dimensions | |
|-----------------------|----|
| Covariance Parameters | 2 |
| Columns in X | 19 |
| Columns in Z | 16 |
| Subjects | 1 |
| Max Obs per Subject | 93 |

Program: A Bio2.sas Created: 02APR2020 7:35 POSTLOCK 

## Appendix 16.1.9.2.2 Statistical Methods and Analysis Output Supporting Table 14.2.3 Supporting Table 14.2.3

The Mixed Procedure

#### Parameter Code=TVEMEMAX

| Number | of | Observations | Read | 93 |
|--------|----|--------------|----------|----|
| Number | of | Observations | Used | 93 |
| Number | of | Observations | Not Used | 0 |

| Iteration History | | |
|--------------------|-------|---------------------------|
| Iteration Evaluati | ons - | -2 Res Log Like Criterion |
| 0 | 1 | 1262.49257037 |
| 1 | 3 | 1199.660352590.00000852 |
| 2 | 1 | 1199.655675450.00000003 |
| 3 | 1 | 1199.655660030.00000000 |

Convergence criteria met.

## Covariance Parameter Estimates

| Cov Parm | Estimate |
|----------------|----------|
| SUBJID (ARMCD) | 414683 |
| Residual | 139616 |

## Fit Statistics

| -2 Res Log Likelihood | 1199.7 |
|--------------------------|--------|
| AIC (Smaller is Better) | 1203.7 |
| AICC (Smaller is Better) | 1203.8 |
| BIC (Smaller is Better) | 1205.2 |

 Program: A Bio2.sas Created: 02APR2020 7:35 POSTLOCK

The Mixed Procedure

Parameter Code=TVEMEMAX

Type 3 Tests of Fixed Effects

| NumDen | | | | |
|--------|---------|----|------|--------------|
| | Effect | DF | DF F | Value Pr > F |
| | TRTPN | 5 | 67 | 2.550.0361 |
| | APERIOD | 5 | 67 | 2.300.0541 |
| | ARMCD | 5 | 10 | 0.580.7139 |

## Coefficients for Oxy 30 vs Placebo Planned Planned

| Planned | Planned |
|---------|-----------|
| Arm | Treatment |

| | | Arm | Treatment | |
|-----------|--------|--------|-----------|------|
| Effect | APERIO | ) Code | (N) | Row1 |
| Intercept | | | | |
| TRTPN | | | 1 | |
| TRTPN | | | 2 | |
| TRTPN | | | 3 | |
| TRTPN | | | 4 | 1 |
| TRTPN | | | 5 | |
| TRTPN | | | 6 | -1 |
| APERIOD | P1 | | | |
| APERIOD | P2 | | | |
| APERIOD | Р3 | | | |
| APERIOD | P4 | | | |
| APERIOD | P5 | | | |
| APERIOD | P6 | | | |
| ARMCD | | ABCEDF | | |
| ARMCD | | BEAFCD | | |

Program: A Bio2.sas Created: 02APR2020 7:35 POSTLOCK 

#### The Mixed Procedure

#### Parameter Code=TVEMEMAX

### Coefficients for Oxy 30 vs Placebo

## Planned Planned Arm Treatment

| | 212111 | I I Ca chichi c | |
|--------|--------------|-----------------|------|
| Effect | APERIOD Code | (N) | Row1 |
| ARMCD | CADBFE | | |
| ARMCD | DCFAEB | | |
| ARMCD | EFBDAC | | |
| ARMCD | FDECBA | | |

## Coefficients for Oxy 60 vs Placebo

#### Planned Planned

| | | Arm | Treatmen | t |
|-----------|--------|--------|----------|------|
| Effect | APERIO | D Code | (N) | Row1 |
| Intercept | 5 | | | |
| TRTPN | | | 1 | |
| TRTPN | | | 2 | |
| TRTPN | | | 3 | |
| TRTPN | | | 4 | |
| TRTPN | | | 5 | 1 |
| TRTPN | | | 6 | -1 |
| APERIOD | P1 | | | |
| APERIOD | P2 | | | |
| APERIOD | P3 | | | |
| APERIOD | P4 | | | |
| APERIOD | P5 | | | |
| APERIOD | P6 | | | |
| ARMCD | | ABCEDF | | |
| ARMCD | | BEAFCD | | |

Program: A\_Bio2.sas Created: 02APR2020 7:35 POSTLOCK


#### The Mixed Procedure

#### Parameter Code=TVEMEMAX

### Coefficients for Oxy 60 vs Placebo

## Planned Planned Arm Treatment

| | 212111 | I I Ca chichi c | |
|--------|--------------|-----------------|------|
| Effect | APERIOD Code | (N) | Row1 |
| ARMCD | CADBFE | | |
| ARMCD | DCFAEB | | |
| ARMCD | EFBDAC | | |
| ARMCD | FDECBA | | |

## Coefficients for Bel 300 vs Oxy 30

#### Planned Planned

| | | Arm | Treatment | ī. |
|-----------|--------|--------|-----------|------|
| Effect | APERIO | ) Code | (N) | Row1 |
| Intercept | | | | |
| TRTPN | | | 1 | 1 |
| TRTPN | | | 2 | |
| TRTPN | | | 3 | |
| TRTPN | | | 4 | -1 |
| TRTPN | | | 5 | |
| TRTPN | | | 6 | |
| APERIOD | P1 | | | |
| APERIOD | P2 | | | |
| APERIOD | Р3 | | | |
| APERIOD | P4 | | | |
| APERIOD | P5 | | | |
| APERIOD | P6 | | | |
| ARMCD | | ABCEDF | | |
| ARMCD | | BEAFCD | | |

Program: A Bio2.sas Created: 02APR2020 7:35 POSTLOCK

#### The Mixed Procedure

#### Parameter Code=TVEMEMAX

### Coefficients for Bel 300 vs Oxy 30

### Planned Planned

| | Arm | Treatment | |
|--------|--------------|-----------|------|
| Effect | APERIOD Code | (N) | Row1 |
| ARMCD | CADBFE | | |
| ARMCD | DCFAEB | | |
| ARMCD | EFBDAC | | |
| ARMCD | FDECBA | | |

## Coefficients for Bel 300 vs Oxy 60

#### Planned Planned

| | | Arm | Treatment | |
|-----------|--------|--------|-----------|------|
| Effect | APERIO | ) Code | (N) | Row1 |
| Intercept | | | | |
| TRTPN | | | 1 | 1 |
| TRTPN | | | 2 | |
| TRTPN | | | 3 | |
| TRTPN | | | 4 | |
| TRTPN | | | 5 | -1 |
| TRTPN | | | 6 | |
| APERIOD | P1 | | | |
| APERIOD | P2 | | | |
| APERIOD | Р3 | | | |
| APERIOD | P4 | | | |
| APERIOD | P5 | | | |
| APERIOD | P6 | | | |
| ARMCD | | ABCEDF | | |
| ARMCD | | BEAFCD | | |

Program: A\_Bio2.sas Created: 02APR2020 7:35 POSTLOCK

#### The Mixed Procedure

#### Parameter Code=TVEMEMAX

## Coefficients for Bel 300 vs Oxy 60

## Planned Planned Arm Treatment

| | 212111 | I I Ca chichi c | |
|--------|--------------|-----------------|------|
| Effect | APERIOD Code | (N) | Row1 |
| ARMCD | CADBFE | | |
| ARMCD | DCFAEB | | |
| ARMCD | EFBDAC | | |
| ARMCD | FDECBA | | |

## Coefficients for Bel 600 vs Oxy 30

#### Planned Planned

| | | Arm | Treatme | ent |
|-----------|--------|--------|---------|------|
| Effect | APERIO | ) Code | (N) | Row1 |
| Intercept | t | | | |
| TRTPN | | | 1 | |
| TRTPN | | | 2 | 1 |
| TRTPN | | | 3 | |
| TRTPN | | | 4 | -1 |
| TRTPN | | | 5 | |
| TRTPN | | | 6 | |
| APERIOD | P1 | | | |
| APERIOD | P2 | | | |
| APERIOD | Р3 | | | |
| APERIOD | P4 | | | |
| APERIOD | P5 | | | |
| APERIOD | P6 | | | |
| ARMCD | | ABCEDF | | |
| ARMCD | | BEAFCD | | |

Program: A Bio2.sas Created: 02APR2020 7:35 POSTLOCK

#### The Mixed Procedure

#### Parameter Code=TVEMEMAX

### Coefficients for Bel 600 vs Oxy 30

## Planned Planned Arm Treatment

| | 212111 | I I Ca chichi c | |
|--------|--------------|-----------------|------|
| Effect | APERIOD Code | (N) | Row1 |
| ARMCD | CADBFE | | |
| ARMCD | DCFAEB | | |
| ARMCD | EFBDAC | | |
| ARMCD | FDECBA | | |

## Coefficients for Bel 600 vs Oxy 60

#### Planned Planned

| | | Arm | Treatment | ; |
|-----------|--------|--------|-----------|------|
| Effect | APERIO | ) Code | (N) | Row1 |
| Intercept | | | | |
| TRTPN | | | 1 | |
| TRTPN | | | 2 | 1 |
| TRTPN | | | 3 | |
| TRTPN | | | 4 | |
| TRTPN | | | 5 | -1 |
| TRTPN | | | 6 | |
| APERIOD | P1 | | | |
| APERIOD | P2 | | | |
| APERIOD | Р3 | | | |
| APERIOD | P4 | | | |
| APERIOD | P5 | | | |
| APERIOD | P6 | | | |
| ARMCD | | ABCEDF | | |
| ARMCD | | BEAFCD | | |

Program: A\_Bio2.sas Created: 02APR2020 7:35 POSTLOCK

#### The Mixed Procedure

#### Parameter Code=TVEMEMAX

## Coefficients for Bel 600 vs Oxy 60

#### Planned Planned

| | Arm | Treatment | |
|--------|--------------|-----------|------|
| Effect | APERIOD Code | (N) | Row1 |
| ARMCD | CADBFE | | |
| ARMCD | DCFAEB | | |
| ARMCD | EFBDAC | | |
| ARMCD | FDECBA | | |

## Coefficients for Bel 900 vs Oxy 30

## Planned Planned

| | I | Arm | Treatment | |
|-----------|-----------|--------|-----------|------|
| Effect | APERIOD ( | Code | (N) | Row1 |
| Intercept | t | | | |
| TRTPN | | | 1 | |
| TRTPN | | | 2 | |
| TRTPN | | | 3 | 1 |
| TRTPN | | | 4 | -1 |
| TRTPN | | | 5 | |
| TRTPN | | | 6 | |
| APERIOD | P1 | | | |
| APERIOD | P2 | | | |
| APERIOD | Р3 | | | |
| APERIOD | P4 | | | |
| APERIOD | P5 | | | |
| APERIOD | P6 | | | |
| ARMCD | I | ABCEDF | | |
| ARMCD | I | BEAFCD | | |

Program: A\_Bio2.sas Created: 02APR2020 7:35 POSTLOCK

#### The Mixed Procedure

#### Parameter Code=TVEMEMAX

### Coefficients for Bel 900 vs Oxy 30

## Planned Planned Arm Treatment

| | 231 | 111 | I I Ca cincii c | |
|--------|------------|------|-----------------|------|
| Effect | APERIOD Co | de | (N) | Row1 |
| ARMCD | CA | DBFE | | |
| ARMCD | DC | FAEB | | |
| ARMCD | EF | BDAC | | |
| ARMCD | FD | ECBA | | |

## Coefficients for Bel 900 vs Oxy 60

#### Planned Planned

| | Ī | Arm | Treatment | |
|-----------|---------|--------|-----------|------|
| Effect | APERIOD | Code | (N) | Row1 |
| Intercept | Ī. | | | |
| TRTPN | | | 1 | |
| TRTPN | | | 2 | |
| TRTPN | | | 3 | 1 |
| TRTPN | | | 4 | |
| TRTPN | | | 5 | -1 |
| TRTPN | | | 6 | |
| APERIOD | P1 | | | |
| APERIOD | P2 | | | |
| APERIOD | Р3 | | | |
| APERIOD | P4 | | | |
| APERIOD | P5 | | | |
| APERIOD | P6 | | | |
| ARMCD | Ž | ABCEDF | | |
| ARMCD | Ι | BEAFCD | | |

#### The Mixed Procedure

#### Parameter Code=TVEMEMAX

## Coefficients for Bel 900 vs Oxy 60

## Planned Planned Arm Treatment

| | 21111 | I I Ca chich c | |
|--------|--------------|----------------|------|
| Effect | APERIOD Code | (N) | Row1 |
| ARMCD | CADBFE | | |
| ARMCD | DCFAEB | | |
| ARMCD | EFBDAC | | |
| ARMCD | FDECBA | | |

## Coefficients for Bel 300 vs Placebo

#### Planned Planned

| | | Arm | Treatment | ; |
|-----------|--------|--------|-----------|------|
| Effect | APERIO | Code | (N) | Row1 |
| Intercept | ; | | | |
| TRTPN | | | 1 | 1 |
| TRTPN | | | 2 | |
| TRTPN | | | 3 | |
| TRTPN | | | 4 | |
| TRTPN | | | 5 | |
| TRTPN | | | 6 | -1 |
| APERIOD | P1 | | | |
| APERIOD | P2 | | | |
| APERIOD | Р3 | | | |
| APERIOD | P4 | | | |
| APERIOD | P5 | | | |
| APERIOD | P6 | | | |
| ARMCD | | ABCEDF | | |
| ARMCD | | BEAFCD | | |

Program: A Bio2.sas Created: 02APR2020 7:35 POSTLOCK 

#### The Mixed Procedure

#### Parameter Code=TVEMEMAX

## Coefficients for Bel 300 vs Placebo

## Planned Planned Arm Treatment

| Effect | APERIOD Code | (N) | Row1 |
|--------|--------------|-----|------|
| ARMCD | CADBFE | | |
| ARMCD | DCFAEB | | |
| ARMCD | EFBDAC | | |
| ARMCD | FDECBA | | |

## Coefficients for Bel 600 vs Placebo

#### Planned Planned

| | | Arm | Treatment | |
|-----------|--------|--------|-----------|------|
| Effect | APERIO | O Code | (N) | Row1 |
| Intercept | | | | |
| TRTPN | | | 1 | |
| TRTPN | | | 2 | 1 |
| TRTPN | | | 3 | |
| TRTPN | | | 4 | |
| TRTPN | | | 5 | |
| TRTPN | | | 6 | -1 |
| APERIOD | P1 | | | |
| APERIOD | P2 | | | |
| APERIOD | Р3 | | | |
| APERIOD | P4 | | | |
| APERIOD | P5 | | | |
| APERIOD | P6 | | | |
| ARMCD | | ABCEDF | | |
| ARMCD | | BEAFCD | | |

Program: A\_Bio2.sas Created: 02APR2020 7:35 POSTLOCK

#### The Mixed Procedure

### Parameter Code=TVEMEMAX

## Coefficients for Bel 600 vs Placebo

## Planned Planned Arm Treatment

| | ALIII | Treatment | |
|--------|--------------|-----------|------|
| Effect | APERIOD Code | (N) | Row1 |
| ARMCD | CADBFE | | |
| ARMCD | DCFAEB | | |
| ARMCD | EFBDAC | | |
| ARMCD | FDECBA | | |

#### Coefficients for Bel 900 vs Placebo

#### Planned Planned

| | | Arm | Treatment | |
|-----------|--------|--------|-----------|------|
| Effect | APERIO | O Code | (N) | Row1 |
| Intercept | | | | |
| TRTPN | | | 1 | |
| TRTPN | | | 2 | |
| TRTPN | | | 3 | 1 |
| TRTPN | | | 4 | |
| TRTPN | | | 5 | |
| TRTPN | | | 6 | -1 |
| APERIOD | P1 | | | |
| APERIOD | P2 | | | |
| APERIOD | Р3 | | | |
| APERIOD | P4 | | | |
| APERIOD | P5 | | | |
| APERIOD | P6 | | | |
| ARMCD | | ABCEDF | | |
| ARMCD | | BEAFCD | | |

## Appendix 16.1.9.2.2 Statistical Methods and Analysis Output Supporting Table 14.2.3 Supporting Table 14.2.3

#### The Mixed Procedure

#### Parameter Code=TVEMEMAX

#### Coefficients for Bel 900 vs Placebo

## Planned Planned

| | Arm | Treatment | |
|--------|--------------|-----------|------|
| Effect | APERIOD Code | (N) | Row1 |
| ARMCD | CADBFE | | |
| ARMCD | DCFAEB | | |
| ARMCD | EFBDAC | | |
| ARMCD | FDECBA | | |

#### Estimates

#### Standard

| Labe | el | | | | Estimate | Error DF t | Value | Pr > t | Alpha | Lower | Upper |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Оху | 30 7 | vs ] | Place | ebo | 85.6321 | 135.3567 | 0.63 | 0.5291 | 0.05 | -184.52 | 355.79 |
| Оху | 60 7 | vs 1 | Place | ebo | -187.67 | 132.6567 | -1.41 | 0.1618 | 0.05 | -452.45 | 77.1076 |
| Bel | 300 | vs | Оху | 30 | 134.18 | 137.0467 | 0.98 | 0.3310 | 0.05 | -139.36 | 407.72 |
| Bel | 300 | vs | Оху | 60 | 407.48 | 135.3467 | 3.01 | 0.0037 | 0.05 | 137.34 | 677.63 |
| Bel | 600 | vs | Оху | 30 | -38.2811 | 135.4267 | -0.28 | 0.7783 | 0.05 | -308.59 | 232.03 |
| Bel | 600 | vs | Оху | 60 | 235.02 | 132.6467 | 1.77 | 0.0810 | 0.05 | -29.7354 | 499.78 |
| Bel | 900 | vs | Оху | 30 | 134.25 | 137.0367 | 0.98 | 0.3308 | 0.05 | -139.26 | 407.76 |
| Bel | 900 | vs | Оху | 60 | 407.55 | 135.4267 | 3.01 | 0.0037 | 0.05 | 137.25 | 677.85 |
| Bel | 300 | vs | Plac | cebo | 219.81 | 135.2667 | 1.63 | 0.1088 | 0.05 | -50.1648 | 489.79 |
| Bel | 600 | vs | Plac | cebo | 47.3510 | 132.3867 | 0.36 | 0.7217 | 0.05 | -216.87 | 311.58 |
| Bel | 900 | VS | Plac | cebo | 219.88 | 135.3567 | 1.62 | 0.1090 | 0.05 | -50.2740 | 490.04 |

Program: A Bio2.sas Created: 02APR2020 7:35 POSTLOCK 

## Appendix 16.1.9.2.2 Statistical Methods and Analysis Output Supporting Table 14.2.3 Supporting Table 14.2.3

#### The Mixed Procedure

#### Parameter Code=TVEMEMAX

### Least Squares Means

| | Planned | | _ | | | | | |
|---|---|---|---|---|---|---|---|---|
| | Treatment | | Standard | | | | | |
| Effect | (N) | Estimate | Error DF t | Value | Pr > t | Alpha | Lower | Upper |
| TRTPN | 1 | 1937.48 | 190.8867 | 10.15 | <.000 | 1 0.1 | 1619.11 | 2255.84 |
| TRTPN | 2 | 1765.02 | 188.9667 | 9.34 | <.000 | 1 0.1 | 1449.85 | 2080.19 |
| TRTPN | 3 | 1937.55 | 190.9367 | 10.15 | <.000 | 1 0.1 | 1619.09 | 2256.01 |
| TRTPN | 4 | 1803.30 | 190.9367 | 9.44 | <.000 | 1 0.1 | 1484.84 | 2121.76 |
| TRTPN | 5 | 1529.99 | 188.9667 | 8.10 | <.000 | 1 0.1 | 1214.82 | 1845.16 |
| TRTPN | 6 | 1717.67 | 188.9667 | 9.09 | <.000 | 1 0.1 | 1402.50 | 2032.83 |

## Differences of Least Squares Means

| | Planned | Planned | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| | Treatment | Treatment | | Standard | | | | | |
| Effect | (N) | (N) | Estimate | Error DF t | Value P | r > t | Alpha | Lower | Upper |
| TRTPN | 1 | 2 | 172.46 | 135.6267 | 1.27 | 0.2079 | 0.1 | -53.7416 | 398.66 |
| TRTPN | 1 | 3 | -0.06905 | 137.0267 | -0.00 | 0.9996 | 0.1 | -228.61 | 228.47 |
| TRTPN | 1 | 4 | 134.18 | 137.0467 | 0.98 | 0.3310 | 0.1 | -94.3961 | 362.75 |
| TRTPN | 1 | 5 | 407.48 | 135.3467 | 3.01 | 0.0037 | 0.1 | 181.74 | 633.22 |
| TRTPN | 1 | 6 | 219.81 | 135.2667 | 1.63 | 0.1088 | 0.1 | -5.7877 | 445.41 |
| TRTPN | 2 | 3 | -172.53 | 135.4467 | -1.27 | 0.2071 | 0.1 | -398.44 | 53.3775 |
| TRTPN | 2 | 4 | -38.2811 | 135.4267 | -0.28 | 0.7783 | 0.1 | -264.16 | 187.59 |
| TRTPN | 2 | 5 | 235.02 | 132.6467 | 1.77 | 0.0810 | 0.1 | 13.7839 | 456.26 |
| TRTPN | 2 | 6 | 47.3510 | 132.3867 | 0.36 | 0.7217 | 0.1 | -173.44 | 268.14 |
| TRTPN | 3 | 4 | 134.25 | 137.0367 | 0.98 | 0.3308 | 0.1 | -94.3054 | 362.80 |
| TRTPN | 3 | 5 | 407.55 | 135.4267 | 3.01 | 0.0037 | 0.1 | 181.68 | 633.42 |
| TRTPN | 3 | 6 | 219.88 | 135.3567 | 1.62 | 0.1090 | 0.1 | -5.8676 | 445.63 |
| TRTPN | 4 | 5 | 273.30 | 135.4267 | 2.02 | 0.0476 | 0.1 | 47.4358 | 499.17 |

Program: A Bio2.sas Created: 02APR2020 7:35 POSTLOCK 

## Appendix 16.1.9.2.2 Statistical Methods and Analysis Output Supporting Table 14.2.3 Supporting Table 14.2.3

The Mixed Procedure

#### Parameter Code=TVEMEMAX

## Differences of Least Squares Means

| | Planned | Planned | | | - | | | | |
|---|---|---|---|---|---|---|---|---|---|
| | Treatment | Treatment | ( | Standard | | | | | |
| Effec | t (N) | (N) | Estimate | Error DF t | Value Pr | > t A | lpha | Lower | Upper |
| TRTPN | 4 | 6 | 85.6321 | 135.3567 | 0.63 | 0.5291 | 0.1 | -140.12 | 311.38 |
| TRTPN | 5 | 6 | -187.67 | 132.6567 | -1.41 | 0.1618 | 0.1 | -408.933 | 33.5848 |

Program: A\_Bio2.sas Created: 02APR2020 7:35 POSTLOCK 
### Appendix 16.1.9.2.3 Statistical Methods and Analysis Output Supporting Table 14.2.4 Supporting Table 14.2.4

#### The Mixed Procedure

#### Parameter Code=MVMIPM

#### Model Information

| Data Set | WORK.ADXV |
|---------------------------|-------------------|
| Dependent Variable | AVAL |
| Covariance Structure | Compound Symmetry |
| Subject Effect | SUBJID |
| Estimation Method | REML |
| Residual Variance Method | Profile |
| Fixed Effects SE Method | Model-Based |
| Degrees of Freedom Method | Between-Within |

#### Class Level Information

| Class Le | evelsValues |
|---|---|
| SUBJID | 151001 1002 1003 1004 1005 1006 1007 1008 1010 1012 1013 1014 1015 1016 1017 |
| TRTPN | 6Bel300 Bel600 Bel900 Oxy30 Oxy60 Plac |
| APERIOD | 6P1 P2 P3 P4 P5 P6 |
| ARMCD | 6ABCEDF BEAFCD CADBFE DCFAEB EFBDAC FDECBA |
| ΑΤΡΤΝ | 60 0 5 1 2 3 4 |

| Dimensions | | |
|-------------|------------|----|
| Covariance | Parameters | 2 |
| Columns in | Χ | 55 |
| Columns in | Z | 0 |
| Subjects | | 15 |
| Max Obs per | Subject | 36 |

Program: A Bio3.sas Created: 02APR2020 7:35 POSTLOCK 

#### Appendix 16.1.9.2.3 Statistical Methods and Analysis Output Supporting Table 14.2.4 Supporting Table 14.2.4

The Mixed Procedure

#### Parameter Code=MVMIPM

| | Nι | umber of Obse | rvations | |
|--------|----|---------------|----------|-----|
| Number | of | Observations | Read | 527 |
| Number | of | Observations | Used | 527 |
| Number | of | Observations | Not Used | 0 |

| Iteration History | | | | | |
|---|---|---|---|---|---|
| Iteration Evaluati | ons -2 | Res | Log | Like | Criterion |
| 0 | 1 | 9845 | .227 | 56633 | _ |
| 1 | 2 | 9742 | .184 | 66751 | 0.00000000 |

Convergence criteria met.

Covariance Parameter
Estimates

Cov Parm Subject Estimate
CS SUBJID 12122276
Residual 26084275

| Fit Statistics | |
|--------------------------|--------|
| -2 Res Log Likelihood | 9742.2 |
| AIC (Smaller is Better) | 9746.2 |
| AICC (Smaller is Better) | 9746.2 |
| BIC (Smaller is Better) | 9747.6 |

Program: A Bio3.sas Created: 02APR2020 7:35 POSTLOCK 

#### Appendix 16.1.9.2.3 Statistical Methods and Analysis Output Supporting Table 14.2.4 Supporting Table 14.2.4

The Mixed Procedure

Parameter Code=MVMIPM

Null Model Likelihood Ratio Test

DF Chi-Square Pr > ChiSq 1 103.04 <.0001

Type 3 Tests of Fixed Effects

| | n uiii i | Jen | |
|-------------|----------|------|--------------|
| Effect | DF | DF F | Value Pr > F |
| TRTPN | 5 | 70 | 7.48<.0001 |
| APERIOD | 5 | 70 | 5.760.0002 |
| ARMCD | 5 | 9 | 0.870.5343 |
| TRTPN*ATPTN | 304 | 407 | 2.210.0003 |

#### Least Squares Means

| | Planned | Analysis | | | | | |
|---|---|---|---|---|---|---|---|
| | Treatment | Timepoint | : | Standard | | | |
| Effect | (N) | (N) | Estimate | Error DFt | Value P | r > t | Alpha Lower Upper |
| TRTPN*ATPTN | NBel300 | 0 | 20100 | 1607.72407 | 12.50 | <.0001 | 0.051694023261 |
| TRTPN*ATPTN | NBel300 | 0.5 | 21760 | 1607.72407 | 13.53 | <.0001 | 0.051859924920 |
| TRTPN*ATPTN | NBel300 | 1 | 19847 | 1607.72407 | 12.35 | <.0001 | 0.051668723008 |
| TRTPN*ATPTN | NBel300 | 2 | 19992 | 1607.72407 | 12.43 | <.0001 | 0.051683123152 |
| TRTPN*ATPTN | NBel300 | 3 | 15579 | 1607.72407 | 9.69 | <.0001 | 0.051241818739 |
| TRTPN*ATPTN | NBel300 | 4 | 16134 | 1607.72407 | 10.04 | <.0001 | 0.051297419295 |
| TRTPN*ATPTN | NBel600 | 0 | 19868 | 1646.63407 | 12.07 | <.0001 | 0.051663123105 |
| TRTPN*ATPTN | NBel600 | 0.5 | 20768 | 1646.63407 | 12.61 | <.0001 | 0.051753124005 |
| TRTPN*ATPTN | NBel600 | 1 | 19400 | 1607.76407 | 12.07 | <.0001 | 0.051624022561 |
| TRTPN*ATPTN | NBe1600 | 2 | 17831 | 1607.76407 | 11.09 | <.0001 | 0.051467020991 |

Program: A Bio3.sas Created: 02APR2020 7:35 POSTLOCK

Appendix 16.1.9.2.3
Statistical Methods and Analysis Output Supporting Table 14.2.4
Supporting Table 14.2.4

The Mixed Procedure

Parameter Code=MVMIPM

Least Squares Means

| | | | 20000 09 | aaroo moamo | | | |
|---|---|---|---|---|---|---|---|
| | Planned | Analysis | | | | | |
| | Treatment | Timepoint | | Standard | | | |
| Effect | (N) | (N) | Estimate | Error DFt | | : > t i | Alpha Lower Upper |
| TRTPN*ATPTN | Bel600 | 3 | 17241 | 1607.76407 | 10.72 | <.0001 | 0.051408120402 |
| TRTPN*ATPTN | Bel600 | 4 | 17258 | 1607.76407 | 10.73 | <.0001 | 0.051409720418 |
| TRTPN*ATPTN | Bel900 | 0 | 21445 | 1646.60407 | 13.02 | <.0001 | 0.051820824682 |
| TRTPN*ATPTN | Bel900 | 0.5 | 22890 | 1607.73407 | 14.24 | <.0001 | 0.051973026051 |
| TRTPN*ATPTN | Bel900 | 1 | 20071 | 1607.73407 | 12.48 | <.0001 | 0.051691023231 |
| TRTPN*ATPTN | Bel900 | 2 | 18313 | 1607.73407 | 11.39 | <.0001 | 0.051515221473 |
| TRTPN*ATPTN | Bel900 | 3 | 17633 | 1607.73407 | 10.97 | <.0001 | 0.051447220793 |
| TRTPN*ATPTN | Bel900 | 4 | 16584 | 1607.73407 | 10.32 | <.0001 | 0.051342419745 |
| TRTPN*ATPTN | 0xy30 | 0 | 20238 | 1691.50407 | 11.96 | <.0001 | 0.051691323563 |
| TRTPN*ATPTN | 0xy30 | 0.5 | 17966 | 1691.50407 | 10.62 | <.0001 | 0.051464121291 |
| TRTPN*ATPTN | Oxy30 | 1 | 16113 | 1646.66407 | 9.79 | <.0001 | 0.051287619350 |
| TRTPN*ATPTN | Oxy30 | 2 | 16969 | 1607.77407 | 10.55 | <.0001 | 0.051380820129 |
| TRTPN*ATPTN | Oxy30 | 3 | 18564 | 1607.77407 | 11.55 | <.0001 | 0.051540321724 |
| TRTPN*ATPTN | Oxy30 | 4 | 18784 | 1607.77407 | 11.68 | <.0001 | 0.051562421945 |
| TRTPN*ATPTN | Oxy60 | 0 | 19149 | 1692.33407 | 11.32 | <.0001 | 0.051582322476 |
| TRTPN*ATPTN | Oxy60 | 0.5 | 16780 | 1692.33407 | 9.92 | <.0001 | 0.051345320106 |
| TRTPN*ATPTN | Oxy60 | 1 | 14484 | 1648.55407 | 8.79 | <.0001 | 0.051124317724 |
| TRTPN*ATPTN | Oxy60 | 2 | 13262 | 1607.78407 | 8.25 | <.0001 | 0.051010116422 |
| TRTPN*ATPTN | Oxy60 | 3 | 13811 | 1607.78407 | 8.59 | <.0001 | 0.051065016972 |
| TRTPN*ATPTN | Oxy60 | 4 | 13931 | 1607.78407 | 8.66 | <.0001 | 0.051077117092 |
| TRTPN*ATPTN | Plac | 0 | 18548 | 1607.72407 | 11.54 | <.0001 | 0.051538821709 |
| TRTPN*ATPTN | Plac | 0.5 | 20129 | 1607.72407 | 12.52 | <.0001 | 0.051696823289 |
| TRTPN*ATPTN | Plac | 1 | 21018 | 1607.72407 | 13.07 | <.0001 | 0.051785724178 |
| TRTPN*ATPTN | Plac | 2 | 17212 | 1607.72407 | 10.71 | <.0001 | 0.051405220373 |

Program: A\_Bio3.sas Created: 02APR2020 7:35 POSTLOCK 

### Appendix 16.1.9.2.3 Statistical Methods and Analysis Output Supporting Table 14.2.4 Supporting Table 14.2.4

The Mixed Procedure

Parameter Code=MVMIPM

Least Squares Means

| | Planned | Analysis | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| | Treatment | Timepoint | : | Standard | | | | | |
| Effect | (N) | (N) | Estimate | Error | DF t | Value Pr | > t | Alpha Lower Upp | eı |
| TRTPN*ATPTN | Plac | 3 | 17014 | 1607.72 | 407 | 10.58 | <.0001 | 1 0.0513854201 | 75 |
| TRTPN*ATPTN | Plac | 4 | 18407 | 1607.72 | 407 | 11.45 | < .0001 | 1 0 0515247215 | 568 |

#### Differences of Least Squares Means

| | | | 2 | | or roupe . | quares mean. | - | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | Planned | Analysis | Planned | Analysis | | | | | | | |
| | Treatment | Timepoint | Treatment | Timepoint | | Standard | | | | | |
| Effect | (N) | (N) | (N) | (N) | Estimate | Error DF t | : Value Pr | c > t | Alpha | Lower | Upper |
| TRTPN*ATPTN | Bel300 | 0 | Be1300 | 0.5 | -1659.32 | 1864.91407 | -0.89 | 0.3741 | 0.05 | -5325.39 | 2006.74 |
| TRTPN*ATPTN | Bel300 | 0 | Be1300 | 1 | 252.85 | 1864.91407 | 0.14 | 0.8922 | 0.05 | -3413.21 | 3918.92 |
| TRTPN*ATPTN | Bel300 | 0 | Be1300 | 2 | 108.37 | 1864.91407 | 0.06 | 0.9537 | 0.05 | -3557.70 | 3774.43 |
| TRTPN*ATPTN | 1Bel300 | 0 | Be1300 | 3 | 4521.35 | 1864.91407 | 2.42 | 0.0158 | 0.05 | 855.29 | 8187.42 |
| TRTPN*ATPTN | 1Bel300 | 0 | Be1300 | 4 | 3966.17 | 1864.91407 | 2.13 | 0.0340 | 0.05 | 300.11 | 7632.24 |
| TRTPN*ATPTN | 1Bel300 | 0 | Be1600 | 0 | 232.42 | 1899.90407 | 0.12 | 0.9027 | 0.05 | -3502.42 | 3967.27 |
| TRTPN*ATPTN | 1Bel300 | 0 | Be1600 | 0.5 | -668.08 | 1899.90407 | -0.35 | 0.7253 | 0.05 | -4402.92 | 3066.77 |
| TRTPN*ATPTN | 1Bel300 | 0 | Be1600 | 1 | 699.98 | 1866.36407 | 0.38 | 0.7078 | 0.05 | -2968.93 | 4368.88 |
| TRTPN*ATPTN | 1Bel300 | 0 | Be1600 | 2 | 2269.65 | 1866.36407 | 1.22 | 0.2247 | 0.05 | -1399.26 | 5938.55 |
| TRTPN*ATPTN | 1Bel300 | 0 | Be1600 | 3 | 2858.87 | 1866.36407 | 1.53 | 0.1264 | 0.05 | -810.04 | 6527.77 |
| TRTPN*ATPTN | 1Bel300 | 0 | Be1600 | 4 | 2842.61 | 1866.36407 | 1.52 | 0.1285 | 0.05 | -826.30 | 6511.51 |
| TRTPN*ATPTN | 1Bel300 | 0 | Be1900 | 0 | -1344.38 | 1899.87407 | -0.71 | 0.4796 | 0.05 | -5079.16 | 2390.40 |
| TRTPN*ATPTN | 1Bel300 | 0 | Be1900 | 0.5 | -2789.80 | 1866.33407 | -1.49 | 0.1357 | 0.05 | -6458.65 | 879.04 |
| TRTPN*ATPTN | Bel300 | 0 | Be1900 | 1 | 29.6690 | 1866.33407 | 0.02 | 0.9873 | 0.05 | -3639.18 | 3698.51 |
| TRTPN*ATPTN | 1Bel300 | 0 | Be1900 | 2 | 1787.42 | 1866.33407 | 0.96 | 0.3388 | 0.05 | -1881.42 | 5456.27 |
| TRTPN*ATPTN | Bel300 | 0 | Be1900 | 3 | 2467.69 | 1866.33407 | 1.32 | 0.1868 | 0.05 | -1201.16 | 6136.53 |
| TRTPN*ATPTN | Bel300 | 0 | Be1900 | 4 | 3516.18 | 1866.33407 | 1.88 | 0.0603 | 0.05 | -152.67 | 7185.02 |

Program: A\_Bio3.sas Created: 02APR2020 7:35 POSTLOCK

### Appendix 16.1.9.2.3 Statistical Methods and Analysis Output Supporting Table 14.2.4 Supporting Table 14.2.4

#### The Mixed Procedure

#### Parameter Code=MVMIPM

#### Differences of Least Squares Means

| | Planned | Analysis | | Analvsis | or heade . | oquares neams | | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| | Treatment | - | | :Timepoint | | Standard | | | | |
| Effect | (N) | (N) | (N) | (N) | Estimate | Error DFt | Value P | r > t . | Alpha Lower | Upper |
| TRTPN*ATPTI | NBel300 | 0 | 0xy30 | 0 | -137.82 | 1938.87407 | -0.07 | 0.9434 | 0.05-3949.28 | 3673.64 |
| TRTPN*ATPTI | NBel300 | 0 | 0xy30 | 0.5 | 2134.33 | 1938.87407 | 1.10 | 0.2716 | 0.05-1677.13 | 5945.78 |
| TRTPN*ATPT | NBel300 | 0 | Oxy30 | 1 | 3987.34 | 1899.93407 | 2.10 | 0.0365 | 0.05 252.43 | 7722.24 |
| TRTPN*ATPT | NBel300 | 0 | Oxy30 | 2 | 3131.59 | 1866.36407 | 1.68 | 0.0941 | 0.05 -537.33 | 6800.51 |
| TRTPN*ATPT | NBel300 | 0 | Oxy30 | 3 | 1536.75 | 1866.36407 | 0.82 | 0.4108 | 0.05-2132.16 | 5205.67 |
| TRTPN*ATPT | NBel300 | 0 | Oxy30 | 4 | 1316.00 | 1866.36407 | 0.71 | 0.4811 | 0.05-2352.92 | 4984.92 |
| TRTPN*ATPT | NBel300 | 0 | Oxy60 | 0 | 950.87 | 1939.56407 | 0.49 | 0.6242 | 0.05-2861.94 | 4763.68 |
| TRTPN*ATPT | NBel300 | 0 | Oxy60 | 0.5 | 3320.72 | 1939.56407 | 1.71 | 0.0876 | 0.05 -492.09 | 7133.53 |
| TRTPN*ATPT | NBe1300 | 0 | Oxy60 | 1 | 5616.58 | 1900.77407 | 2.95 | 0.0033 | 0.05 1880.02 | 9353.14 |
| TRTPN*ATPT | NBel300 | 0 | Oxy60 | 2 | 6838.81 | 1866.36407 | 3.66 | 0.0003 | 0.05 3169.89 | 10508 |
| TRTPN*ATPT | NBel300 | 0 | Oxy60 | 3 | 6289.34 | 1866.36407 | 3.37 | 0.0008 | 0.05 2620.42 | 9958.26 |
| TRTPN*ATPT | NBel300 | 0 | Oxy60 | 4 | 6169.20 | 1866.36407 | 3.31 | 0.0010 | 0.05 2500.29 | 9838.12 |
| TRTPN*ATPT | NBe1300 | 0 | Plac | 0 | 1552.01 | 1865.61407 | 0.83 | 0.4059 | 0.05-2115.42 | 5219.44 |
| TRTPN*ATPT | NBe1300 | 0 | Plac | 0.5 | -28.3753 | 1865.61407 | -0.02 | 0.9879 | 0.05-3695.80 | 3639.05 |
| TRTPN*ATPT | NBel300 | 0 | Plac | 1 | -917.63 | 1865.61407 | -0.49 | 0.6231 | 0.05-4585.06 | 2749.79 |
| TRTPN*ATPT | NBe1300 | 0 | Plac | 2 | 2887.83 | 1865.61407 | 1.55 | 0.1224 | 0.05 -779.60 | 6555.26 |
| TRTPN*ATPT | NBel300 | 0 | Plac | 3 | 3085.85 | 1865.61407 | 1.65 | 0.0989 | 0.05 -581.58 | 6753.28 |
| TRTPN*ATPT | NBel300 | 0 | Plac | 4 | 1693.01 | 1865.61407 | 0.91 | 0.3647 | 0.05-1974.42 | 5360.43 |
| TRTPN*ATPT | NBe1300 | 0.5 | Be1300 | 1 | 1912.18 | 1864.91407 | 1.03 | 0.3058 | 0.05-1753.89 | 5578.24 |
| TRTPN*ATPT | NBe1300 | 0.5 | Be1300 | 2 | 1767.69 | 1864.91407 | 0.95 | 0.3438 | 0.05-1898.38 | 5433.75 |
| TRTPN*ATPT | NBel300 | 0.5 | Be1300 | 3 | 6180.67 | 1864.91407 | 3.31 | 0.0010 | 0.05 2514.61 | 9846.74 |
| TRTPN*ATPT | NBe1300 | 0.5 | Be1300 | 4 | 5625.50 | 1864.91407 | 3.02 | 0.0027 | 0.05 1959.43 | 9291.56 |
| TRTPN*ATPT | NBel300 | 0.5 | Be1600 | 0 | 1891.74 | 1899.90407 | 1.00 | 0.3200 | 0.05-1843.10 | 5626.59 |
| TRTPN*ATPT | NBel300 | 0.5 | Be1600 | 0.5 | 991.25 | 1899.90407 | 0.52 | 0.6021 | 0.05-2743.60 | 4726.09 |
| TRTPN*ATPT | NBe1300 | 0.5 | Be1600 | 1 | 2359.30 | 1866.36407 | 1.26 | 0.2069 | 0.05-1309.61 | 6028.20 |

Program: A\_Bio3.sas Created: 02APR2020 7:35 POSTLOCK


Appendix 16.1.9.2.3
Statistical Methods and Analysis Output Supporting Table 14.2.4
Supporting Table 14.2.4

#### The Mixed Procedure

#### Parameter Code=MVMIPM

#### Differences of Least Squares Means

| | <b>5</b> 1 . | | | | or heade i | oquares means | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | Planned | Analysis | | Analysis | | Q1 1 1 | | | | | |
| T. C. C | | - | | Timepoint | | Standard | | | | _ | |
| Effect | (N) | (N) | (N) | (N) | Estimate | Error DF t | | | | Lower | Upper |
| TRTPN*ATPTN | | 0.5 | Be1600 | 2 | | 1866.36407 | 2.11 | | | 260.07 | 7597.88 |
| TRTPN*ATPTN | Bel300 | 0.5 | Be1600 | 3 | 4518.19 | 1866.36407 | 2.42 | 0.0159 | 0.05 | 849.28 | 8187.09 |
| TRTPN*ATPTN | Bel300 | 0.5 | Be1600 | 4 | 4501.93 | 1866.36407 | 2.41 | 0.0163 | 0.05 | 833.02 | 8170.83 |
| TRTPN*ATPTN | Bel300 | 0.5 | Be1900 | 0 | 314.94 | 1899.87407 | 0.17 | 0.8684 | 0.05 | -3419.84 | 4049.73 |
| TRTPN*ATPTN | Bel300 | 0.5 | Be1900 | 0.5 | -1130.48 | 1866.33407 | -0.61 | 0.5450 | 0.05 | -4799.33 | 2538.36 |
| TRTPN*ATPTN | Bel300 | 0.5 | Be1900 | 1 | 1688.99 | 1866.33407 | 0.90 | 0.3660 | 0.05 | -1979.86 | 5357.84 |
| TRTPN*ATPTN | Bel300 | 0.5 | Be1900 | 2 | 3446.74 | 1866.33407 | 1.85 | 0.0655 | 0.05 | -222.10 | 7115.59 |
| TRTPN*ATPTN | Bel300 | 0.5 | Be1900 | 3 | 4127.01 | 1866.33407 | 2.21 | 0.0276 | 0.05 | 458.16 | 7795.85 |
| TRTPN*ATPTN | Bel300 | 0.5 | Be1900 | 4 | 5175.50 | 1866.33407 | 2.77 | 0.0058 | 0.05 | 1506.65 | 8844.34 |
| TRTPN*ATPTN | Bel300 | 0.5 | Oxy30 | 0 | 1521.50 | 1938.87407 | 0.78 | 0.4331 | 0.05 | -2289.96 | 5332.96 |
| TRTPN*ATPTN | Bel300 | 0.5 | Oxy30 | 0.5 | 3793.65 | 1938.87407 | 1.96 | 0.0511 | 0.05 | -17.8074 | 7605.10 |
| TRTPN*ATPTN | Bel300 | 0.5 | 0xy30 | 1 | 5646.66 | 1899.93407 | 2.97 | 0.0031 | 0.05 | 1911.76 | 9381.56 |
| TRTPN*ATPTN | Bel300 | 0.5 | Oxy30 | 2 | 4790.91 | 1866.36407 | 2.57 | 0.0106 | 0.05 | 1121.99 | 8459.83 |
| TRTPN*ATPTN | Bel300 | 0.5 | Oxy30 | 3 | 3196.07 | 1866.36407 | 1.71 | 0.0876 | 0.05 | -472.84 | 6864.99 |
| TRTPN*ATPTN | Bel300 | 0.5 | Oxy30 | 4 | 2975.32 | 1866.36407 | 1.59 | 0.1117 | 0.05 | -693.60 | 6644.24 |
| TRTPN*ATPTN | Bel300 | 0.5 | Oxy60 | 0 | 2610.19 | 1939.56407 | 1.35 | 0.1791 | 0.05 | -1202.62 | 6423.01 |
| TRTPN*ATPTN | Bel300 | 0.5 | Oxy60 | 0.5 | 4980.04 | 1939.56407 | 2.57 | 0.0106 | 0.05 | 1167.23 | 8792.85 |
| TRTPN*ATPTN | Bel300 | 0.5 | Oxy60 | 1 | 7275.90 | 1900.77407 | 3.83 | 0.0001 | 0.05 | 3539.34 | 11012 |
| TRTPN*ATPTN | Bel300 | 0.5 | Oxy60 | 2 | 8498.13 | 1866.36407 | 4.55 | <.0001 | 0.05 | 4829.22 | 12167 |
| TRTPN*ATPTN | Bel300 | 0.5 | Oxy60 | 3 | 7948.66 | 1866.36407 | 4.26 | <.0001 | 0.05 | 4279.74 | 11618 |
| TRTPN*ATPTN | Bel300 | 0.5 | Oxy60 | 4 | 7828.52 | 1866.36407 | 4.19 | <.0001 | 0.05 | 4159.61 | 11497 |
| TRTPN*ATPTN | Bel300 | 0.5 | Plac | 0 | 3211.33 | 1865.61407 | 1.72 | 0.0860 | 0.05 | -456.10 | 6878.76 |
| TRTPN*ATPTN | Bel300 | 0.5 | Plac | 0.5 | 1630.95 | 1865.61407 | 0.87 | 0.3825 | 0.05 | -2036.48 | 5298.37 |
| TRTPN*ATPTN | Bel300 | 0.5 | Plac | 1 | 741.69 | 1865.61407 | 0.40 | 0.6912 | 0.05 | -2925.74 | 4409.12 |
| TRTPN*ATPTN | Bel300 | 0.5 | Plac | 2 | 4547.15 | 1865.61407 | 2.44 | 0.0152 | 0.05 | 879.72 | 8214.58 |

Program: A Bio3.sas Created: 02APR2020 7:35 POSTLOCK 

### Appendix 16.1.9.2.3 Statistical Methods and Analysis Output Supporting Table 14.2.4 Supporting Table 14.2.4

#### The Mixed Procedure

#### Parameter Code=MVMIPM

#### Differences of Least Squares Means

| | D1 1 | 7 1 ' | | | or bease i | oquares means | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | Planned | Analysis | | Analysis<br>Timepoint | | Standard | | | | | |
| Effect | (N) | (N) | (N) | (N) | Estimate | Error DF t | 1/2 ] 110 P: | r > 1+1 | 7.lnha | Lower | Upper |
| TRTPN*ATPT | ` ' | 0.5 | | 3 | | 1865.61407 | 2.54 | 0.0113 | | 1077.74 | 8412.60 |
| | | | Plac | | | | | | | | |
| TRTPN*ATPT | | 0.5 | Plac | 4 | | 1865.61407 | 1.80 | 0.0731 | | -315.10 | 7019.76 |
| TRTPN*ATPT | | 1 | Be1300 | 2 | | 1864.91407 | -0.08 | | | | 3521.58 |
| TRTPN*ATPT | | 1 | Be1300 | 3 | | 1864.91407 | 2.29 | 0.0226 | 0.05 | 602.43 | 7934.56 |
| TRTPN*ATPT | N Bel300 | 1 | Be1300 | 4 | 3713.32 | 1864.91407 | 1.99 | 0.0471 | 0.05 | 47.2543 | 7379.39 |
| TRTPN*ATPT | NBe1300 | 1 | Be1600 | 0 | -20.4327 | 1899.90407 | -0.01 | 0.9914 | 0.05- | -3755.28 | 3714.41 |
| TRTPN*ATPT | N Bel300 | 1 | Be1600 | 0.5 | -920.93 | 1899.90407 | -0.48 | 0.6281 | 0.05- | -4655.78 | 2813.92 |
| TRTPN*ATPT | N Bel300 | 1 | Be1600 | 1 | 447.12 | 1866.36407 | 0.24 | 0.8108 | 0.05- | -3221.78 | 4116.03 |
| TRTPN*ATPT | N Bel300 | 1 | Be1600 | 2 | 2016.79 | 1866.36407 | 1.08 | 0.2805 | 0.05- | -1652.11 | 5685.70 |
| TRTPN*ATPT | N Bel300 | 1 | Be1600 | 3 | 2606.01 | 1866.36407 | 1.40 | 0.1634 | 0.05- | -1062.89 | 6274.92 |
| TRTPN*ATPT | N Bel300 | 1 | Be1600 | 4 | 2589.75 | 1866.36407 | 1.39 | 0.1660 | 0.05- | -1079.15 | 6258.66 |
| TRTPN*ATPT | N Bel300 | 1 | Be1900 | 0 | -1597.23 | 1899.87407 | -0.84 | 0.4010 | 0.05- | -5332.01 | 2137.55 |
| TRTPN*ATPT | N Bel300 | 1 | Be1900 | 0.5 | -3042.66 | 1866.33407 | -1.63 | 0.1038 | 0.05- | -6711.50 | 626.19 |
| TRTPN*ATPT | N Bel300 | 1 | Be1900 | 1 | -223.19 | 1866.33407 | -0.12 | 0.9049 | 0.05- | -3892.03 | 3445.66 |
| TRTPN*ATPT | N Bel300 | 1 | Be1900 | 2 | 1534.57 | 1866.33407 | 0.82 | 0.4114 | 0.05- | -2134.28 | 5203.41 |
| TRTPN*ATPT | N Bel300 | 1 | Be1900 | 3 | 2214.83 | 1866.33407 | 1.19 | 0.2360 | 0.05- | -1454.01 | 5883.68 |
| TRTPN*ATPT | N Bel300 | 1 | Be1900 | 4 | 3263.32 | 1866.33407 | 1.75 | 0.0811 | 0.05 | -405.52 | 6932.17 |
| TRTPN*ATPT | N Bel300 | 1 | Oxy30 | 0 | -390.68 | 1938.87407 | -0.20 | 0.8404 | 0.05- | -4202.13 | 3420.78 |
| TRTPN*ATPT | N Bel300 | 1 | Oxy30 | 0.5 | 1881.47 | 1938.87407 | 0.97 | 0.3324 | 0.05- | -1929.98 | 5692.93 |
| TRTPN*ATPT | N Bel300 | 1 | Oxy30 | 1 | 3734.48 | 1899.93407 | 1.97 | 0.0500 | 0.05 | -0.4199 | 7469.38 |
| TRTPN*ATPT | N Bel300 | 1 | Oxy30 | 2 | 2878.74 | 1866.36407 | 1.54 | 0.1237 | 0.05 | -790.18 | 6547.65 |
| TRTPN*ATPT | N Bel300 | 1 | Oxy30 | 3 | 1283.90 | 1866.36407 | 0.69 | 0.4919 | 0.05- | -2385.02 | 4952.82 |
| TRTPN*ATPT | N Bel300 | 1 | 0xy30 | 4 | 1063.15 | 1866.36407 | 0.57 | 0.5692 | 0.05- | -2605.77 | 4732.06 |
| TRTPN*ATPT | N Bel300 | 1 | 0xy60 | 0 | 698.02 | 1939.56407 | 0.36 | 0.7191 | 0.05- | -3114.79 | 4510.83 |
| TRTPN*ATPT | N Bel300 | 1 | Oxy60 | 0.5 | 3067.86 | 1939.56407 | 1.58 | 0.1145 | 0.05 | -744.95 | 6880.67 |
| | | | _ | | | | | | | | |

Program: A\_Bio3.sas Created: 02APR2020 7:35 POSTLOCK

### Appendix 16.1.9.2.3 Statistical Methods and Analysis Output Supporting Table 14.2.4 Supporting Table 14.2.4

#### The Mixed Procedure

#### Parameter Code=MVMIPM

#### Differences of Least Squares Means

| | D1 | 3 3 ! | | | or bease i | oquares neams | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | Planned | Analysis | | Analysis | | 0.1 | | | | | |
| | | - | Treatment | - | | Standard | | | | _ | |
| Effect | (N) | (N) | (N) | (N) | Estimate | Error DF t | | | | Lower | Upper |
| TRTPN*ATPTN | | 1 | Oxy60 | 1 | | 1900.77407 | 2.82 | 0.0050 | | | 9100.29 |
| TRTPN*ATPTN | Bel300 | 1 | Oxy60 | 2 | 6585.96 | 1866.36407 | 3.53 | 0.0005 | 0.05 | 2917.04 | 10255 |
| TRTPN*ATPTN | Be1300 | 1 | Oxy60 | 3 | 6036.48 | 1866.36407 | 3.23 | 0.0013 | 0.05 | 2367.57 | 9705.40 |
| TRTPN*ATPTN | Be1300 | 1 | Oxy60 | 4 | 5916.35 | 1866.36407 | 3.17 | 0.0016 | 0.05 | 2247.43 | 9585.27 |
| TRTPN*ATPTN | Be1300 | 1 | Plac | 0 | 1299.16 | 1865.61407 | 0.70 | 0.4866 | 0.05 - | -2368.27 | 4966.59 |
| TRTPN*ATPTN | Bel300 | 1 | Plac | 0.5 | -281.23 | 1865.61407 | -0.15 | 0.8803 | 0.05- | -3948.66 | 3386.20 |
| TRTPN*ATPTN | Be1300 | 1 | Plac | 1 | -1170.49 | 1865.61407 | -0.63 | 0.5307 | 0.05 - | -4837.92 | 2496.94 |
| TRTPN*ATPTN | Bel300 | 1 | Plac | 2 | 2634.97 | 1865.61407 | 1.41 | 0.1586 | 0.05- | -1032.46 | 6302.40 |
| TRTPN*ATPTN | Bel300 | 1 | Plac | 3 | 2832.99 | 1865.61407 | 1.52 | 0.1297 | 0.05 | -834.43 | 6500.42 |
| TRTPN*ATPTN | Be1300 | 1 | Plac | 4 | 1440.15 | 1865.61407 | 0.77 | 0.4406 | 0.05- | -2227.28 | 5107.58 |
| TRTPN*ATPTN | Bel300 | 2 | Bel300 | 3 | 4412.99 | 1864.91407 | 2.37 | 0.0184 | 0.05 | 746.92 | 8079.05 |
| TRTPN*ATPTN | Bel300 | 2 | Be1300 | 4 | 3857.81 | 1864.91407 | 2.07 | 0.0392 | 0.05 | 191.74 | 7523.88 |
| TRTPN*ATPTN | Bel300 | 2 | Be1600 | 0 | 124.06 | 1899.90407 | 0.07 | 0.9480 | 0.05 - | -3610.79 | 3858.90 |
| TRTPN*ATPTN | Bel300 | 2 | Be1600 | 0.5 | -776.44 | 1899.90407 | -0.41 | 0.6830 | 0.05 - | 4511.29 | 2958.41 |
| TRTPN*ATPTN | Bel300 | 2 | Be1600 | 1 | 591.61 | 1866.36407 | 0.32 | 0.7514 | 0.05- | -3077.29 | 4260.52 |
| TRTPN*ATPTN | Bel300 | 2 | Be1600 | 2 | 2161.28 | 1866.36407 | 1.16 | 0.2475 | 0.05 - | -1507.62 | 5830.19 |
| TRTPN*ATPTN | Bel300 | 2 | Be1600 | 3 | 2750.50 | 1866.36407 | 1.47 | 0.1413 | 0.05 | -918.40 | 6419.41 |
| TRTPN*ATPTN | Bel300 | 2 | Be1600 | 4 | 2734.24 | 1866.36407 | 1.47 | 0.1437 | 0.05 | -934.66 | 6403.15 |
| TRTPN*ATPTN | Bel300 | 2 | Be1900 | 0 | -1452.74 | 1899.87407 | -0.76 | 0.4449 | 0.05 - | -5187.53 | 2282.04 |
| TRTPN*ATPTN | Bel300 | 2 | Be1900 | 0.5 | -2898.17 | 1866.33407 | -1.55 | 0.1212 | 0.05- | -6567.01 | 770.68 |
| TRTPN*ATPTN | Bel300 | 2 | Be1900 | 1 | -78.6961 | 1866.33407 | -0.04 | 0.9664 | 0.05 - | -3747.54 | 3590.15 |
| TRTPN*ATPTN | Bel300 | 2 | Be1900 | 2 | 1679.06 | 1866.33407 | 0.90 | 0.3688 | 0.05 - | -1989.79 | 5347.90 |
| TRTPN*ATPTN | Bel300 | 2 | Be1900 | 3 | 2359.32 | 1866.33407 | 1.26 | 0.2069 | 0.05- | -1309.52 | 6028.17 |
| TRTPN*ATPTN | Be1300 | 2 | Be1900 | 4 | 3407.81 | 1866.33407 | 1.83 | 0.0686 | 0.05 | -261.03 | 7076.66 |
| TRTPN*ATPTN | Bel300 | 2 | 0xy30 | 0 | -246.19 | 1938.87407 | -0.13 | 0.8990 | 0.05- | -4057.64 | 3565.27 |

Program: A Bio3.sas Created: 02APR2020 7:35 POSTLOCK 

### Appendix 16.1.9.2.3 Statistical Methods and Analysis Output Supporting Table 14.2.4 Supporting Table 14.2.4

#### The Mixed Procedure

#### Parameter Code=MVMIPM

#### Differences of Least Squares Means

| | D1 1 | 3 | | | or bease . | oquares means | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | Planned | Analysis | Planned<br>Treatment | Analysis | | Standard | | | | | |
| Effect. | (N) | (N) | (N) | (N) | Estimate | Error DF t | 772 luo D | v > 1+1 | 7. lmha | Lower | Upper |
| TRTPN*ATPTN | . , | 2 | . , | 0.5 | | 1938.87407 | 1.04 | 0.2967 | | L785.49 | 5837.42 |
| | | | Oxy30 | | | | | | | | |
| TRTPN*ATPTN | | 2 | Oxy30 | 1 | | 1899.93407 | 2.04 | 0.0418 | | 144.07 | 7613.87 |
| TRTPN*ATPTN | | 2 | Oxy30 | 2 | | 1866.36407 | 1.62 | | | -645.69 | 6692.14 |
| TRTPN*ATPTN | | 2 | Oxy30 | 3 | | 1866.36407 | 0.77 | 0.4445 | | 2240.53 | 5097.31 |
| TRTPN*ATPTN | | 2 | 0xy30 | 4 | | 1866.36407 | 0.65 | 0.5180 | | | 4876.55 |
| TRTPN*ATPTN | | 2 | Oxy60 | 0 | | 1939.56407 | 0.43 | | | 2970.30 | 4655.32 |
| TRTPN*ATPTN | 1Bel300 | 2 | Oxy60 | 0.5 | 3212.35 | 1939.56407 | 1.66 | 0.0984 | 0.05 - | -600.46 | 7025.16 |
| TRTPN*ATPTN | 1Bel300 | 2 | Oxy60 | 1 | 5508.22 | 1900.77407 | 2.90 | 0.0040 | 0.05 1 | L771.65 | 9244.78 |
| TRTPN*ATPTN | NBe1300 | 2 | Oxy60 | 2 | 6730.45 | 1866.36407 | 3.61 | 0.0003 | 0.05 3 | 3061.53 | 10399 |
| TRTPN*ATPTN | NBel300 | 2 | Oxy60 | 3 | 6180.97 | 1866.36407 | 3.31 | 0.0010 | 0.05 2 | 2512.06 | 9849.89 |
| TRTPN*ATPTN | NBel300 | 2 | Oxy60 | 4 | 6060.84 | 1866.36407 | 3.25 | 0.0013 | 0.05 2 | 2391.92 | 9729.76 |
| TRTPN*ATPTN | NBel300 | 2 | Plac | 0 | 1443.65 | 1865.61407 | 0.77 | 0.4395 | 0.05-2 | 2223.78 | 5111.08 |
| TRTPN*ATPTN | NBel300 | 2 | Plac | 0.5 | -136.74 | 1865.61407 | -0.07 | 0.9416 | 0.05 -3 | 3804.17 | 3530.69 |
| TRTPN*ATPTN | NBel300 | 2 | Plac | 1 | -1026.00 | 1865.61407 | -0.55 | 0.5827 | 0.05-4 | 1693.43 | 2641.43 |
| TRTPN*ATPTN | NBel300 | 2 | Plac | 2 | 2779.46 | 1865.61407 | 1.49 | 0.1370 | 0.05 - | -887.97 | 6446.89 |
| TRTPN*ATPTN | 1Bel300 | 2 | Plac | 3 | 2977.48 | 1865.61407 | 1.60 | 0.1113 | 0.05 - | -689.95 | 6644.91 |
| TRTPN*ATPTN | NBel300 | 2 | Plac | 4 | 1584.64 | 1865.61407 | 0.85 | 0.3962 | 0.05-2 | 2082.79 | 5252.07 |
| TRTPN*ATPTN | NBel300 | 3 | Be1300 | 4 | -555.18 | 1864.91407 | -0.30 | 0.7661 | 0.05-4 | 1221.24 | 3110.89 |
| TRTPN*ATPTN | NBel300 | 3 | Be1600 | 0 | -4288.93 | 1899.90407 | -2.26 | 0.0245 | 0.05-8 | 3023.78 | -554.08 |
| TRTPN*ATPTN | NBel300 | 3 | Be1600 | 0.5 | -5189.43 | 1899.90407 | -2.73 | 0.0066 | 0.05-8 | 3924.27 | -1454.58 |
| TRTPN*ATPTN | JBel300 | 3 | Be1600 | 1 | -3821.38 | 1866.36407 | -2.05 | 0.0413 | 0.05-7 | 7490.28 | -152.47 |
| TRTPN*ATPTN | 1Bel300 | 3 | Be1600 | 2 | | 1866.36407 | -1.21 | 0.2283 | | | 1417.20 |
| TRTPN*ATPTN | | 3 | Be1600 | 3 | | 1866.36407 | -0.89 | 0.3736 | | | 2006.42 |
| TRTPN*ATPTN | | 3 | Be1600 | 4 | | 1866.36407 | -0.90 | | | | 1990.16 |
| TRTPN*ATPTN | | 3 | Be1000 | 0 | | 1899.87407 | -3.09 | | | | -2130.95 |
| TIVILIN WILLI | 4 DCTOO | J | DCIJUU | U | 5005.75 | 1077.07.107 | 3.03 | 0.0022 | 0.00 -3 | ,000.JI | 2130.93 |

Program: A Bio3.sas Created: 02APR2020 7:35 POSTLOCK 

## Appendix 16.1.9.2.3 Statistical Methods and Analysis Output Supporting Table 14.2.4 Supporting Table 14.2.4

#### The Mixed Procedure

#### Parameter Code=MVMIPM

#### Differences of Least Squares Means

| | D1 1 | 7 1 ' : | | | or bease i | oquares means | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | Planned | Analysis | | Analysis<br>Timepoint | | Standard | | | | | |
| Effect | (N) | (N) | (N) | (N) | Estimate | Error DF t | Walua Di | · > + | Alnha | Lower | Upper |
| TRTPN*ATPT | ` ' | 3 | Bel900 | 0.5 | | 1866.33407 | -3.92 | 0.0001 | | | -3642.31 |
| TRTPN*ATPT | | 3 | | | | 1866.33407 | -2.41 | 0.0165 | | | -822.84 |
| | | - | Be1900 | 1 | | | | | | | |
| TRTPN*ATPT | | 3 | Be1900 | 2 | | 1866.33407 | -1.46 | | 0.05 -6 | | 934.92 |
| TRTPN*ATPT | | 3 | Be1900 | 3 | | 1866.33407 | -1.10 | 0.2718 | | | 1615.18 |
| TRTPN*ATPT | | 3 | Be1900 | 4 | | 1866.33407 | -0.54 | 0.5905 | | | 2663.67 |
| TRTPN*ATPT | | 3 | Oxy30 | 0 | | 1938.87407 | -2.40 | | | | -847.72 |
| TRTPN*ATPT | N Bel300 | 3 | 0xy30 | 0.5 | | 1938.87407 | -1.23 | 0.2190 | | | 1424.43 |
| TRTPN*ATPT | N Bel300 | 3 | Oxy30 | 1 | -534.02 | 1899.93407 | -0.28 | 0.7788 | 0.05-4 | 1268.92 | 3200.88 |
| TRTPN*ATPT | N Bel300 | 3 | Oxy30 | 2 | -1389.76 | 1866.36407 | -0.74 | 0.4569 | 0.05-5 | 058.68 | 2279.16 |
| TRTPN*ATPT | N Bel300 | 3 | Oxy30 | 3 | -2984.60 | 1866.36407 | -1.60 | 0.1106 | 0.05-6 | 653.52 | 684.32 |
| TRTPN*ATPT | N Bel300 | 3 | Oxy30 | 4 | -3205.35 | 1866.36407 | -1.72 | 0.0867 | 0.05-6 | 874.27 | 463.57 |
| TRTPN*ATPT | N Bel300 | 3 | Oxy60 | 0 | -3570.48 | 1939.56407 | -1.84 | 0.0664 | 0.05-7 | 383.29 | 242.33 |
| TRTPN*ATPT | N Bel300 | 3 | Oxy60 | 0.5 | -1200.64 | 1939.56407 | -0.62 | 0.5362 | 0.05-5 | 013.45 | 2612.18 |
| TRTPN*ATPT | NBel300 | 3 | Oxy60 | 1 | 1095.23 | 1900.77407 | 0.58 | 0.5648 | 0.05-2 | 2641.33 | 4831.79 |
| TRTPN*ATPT | N Bel300 | 3 | Oxy60 | 2 | 2317.46 | 1866.36407 | 1.24 | 0.2151 | 0.05-1 | 351.46 | 5986.38 |
| TRTPN*ATPT | N Bel300 | 3 | Oxy60 | 3 | 1767.99 | 1866.36407 | 0.95 | 0.3441 | 0.05-1 | 900.93 | 5436.90 |
| TRTPN*ATPT | N Bel300 | 3 | Oxy60 | 4 | 1647.85 | 1866.36407 | 0.88 | 0.3778 | 0.05-2 | 2021.07 | 5316.77 |
| TRTPN*ATPT | N Bel300 | 3 | Plac | 0 | -2969.34 | 1865.61407 | -1.59 | 0.1122 | 0.05-6 | 636.77 | 698.09 |
| TRTPN*ATPT | N Bel300 | 3 | Plac | 0.5 | -4549.73 | 1865.61407 | -2.44 | 0.0152 | 0.05-8 | 3217.16 | -882.30 |
| TRTPN*ATPT | N Bel300 | 3 | Plac | 1 | -5438.99 | 1865.61407 | -2.92 | 0.0037 | 0.05-9 | 106.42 | -1771.56 |
| TRTPN*ATPT | N Bel300 | 3 | Plac | 2 | -1633.53 | 1865.61407 | -0.88 | 0.3818 | 0.05-5 | 300.95 | 2033.90 |
| TRTPN*ATPT | N Bel300 | 3 | Plac | 3 | -1435.50 | 1865.61407 | -0.77 | 0.4421 | 0.05-5 | 102.93 | 2231.93 |
| TRTPN*ATPT | N Bel300 | 3 | Plac | 4 | -2828.35 | 1865.61407 | -1.52 | 0.1303 | 0.05-6 | 495.78 | 839.08 |
| TRTPN*ATPT | N Bel300 | 4 | Be1600 | 0 | -3733.75 | 1899.90407 | -1.97 | 0.0501 | 0.05-7 | 468.60 | 1.0934 |
| TRTPN*ATPT | N Bel300 | 4 | Be1600 | 0.5 | -4634.25 | 1899.90407 | -2.44 | 0.0151 | 0.05-8 | 369.10 | -899.40 |

Program: A Bio3.sas Created: 02APR2020 7:35 POSTLOCK 

### Appendix 16.1.9.2.3 Statistical Methods and Analysis Output Supporting Table 14.2.4 Supporting Table 14.2.4

#### The Mixed Procedure

#### Parameter Code=MVMIPM

#### Differences of Least Squares Means

| | | | | | or nease r | squares neams | | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| | Planned | Analysis | | Analysis | | | | | | |
| | | - | Treatment | - | | Standard | | | | |
| Effect | (N) | (N) | (N) | (N) | Estimate | Error DFt | | | - | -11- |
| TRTPN*ATPTN | Be1300 | 4 | Be1600 | 1 | -3266.20 | 1866.36407 | -1.75 | | 0.05-6935. | |
| TRTPN*ATPTN | Be1300 | 4 | Be1600 | 2 | -1696.53 | 1866.36407 | -0.91 | 0.3639 | 0.05-5365. | 13 1972.38 |
| TRTPN*ATPTN | Bel300 | 4 | Be1600 | 3 | -1107.31 | 1866.36407 | -0.59 | 0.5533 | 0.05-4776.2 | 21 2561.60 |
| TRTPN*ATPTN | Bel300 | 4 | Be1600 | 4 | -1123.57 | 1866.36407 | -0.60 | 0.5475 | 0.05-4792. | 47 2545.34 |
| TRTPN*ATPTN | Bel300 | 4 | Be1900 | 0 | -5310.55 | 1899.87407 | -2.80 | 0.0054 | 0.05-9045. | 33 -1575.77 |
| TRTPN*ATPTN | Bel300 | 4 | Be1900 | 0.5 | -6755.98 | 1866.33407 | -3.62 | 0.0003 | 0.05 -1042 | 25 - 3087.13 |
| TRTPN*ATPTN | Bel300 | 4 | Be1900 | 1 | -3936.51 | 1866.33407 | -2.11 | 0.0355 | 0.05-7605. | 35 -267.66 |
| TRTPN*ATPTN | Bel300 | 4 | Be1900 | 2 | -2178.75 | 1866.33407 | -1.17 | 0.2437 | 0.05-5847. | 60 1490.09 |
| TRTPN*ATPTN | Bel300 | 4 | Be1900 | 3 | -1498.49 | 1866.33407 | -0.80 | 0.4225 | 0.05-5167. | 33 2170.36 |
| TRTPN*ATPTN | Bel300 | 4 | Be1900 | 4 | -450.00 | 1866.33407 | -0.24 | 0.8096 | 0.05-4118. | 34 3218.85 |
| TRTPN*ATPTN | Bel300 | 4 | 0xy30 | 0 | -4104.00 | 1938.87407 | -2.12 | 0.0349 | 0.05-7915. | 45 -292.54 |
| TRTPN*ATPTN | Bel300 | 4 | Oxy30 | 0.5 | -1831.85 | 1938.87407 | -0.94 | 0.3453 | 0.05-5643. | 30 1979.61 |
| TRTPN*ATPTN | Bel300 | 4 | Oxy30 | 1 | 21.1604 | 1899.93407 | 0.01 | 0.9911 | 0.05-3713. | 74 3756.06 |
| TRTPN*ATPTN | Bel300 | 4 | Oxy30 | 2 | -834.58 | 1866.36407 | -0.45 | 0.6550 | 0.05-4503. | 50 2834.33 |
| TRTPN*ATPTN | Bel300 | 4 | 0xy30 | 3 | -2429.42 | 1866.36407 | -1.30 | 0.1938 | 0.05-6098. | 34 1239.50 |
| TRTPN*ATPTN | Bel300 | 4 | Oxy30 | 4 | -2650.17 | 1866.36407 | -1.42 | 0.1564 | 0.05-6319. | 09 1018.74 |
| TRTPN*ATPTN | Bel300 | 4 | Oxy60 | 0 | -3015.30 | 1939.56407 | -1.55 | 0.1208 | 0.05-6828. | 11 797.51 |
| TRTPN*ATPTN | Bel300 | 4 | Oxy60 | 0.5 | -645.46 | 1939.56407 | -0.33 | 0.7395 | 0.05-4458. | 27 3167.35 |
| TRTPN*ATPTN | Bel300 | 4 | Oxy60 | 1 | 1650.41 | 1900.77407 | 0.87 | 0.3858 | 0.05-2086. | 16 5386.97 |
| TRTPN*ATPTN | Bel300 | 4 | Oxy60 | 2 | 2872.64 | 1866.36407 | 1.54 | 0.1245 | 0.05 -796.2 | 28 6541.55 |
| TRTPN*ATPTN | Be1300 | 4 | Oxy60 | 3 | 2323.16 | 1866.36407 | 1.24 | 0.2139 | 0.05-1345. | 75 5992.08 |
| TRTPN*ATPTN | Bel300 | 4 | Oxy60 | 4 | 2203.03 | 1866.36407 | 1.18 | 0.2385 | 0.05-1465. | 39 5871.95 |
| TRTPN*ATPTN | Bel300 | 4 | Plac | 0 | -2414.16 | 1865.61407 | -1.29 | 0.1964 | 0.05-6081. | 59 1253.27 |
| TRTPN*ATPTN | Be1300 | 4 | Plac | 0.5 | -3994.55 | 1865.61407 | -2.14 | 0.0329 | 0.05-7661. | 98 -327.12 |
| TRTPN*ATPTN | Be1300 | 4 | Plac | 1 | -4883.81 | 1865.61407 | -2.62 | 0.0092 | 0.05-8551. | 24 -1216.38 |

Program: A Bio3.sas Created: 02APR2020 7:35 POSTLOCK 

### Appendix 16.1.9.2.3 Statistical Methods and Analysis Output Supporting Table 14.2.4 Supporting Table 14.2.4

#### The Mixed Procedure

#### Parameter Code=MVMIPM

#### Differences of Least Squares Means

| | Planned | Analysis | Planned | Analysis | 01 10000 . | oquares means | | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| | Treatment | Timepoint | Treatment | Timepoint | | Standard | | | | |
| Effect | (N) | (N) | (N) | (N) | Estimate | Error DFt | Value Pr | r > t 2 | Alpha Lower | Upper |
| TRTPN*ATPTN | Bel300 | 4 | Plac | 2 | -1078.35 | 1865.61407 | -0.58 | 0.5636 | 0.05-4745.78 | 2589.08 |
| TRTPN*ATPTN | Bel300 | 4 | Plac | 3 | -880.33 | 1865.61407 | -0.47 | 0.6373 | 0.05-4547.75 | 2787.10 |
| TRTPN*ATPTN | Bel300 | 4 | Plac | 4 | -2273.17 | 1865.61407 | -1.22 | 0.2238 | 0.05-5940.60 | 1394.26 |
| TRTPN*ATPTN | Bel600 | 0 | Be1600 | 0.5 | -900.50 | 1930.37407 | -0.47 | 0.6411 | 0.05-4695.24 | 2894.24 |
| TRTPN*ATPTN | 1Bel600 | 0 | Be1600 | 1 | 467.56 | 1899.21407 | 0.25 | 0.8057 | 0.05-3265.93 | 4201.04 |
| TRTPN*ATPTN | 1Bel600 | 0 | Be1600 | 2 | 2037.23 | 1899.21407 | 1.07 | 0.2841 | 0.05-1696.26 | 5770.71 |
| TRTPN*ATPTN | Bel600 | 0 | Be1600 | 3 | 2626.45 | 1899.21407 | 1.38 | 0.1674 | 0.05 -1107.04 | 6359.93 |
| TRTPN*ATPTN | 1Bel600 | 0 | Be1600 | 4 | 2610.19 | 1899.21407 | 1.37 | 0.1701 | 0.05-1123.30 | 6343.67 |
| TRTPN*ATPTN | Bel600 | 0 | Be1900 | 0 | -1576.80 | 1933.90407 | -0.82 | 0.4154 | 0.05-5378.48 | 2224.88 |
| TRTPN*ATPTN | Bel600 | 0 | Be1900 | 0.5 | -3022.23 | 1899.91407 | -1.59 | 0.1124 | 0.05-6757.09 | 712.64 |
| TRTPN*ATPTN | 1Bel600 | 0 | Be1900 | 1 | -202.75 | 1899.91407 | -0.11 | 0.9151 | 0.05-3937.62 | 3532.11 |
| TRTPN*ATPTN | 1Bel600 | 0 | Be1900 | 2 | 1555.00 | 1899.91407 | 0.82 | 0.4136 | 0.05-2179.86 | 5289.86 |
| TRTPN*ATPTN | Bel600 | 0 | Be1900 | 3 | 2235.27 | 1899.91407 | 1.18 | 0.2401 | 0.05-1499.60 | 5970.13 |
| TRTPN*ATPTN | 1Bel600 | 0 | Be1900 | 4 | 3283.75 | 1899.91407 | 1.73 | 0.0847 | 0.05 -451.11 | 7018.62 |
| TRTPN*ATPTN | 1Bel600 | 0 | 0xy30 | 0 | -370.24 | 1971.65407 | -0.19 | 0.8511 | 0.05-4246.13 | 3505.65 |
| TRTPN*ATPTN | 1Bel600 | 0 | 0xy30 | 0.5 | 1901.91 | 1971.65407 | 0.96 | 0.3353 | 0.05-1973.99 | 5777.80 |
| TRTPN*ATPTN | 1Bel600 | 0 | 0xy30 | 1 | 3754.91 | 1933.14407 | 1.94 | 0.0528 | 0.05-45.2754 | 7555.10 |
| TRTPN*ATPTN | 1Bel600 | 0 | 0xy30 | 2 | 2899.17 | 1899.96407 | 1.53 | 0.1278 | 0.05 -835.79 | 6634.13 |
| TRTPN*ATPTN | 1Bel600 | 0 | 0xy30 | 3 | 1304.33 | 1899.96407 | 0.69 | 0.4928 | 0.05-2430.63 | 5039.29 |
| TRTPN*ATPTN | 1Bel600 | 0 | 0xy30 | 4 | 1083.58 | 1899.96407 | 0.57 | 0.5688 | 0.05-2651.38 | 4818.53 |
| TRTPN*ATPTN | 1Bel600 | 0 | Oxy60 | 0 | 718.45 | 1973.27407 | 0.36 | 0.7160 | 0.05-3160.62 | 4597.53 |
| TRTPN*ATPTN | 1Bel600 | 0 | Oxy60 | 0.5 | 3088.30 | 1973.27407 | 1.57 | 0.1183 | 0.05 -790.78 | 6967.37 |
| TRTPN*ATPTN | 1Bel600 | 0 | Oxy60 | 1 | 5384.16 | 1935.61407 | 2.78 | 0.0057 | 0.05 1579.12 | 9189.20 |
| TRTPN*ATPTN | 1Bel600 | 0 | Oxy60 | 2 | 6606.39 | 1900.72407 | 3.48 | 0.0006 | 0.05 2869.93 | 10343 |
| TRTPN*ATPTN | 1Bel600 | 0 | Oxy60 | 3 | 6056.92 | 1900.72407 | 3.19 | 0.0016 | 0.05 2320.46 | 9793.38 |

Program: A\_Bio3.sas Created: 02APR2020 7:35 POSTLOCK

Appendix 16.1.9.2.3
Statistical Methods and Analysis Output Supporting Table 14.2.4
Supporting Table 14.2.4

#### The Mixed Procedure

#### Parameter Code=MVMIPM

#### Differences of Least Squares Means

| | | | D11 | . ICICIICCO I | or nease i | oquares means | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | Planned | Analysis | Planned | Analysis | | | | | | | |
| | Treatment | Timepoint | Treatment | Timepoint | | Standard | | | | | |
| Effect | (N) | (N) | (N) | (N) | Estimate | Error DF t | | | | Lower | Upper |
| TRTPN*ATPTN | Be1600 | 0 | Oxy60 | 4 | 5936.78 | 1900.72407 | 3.12 | 0.0019 | | 2200.32 | 9673.24 |
| TRTPN*ATPTN | Be1600 | 0 | Plac | 0 | 1319.59 | 1899.90407 | 0.69 | 0.4877 | 0.05- | -2415.26 | 5054.44 |
| TRTPN*ATPTN | Be1600 | 0 | Plac | 0.5 | -260.80 | 1899.90407 | -0.14 | 0.8909 | 0.05- | -3995.64 | 3474.05 |
| TRTPN*ATPTN | Be1600 | 0 | Plac | 1 | -1150.06 | 1899.90407 | -0.61 | 0.5453 | 0.05- | -4884.90 | 2584.79 |
| TRTPN*ATPTN | Be1600 | 0 | Plac | 2 | 2655.41 | 1899.90407 | 1.40 | 0.1630 | 0.05- | -1079.44 | 6390.25 |
| TRTPN*ATPTN | Bel600 | 0 | Plac | 3 | 2853.43 | 1899.90407 | 1.50 | 0.1339 | 0.05 | -881.42 | 6588.27 |
| TRTPN*ATPTN | Bel600 | 0 | Plac | 4 | 1460.58 | 1899.90407 | 0.77 | 0.4425 | 0.05- | -2274.26 | 5195.43 |
| TRTPN*ATPTN | Bel600 | 0.5 | Be1600 | 1 | 1368.05 | 1899.21407 | 0.72 | 0.4717 | 0.05- | -2365.43 | 5101.54 |
| TRTPN*ATPTN | Bel600 | 0.5 | Be1600 | 2 | 2937.73 | 1899.21407 | 1.55 | 0.1227 | 0.05 | -795.76 | 6671.21 |
| TRTPN*ATPTN | Be1600 | 0.5 | Be1600 | 3 | 3526.94 | 1899.21407 | 1.86 | 0.0640 | 0.05 | -206.54 | 7260.43 |
| TRTPN*ATPTN | Be1600 | 0.5 | Be1600 | 4 | 3510.68 | 1899.21407 | 1.85 | 0.0653 | 0.05 | -222.80 | 7244.17 |
| TRTPN*ATPTN | Be1600 | 0.5 | Be1900 | 0 | -676.30 | 1933.90407 | -0.35 | 0.7267 | 0.05- | -4477.98 | 3125.38 |
| TRTPN*ATPTN | Be1600 | 0.5 | Be1900 | 0.5 | -2121.73 | 1899.91407 | -1.12 | 0.2648 | 0.05- | -5856.59 | 1613.13 |
| TRTPN*ATPTN | Be1600 | 0.5 | Be1900 | 1 | 697.74 | 1899.91407 | 0.37 | 0.7136 | 0.05- | -3037.12 | 4432.61 |
| TRTPN*ATPTN | Be1600 | 0.5 | Be1900 | 2 | 2455.50 | 1899.91407 | 1.29 | 0.1969 | 0.05- | -1279.36 | 6190.36 |
| TRTPN*ATPTN | Be1600 | 0.5 | Be1900 | 3 | 3135.76 | 1899.91407 | 1.65 | 0.0996 | 0.05 | -599.10 | 6870.63 |
| TRTPN*ATPTN | Be1600 | 0.5 | Be1900 | 4 | 4184.25 | 1899.91407 | 2.20 | 0.0282 | 0.05 | 449.39 | 7919.11 |
| TRTPN*ATPTN | Bel600 | 0.5 | 0xy30 | 0 | 530.25 | 1971.65407 | 0.27 | 0.7881 | 0.05- | -3345.64 | 4406.15 |
| TRTPN*ATPTN | Be1600 | 0.5 | 0xy30 | 0.5 | 2802.40 | 1971.65407 | 1.42 | 0.1560 | 0.05- | -1073.49 | 6678.29 |
| TRTPN*ATPTN | Bel600 | 0.5 | 0xy30 | 1 | 4655.41 | 1933.14407 | 2.41 | 0.0165 | 0.05 | 855.22 | 8455.60 |
| TRTPN*ATPTN | Bel600 | 0.5 | 0xy30 | 2 | 3799.67 | 1899.96407 | 2.00 | 0.0462 | 0.05 | 64.7109 | 7534.62 |
| TRTPN*ATPTN | Be1600 | 0.5 | 0xy30 | 3 | 2204.83 | 1899.96407 | 1.16 | 0.2465 | 0.05- | -1530.13 | 5939.78 |
| TRTPN*ATPTN | Bel600 | 0.5 | 0xy30 | 4 | 1984.08 | 1899.96407 | 1.04 | 0.2970 | 0.05- | -1750.88 | 5719.03 |
| TRTPN*ATPTN | Bel600 | 0.5 | Oxy60 | 0 | 1618.95 | 1973.27407 | 0.82 | 0.4124 | 0.05- | -2260.13 | 5498.03 |
| TRTPN*ATPTN | Bel600 | 0.5 | Oxy60 | 0.5 | 3988.79 | 1973.27407 | 2.02 | 0.0439 | 0.05 | 109.72 | 7867.87 |

Program: A\_Bio3.sas Created: 02APR2020 7:35 POSTLOCK


Appendix 16.1.9.2.3
Statistical Methods and Analysis Output Supporting Table 14.2.4
Supporting Table 14.2.4

#### The Mixed Procedure

#### Parameter Code=MVMIPM

#### Differences of Least Squares Means

| | | | בב | . ICICIICCO I | or nease t | quares neams | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | Planned | Analysis | | Analysis | | | | | | | |
| | Treatment | Timepoint | Treatment | Timepoint | | Standard | | | | | |
| Effect | (N) | (N) | (N) | (N) | Estimate | Error DF t | | | - | Lower | Upper |
| TRTPN*ATPTN | Be1600 | 0.5 | Oxy60 | 1 | 6284.66 | 1935.61407 | 3.25 | 0.0013 | | 2479.62 | 10090 |
| TRTPN*ATPTN | Be1600 | 0.5 | Oxy60 | 2 | 7506.89 | 1900.72407 | 3.95 | <.0001 | 0.05 | 3770.43 | 11243 |
| TRTPN*ATPTN | Be1600 | 0.5 | Oxy60 | 3 | 6957.41 | 1900.72407 | 3.66 | 0.0003 | 0.05 | 3220.95 | 10694 |
| TRTPN*ATPTN | Be1600 | 0.5 | Oxy60 | 4 | 6837.28 | 1900.72407 | 3.60 | 0.0004 | 0.05 | 3100.82 | 10574 |
| TRTPN*ATPTN | Bel600 | 0.5 | Plac | 0 | 2220.09 | 1899.90407 | 1.17 | 0.2433 | 0.05- | 1514.76 | 5954.93 |
| TRTPN*ATPTN | Bel600 | 0.5 | Plac | 0.5 | 639.70 | 1899.90407 | 0.34 | 0.7365 | 0.05- | 3095.15 | 4374.55 |
| TRTPN*ATPTN | Bel600 | 0.5 | Plac | 1 | -249.56 | 1899.90407 | -0.13 | 0.8956 | 0.05- | 3984.41 | 3485.29 |
| TRTPN*ATPTN | Bel600 | 0.5 | Plac | 2 | 3555.90 | 1899.90407 | 1.87 | 0.0620 | 0.05 | -178.94 | 7290.75 |
| TRTPN*ATPTN | Bel600 | 0.5 | Plac | 3 | 3753.92 | 1899.90407 | 1.98 | 0.0488 | 0.05 | 19.0786 | 7488.77 |
| TRTPN*ATPTN | Bel600 | 0.5 | Plac | 4 | 2361.08 | 1899.90407 | 1.24 | 0.2147 | 0.05- | 1373.77 | 6095.93 |
| TRTPN*ATPTN | Bel600 | 1 | Be1600 | 2 | 1569.67 | 1864.91407 | 0.84 | 0.4005 | 0.05- | 2096.39 | 5235.74 |
| TRTPN*ATPTN | Bel600 | 1 | Be1600 | 3 | 2158.89 | 1864.91407 | 1.16 | 0.2477 | 0.05- | 1507.18 | 5824.96 |
| TRTPN*ATPTN | Bel600 | 1 | Be1600 | 4 | 2142.63 | 1864.91407 | 1.15 | 0.2513 | 0.05- | 1523.44 | 5808.70 |
| TRTPN*ATPTN | Bel600 | 1 | Be1900 | 0 | -2044.36 | 1900.65407 | -1.08 | 0.2827 | 0.05- | 5780.66 | 1691.95 |
| TRTPN*ATPTN | Bel600 | 1 | Be1900 | 0.5 | -3489.78 | 1866.36407 | -1.87 | 0.0622 | 0.05- | 7158.69 | 179.13 |
| TRTPN*ATPTN | Bel600 | 1 | Be1900 | 1 | -670.31 | 1866.36407 | -0.36 | 0.7197 | 0.05- | 4339.22 | 2998.60 |
| TRTPN*ATPTN | Bel600 | 1 | Be1900 | 2 | 1087.45 | 1866.36407 | 0.58 | 0.5604 | 0.05- | 2581.47 | 4756.36 |
| TRTPN*ATPTN | Bel600 | 1 | Be1900 | 3 | 1767.71 | 1866.36407 | 0.95 | 0.3441 | 0.05- | 1901.20 | 5436.62 |
| TRTPN*ATPTN | Bel600 | 1 | Be1900 | 4 | 2816.20 | 1866.36407 | 1.51 | 0.1321 | 0.05 | -852.71 | 6485.11 |
| TRTPN*ATPTN | Bel600 | 1 | 0xy30 | 0 | -837.80 | 1939.83407 | -0.43 | 0.6660 | 0.05- | 4651.14 | 2975.54 |
| TRTPN*ATPTN | Bel600 | 1 | Oxy30 | 0.5 | 1434.35 | 1939.83407 | 0.74 | 0.4601 | 0.05- | 2378.99 | 5247.69 |
| TRTPN*ATPTN | Bel600 | 1 | 0xy30 | 1 | 3287.36 | 1900.00407 | 1.73 | 0.0844 | 0.05 | -447.69 | 7022.40 |
| TRTPN*ATPTN | Bel600 | 1 | Oxy30 | 2 | 2431.61 | 1865.62407 | 1.30 | 0.1932 | 0.05- | 1235.83 | 6099.06 |
| TRTPN*ATPTN | Be1600 | 1 | 0xy30 | 3 | 836.78 | 1865.62407 | 0.45 | 0.6540 | 0.05- | 2830.67 | 4504.22 |
| TRTPN*ATPTN | Bel600 | 1 | 0xy30 | 4 | 616.02 | 1865.62407 | 0.33 | 0.7414 | 0.05- | 3051.42 | 4283.47 |

Program: A\_Bio3.sas Created: 02APR2020 7:35 POSTLOCK


### Appendix 16.1.9.2.3 Statistical Methods and Analysis Output Supporting Table 14.2.4 Supporting Table 14.2.4

#### The Mixed Procedure

#### Parameter Code=MVMIPM

#### Differences of Least Squares Means

| | Planned | Analysis | | Analvsis | or bease . | oquares neams | | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| | Treatment | _ | | . Timepoint | | Standard | | | | |
| Effect | (N) | (N) | (N) | (N) | Estimate | Error DFt | Value P | r > t . | Alpha Lower | Upper |
| TRTPN*ATPT | N Bel600 | 1 | Oxy60 | 0 | 250.90 | 1940.37407 | 0.13 | 0.8972 | 0.05-3563.50 | 4065.30 |
| TRTPN*ATPT | N Bel600 | 1 | Oxy60 | 0.5 | 2620.74 | 1940.37407 | 1.35 | 0.1776 | 0.05-1193.66 | 6435.14 |
| TRTPN*ATPT | N Bel600 | 1 | Oxy60 | 1 | 4916.60 | 1901.48407 | 2.59 | 0.0101 | 0.05 1178.66 | 8654.55 |
| TRTPN*ATPTI | NBel600 | 1 | Oxy60 | 2 | 6138.83 | 1866.33407 | 3.29 | 0.0011 | 0.05 2469.98 | 9807.69 |
| TRTPN*ATPTI | NBel600 | 1 | Oxy60 | 3 | 5589.36 | 1866.33407 | 2.99 | 0.0029 | 0.05 1920.50 | 9258.22 |
| TRTPN*ATPTI | NBel600 | 1 | Oxy60 | 4 | 5469.23 | 1866.33407 | 2.93 | 0.0036 | 0.05 1800.37 | 9138.08 |
| TRTPN*ATPT | N Bel600 | 1 | Plac | 0 | 852.03 | 1866.36407 | 0.46 | 0.6483 | 0.05-2816.87 | 4520.94 |
| TRTPN*ATPT | N Bel600 | 1 | Plac | 0.5 | -728.35 | 1866.36407 | -0.39 | 0.6966 | 0.05-4397.26 | 2940.55 |
| TRTPN*ATPT | N Bel600 | 1 | Plac | 1 | -1617.61 | 1866.36407 | -0.87 | 0.3866 | 0.05-5286.52 | 2051.29 |
| TRTPN*ATPT | N Bel600 | 1 | Plac | 2 | 2187.85 | 1866.36407 | 1.17 | 0.2418 | 0.05-1481.05 | 5856.75 |
| TRTPN*ATPT | N Bel600 | 1 | Plac | 3 | 2385.87 | 1866.36407 | 1.28 | 0.2019 | 0.05-1283.03 | 6054.78 |
| TRTPN*ATPT | N Bel600 | 1 | Plac | 4 | 993.03 | 1866.36407 | 0.53 | 0.5950 | 0.05-2675.88 | 4661.93 |
| TRTPN*ATPT | N Bel600 | 2 | Be1600 | 3 | 589.22 | 1864.91407 | 0.32 | 0.7522 | 0.05-3076.85 | 4255.28 |
| TRTPN*ATPT | N Bel600 | 2 | Be1600 | 4 | 572.96 | 1864.91407 | 0.31 | 0.7588 | 0.05-3093.11 | 4239.02 |
| TRTPN*ATPT | N Bel600 | 2 | Be1900 | 0 | -3614.03 | 1900.65407 | -1.90 | 0.0579 | 0.05-7350.33 | 122.28 |
| TRTPN*ATPT | N Bel600 | 2 | Be1900 | 0.5 | -5059.45 | 1866.36407 | -2.71 | 0.0070 | 0.05-8728.37 | -1390.54 |
| TRTPN*ATPT | N Bel600 | 2 | Be1900 | 1 | -2239.98 | 1866.36407 | -1.20 | 0.2308 | 0.05-5908.89 | 1428.93 |
| TRTPN*ATPT | N Bel600 | 2 | Be1900 | 2 | -482.23 | 1866.36407 | -0.26 | 0.7962 | 0.05-4151.14 | 3186.69 |
| TRTPN*ATPT | N Bel600 | 2 | Be1900 | 3 | 198.04 | 1866.36407 | 0.11 | 0.9155 | 0.05-3470.87 | 3866.95 |
| TRTPN*ATPT | N Bel600 | 2 | Be1900 | 4 | 1246.53 | 1866.36407 | 0.67 | 0.5046 | 0.05-2422.39 | 4915.44 |
| TRTPN*ATPT | N Bel600 | 2 | 0xy30 | 0 | -2407.47 | 1939.83407 | -1.24 | 0.2153 | 0.05-6220.81 | 1405.87 |
| TRTPN*ATPT | N Bel600 | 2 | 0xy30 | 0.5 | -135.32 | 1939.83407 | -0.07 | 0.9444 | 0.05-3948.66 | |
| TRTPN*ATPT | N Bel600 | 2 | 0xy30 | 1 | 1717.69 | 1900.00407 | 0.90 | 0.3665 | 0.05-2017.36 | 5452.73 |
| TRTPN*ATPT | NBel600 | 2 | 0xy30 | 2 | 861.94 | 1865.62407 | 0.46 | 0.6443 | 0.05-2805.51 | 4529.39 |
| TRTPN*ATPTI | NBel600 | 2 | 0xy30 | 3 | -732.90 | 1865.62407 | -0.39 | 0.6946 | 0.05-4400.34 | 2934.55 |

Program: A\_Bio3.sas Created: 02APR2020 7:35 POSTLOCK 

### Appendix 16.1.9.2.3 Statistical Methods and Analysis Output Supporting Table 14.2.4 Supporting Table 14.2.4

#### The Mixed Procedure

#### Parameter Code=MVMIPM

#### Differences of Least Squares Means

| | | | | | or nease . | squares neams | | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| | Planned | Analysis | | Analysis | | | | | | |
| | Treatment | Timepoint | Treatment | Timepoint | | Standard | | | | |
| Effect | (N) | (N) | (N) | (N) | Estimate | Error DFt | | | - | Upper |
| TRTPN*ATPTN | Be1600 | 2 | 0xy30 | 4 | -953.65 | 1865.62407 | -0.51 | 0.6095 | 0.05-4621.10 | 2713.80 |
| TRTPN*ATPTN | Be1600 | 2 | Oxy60 | 0 | -1318.78 | 1940.37407 | -0.68 | 0.4971 | 0.05-5133.18 | 2495.63 |
| TRTPN*ATPTN | Be1600 | 2 | Oxy60 | 0.5 | 1051.07 | 1940.37407 | 0.54 | 0.5883 | 0.05-2763.33 | 4865.47 |
| TRTPN*ATPTN | Be1600 | 2 | Oxy60 | 1 | 3346.93 | 1901.48407 | 1.76 | 0.0791 | 0.05 -391.02 | 7084.88 |
| TRTPN*ATPTN | Be1600 | 2 | Oxy60 | 2 | 4569.16 | 1866.33407 | 2.45 | 0.0148 | 0.05 900.31 | 8238.02 |
| TRTPN*ATPTN | Bel600 | 2 | Oxy60 | 3 | 4019.69 | 1866.33407 | 2.15 | 0.0318 | 0.05 350.83 | 7688.54 |
| TRTPN*ATPTN | Be1600 | 2 | Oxy60 | 4 | 3899.55 | 1866.33407 | 2.09 | 0.0373 | 0.05 230.70 | 7568.41 |
| TRTPN*ATPTN | Bel600 | 2 | Plac | 0 | -717.64 | 1866.36407 | -0.38 | 0.7008 | 0.05-4386.54 | 2951.27 |
| TRTPN*ATPTN | Be1600 | 2 | Plac | 0.5 | -2298.02 | 1866.36407 | -1.23 | 0.2189 | 0.05-5966.93 | 1370.88 |
| TRTPN*ATPTN | Bel600 | 2 | Plac | 1 | -3187.28 | 1866.36407 | -1.71 | 0.0884 | 0.05-6856.19 | 481.62 |
| TRTPN*ATPTN | Bel600 | 2 | Plac | 2 | 618.18 | 1866.36407 | 0.33 | 0.7406 | 0.05-3050.73 | 4287.08 |
| TRTPN*ATPTN | Bel600 | 2 | Plac | 3 | 816.20 | 1866.36407 | 0.44 | 0.6621 | 0.05-2852.71 | 4485.10 |
| TRTPN*ATPTN | Bel600 | 2 | Plac | 4 | -576.64 | 1866.36407 | -0.31 | 0.7575 | 0.05-4245.55 | 3092.26 |
| TRTPN*ATPTN | Bel600 | 3 | Be1600 | 4 | -16.2605 | 1864.91407 | -0.01 | 0.9930 | 0.05-3682.33 | 3649.81 |
| TRTPN*ATPTN | Bel600 | 3 | Be1900 | 0 | -4203.25 | 1900.65407 | -2.21 | 0.0276 | 0.05-7939.55 | -466.94 |
| TRTPN*ATPTN | Bel600 | 3 | Be1900 | 0.5 | -5648.67 | 1866.36407 | -3.03 | 0.0026 | 0.05-9317.58 | -1979.76 |
| TRTPN*ATPTN | Bel600 | 3 | Be1900 | 1 | -2829.20 | 1866.36407 | -1.52 | 0.1303 | 0.05-6498.11 | 839.71 |
| TRTPN*ATPTN | Bel600 | 3 | Be1900 | 2 | -1071.44 | 1866.36407 | -0.57 | 0.5662 | 0.05-4740.36 | 2597.47 |
| TRTPN*ATPTN | Bel600 | 3 | Be1900 | 3 | -391.18 | 1866.36407 | -0.21 | 0.8341 | 0.05-4060.09 | 3277.73 |
| TRTPN*ATPTN | Bel600 | 3 | Be1900 | 4 | 657.31 | 1866.36407 | 0.35 | 0.7249 | 0.05-3011.60 | 4326.22 |
| TRTPN*ATPTN | Bel600 | 3 | 0xy30 | 0 | -2996.69 | 1939.83407 | -1.54 | 0.1232 | 0.05-6810.03 | 816.65 |
| TRTPN*ATPTN | Bel600 | 3 | 0xy30 | 0.5 | -724.54 | 1939.83407 | -0.37 | 0.7090 | 0.05-4537.88 | 3088.80 |
| TRTPN*ATPTN | Bel600 | 3 | 0xy30 | 1 | 1128.47 | 1900.00407 | 0.59 | 0.5529 | 0.05-2606.58 | 4863.51 |
| TRTPN*ATPTN | Bel600 | 3 | 0xy30 | 2 | 272.72 | 1865.62407 | 0.15 | 0.8838 | 0.05-3394.72 | 3940.17 |
| TRTPN*ATPTN | Bel600 | 3 | 0xy30 | 3 | -1322.11 | 1865.62407 | -0.71 | 0.4789 | 0.05-4989.56 | 2345.33 |

Program: A Bio3.sas Created: 02APR2020 7:35 POSTLOCK 

### Appendix 16.1.9.2.3 Statistical Methods and Analysis Output Supporting Table 14.2.4 Supporting Table 14.2.4

#### The Mixed Procedure

#### Parameter Code=MVMIPM

#### Differences of Least Squares Means

| | Planned | Analysis | Planned | Analysis | | 100200 | | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| | Treatment | Timepoint | Treatment | Timepoint | | Standard | | | | |
| Effect | (N) | (N) | (N) | (N) | Estimate | Error DFt | Value Pr | r > t | Alpha Lower | Upper |
| TRTPN*ATPTN | 1Bel600 | 3 | Oxy30 | 4 | -1542.87 | 1865.62407 | -0.83 | 0.4087 | 0.05-5210.31 | 2124.58 |
| TRTPN*ATPTN | 1Bel600 | 3 | Oxy60 | 0 | -1907.99 | 1940.37407 | -0.98 | 0.3260 | 0.05-5722.39 | 1906.41 |
| TRTPN*ATPTN | 1Bel600 | 3 | Oxy60 | 0.5 | 461.85 | 1940.37407 | 0.24 | 0.8120 | 0.05-3352.55 | 4276.25 |
| TRTPN*ATPTN | 1Bel600 | 3 | Oxy60 | 1 | 2757.71 | 1901.48407 | 1.45 | 0.1477 | 0.05 -980.23 | 6495.66 |
| TRTPN*ATPTN | 1Bel600 | 3 | Oxy60 | 2 | 3979.94 | 1866.33407 | 2.13 | 0.0336 | 0.05 311.09 | 7648.80 |
| TRTPN*ATPTN | NBe1600 | 3 | Oxy60 | 3 | 3430.47 | 1866.33407 | 1.84 | 0.0668 | 0.05 -238.39 | 7099.33 |
| TRTPN*ATPTN | 1Bel600 | 3 | Oxy60 | 4 | 3310.34 | 1866.33407 | 1.77 | 0.0769 | 0.05 -358.52 | 6979.19 |
| TRTPN*ATPTN | NBe1600 | 3 | Plac | 0 | -1306.86 | 1866.36407 | -0.70 | 0.4842 | 0.05-4975.76 | 2362.05 |
| TRTPN*ATPTN | 1Bel600 | 3 | Plac | 0.5 | -2887.24 | 1866.36407 | -1.55 | 0.1226 | 0.05-6556.15 | 781.66 |
| TRTPN*ATPTN | 1Bel600 | 3 | Plac | 1 | -3776.50 | 1866.36407 | -2.02 | 0.0437 | 0.05-7445.41 | -107.60 |
| TRTPN*ATPTN | NBe1600 | 3 | Plac | 2 | 28.9600 | 1866.36407 | 0.02 | 0.9876 | 0.05-3639.94 | 3697.86 |
| TRTPN*ATPTN | NBe1600 | 3 | Plac | 3 | 226.98 | 1866.36407 | 0.12 | 0.9033 | 0.05-3441.92 | 3895.89 |
| TRTPN*ATPTN | 1Bel600 | 3 | Plac | 4 | -1165.86 | 1866.36407 | -0.62 | 0.5325 | 0.05-4834.77 | 2503.04 |
| TRTPN*ATPTN | NBe1600 | 4 | Be1900 | 0 | -4186.98 | 1900.65407 | -2.20 | 0.0282 | 0.05-7923.29 | -450.68 |
| TRTPN*ATPTN | 1Bel600 | 4 | Be1900 | 0.5 | -5632.41 | 1866.36407 | -3.02 | 0.0027 | 0.05-9301.32 | -1963.50 |
| TRTPN*ATPTN | NBe1600 | 4 | Be1900 | 1 | -2812.94 | 1866.36407 | -1.51 | 0.1325 | 0.05-6481.85 | 855.97 |
| TRTPN*ATPTN | 1Bel600 | 4 | Be1900 | 2 | -1055.18 | 1866.36407 | -0.57 | 0.5721 | 0.05-4724.10 | 2613.73 |
| TRTPN*ATPTN | 1Bel600 | 4 | Be1900 | 3 | -374.92 | 1866.36407 | -0.20 | 0.8409 | 0.05-4043.83 | 3293.99 |
| TRTPN*ATPTN | NBe1600 | 4 | Be1900 | 4 | 673.57 | 1866.36407 | 0.36 | 0.7184 | 0.05-2995.34 | 4342.48 |
| TRTPN*ATPTN | 1Bel600 | 4 | 0xy30 | 0 | -2980.43 | 1939.83407 | -1.54 | 0.1252 | 0.05-6793.77 | 832.91 |
| TRTPN*ATPTN | 1Bel600 | 4 | 0xy30 | 0.5 | -708.28 | 1939.83407 | -0.37 | 0.7152 | 0.05-4521.62 | 3105.06 |
| TRTPN*ATPTN | NBe1600 | 4 | 0xy30 | 1 | 1144.73 | 1900.00407 | 0.60 | 0.5472 | 0.05-2590.32 | 4879.77 |
| TRTPN*ATPTN | 1Bel600 | 4 | 0xy30 | 2 | 288.98 | 1865.62407 | 0.15 | 0.8770 | 0.05-3378.46 | 3956.43 |
| TRTPN*ATPTN | 1Bel600 | 4 | 0xy30 | 3 | -1305.85 | 1865.62407 | -0.70 | 0.4844 | 0.05-4973.30 | 2361.59 |
| TRTPN*ATPTN | NBe1600 | 4 | 0xy30 | 4 | -1526.61 | 1865.62407 | -0.82 | 0.4137 | 0.05-5194.05 | 2140.84 |

Program: A\_Bio3.sas Created: 02APR2020 7:35 POSTLOCK

#### Appendix 16.1.9.2.3 Statistical Methods and Analysis Output Supporting Table 14.2.4 Supporting Table 14.2.4

#### The Mixed Procedure

#### Parameter Code=MVMIPM

#### Differences of Least Squares Means

| | Planned | Analysis | | Analvsis | or hease . | oquares means | | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| | | - | | t Timepoint | | Standard | | | | |
| Effect | (N) | (N) | (N) | (N) | Estimate | Error DFt | Value P | r > t . | Alpha Lower | Upper |
| TRTPN*ATPT | N Bel600 | 4 | Oxy60 | 0 | -1891.73 | 1940.37407 | -0.97 | 0.3302 | 0.05-5706.13 | 1922.67 |
| TRTPN*ATPTI | N Bel600 | 4 | Oxy60 | 0.5 | 478.11 | 1940.37407 | 0.25 | 0.8055 | 0.05-3336.29 | 4292.51 |
| TRTPN*ATPT | N Bel600 | 4 | Oxy60 | 1 | 2773.97 | 1901.48407 | 1.46 | 0.1454 | 0.05 -963.97 | 6511.92 |
| TRTPN*ATPTI | NBel600 | 4 | Oxy60 | 2 | 3996.20 | 1866.33407 | 2.14 | 0.0329 | 0.05 327.35 | 7665.06 |
| TRTPN*ATPT | N Bel600 | 4 | Oxy60 | 3 | 3446.73 | 1866.33407 | 1.85 | 0.0655 | 0.05 -222.12 | 7115.59 |
| TRTPN*ATPT | N Bel600 | 4 | Oxy60 | 4 | 3326.60 | 1866.33407 | 1.78 | 0.0754 | 0.05 -342.26 | 6995.45 |
| TRTPN*ATPTI | NBel600 | 4 | Plac | 0 | -1290.60 | 1866.36407 | -0.69 | 0.4896 | 0.05-4959.50 | 2378.31 |
| TRTPN*ATPTI | NBel600 | 4 | Plac | 0.5 | -2870.98 | 1866.36407 | -1.54 | 0.1248 | 0.05-6539.89 | 797.92 |
| TRTPN*ATPTI | N Bel600 | 4 | Plac | 1 | -3760.24 | 1866.36407 | -2.01 | 0.0446 | 0.05-7429.15 | -91.3370 |
| TRTPN*ATPTI | N Bel600 | 4 | Plac | 2 | 45.2205 | 1866.36407 | 0.02 | 0.9807 | 0.05-3623.68 | 3714.13 |
| TRTPN*ATPTI | N Bel600 | 4 | Plac | 3 | 243.24 | 1866.36407 | 0.13 | 0.8964 | 0.05-3425.66 | 3912.15 |
| TRTPN*ATPTI | NBel600 | 4 | Plac | 4 | -1149.60 | 1866.36407 | -0.62 | 0.5383 | 0.05-4818.51 | 2519.30 |
| TRTPN*ATPT | N Bel900 | 0 | Be1900 | 0.5 | -1445.43 | 1899.15407 | -0.76 | 0.4470 | 0.05-5178.80 | 2287.94 |
| TRTPN*ATPT | N Bel900 | 0 | Be1900 | 1 | 1374.05 | 1899.15407 | 0.72 | 0.4698 | 0.05-2359.32 | 5107.42 |
| TRTPN*ATPT | N Bel900 | 0 | Be1900 | 2 | 3131.80 | 1899.15407 | 1.65 | 0.0999 | 0.05 -601.57 | 6865.17 |
| TRTPN*ATPT | N Bel900 | 0 | Be1900 | 3 | 3812.07 | 1899.15407 | 2.01 | 0.0454 | 0.05 78.6944 | 7545.44 |
| TRTPN*ATPT | N Bel900 | 0 | Be1900 | 4 | 4860.55 | 1899.15407 | 2.56 | 0.0108 | 0.05 1127.18 | 8593.93 |
| TRTPN*ATPTI | N Bel900 | 0 | Oxy30 | 0 | 1206.56 | 1972.55407 | 0.61 | 0.5411 | 0.05-2671.09 | 5084.21 |
| TRTPN*ATPT | N Bel900 | 0 | Oxy30 | 0.5 | 3478.71 | 1972.55407 | 1.76 | 0.0786 | 0.05 -398.94 | 7356.35 |
| TRTPN*ATPT | N Bel900 | 0 | Oxy30 | 1 | 5331.71 | 1933.93407 | 2.76 | 0.0061 | 0.05 1529.98 | 9133.44 |
| TRTPN*ATPTI | N Bel900 | 0 | Oxy30 | 2 | 4475.97 | 1900.64407 | 2.35 | 0.0190 | 0.05 739.68 | 8212.26 |
| TRTPN*ATPT | N Bel900 | 0 | Oxy30 | 3 | 2881.13 | 1900.64407 | 1.52 | 0.1303 | 0.05 -855.16 | 6617.42 |
| TRTPN*ATPT | N Bel900 | 0 | Oxy30 | 4 | 2660.38 | 1900.64407 | 1.40 | 0.1624 | 0.05-1075.92 | 6396.67 |
| TRTPN*ATPTI | N Bel900 | 0 | Oxy60 | 0 | 2295.25 | 1970.63407 | 1.16 | 0.2448 | 0.05-1578.63 | 6169.13 |
| TRTPN*ATPTI | N Bel900 | 0 | Oxy60 | 0.5 | 4665.10 | 1970.63407 | 2.37 | 0.0184 | 0.05 791.22 | 8538.98 |

Program: A Bio3.sas Created: 02APR2020 7:35 POSTLOCK 

### Appendix 16.1.9.2.3 Statistical Methods and Analysis Output Supporting Table 14.2.4 Supporting Table 14.2.4

#### The Mixed Procedure

#### Parameter Code=MVMIPM

#### Differences of Least Squares Means

| | Planned | Analysis | Planned | Analysis | 01 10000 . | squares means | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | Treatmen | t Timepoint | Treatment | t Timepoint | | Standard | | | | | |
| Effect | (N) | (N) | (N) | (N) | Estimate | Error DFt | Value P | r > t | Alpha | Lower | Upper |
| TRTPN*ATPT | N Bel900 | 0 | Oxy60 | 1 | 6960.96 | 1933.11407 | 3.60 | 0.0004 | 0.05 | 3160.84 | 10761 |
| TRTPN*ATPT | N Bel900 | 0 | Oxy60 | 2 | 8183.19 | 1899.14407 | 4.31 | <.0001 | 0.05 | 4449.84 | 11917 |
| TRTPN*ATPT | NBel900 | 0 | Oxy60 | 3 | 7633.72 | 1899.14407 | 4.02 | <.0001 | 0.05 | 3900.36 | 11367 |
| TRTPN*ATPT | N Bel900 | 0 | Oxy60 | 4 | 7513.58 | 1899.14407 | 3.96 | <.0001 | 0.05 | 3780.23 | 11247 |
| TRTPN*ATPT | NBel900 | 0 | Plac | 0 | 2896.39 | 1899.87407 | 1.52 | 0.1282 | 0.05 | -838.39 | 6631.17 |
| TRTPN*ATPT | NBel900 | 0 | Plac | 0.5 | 1316.00 | 1899.87407 | 0.69 | 0.4889 | 0.05 | -2418.78 | 5050.78 |
| TRTPN*ATPT | N Bel900 | 0 | Plac | 1 | 426.74 | 1899.87407 | 0.22 | 0.8224 | 0.05 | -3308.04 | 4161.53 |
| TRTPN*ATPT | NBel900 | 0 | Plac | 2 | 4232.21 | 1899.87407 | 2.23 | 0.0265 | 0.05 | 497.42 | 7966.99 |
| TRTPN*ATPT | N Bel900 | 0 | Plac | 3 | 4430.23 | 1899.87407 | 2.33 | 0.0202 | 0.05 | 695.44 | 8165.01 |
| TRTPN*ATPT | N Bel900 | 0 | Plac | 4 | 3037.38 | 1899.87407 | 1.60 | 0.1107 | 0.05 | -697.40 | 6772.17 |
| TRTPN*ATPT | NBel900 | 0.5 | Be1900 | 1 | 2819.47 | 1864.91407 | 1.51 | 0.1313 | 0.05 | -846.59 | 6485.54 |
| TRTPN*ATPT | NBel900 | 0.5 | Be1900 | 2 | 4577.23 | 1864.91407 | 2.45 | 0.0145 | 0.05 | 911.16 | 8243.29 |
| TRTPN*ATPT | N Bel900 | 0.5 | Be1900 | 3 | 5257.49 | 1864.91407 | 2.82 | 0.0051 | 0.05 | 1591.43 | 8923.56 |
| TRTPN*ATPT | N Bel900 | 0.5 | Be1900 | 4 | 6305.98 | 1864.91407 | 3.38 | 0.0008 | 0.05 | 2639.92 | 9972.05 |
| TRTPN*ATPT | NBel900 | 0.5 | Oxy30 | 0 | 2651.98 | 1938.86407 | 1.37 | 0.1721 | 0.05 | -1159.45 | 6463.42 |
| TRTPN*ATPT | N Bel900 | 0.5 | Oxy30 | 0.5 | 4924.13 | 1938.86407 | 2.54 | 0.0115 | 0.05 | 1112.69 | 8735.57 |
| TRTPN*ATPT | NBel900 | 0.5 | Oxy30 | 1 | 6777.14 | 1899.92407 | 3.57 | 0.0004 | 0.05 | 3042.26 | 10512 |
| TRTPN*ATPT | NBel900 | 0.5 | Oxy30 | 2 | 5921.40 | 1866.35407 | 3.17 | 0.0016 | 0.05 | 2252.51 | 9590.28 |
| TRTPN*ATPT | N Bel900 | 0.5 | Oxy30 | 3 | 4326.56 | 1866.35407 | 2.32 | 0.0209 | 0.05 | 657.67 | 7995.44 |
| TRTPN*ATPT | NBel900 | 0.5 | Oxy30 | 4 | 4105.80 | 1866.35407 | 2.20 | 0.0284 | 0.05 | 436.92 | 7774.69 |
| TRTPN*ATPT | NBel900 | 0.5 | Oxy60 | 0 | 3740.68 | 1937.93407 | 1.93 | 0.0543 | 0.05 | -68.9214 | 7550.28 |
| TRTPN*ATPT | N Bel900 | 0.5 | Oxy60 | 0.5 | 6110.52 | 1937.93407 | 3.15 | 0.0017 | 0.05 | 2300.92 | 9920.12 |
| TRTPN*ATPT | NBel900 | 0.5 | Oxy60 | 1 | 8406.39 | 1900.81407 | 4.42 | <.0001 | 0.05 | 4669.76 | 12143 |
| TRTPN*ATPT | NBel900 | 0.5 | Oxy60 | 2 | 9628.62 | 1865.66407 | 5.16 | <.0001 | 0.05 | 5961.08 | 13296 |
| TRTPN*ATPT | NBel900 | 0.5 | Oxy60 | 3 | 9079.14 | 1865.66407 | 4.87 | <.0001 | 0.05 | 5411.61 | 12747 |

Program: A\_Bio3.sas Created: 02APR2020 7:35 POSTLOCK

Appendix 16.1.9.2.3
Statistical Methods and Analysis Output Supporting Table 14.2.4
Supporting Table 14.2.4

#### The Mixed Procedure

#### Parameter Code=MVMIPM

#### Differences of Least Squares Means

| | | | | | or nease . | oquares means | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | Planned | Analysis | | Analysis | | | | | | | |
| | Treatment | - | Treatment | Timepoint | | Standard | | | | | |
| Effect | (N) | (N) | (N) | (N) | Estimate | Error DFt | | | | Lower | Upper |
| TRTPN*ATPTN | Be1900 | 0.5 | Oxy60 | 4 | 8959.01 | 1865.66407 | 4.80 | <.0001 | 0.05 | 5291.47 | 12627 |
| TRTPN*ATPTN | Be1900 | 0.5 | Plac | 0 | 4341.82 | 1866.33407 | 2.33 | 0.0205 | 0.05 | 672.97 | 8010.66 |
| TRTPN*ATPTN | Bel900 | 0.5 | Plac | 0.5 | 2761.43 | 1866.33407 | 1.48 | 0.1398 | 0.05 | -907.42 | 6430.27 |
| TRTPN*ATPTN | Be1900 | 0.5 | Plac | 1 | 1872.17 | 1866.33407 | 1.00 | 0.3164 | 0.05- | -1796.68 | 5541.02 |
| TRTPN*ATPTN | Bel900 | 0.5 | Plac | 2 | 5677.63 | 1866.33407 | 3.04 | 0.0025 | 0.05 | 2008.79 | 9346.48 |
| TRTPN*ATPTN | Bel900 | 0.5 | Plac | 3 | 5875.65 | 1866.33407 | 3.15 | 0.0018 | 0.05 | 2206.81 | 9544.50 |
| TRTPN*ATPTN | Bel900 | 0.5 | Plac | 4 | 4482.81 | 1866.33407 | 2.40 | 0.0168 | 0.05 | 813.96 | 8151.66 |
| TRTPN*ATPTN | Bel900 | 1 | Be1900 | 2 | 1757.75 | 1864.91407 | 0.94 | 0.3465 | 0.05- | -1908.31 | 5423.82 |
| TRTPN*ATPTN | Bel900 | 1 | Be1900 | 3 | 2438.02 | 1864.91407 | 1.31 | 0.1918 | 0.05- | -1228.05 | 6104.08 |
| TRTPN*ATPTN | Bel900 | 1 | Be1900 | 4 | 3486.51 | 1864.91407 | 1.87 | 0.0623 | 0.05 | -179.56 | 7152.57 |
| TRTPN*ATPTN | Bel900 | 1 | 0xy30 | 0 | -167.49 | 1938.86407 | -0.09 | 0.9312 | 0.05- | -3978.93 | 3643.95 |
| TRTPN*ATPTN | Be1900 | 1 | 0xy30 | 0.5 | 2104.66 | 1938.86407 | 1.09 | 0.2783 | 0.05- | -1706.78 | 5916.10 |
| TRTPN*ATPTN | Bel900 | 1 | 0xy30 | 1 | 3957.67 | 1899.92407 | 2.08 | 0.0379 | 0.05 | 222.79 | 7692.54 |
| TRTPN*ATPTN | Be1900 | 1 | 0xy30 | 2 | 3101.92 | 1866.35407 | 1.66 | 0.0973 | 0.05 | -566.96 | 6770.81 |
| TRTPN*ATPTN | Bel900 | 1 | 0xy30 | 3 | 1507.08 | 1866.35407 | 0.81 | 0.4198 | 0.05- | -2161.80 | 5175.97 |
| TRTPN*ATPTN | Bel900 | 1 | 0xy30 | 4 | 1286.33 | 1866.35407 | 0.69 | 0.4911 | 0.05- | -2382.56 | 4955.22 |
| TRTPN*ATPTN | Be1900 | 1 | Oxy60 | 0 | 921.20 | 1937.93407 | 0.48 | 0.6348 | 0.05- | -2888.39 | 4730.80 |
| TRTPN*ATPTN | Bel900 | 1 | Oxy60 | 0.5 | 3291.05 | 1937.93407 | 1.70 | 0.0902 | 0.05 | -518.55 | 7100.65 |
| TRTPN*ATPTN | Bel900 | 1 | Oxy60 | 1 | 5586.91 | 1900.81407 | 2.94 | 0.0035 | 0.05 | 1850.29 | 9323.53 |
| TRTPN*ATPTN | Be1900 | 1 | Oxy60 | 2 | 6809.14 | 1865.66407 | 3.65 | 0.0003 | 0.05 | 3141.61 | 10477 |
| TRTPN*ATPTN | Bel900 | 1 | Oxy60 | 3 | 6259.67 | 1865.66407 | 3.36 | 0.0009 | 0.05 | 2592.14 | 9927.20 |
| TRTPN*ATPTN | Be1900 | 1 | Oxy60 | 4 | 6139.53 | 1865.66407 | 3.29 | 0.0011 | 0.05 | 2472.00 | 9807.07 |
| TRTPN*ATPTN | Be1900 | 1 | Plac | 0 | 1522.34 | 1866.33407 | 0.82 | 0.4152 | 0.05- | -2146.50 | 5191.19 |
| TRTPN*ATPTN | Be1900 | 1 | Plac | 0.5 | -58.0443 | 1866.33407 | -0.03 | 0.9752 | 0.05- | -3726.89 | 3610.80 |
| TRTPN*ATPTN | Bel900 | 1 | Plac | 1 | -947.30 | 1866.33407 | -0.51 | 0.6120 | 0.05- | -4616.15 | 2721.54 |

Program: A Bio3.sas Created: 02APR2020 7:35 POSTLOCK 

## Appendix 16.1.9.2.3 Statistical Methods and Analysis Output Supporting Table 14.2.4 Supporting Table 14.2.4

#### The Mixed Procedure

#### Parameter Code=MVMIPM

#### Differences of Least Squares Means

| | <b>5</b> 1 1 | | | | or heade . | oquares means | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | Planned | Analysis | | Analysis | | Q1 1 1 | | | | | |
| 766 | | - | | Timepoint | | Standard | | | - 1 1 | _ | |
| Effect | (N) | (N) | (N) | (N) | Estimate | Error DF t | | | | Lower | Upper |
| TRTPN*ATPTN | Be1900 | 1 | Plac | 2 | | 1866.33407 | 1.53 | 0.1264 | | -810.69 | 6527.00 |
| TRTPN*ATPTN | Bel900 | 1 | Plac | 3 | 3056.18 | 1866.33407 | 1.64 | 0.1023 | 0.05 | -612.67 | 6725.03 |
| TRTPN*ATPTN | Bel900 | 1 | Plac | 4 | 1663.34 | 1866.33407 | 0.89 | 0.3733 | 0.05- | -2005.51 | 5332.18 |
| TRTPN*ATPTN | Bel900 | 2 | Be1900 | 3 | 680.26 | 1864.91407 | 0.36 | 0.7155 | 0.05- | -2985.80 | 4346.33 |
| TRTPN*ATPTN | Bel900 | 2 | Be1900 | 4 | 1728.75 | 1864.91407 | 0.93 | 0.3545 | 0.05- | -1937.31 | 5394.82 |
| TRTPN*ATPTN | Bel900 | 2 | Oxy30 | 0 | -1925.24 | 1938.86407 | -0.99 | 0.3213 | 0.05- | -5736.68 | 1886.19 |
| TRTPN*ATPTN | Be1900 | 2 | Oxy30 | 0.5 | 346.90 | 1938.86407 | 0.18 | 0.8581 | 0.05- | -3464.53 | 4158.34 |
| TRTPN*ATPTN | Bel900 | 2 | 0xy30 | 1 | 2199.91 | 1899.92407 | 1.16 | 0.2476 | 0.05- | -1534.96 | 5934.79 |
| TRTPN*ATPTN | Be1900 | 2 | Oxy30 | 2 | 1344.17 | 1866.35407 | 0.72 | 0.4718 | 0.05- | -2324.72 | 5013.06 |
| TRTPN*ATPTN | Bel900 | 2 | 0xy30 | 3 | -250.67 | 1866.35407 | -0.13 | 0.8932 | 0.05- | -3919.56 | 3418.22 |
| TRTPN*ATPTN | Bel900 | 2 | Oxy30 | 4 | -471.42 | 1866.35407 | -0.25 | 0.8007 | 0.05- | -4140.31 | 3197.46 |
| TRTPN*ATPTN | Bel900 | 2 | Oxy60 | 0 | -836.55 | 1937.93407 | -0.43 | 0.6662 | 0.05- | -4646.15 | 2973.05 |
| TRTPN*ATPTN | Bel900 | 2 | Oxy60 | 0.5 | 1533.29 | 1937.93407 | 0.79 | 0.4293 | 0.05- | -2276.31 | 5342.89 |
| TRTPN*ATPTN | Bel900 | 2 | Oxy60 | 1 | 3829.16 | 1900.81407 | 2.01 | 0.0446 | 0.05 | 92.5345 | 7565.78 |
| TRTPN*ATPTN | Bel900 | 2 | Oxy60 | 2 | 5051.39 | 1865.66407 | 2.71 | 0.0071 | 0.05 | 1383.85 | 8718.92 |
| TRTPN*ATPTN | Be1900 | 2 | Oxy60 | 3 | 4501.91 | 1865.66407 | 2.41 | 0.0163 | 0.05 | 834.38 | 8169.45 |
| TRTPN*ATPTN | Be1900 | 2 | Oxy60 | 4 | 4381.78 | 1865.66407 | 2.35 | 0.0193 | 0.05 | 714.25 | 8049.31 |
| TRTPN*ATPTN | Be1900 | 2 | Plac | 0 | -235.41 | 1866.33407 | -0.13 | 0.8997 | 0.05- | -3904.26 | 3433.43 |
| TRTPN*ATPTN | Be1900 | 2 | Plac | 0.5 | -1815.80 | 1866.33407 | -0.97 | 0.3312 | 0.05- | -5484.64 | 1853.05 |
| TRTPN*ATPTN | Be1900 | 2 | Plac | 1 | -2705.06 | 1866.33407 | -1.45 | 0.1480 | 0.05- | -6373.90 | 963.79 |
| TRTPN*ATPTN | Be1900 | 2 | Plac | 2 | 1100.40 | 1866.33407 | 0.59 | 0.5558 | 0.05- | -2568.44 | 4769.25 |
| TRTPN*ATPTN | Be1900 | 2 | Plac | 3 | 1298.43 | 1866.33407 | 0.70 | 0.4870 | 0.05- | -2370.42 | 4967.27 |
| TRTPN*ATPTN | Be1900 | 2 | Plac | 4 | -94.4181 | 1866.33407 | -0.05 | 0.9597 | 0.05- | -3763.26 | 3574.43 |
| TRTPN*ATPTN | Bel900 | 3 | Be1900 | 4 | 1048.49 | 1864.91407 | 0.56 | 0.5743 | 0.05- | -2617.58 | 4714.55 |
| TRTPN*ATPTN | Be1900 | 3 | Oxy30 | 0 | -2605.51 | 1938.86407 | -1.34 | 0.1798 | 0.05- | -6416.95 | 1205.93 |

Program: A\_Bio3.sas Created: 02APR2020 7:35 POSTLOCK


### Appendix 16.1.9.2.3 Statistical Methods and Analysis Output Supporting Table 14.2.4 Supporting Table 14.2.4

#### The Mixed Procedure

#### Parameter Code=MVMIPM

#### Differences of Least Squares Means

| | Planned | Analysis | | Analysis | or hease . | squares means | | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| | | 4 | | t Timepoint | | Standard | | | | |
| Effect | (N) | (N) | (N) | (N) | Estimate | Error DFt | Value P | r > t | Alpha Lower | Upper |
| TRTPN*ATPT | NBel900 | 3 | Oxy30 | 0.5 | -333.36 | 1938.86407 | -0.17 | 0.8636 | 0.05-4144.80 | 3478.08 |
| TRTPN*ATPT | NBel900 | 3 | Oxy30 | 1 | 1519.65 | 1899.92407 | 0.80 | 0.4243 | 0.05-2215.23 | 5254.52 |
| TRTPN*ATPT | NBel900 | 3 | Oxy30 | 2 | 663.90 | 1866.35407 | 0.36 | 0.7222 | 0.05-3004.98 | 4332.79 |
| TRTPN*ATPT | N Bel900 | 3 | Oxy30 | 3 | -930.93 | 1866.35407 | -0.50 | 0.6182 | 0.05-4599.82 | 2737.95 |
| TRTPN*ATPT | N Bel900 | 3 | Oxy30 | 4 | -1151.69 | 1866.35407 | -0.62 | 0.5375 | 0.05-4820.57 | 2517.20 |
| TRTPN*ATPT | N Bel900 | 3 | Oxy60 | 0 | -1516.81 | 1937.93407 | -0.78 | 0.4343 | 0.05-5326.41 | 2292.79 |
| TRTPN*ATPT | N Bel900 | 3 | Oxy60 | 0.5 | 853.03 | 1937.93407 | 0.44 | 0.6600 | 0.05-2956.57 | 4662.63 |
| TRTPN*ATPT | N Bel900 | 3 | Oxy60 | 1 | 3148.89 | 1900.81407 | 1.66 | 0.0984 | 0.05 -587.73 | 6885.52 |
| TRTPN*ATPT | N Bel900 | 3 | Oxy60 | 2 | 4371.12 | 1865.66407 | 2.34 | 0.0196 | 0.05 703.59 | 8038.66 |
| TRTPN*ATPT | N Bel900 | 3 | Oxy60 | 3 | 3821.65 | 1865.66407 | 2.05 | 0.0412 | 0.05 154.12 | 7489.18 |
| TRTPN*ATPT | N Bel900 | 3 | Oxy60 | 4 | 3701.52 | 1865.66407 | 1.98 | 0.0479 | 0.05 33.9823 | 7369.05 |
| TRTPN*ATPT | N Bel900 | 3 | Plac | 0 | -915.68 | 1866.33407 | -0.49 | 0.6240 | 0.05-4584.52 | 2753.17 |
| TRTPN*ATPT | N Bel900 | 3 | Plac | 0.5 | -2496.06 | 1866.33407 | -1.34 | 0.1818 | 0.05-6164.91 | 1172.78 |
| TRTPN*ATPT | N Bel900 | 3 | Plac | 1 | -3385.32 | 1866.33407 | -1.81 | 0.0704 | 0.05-7054.17 | 283.52 |
| TRTPN*ATPT | N Bel900 | 3 | Plac | 2 | 420.14 | 1866.33407 | 0.23 | 0.8220 | 0.05-3248.71 | 4088.99 |
| TRTPN*ATPT | N Bel900 | 3 | Plac | 3 | 618.16 | 1866.33407 | 0.33 | 0.7407 | 0.05-3050.68 | 4287.01 |
| TRTPN*ATPT | N Bel900 | 3 | Plac | 4 | -774.68 | 1866.33407 | -0.42 | 0.6783 | 0.05-4443.53 | 2894.16 |
| TRTPN*ATPT | N Bel900 | 4 | Oxy30 | 0 | -3654.00 | 1938.86407 | -1.88 | 0.0602 | 0.05-7465.44 | 157.44 |
| TRTPN*ATPT | N Bel900 | 4 | Oxy30 | 0.5 | -1381.85 | 1938.86407 | -0.71 | 0.4764 | 0.05-5193.29 | 2429.59 |
| TRTPN*ATPT | N Bel900 | 4 | Oxy30 | 1 | 471.16 | 1899.92407 | 0.25 | 0.8043 | 0.05-3263.72 | 4206.03 |
| TRTPN*ATPT | N Bel900 | 4 | Oxy30 | 2 | -384.59 | 1866.35407 | -0.21 | 0.8368 | 0.05-4053.47 | 3284.30 |
| TRTPN*ATPT | N Bel900 | 4 | Oxy30 | 3 | -1979.42 | 1866.35407 | -1.06 | 0.2895 | 0.05-5648.31 | 1689.46 |
| TRTPN*ATPT | NBel900 | 4 | Oxy30 | 4 | -2200.18 | 1866.35407 | -1.18 | 0.2391 | 0.05-5869.06 | 1468.71 |
| TRTPN*ATPT | NBel900 | 4 | Oxy60 | 0 | -2565.30 | 1937.93407 | -1.32 | 0.1863 | 0.05-6374.90 | 1244.30 |
| TRTPN*ATPT | NBel900 | 4 | Oxy60 | 0.5 | -195.46 | 1937.93407 | -0.10 | 0.9197 | 0.05-4005.06 | 3614.14 |

Program: A\_Bio3.sas Created: 02APR2020 7:35 POSTLOCK 

### Appendix 16.1.9.2.3 Statistical Methods and Analysis Output Supporting Table 14.2.4 Supporting Table 14.2.4

#### The Mixed Procedure

#### Parameter Code=MVMIPM

#### Differences of Least Squares Means

| | | | | | or heade i | oquares means | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | Planned | Analysis | | Analysis | | | | | | | |
| | | - | Treatment | - | | Standard | | | | | |
| Effect | (N) | (N) | (N) | (N) | Estimate | Error DFt | | | | Lower | Upper |
| TRTPN*ATPTN | Be1900 | 4 | Oxy60 | 1 | 2100.40 | 1900.81407 | 1.11 | 0.2698 | 0.05-1 | 636.22 | 5837.03 |
| TRTPN*ATPTN | Be1900 | 4 | Oxy60 | 2 | | 1865.66407 | 1.78 | 0.0757 | 0.05 - | 344.90 | 6990.17 |
| TRTPN*ATPTN | Be1900 | 4 | Oxy60 | 3 | 2773.16 | 1865.66407 | 1.49 | 0.1379 | 0.05 - | 894.37 | 6440.69 |
| TRTPN*ATPTN | Be1900 | 4 | Oxy60 | 4 | 2653.03 | 1865.66407 | 1.42 | 0.1558 | 0.05-1 | 014.51 | 6320.56 |
| TRTPN*ATPTN | Be1900 | 4 | Plac | 0 | -1964.16 | 1866.33407 | -1.05 | 0.2932 | 0.05-5 | 633.01 | 1704.68 |
| TRTPN*ATPTN | Bel900 | 4 | Plac | 0.5 | -3544.55 | 1866.33407 | -1.90 | 0.0582 | 0.05-7 | 213.40 | 124.29 |
| TRTPN*ATPTN | Be1900 | 4 | Plac | 1 | -4433.81 | 1866.33407 | -2.38 | 0.0180 | 0.05-8 | 3102.66 | -764.97 |
| TRTPN*ATPTN | Bel900 | 4 | Plac | 2 | -628.35 | 1866.33407 | -0.34 | 0.7365 | 0.05-4 | 1297.19 | 3040.50 |
| TRTPN*ATPTN | Be1900 | 4 | Plac | 3 | -430.33 | 1866.33407 | -0.23 | 0.8178 | 0.05-4 | 1099.17 | 3238.52 |
| TRTPN*ATPTN | Bel900 | 4 | Plac | 4 | -1823.17 | 1866.33407 | -0.98 | 0.3292 | 0.05-5 | 492.02 | 1845.67 |
| TRTPN*ATPTN | Oxy30 | 0 | Oxy30 | 0.5 | 2272.15 | 2003.24407 | 1.13 | 0.2574 | 0.05-1 | 665.84 | 6210.13 |
| TRTPN*ATPTN | Oxy30 | 0 | Oxy30 | 1 | 4125.16 | 1968.65407 | 2.10 | 0.0368 | 0.05 | 255.17 | 7995.14 |
| TRTPN*ATPTN | Oxy30 | 0 | Oxy30 | 2 | 3269.41 | 1939.06407 | 1.69 | 0.0925 | 0.05 - | 542.40 | 7081.23 |
| TRTPN*ATPTN | Oxy30 | 0 | Oxy30 | 3 | 1674.57 | 1939.06407 | 0.86 | 0.3883 | 0.05-2 | 2137.24 | 5486.39 |
| TRTPN*ATPTN | Oxy30 | 0 | Oxy30 | 4 | 1453.82 | 1939.06407 | 0.75 | 0.4538 | 0.05-2 | 357.99 | 5265.63 |
| TRTPN*ATPTN | Oxy30 | 0 | Oxy60 | 0 | 1088.69 | 2010.59407 | 0.54 | 0.5885 | 0.05-2 | 2863.74 | 5041.13 |
| TRTPN*ATPTN | Oxy30 | 0 | Oxy60 | 0.5 | 3458.54 | 2010.59407 | 1.72 | 0.0862 | 0.05 - | 493.90 | 7410.98 |
| TRTPN*ATPTN | Oxy30 | 0 | Oxy60 | 1 | 5754.40 | 1975.27407 | 2.91 | 0.0038 | 0.05 1 | 871.40 | 9637.40 |
| TRTPN*ATPTN | Oxy30 | 0 | Oxy60 | 2 | 6976.63 | 1940.65407 | 3.59 | 0.0004 | 0.05 3 | 3161.68 | 10792 |
| TRTPN*ATPTN | Oxy30 | 0 | Oxy60 | 3 | 6427.16 | 1940.65407 | 3.31 | 0.0010 | 0.05 2 | 2612.20 | 10242 |
| TRTPN*ATPTN | Oxy30 | 0 | Oxy60 | 4 | 6307.02 | 1940.65407 | 3.25 | 0.0013 | 0.05 2 | 2492.07 | 10122 |
| TRTPN*ATPTN | Oxy30 | 0 | Plac | 0 | 1689.83 | 1938.87407 | 0.87 | 0.3840 | 0.05-2 | 2121.62 | 5501.29 |
| TRTPN*ATPTN | Oxy30 | 0 | Plac | 0.5 | 109.45 | 1938.87407 | 0.06 | 0.9550 | 0.05-3 | 3702.01 | 3920.90 |
| TRTPN*ATPTN | Oxy30 | 0 | Plac | 1 | -779.81 | 1938.87407 | -0.40 | 0.6877 | 0.05-4 | 1591.27 | 3031.64 |
| TRTPN*ATPTN | Оху30 | 0 | Plac | 2 | 3025.65 | 1938.87407 | 1.56 | 0.1194 | 0.05 - | 785.81 | 6837.10 |

Program: A Bio3.sas Created: 02APR2020 7:35 POSTLOCK


## Appendix 16.1.9.2.3 Statistical Methods and Analysis Output Supporting Table 14.2.4 Supporting Table 14.2.4

#### The Mixed Procedure

#### Parameter Code=MVMIPM

#### Differences of Least Squares Means

| | D1 | 20.03.01 | | | or heade . | oquares means | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | Planned | Analysis | | Analysis<br>Timepoint | _ | Standard | | | | | |
| Effect | (N) | (N) | (N) | (N) | Estimate | Error DF t | 772 ] 110 D | ~ \ l+l | 7 l nha | Lower | Upper |
| | , , | 0 | Plac | 3 | | 1938.87407 | 1.66 | | | -587.79 | |
| TRTPN*ATPT | - | • | | - | | | | | | | |
| TRTPN*ATPT | 4 | 0 | Plac | 4 | | 1938.87407 | 0.94 | | | -1980.63 | 5642.28 |
| TRTPN*ATPT | 4 | 0.5 | Oxy30 | 1 | | 1968.65407 | 0.94 | | | -2016.98 | |
| TRTPN*ATPT | 4 | 0.5 | Oxy30 | 2 | | 1939.06407 | 0.51 | 0.6073 | | -2814.55 | |
| TRTPN*ATPT | 4 | 0.5 | Oxy30 | 3 | | 1939.06407 | -0.31 | 0.7581 | | -4409.39 | 3214.24 |
| TRTPN*ATPT | 4 | 0.5 | 0xy30 | 4 | | 1939.06407 | -0.42 | | | -4630.14 | |
| TRTPN*ATPT | и Оху30 | 0.5 | Oxy60 | 0 | -1183.45 | 2010.59407 | -0.59 | 0.5564 | 0.05- | -5135.89 | 2768.98 |
| TRTPN*ATPT | N Оху30 | 0.5 | Oxy60 | 0.5 | 1186.39 | 2010.59407 | 0.59 | 0.5555 | 0.05- | -2766.05 | 5138.83 |
| TRTPN*ATPT | и Оху30 | 0.5 | Oxy60 | 1 | 3482.25 | 1975.27407 | 1.76 | 0.0787 | 0.05 | -400.75 | 7365.26 |
| TRTPN*ATPT | и Оху30 | 0.5 | Oxy60 | 2 | 4704.48 | 1940.65407 | 2.42 | 0.0158 | 0.05 | 889.53 | 8519.44 |
| TRTPN*ATPT | NOxy30 | 0.5 | Oxy60 | 3 | 4155.01 | 1940.65407 | 2.14 | 0.0329 | 0.05 | 340.05 | 7969.97 |
| TRTPN*ATPT | NOxy30 | 0.5 | Oxy60 | 4 | 4034.88 | 1940.65407 | 2.08 | 0.0382 | 0.05 | 219.92 | 7849.83 |
| TRTPN*ATPT | NOxy30 | 0.5 | Plac | 0 | -582.32 | 1938.87407 | -0.30 | 0.7641 | 0.05- | -4393.77 | 3229.14 |
| TRTPN*ATPT | NOxy30 | 0.5 | Plac | 0.5 | -2162.70 | 1938.87407 | -1.12 | 0.2653 | 0.05- | -5974.16 | 1648.75 |
| TRTPN*ATPT | N Oxy30 | 0.5 | Plac | 1 | -3051.96 | 1938.87407 | -1.57 | 0.1162 | 0.05- | -6863.42 | 759.49 |
| TRTPN*ATPT | N Oxy30 | 0.5 | Plac | 2 | 753.50 | 1938.87407 | 0.39 | 0.6978 | 0.05- | -3057.96 | 4564.96 |
| TRTPN*ATPT | N Oxv30 | 0.5 | Plac | 3 | 951.52 | 1938.87407 | 0.49 | 0.6239 | 0.05- | -2859.93 | 4762.98 |
| TRTPN*ATPT | N Oxv30 | 0.5 | Plac | 4 | -441.32 | 1938.87407 | -0.23 | 0.8201 | 0.05- | -4252.78 | 3370.13 |
| TRTPN*ATPT | N Oxv30 | 1 | Oxy30 | 2 | -855.74 | 1899.26407 | -0.45 | 0.6525 | 0.05- | -4589.34 | 2877.85 |
| TRTPN*ATPT | N Oxv30 | 1 | 0xy30 | 3 | -2450.58 | 1899.26407 | -1.29 | 0.1977 | 0.05- | -6184.17 | 1283.01 |
| TRTPN*ATPT | 4 | 1 | Oxy30 | 4 | | 1899.26407 | -1.41 | 0.1603 | | -6404.93 | 1062.26 |
| TRTPN*ATPT | 4 | 1 | Oxy60 | 0 | | 1972.42407 | -1.54 | | | -6913.87 | 840.94 |
| TRTPN*ATPT | 4 | 1 | Oxy60 | 0.5 | | 1972.42407 | -0.34 | 0.7356 | | -4544.02 | 3210.79 |
| TRTPN*ATPT | - | 1 | Oxy60 | 1 | | 1935.67407 | 0.84 | 0.4005 | | -2175.91 | |
| TRTPN*ATPT | 4 | 1 | Oxy60 | 2 | | 1900.76407 | 1.50 | | | -885.06 | |
| INIEN.AILI | IN OVÄNO | T | OAYOU | 4 | 2001.40 | 1900.70407 | 1.30 | 0.1343 | 0.05 | -003.00 | 0300.02 |

Program: A\_Bio3.sas Created: 02APR2020 7:35 POSTLOCK


Appendix 16.1.9.2.3
Statistical Methods and Analysis Output Supporting Table 14.2.4
Supporting Table 14.2.4

#### The Mixed Procedure

#### Parameter Code=MVMIPM

#### Differences of Least Squares Means

| | Planned | Analysis | | Analvsis | or bease . | oquares neams | | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| | Treatment | _ | | Timepoint | | Standard | | | | |
| Effect | (N) | (N) | (N) | (N) | Estimate | Error DFt | Value Pa | r > t . | Alpha Lower | Upper |
| TRTPN*ATPT | 10xy30 | 1 | Oxy60 | 3 | 2302.00 | 1900.76407 | 1.21 | 0.2266 | 0.05-1434.54 | 6038.54 |
| TRTPN*ATPT | N 0xy30 | 1 | Oxy60 | 4 | 2181.87 | 1900.76407 | 1.15 | 0.2517 | 0.05-1554.67 | 5918.41 |
| TRTPN*ATPT | N 0xy30 | 1 | Plac | 0 | -2435.32 | 1899.93407 | -1.28 | 0.2006 | 0.05-6170.22 | 1299.58 |
| TRTPN*ATPT | NOxy30 | 1 | Plac | 0.5 | -4015.71 | 1899.93407 | -2.11 | 0.0352 | 0.05-7750.61 | -280.81 |
| TRTPN*ATPT | N 0xy30 | 1 | Plac | 1 | -4904.97 | 1899.93407 | -2.58 | 0.0102 | 0.05-8639.87 | -1170.07 |
| TRTPN*ATPT | N 0xy30 | 1 | Plac | 2 | -1099.51 | 1899.93407 | -0.58 | 0.5631 | 0.05-4834.41 | 2635.39 |
| TRTPN*ATPT | N 0xy30 | 1 | Plac | 3 | -901.49 | 1899.93407 | -0.47 | 0.6354 | 0.05-4636.39 | 2833.41 |
| TRTPN*ATPT | N 0xy30 | 1 | Plac | 4 | -2294.33 | 1899.93407 | -1.21 | 0.2279 | 0.05-6029.23 | 1440.57 |
| TRTPN*ATPT | 0 EyxO | 2 | Oxy30 | 3 | -1594.84 | 1864.91407 | -0.86 | 0.3930 | 0.05-5260.90 | 2071.23 |
| TRTPN*ATPT | 0 EyxO V | 2 | Oxy30 | 4 | -1815.59 | 1864.91407 | -0.97 | 0.3309 | 0.05-5481.66 | 1850.47 |
| TRTPN*ATPT | 0 EyxO V | 2 | Oxy60 | 0 | -2180.72 | 1939.53407 | -1.12 | 0.2615 | 0.05-5993.46 | 1632.03 |
| TRTPN*ATPT | 4 | 2 | Oxy60 | 0.5 | 189.13 | 1939.53407 | 0.10 | 0.9224 | 0.05-3623.62 | 4001.87 |
| TRTPN*ATPT | 0 EyxO | 2 | Oxy60 | 1 | 2484.99 | 1901.48407 | 1.31 | 0.1920 | 0.05-1252.95 | 6222.93 |
| TRTPN*ATPT | 0 EyxO | 2 | Oxy60 | 2 | 3707.22 | 1866.32407 | 1.99 | 0.0477 | 0.05 38.3874 | 7376.05 |
| TRTPN*ATPT | 0 EyxO | 2 | Oxy60 | 3 | 3157.75 | 1866.32407 | 1.69 | 0.0914 | 0.05 -511.09 | 6826.58 |
| TRTPN*ATPT | 0 EyxO | 2 | Oxy60 | 4 | 3037.61 | 1866.32407 | 1.63 | 0.1044 | 0.05 -631.22 | 6706.45 |
| TRTPN*ATPT | 0 EyxO | 2 | Plac | 0 | -1579.58 | 1866.36407 | -0.85 | 0.3979 | 0.05-5248.50 | 2089.34 |
| TRTPN*ATPT | 0 EyxO V | 2 | Plac | 0.5 | -3159.97 | 1866.36407 | -1.69 | 0.0912 | 0.05-6828.88 | 508.95 |
| TRTPN*ATPT | 0 EyxO | 2 | Plac | 1 | -4049.23 | 1866.36407 | -2.17 | 0.0306 | 0.05-7718.14 | -380.31 |
| TRTPN*ATPT | 0 EyxO | 2 | Plac | 2 | -243.76 | 1866.36407 | -0.13 | 0.8961 | 0.05-3912.68 | 3425.15 |
| TRTPN*ATPT | 0 EyxO V | 2 | Plac | 3 | -45.7422 | 1866.36407 | -0.02 | 0.9805 | 0.05-3714.66 | 3623.18 |
| TRTPN*ATPT | 0 EyxO | 2 | Plac | 4 | -1438.59 | 1866.36407 | -0.77 | 0.4413 | 0.05-5107.50 | 2230.33 |
| TRTPN*ATPT | 0 EyxO | 3 | Oxy30 | 4 | -220.75 | 1864.91407 | -0.12 | 0.9058 | 0.05-3886.82 | 3445.31 |
| TRTPN*ATPT | NOxy30 | 3 | Oxy60 | 0 | | 1939.53407 | -0.30 | 0.7628 | 0.05-4398.63 | 3226.87 |
| TRTPN*ATPT | 0 EyxO | 3 | Oxy60 | 0.5 | 1783.96 | 1939.53407 | 0.92 | 0.3582 | 0.05-2028.78 | 5596.71 |

Program: A Bio3.sas Created: 02APR2020 7:35 POSTLOCK 

Appendix 16.1.9.2.3
Statistical Methods and Analysis Output Supporting Table 14.2.4
Supporting Table 14.2.4

#### The Mixed Procedure

#### Parameter Code=MVMIPM

#### Differences of Least Squares Means

| | | | בב | TCTCTCCO | or nease i | oquares means | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | Planned | Analysis | | Analysis | | | | | | | |
| | Treatment | Timepoint | Treatment | Timepoint | | Standard | | | | | |
| Effect | (N) | (N) | (N) | (N) | Estimate | Error DF t | | r > t 1 | Alpha | Lower | Upper |
| TRTPN*ATPTN | IOxy30 | 3 | Oxy60 | 1 | 4079.83 | 1901.48407 | 2.15 | 0.0325 | 0.05 | 341.89 | 7817.77 |
| TRTPN*ATPTN | 10xy30 | 3 | Oxy60 | 2 | 5302.06 | 1866.32407 | 2.84 | 0.0047 | 0.05 | 1633.23 | 8970.89 |
| TRTPN*ATPTN | 10xy30 | 3 | Oxy60 | 3 | 4752.59 | 1866.32407 | 2.55 | 0.0112 | 0.05 | 1083.75 | 8421.42 |
| TRTPN*ATPTN | 10xy30 | 3 | Oxy60 | 4 | 4632.45 | 1866.32407 | 2.48 | 0.0135 | 0.05 | 963.62 | 8301.28 |
| TRTPN*ATPTN | 10xy30 | 3 | Plac | 0 | 15.2591 | 1866.36407 | 0.01 | 0.9935 | 0.05- | -3653.66 | 3684.18 |
| TRTPN*ATPTN | 10xy30 | 3 | Plac | 0.5 | -1565.13 | 1866.36407 | -0.84 | 0.4022 | 0.05- | -5234.05 | 2103.79 |
| TRTPN*ATPTN | 10xy30 | 3 | Plac | 1 | -2454.39 | 1866.36407 | -1.32 | 0.1892 | 0.05- | -6123.31 | 1214.53 |
| TRTPN*ATPTN | 10xy30 | 3 | Plac | 2 | 1351.07 | 1866.36407 | 0.72 | 0.4695 | 0.05- | -2317.84 | 5019.99 |
| TRTPN*ATPTN | 10xy30 | 3 | Plac | 3 | 1549.10 | 1866.36407 | 0.83 | 0.4070 | 0.05- | -2119.82 | 5218.01 |
| TRTPN*ATPTN | 10xy30 | 3 | Plac | 4 | 156.25 | 1866.36407 | 0.08 | 0.9333 | 0.05- | -3512.67 | 3825.17 |
| TRTPN*ATPTN | 10xy30 | 4 | Oxy60 | 0 | -365.13 | 1939.53407 | -0.19 | 0.8508 | 0.05- | 4177.87 | 3447.62 |
| TRTPN*ATPTN | 10xy30 | 4 | Oxy60 | 0.5 | 2004.72 | 1939.53407 | 1.03 | 0.3019 | 0.05- | -1808.03 | 5817.46 |
| TRTPN*ATPTN | 10xy30 | 4 | Oxy60 | 1 | 4300.58 | 1901.48407 | 2.26 | 0.0242 | 0.05 | 562.64 | 8038.52 |
| TRTPN*ATPTN | 10xy30 | 4 | Oxy60 | 2 | 5522.81 | 1866.32407 | 2.96 | 0.0033 | 0.05 | 1853.98 | 9191.64 |
| TRTPN*ATPTN | 10xy30 | 4 | Oxy60 | 3 | 4973.34 | 1866.32407 | 2.66 | 0.0080 | 0.05 | 1304.50 | 8642.17 |
| TRTPN*ATPTN | 10xy30 | 4 | Oxy60 | 4 | 4853.20 | 1866.32407 | 2.60 | 0.0097 | 0.05 | 1184.37 | 8522.04 |
| TRTPN*ATPTN | 10xy30 | 4 | Plac | 0 | 236.01 | 1866.36407 | 0.13 | 0.8994 | 0.05- | -3432.91 | 3904.93 |
| TRTPN*ATPTN | Oxy30 | 4 | Plac | 0.5 | -1344.38 | 1866.36407 | -0.72 | 0.4717 | 0.05- | -5013.29 | 2324.54 |
| TRTPN*ATPTN | 10xy30 | 4 | Plac | 1 | -2233.63 | 1866.36407 | -1.20 | 0.2321 | 0.05- | -5902.55 | 1435.28 |
| TRTPN*ATPTN | 10xy30 | 4 | Plac | 2 | 1571.83 | 1866.36407 | 0.84 | 0.4002 | 0.05- | -2097.09 | 5240.75 |
| TRTPN*ATPTN | Oxy30 | 4 | Plac | 3 | 1769.85 | 1866.36407 | 0.95 | 0.3435 | 0.05- | -1899.07 | 5438.77 |
| TRTPN*ATPTN | 10xy30 | 4 | Plac | 4 | 377.01 | 1866.36407 | 0.20 | 0.8400 | 0.05- | -3291.91 | 4045.92 |
| TRTPN*ATPTN | Oxy60 | 0 | Oxy60 | 0.5 | 2369.84 | 2003.24407 | 1.18 | 0.2375 | 0.05- | -1568.14 | 6307.83 |
| TRTPN*ATPTN | IOxy60 | 0 | Oxy60 | 1 | 4665.71 | 1971.54407 | 2.37 | 0.0184 | 0.05 | 790.04 | 8541.38 |
| TRTPN*ATPTN | 10xy60 | 0 | Oxy60 | 2 | 5887.94 | 1937.96407 | 3.04 | 0.0025 | 0.05 | 2078.28 | 9697.60 |

Program: A Bio3.sas Created: 02APR2020 7:35 POSTLOCK 

Appendix 16.1.9.2.3
Statistical Methods and Analysis Output Supporting Table 14.2.4
Supporting Table 14.2.4

#### The Mixed Procedure

#### Parameter Code=MVMIPM

#### Differences of Least Squares Means

| | Planned | Analysis | | Analysis | or bease . | squares means | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | Treatment | - | | t Timepoint | : | Standard | | | | | |
| Effect | (N) | (N) | (N) | (N) | Estimate | Error DFt | Value P | r > t | Alpha | Lower | Upper |
| TRTPN*ATPTI | N 0xy60 | 0 | Oxy60 | 3 | 5338.46 | 1937.96407 | 2.75 | 0.0061 | 0.05 1 | 1528.80 | 9148.12 |
| TRTPN*ATPT | NOxy60 | 0 | Oxy60 | 4 | 5218.33 | 1937.96407 | 2.69 | 0.0074 | 0.05 1 | 408.67 | 9027.99 |
| TRTPN*ATPT | NOxy60 | 0 | Plac | 0 | 601.14 | 1939.56407 | 0.31 | 0.7568 | 0.05-3 | 3211.67 | 4413.95 |
| TRTPN*ATPT | NOxy60 | 0 | Plac | 0.5 | -979.25 | 1939.56407 | -0.50 | 0.6139 | 0.05-4 | 1792.06 | 2833.56 |
| TRTPN*ATPT | NOxy60 | 0 | Plac | 1 | -1868.51 | 1939.56407 | -0.96 | 0.3359 | 0.05-5 | 5681.32 | 1944.30 |
| TRTPN*ATPT | NOxy60 | 0 | Plac | 2 | 1936.95 | 1939.56407 | 1.00 | 0.3186 | 0.05-1 | 1875.86 | 5749.76 |
| TRTPN*ATPT | NOxy60 | 0 | Plac | 3 | 2134.98 | 1939.56407 | 1.10 | 0.2717 | 0.05-1 | 677.84 | 5947.79 |
| TRTPN*ATPT | NOxy60 | 0 | Plac | 4 | 742.13 | 1939.56407 | 0.38 | 0.7022 | 0.05-3 | 3070.68 | 4554.94 |
| TRTPN*ATPT | NOxy60 | 0.5 | Oxy60 | 1 | 2295.86 | 1971.54407 | 1.16 | 0.2449 | 0.05-1 | 1579.81 | 6171.53 |
| TRTPN*ATPT | NOxy60 | 0.5 | Oxy60 | 2 | 3518.09 | 1937.96407 | 1.82 | 0.0702 | 0.05 - | -291.57 | 7327.75 |
| TRTPN*ATPT | NOxy60 | 0.5 | Oxy60 | 3 | 2968.62 | 1937.96407 | 1.53 | 0.1263 | 0.05 - | -841.04 | 6778.28 |
| TRTPN*ATPT | NOxy60 | 0.5 | Oxy60 | 4 | 2848.49 | 1937.96407 | 1.47 | 0.1424 | 0.05 - | -961.17 | 6658.15 |
| TRTPN*ATPT | NOxy60 | 0.5 | Plac | 0 | -1768.71 | 1939.56407 | -0.91 | 0.3624 | 0.05-5 | 5581.52 | 2044.11 |
| TRTPN*ATPT | NOxy60 | 0.5 | Plac | 0.5 | -3349.09 | 1939.56407 | -1.73 | 0.0850 | 0.05-7 | 7161.90 | 463.72 |
| TRTPN*ATPT | NOxy60 | 0.5 | Plac | 1 | -4238.35 | 1939.56407 | -2.19 | 0.0294 | 0.05-8 | 3051.16 | -425.54 |
| TRTPN*ATPT | NOxy60 | 0.5 | Plac | 2 | -432.89 | 1939.56407 | -0.22 | 0.8235 | 0.05-4 | 1245.70 | 3379.92 |
| TRTPN*ATPT | NOxy60 | 0.5 | Plac | 3 | -234.87 | 1939.56407 | -0.12 | 0.9037 | 0.05-4 | 1047.68 | 3577.94 |
| TRTPN*ATPT | NOxy60 | 0.5 | Plac | 4 | -1627.71 | 1939.56407 | -0.84 | 0.4018 | 0.05-5 | 5440.52 | 2185.10 |
| TRTPN*ATPT | NOxy60 | 1 | Oxy60 | 2 | 1222.23 | 1899.22407 | 0.64 | 0.5202 | 0.05-2 | 2511.28 | 4955.74 |
| TRTPN*ATPT | NOxy60 | 1 | Oxy60 | 3 | 672.76 | 1899.22407 | 0.35 | 0.7234 | 0.05-3 | 3060.75 | 4406.26 |
| TRTPN*ATPT | NOxy60 | 1 | Oxy60 | 4 | 552.62 | 1899.22407 | 0.29 | 0.7712 | 0.05 -3 | 3180.88 | 4286.13 |
| TRTPN*ATPT | NOxy60 | 1 | Plac | 0 | -4064.57 | 1900.77407 | -2.14 | 0.0331 | 0.05-7 | 7801.13 | -328.01 |
| TRTPN*ATPT | NOxy60 | 1 | Plac | 0.5 | -5644.96 | 1900.77407 | -2.97 | 0.0032 | 0.05-9 | 3381.52 - | -1908.39 |
| TRTPN*ATPT | NOxy60 | 1 | Plac | 1 | -6534.22 | 1900.77407 | -3.44 | 0.0006 | 0.05 | -10271 - | -2797.65 |
| TRTPN*ATPT | NOxy60 | 1 | Plac | 2 | -2728.75 | 1900.77407 | -1.44 | 0.1519 | 0.05-6 | 3465.31 | 1007.81 |

Program: A Bio3.sas Created: 02APR2020 7:35 POSTLOCK 

## Appendix 16.1.9.2.3 Statistical Methods and Analysis Output Supporting Table 14.2.4 Supporting Table 14.2.4

#### The Mixed Procedure

#### Parameter Code=MVMIPM

#### Differences of Least Squares Means

| | D]1 | 71 | | | or bease i | oquares neans | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | Planned | Analysis | | Analysis<br>Timepoint | | Standard | | | | | |
| Effect | (N) | (N) | (N) | (N) | Estimate | Error DF t | 1/2 ] 110 D1 | · > + | Alnha | Lower | Upper |
| TRTPN*ATPT | . , | 1 | Plac | 3 | | 1900.77407 | -1.33 | | | | 1205.83 |
| TRTPN*ATPT | 4 | 1 | Plac | 4 | | 1900.77407 | -2.06 | | | | -187.01 |
| TRTPN*ATPT | 4 | 2 | | 3 | | 1864.91407 | -0.29 | | | | 3116.59 |
| TRTPN*ATPTI | 4 | 2 | 0xy60<br>0xy60 | 4 | | 1864.91407 | -0.29 | | | | 2996.46 |
| | 4 | | 4 | | | | | | | | |
| TRTPN*ATPT | 4 | 2 | Plac | 0 | | 1866.36407 | -2.83 | | | | -1617.88 |
| TRTPN*ATPT | 4 | 2 | Plac | 0.5 | | 1866.36407 | -3.68 | 0.0003 | | | -3198.27 |
| TRTPN*ATPTI | 10xy60 | 2 | Plac | 1 | -7756.45 | 1866.36407 | -4.16 | <.0001 | 0.05 | -11425 | -4087.53 |
| TRTPN*ATPTI | 10xy60 | 2 | Plac | 2 | -3950.98 | 1866.36407 | -2.12 | 0.0349 | 0.05 - | -7619.90 | -282.07 |
| TRTPN*ATPT | 10xy60 | 2 | Plac | 3 | -3752.96 | 1866.36407 | -2.01 | 0.0450 | 0.05- | -7421.88 | -84.0457 |
| TRTPN*ATPTI | 10xy60 | 2 | Plac | 4 | -5145.81 | 1866.36407 | -2.76 | 0.0061 | 0.05- | -8814.72 | -1476.89 |
| TRTPN*ATPT1 | 10xy60 | 3 | Oxy60 | 4 | -120.13 | 1864.91407 | -0.06 | 0.9487 | 0.05- | -3786.20 | 3545.93 |
| TRTPN*ATPT | N 0xy60 | 3 | Plac | 0 | -4737.33 | 1866.36407 | -2.54 | 0.0115 | 0.05- | -8406.24 | -1068.41 |
| TRTPN*ATPT1 | 10xy60 | 3 | Plac | 0.5 | -6317.71 | 1866.36407 | -3.39 | 0.0008 | 0.05- | -9986.63 | -2648.80 |
| TRTPN*ATPT1 | 10xy60 | 3 | Plac | 1 | -7206.97 | 1866.36407 | -3.86 | 0.0001 | 0.05 | -10876 | -3538.06 |
| TRTPN*ATPT1 | 10xy60 | 3 | Plac | 2 | -3401.51 | 1866.36407 | -1.82 | 0.0691 | 0.05- | -7070.43 | 267.41 |
| TRTPN*ATPT | NOxy60 | 3 | Plac | 3 | -3203.49 | 1866.36407 | -1.72 | 0.0868 | 0.05- | -6872.41 | 465.43 |
| TRTPN*ATPT | NOxy60 | 3 | Plac | 4 | -4596.33 | 1866.36407 | -2.46 | 0.0142 | 0.05- | -8265.25 | -927.42 |
| TRTPN*ATPT | NOxy60 | 4 | Plac | 0 | -4617.19 | 1866.36407 | -2.47 | 0.0138 | 0.05- | -8286.11 | -948.27 |
| TRTPN*ATPT | 10xy60 | 4 | Plac | 0.5 | -6197.58 | 1866.36407 | -3.32 | 0.0010 | 0.05- | -9866.50 | -2528.66 |
| TRTPN*ATPT | NOxy60 | 4 | Plac | 1 | -7086.84 | 1866.36407 | -3.80 | 0.0002 | 0.05 | -10756 | -3417.92 |
| TRTPN*ATPT | NOxy60 | 4 | Plac | 2 | -3281.38 | 1866.36407 | -1.76 | 0.0795 | 0.05- | -6950.29 | 387.54 |
| TRTPN*ATPT | 10xy60 | 4 | Plac | 3 | -3083.35 | 1866.36407 | -1.65 | 0.0993 | 0.05- | -6752.27 | 585.56 |
| TRTPN*ATPTI | -<br>NOxy60 | 4 | Plac | 4 | -4476.20 | 1866.36407 | -2.40 | 0.0169 | 0.05- | -8145.12 | -807.28 |
| TRTPN*ATPT | N Plac | 0 | Plac | 0.5 | -1580.39 | 1864.91407 | -0.85 | 0.3973 | 0.05- | -5246.45 | 2085.68 |
| TRTPN*ATPTI | N Plac | 0 | Plac | 1 | -2469.65 | 1864.91407 | -1.32 | 0.1862 | 0.05- | -6135.71 | 1196.42 |

Program: A Bio3.sas Created: 02APR2020 7:35 POSTLOCK


### Appendix 16.1.9.2.3 Statistical Methods and Analysis Output Supporting Table 14.2.4 Supporting Table 14.2.4

#### The Mixed Procedure

#### Parameter Code=MVMIPM

#### Differences of Least Squares Means

| | | | | | | 1 | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | Planned | Analysis | Planned | Analysis | | | | | | | |
| | Treatment | Timepoint | Treatment | Timepoint | : | Standard | | | | | |
| Effect | (N) | (N) | (N) | (N) | Estimate | Error DFt | Value Pr | > t . | Alpha | Lower | Upper |
| TRTPN*ATPTN | Plac | 0 | Plac | 2 | 1335.82 | 1864.91407 | 0.72 | 0.4742 | 0.05 - | 2330.25 | 5001.88 |
| TRTPN*ATPTN | Plac | 0 | Plac | 3 | 1533.84 | 1864.91407 | 0.82 | 0.4113 | 0.05 - | 2132.23 | 5199.90 |
| TRTPN*ATPTN | Plac | 0 | Plac | 4 | 140.99 | 1864.91407 | 0.08 | 0.9398 | 0.05 - | 3525.07 | 3807.06 |
| TRTPN*ATPTN | Plac | 0.5 | Plac | 1 | -889.26 | 1864.91407 | -0.48 | 0.6337 | 0.05 - | 4555.32 | 2776.81 |
| TRTPN*ATPTN | Plac | 0.5 | Plac | 2 | 2916.20 | 1864.91407 | 1.56 | 0.1187 | 0.05 | -749.86 | 6582.27 |
| TRTPN*ATPTN | Plac | 0.5 | Plac | 3 | 3114.22 | 1864.91407 | 1.67 | 0.0957 | 0.05 | -551.84 | 6780.29 |
| TRTPN*ATPTN | Plac | 0.5 | Plac | 4 | 1721.38 | 1864.91407 | 0.92 | 0.3565 | 0.05 - | 1944.68 | 5387.45 |
| TRTPN*ATPTN | Plac | 1 | Plac | 2 | 3805.46 | 1864.91407 | 2.04 | 0.0419 | 0.05 | 139.40 | 7471.53 |
| TRTPN*ATPTN | Plac | 1 | Plac | 3 | 4003.48 | 1864.91407 | 2.15 | 0.0324 | 0.05 | 337.42 | 7669.55 |
| TRTPN*ATPTN | Plac | 1 | Plac | 4 | 2610.64 | 1864.91407 | 1.40 | 0.1623 | 0.05 - | 1055.43 | 6276.71 |
| TRTPN*ATPTN | Plac | 2 | Plac | 3 | 198.02 | 1864.91407 | 0.11 | 0.9155 | 0.05 - | 3468.04 | 3864.09 |
| TRTPN*ATPTN | Plac | 2 | Plac | 4 | -1194.82 | 1864.91407 | -0.64 | 0.5221 | 0.05 - | 4860.89 | 2471.24 |
| TRTPN*ATPTN | Plac | 3 | Plac | 4 | -1392.84 | 1864.91407 | -0.75 | 0.4556 | 0.05 - | 5058.91 | 2273.22 |

### Tests of Effect Slices Analysis

Timepoint Num Den

| Effect | (N) | DF | DF F | Value E | r > | F |
|-----------|--------|-----|------|---------|-------|----|
| TRTPN*ATP | rn 0 | 5 - | 407 | 0.540 | .748 | 30 |
| TRTPN*ATP | rn 0.5 | 5 - | 407 | 2.800 | 0.016 | 58 |
| TRTPN*ATP | rn 1 | 5 - | 407 | 3.650 | 0.003 | 31 |
| TRTPN*ATP | rn 2 | 5 - | 407 | 2.870 | 0.014 | 17 |
| TRTPN*ATP | rn 3 | 5 - | 407 | 1.640 | ).147 | 71 |
| TRTPN*ATP | rn 4 | 5 - | 407 | 1.770 | .117 | 73 |

Program: A\_Bio3.sas Created: 02APR2020 7:35 POSTLOCK

Appendix 16.1.9.2.3
Statistical Methods and Analysis Output Supporting Table 14.2.4
Supporting Table 14.2.4

The Mixed Procedure

Parameter Code=MVMIPM

Program: A\_Bio3.sas Created: 02APR2020 7:35 POSTLOCK 

### Appendix 16.1.9.2.4 Statistical Methods and Analysis Output Supporting Table 14.2.5 Supporting Table 14.2.4

#### The Mixed Procedure

#### Parameter Code=MVMIPM

#### Model Information

| Data Set | WORK.ADXV |
|---------------------------|-------------------|
| Dependent Variable | AVAL |
| Covariance Structure | Compound Symmetry |
| Subject Effect | SUBJID |
| Estimation Method | REML |
| Residual Variance Method | Profile |
| Fixed Effects SE Method | Model-Based |
| Degrees of Freedom Method | Between-Within |

#### Class Level Information

| Class | LevelsValues |
|---|---|
| SUBJID | 161001 1002 1003 1004 1005 1006 1007 1008 1010 1012 1013 1014 1015 1016 1017 1018 |
| TRTPN | 6Bel300 Bel600 Bel900 Oxy30 Oxy60 Plac |
| APERIOD | 6 P1 P2 P3 P4 P5 P6 |
| ARMCD | 6ABCEDF BEAFCD CADBFE DCFAEB EFBDAC FDECBA |
| ATPTN | 60 0.5 1 2 3 4 |

| Dimensi | ons |
|------------------|----------|
| Covariance Param | neters 2 |
| Columns in X | 55 |
| Columns in Z | 0 |
| Subjects | 16 |
| Max Obs per Sub- | ject 36 |

Program: A Bio4.sas Created: 02APR2020 7:36 POSTLOCK 

#### Appendix 16.1.9.2.4 Statistical Methods and Analysis Output Supporting Table 14.2.5 Supporting Table 14.2.4

The Mixed Procedure

#### Parameter Code=MVMIPM

| | Nι | umber of Obse | rvations | |
|--------|----|---------------|----------|-----|
| Number | of | Observations | Read | 545 |
| Number | of | Observations | Used | 545 |
| Number | of | Observations | Not Used | 0 |

#### Iteration History

| Iteration Evaluatio | ons | -2 Res Log Like Criterion |
|---------------------|-----|---------------------------|
| 0 | 1 | 10201.54397027 |
| 1 | 2 | 10095.465159980.00000006 |
| 2 | 1 | 10095.464884110.00000000 |

Convergence criteria met.

Covariance Parameter
Estimates

Cov Parm Subject Estimate
CS SUBJID 11371173
Residual 25636473

# Fit Statistics -2 Res Log Likelihood 10095.5 AIC (Smaller is Better) 10099.5 AICC (Smaller is Better) 10099.5 BIC (Smaller is Better) 10101.0

Program: A Bio4.sas Created: 02APR2020 7:36 POSTLOCK 

### Appendix 16.1.9.2.4 Statistical Methods and Analysis Output Supporting Table 14.2.5 Supporting Table 14.2.4

The Mixed Procedure

Parameter Code=MVMIPM

Null Model Likelihood Ratio Test

DF Chi-Square Pr > ChiSq 1 106.08 <.0001

Type 3 Tests of Fixed Effects

| | n uiii i | Jen | |
|-------------|----------|------|--------------|
| Effect | DF | DF F | Value Pr > F |
| TRTPN | 5 | 72 | 7.88<.0001 |
| APERIOD | 5 | 72 | 5.820.0001 |
| ARMCD | 5 | 10 | 1.340.3239 |
| TRTPN*ATPTN | 304 | 122 | 2.220.0003 |

#### Least Squares Means

| | Planned | Analysis | | | | | |
|---|---|---|---|---|---|---|---|
| | Treatment | Timepoint | | Standard | | | |
| Effect | (N) | (N) | Estimate | Error DF | t ValueP | r > t | Alpha Lower Upper |
| TRTPN*ATPTN | NBel300 | 0 | 19956 | 1566.43422 | 12.74 | <.0001 | 0.051687723035 |
| TRTPN*ATPTN | NBel300 | 0.5 | 21615 | 1566.43422 | 13.80 | <.0001 | 0.051853624694 |
| TRTPN*ATPTN | NBel300 | 1 | 19703 | 1566.43422 | 12.58 | <.0001 | 0.051662422782 |
| TRTPN*ATPTN | NBel300 | 2 | 19848 | 1566.43422 | 12.67 | <.0001 | 0.051676922927 |
| TRTPN*ATPTN | NBel300 | 3 | 15435 | 1566.43422 | 9.85 | <.0001 | 0.051235618514 |
| TRTPN*ATPTN | NBel300 | 4 | 15990 | 1566.43422 | 10.21 | <.0001 | 0.051291119069 |
| TRTPN*ATPTN | NBe1600 | 0 | 19546 | 1565.91422 | 12.48 | <.0001 | 0.051646822624 |
| TRTPN*ATPTN | NBe1600 | 0.5 | 20533 | 1565.91422 | 13.11 | <.0001 | 0.051745523611 |
| TRTPN*ATPTN | NBel600 | 1 | 19148 | 1530.53422 | 12.51 | <.0001 | 0.051614022156 |
| TRTPN*ATPTN | NBel600 | 2 | 17543 | 1530.53422 | 11.46 | <.0001 | 0.051453420551 |

Program: A\_Bio4.sas Created: 02APR2020 7:36 POSTLOCK


Appendix 16.1.9.2.4
Statistical Methods and Analysis Output Supporting Table 14.2.5
Supporting Table 14.2.4

The Mixed Procedure

Parameter Code=MVMIPM

Least Squares Means

| | | | TCGSC DG | laares means | | | |
|---|---|---|---|---|---|---|---|
| | Planned | Analysis | | | | | |
| | Treatment | Timepoint | : | Standard | | | |
| Effect | (N) | (N) | Estimate | | Value Pr | 2 > t | Alpha Lower Upper |
| TRTPN*ATPTN | Be1600 | 3 | 16703 | 1530.53422 | 10.91 | <.0001 | 0.051369519712 |
| TRTPN*ATPTN | Bel600 | 4 | | 1530.53422 | 11.03 | <.0001 | 0.051387819895 |
| TRTPN*ATPTN | Be1900 | 0 | 21316 | 1605.83422 | 13.27 | <.0001 | 0.051816024473 |
| TRTPN*ATPTN | Bel900 | 0.5 | 22751 | 1566.65422 | 14.52 | <.0001 | 0.051967225831 |
| TRTPN*ATPTN | Be1900 | 1 | 19932 | 1566.65422 | 12.72 | <.0001 | 0.051685223011 |
| TRTPN*ATPTN | Be1900 | 2 | 18174 | 1566.65422 | 11.60 | <.0001 | 0.051509421253 |
| TRTPN*ATPTN | Be1900 | 3 | 17494 | 1566.65422 | 11.17 | <.0001 | 0.051441420573 |
| TRTPN*ATPTN | Be1900 | 4 | 16445 | 1566.65422 | 10.50 | <.0001 | 0.051336619525 |
| TRTPN*ATPTN | Oxy30 | 0 | 20087 | 1651.59422 | 12.16 | <.0001 | 0.051684123334 |
| TRTPN*ATPTN | Oxy30 | 0.5 | 17815 | 1651.59422 | 10.79 | <.0001 | 0.051456921061 |
| TRTPN*ATPTN | Oxy30 | 1 | 15960 | 1606.15422 | 9.94 | <.0001 | 0.051280319117 |
| TRTPN*ATPTN | Oxy30 | 2 | 16815 | 1566.67422 | 10.73 | <.0001 | 0.051373619895 |
| TRTPN*ATPTN | Oxy30 | 3 | 18410 | 1566.67422 | 11.75 | <.0001 | 0.051533121490 |
| TRTPN*ATPTN | Oxy30 | 4 | 18631 | 1566.67422 | 11.89 | <.0001 | 0.051555221711 |
| TRTPN*ATPTN | Oxy60 | 0 | 18627 | 1607.20422 | 11.59 | <.0001 | 0.051546821786 |
| TRTPN*ATPTN | Oxy60 | 0.5 | 16395 | 1607.20422 | 10.20 | <.0001 | 0.051323619554 |
| TRTPN*ATPTN | Oxy60 | 1 | 14303 | 1567.67422 | 9.12 | <.0001 | 0.051122217385 |
| TRTPN*ATPTN | Oxy60 | 2 | 13311 | 1530.56422 | 8.70 | <.0001 | 0.051030216319 |
| TRTPN*ATPTN | Oxy60 | 3 | 13978 | 1530.56422 | 9.13 | <.0001 | 0.051096916986 |
| TRTPN*ATPTN | Oxy60 | 4 | 14097 | 1530.56422 | 9.21 | <.0001 | 0.051108817105 |
| TRTPN*ATPTN | Plac | 0 | 18495 | 1530.50422 | 12.08 | <.0001 | 0.051548721503 |
| TRTPN*ATPTN | Plac | 0.5 | 20021 | 1530.50422 | 13.08 | <.0001 | 0.051701223029 |
| TRTPN*ATPTN | Plac | 1 | 20972 | 1530.50422 | 13.70 | <.0001 | 0.051796423981 |
| TRTPN*ATPTN | Plac | 2 | 16906 | 1530.50422 | 11.05 | <.0001 | 0.051389719914 |

Program: A\_Bio4.sas Created: 02APR2020 7:36 POSTLOCK 

Appendix 16.1.9.2.4

Statistical Methods and Analysis Output Supporting Table 14.2.5

Supporting Table 14.2.4

The Mixed Procedure

Parameter Code=MVMIPM

Least Squares Means

Differences of Least Squares Means

Analysis Planned Analysis

Treatment Timepoint Treatment Timepoint Standard Effect (N) (N) (N) (N) Estimate Error DFt Value Pr > |t|Alpha Lower Upper TRTPN\*ATPTN Bel300 Be1300 0.5 -1659.32 1848.84422 -0.90 0.3700 0.05-5293.40 1974.75 TRTPN\*ATPTN Bel300 0 Be1300 252.85 1848.84422 0.14 0.8913 0.05 - 3381.22 3886.93 TRTPN\*ATPTN Bel300 Be1300 108.37 1848.84422 0.06 0.9533 0.05 - 3525.71 3742.44 TRTPN\*ATPTN Bel300 Be1300 4521.35 1848.84422 0.0149 0.05 887.28 8155.43 0 2.45 TRTPN\*ATPTN Bel300 Be1300 3966.17 1848.84422 2.15 0.0325 0.05 332.10 7600.25 TRTPN\*ATPTN Bel300 Be1600 410.18 1852.53422 0.22 0.8249 0.05 - 3231.15 4051.51 -576.54 1852.53422 -0.31 0.7558 0.05-4217.87 3064.79 TRTPN\*ATPTN Bel300 0 Be1600 0.5 0.6578 0.05 - 2774.72 4390.90 TRTPN\*ATPTN Bel300 0 Be1600 808.09 1822.76422 0.44 TRTPN\*ATPTN Bel300 Be1600 2413.31 1822.76422 1.32 0.1862 0.05 - 1169.50 5996.12 TRTPN\*ATPTN Bel300 0 Be1600 3252.96 1822.76422 1.78 0.0750 0.05 -329.85 6835.77 TRTPN\*ATPTN Bel300 0 Be1600 3069.51 1822.76422 1.68 0.0929 0.05 -513.30 6652.32 TRTPN\*ATPTN Bel300 0 Be1900 -1360.31 1883.44422 -0.72 0.4705 0.05 - 5062.40 2341.78 TRTPN\*ATPTN Bel300 Be1900 -2794.98 1850.18422 -1.510.1316 0.05-6431.69 24.4926 1850.18422 TRTPN\*ATPTN Bel300 0 Be1900 0.01 0.9894 0.05 - 3612.22 3661.20 TRTPN\*ATPTN Bel300 0 Bel900 1782.25 1850.18422 0.96 0.3360 0.05-1854.46 5418.96 TRTPN\*ATPTN Bel300 0.1839 0.05-1174.20 6099.22 Be1900 2462.51 1850.18422 1.33 TRTPN\*ATPTN Bel300 Bel900 3511.00 1850.18422 1.90 0.0584 0.05 -125.71 7147.71

Program: A\_Bio4.sas Created: 02APR2020 7:36 POSTLOCK
Appendix 16.1.9.2.4
Statistical Methods and Analysis Output Supporting Table 14.2.5
Supporting Table 14.2.4

# The Mixed Procedure

#### Parameter Code=MVMIPM

# Differences of Least Squares Means

| | Planned | Analysis | | Analvsis | or bease . | oquares means | | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| | Treatment | 4 | | :Timepoint | | Standard | | | | |
| Effect | (N) | (N) | (N) | (N) | Estimate | Error DFt | Value P | r > t . | Alpha Lower | Upper |
| TRTPN*ATPT | NBel300 | 0 | Oxy30 | 0 | -131.08 | 1922.13422 | -0.07 | 0.9457 | 0.05-3909.22 | 3647.07 |
| TRTPN*ATPT | NBel300 | 0 | Oxy30 | 0.5 | 2141.07 | 1922.13422 | 1.11 | 0.2660 | 0.05-1637.08 | 5919.22 |
| TRTPN*ATPT | NBel300 | 0 | Oxy30 | 1 | 3995.79 | 1883.53422 | 2.12 | 0.0345 | 0.05 293.52 | 7698.06 |
| TRTPN*ATPT | NBel300 | 0 | Oxy30 | 2 | 3140.64 | 1850.26422 | 1.70 | 0.0904 | 0.05 -496.23 | 6777.51 |
| TRTPN*ATPT | NBel300 | 0 | Oxy30 | 3 | 1545.80 | 1850.26422 | 0.84 | 0.4039 | 0.05-2091.07 | 5182.67 |
| TRTPN*ATPT | NBel300 | 0 | Oxy30 | 4 | 1325.05 | 1850.26422 | 0.72 | 0.4743 | 0.05-2311.82 | 4961.92 |
| TRTPN*ATPT | NBe1300 | 0 | Oxy60 | 0 | 1329.04 | 1886.80422 | 0.70 | 0.4816 | 0.05-2379.67 | 5037.74 |
| TRTPN*ATPT | NBe1300 | 0 | Oxy60 | 0.5 | 3561.27 | 1886.80422 | 1.89 | 0.0598 | 0.05 -147.43 | 7269.97 |
| TRTPN*ATPT | NBe1300 | 0 | Oxy60 | 1 | 5652.80 | 1852.83422 | 3.05 | 0.0024 | 0.05 2010.86 | 9294.73 |
| TRTPN*ATPT | NBe1300 | 0 | Oxy60 | 2 | 6645.35 | 1822.14422 | 3.65 | 0.0003 | 0.05 3063.75 | 10227 |
| TRTPN*ATPT | NBe1300 | 0 | Oxy60 | 3 | 5978.53 | 1822.14422 | 3.28 | 0.0011 | 0.05 2396.93 | 9560.13 |
| TRTPN*ATPT | NBe1300 | 0 | Oxy60 | 4 | 5859.39 | 1822.14422 | 3.22 | 0.0014 | 0.05 2277.79 | 9440.99 |
| TRTPN*ATPT | NBe1300 | 0 | Plac | 0 | 1461.12 | 1821.91422 | 0.80 | 0.4230 | 0.05-2120.03 | 5042.26 |
| TRTPN*ATPT | NBe1300 | 0 | Plac | 0.5 | -64.5111 | 1821.91422 | -0.04 | 0.9718 | 0.05-3645.65 | 3516.63 |
| TRTPN*ATPT | NBe1300 | 0 | Plac | 1 | -1016.01 | 1821.91422 | -0.56 | 0.5774 | 0.05-4597.16 | 2565.13 |
| TRTPN*ATPT | NBe1300 | 0 | Plac | 2 | 3050.29 | 1821.91422 | 1.67 | 0.0948 | 0.05 -530.86 | 6631.43 |
| TRTPN*ATPT | NBe1300 | 0 | Plac | 3 | 2636.22 | 1821.91422 | 1.45 | 0.1487 | 0.05 -944.92 | 6217.36 |
| TRTPN*ATPT | NBe1300 | 0 | Plac | 4 | 1456.98 | 1821.91422 | 0.80 | 0.4243 | 0.05-2124.16 | 5038.13 |
| TRTPN*ATPT | NBe1300 | 0.5 | Be1300 | 1 | 1912.18 | 1848.84422 | 1.03 | 0.3016 | 0.05-1721.90 | 5546.25 |
| TRTPN*ATPT | NBe1300 | 0.5 | Be1300 | 2 | | 1848.84422 | 0.96 | 0.3396 | 0.05-1866.39 | 5401.76 |
| TRTPN*ATPT | NBe1300 | 0.5 | Be1300 | 3 | 6180.67 | 1848.84422 | 3.34 | 0.0009 | 0.05 2546.60 | 9814.75 |
| TRTPN*ATPTI | NBe1300 | 0.5 | Bel300 | 4 | 5625.50 | 1848.84422 | 3.04 | 0.0025 | 0.05 1991.42 | 9259.57 |
| TRTPN*ATPT | NBe1300 | 0.5 | Be1600 | 0 | | 1852.53422 | 1.12 | 0.2646 | 0.05-1571.83 | 5710.83 |
| TRTPN*ATPT | NBe1300 | 0.5 | Be1600 | 0.5 | 1082.78 | 1852.53422 | 0.58 | 0.5592 | 0.05-2558.55 | 4724.11 |
| TRTPN*ATPT | NBe1300 | 0.5 | Be1600 | 1 | 2467.41 | 1822.76422 | 1.35 | 0.1766 | 0.05-1115.40 | 6050.22 |

Program: A Bio4.sas Created: 02APR2020 7:36 POSTLOCK 

Appendix 16.1.9.2.4
Statistical Methods and Analysis Output Supporting Table 14.2.5
Supporting Table 14.2.4

# The Mixed Procedure

#### Parameter Code=MVMIPM

# Differences of Least Squares Means

| | | | | | or nease . | oquares means | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | Planned | Analysis | | Analysis | | o. 1 1 | | | | | |
| | | - | | Timepoint | | Standard | _ | | | | |
| Effect | (N) | (N) | (N) | (N) | Estimate | Error DF t | | | | Lower | Upper |
| TRTPN*ATPTN | Bel300 | 0.5 | Be1600 | 2 | 4072.63 | 1822.76422 | 2.23 | 0.0260 | 0.05 | 489.82 | 7655.44 |
| TRTPN*ATPTN | Be1300 | 0.5 | Be1600 | 3 | 4912.28 | 1822.76422 | 2.69 | 0.0073 | 0.05 | 1329.47 | 8495.09 |
| TRTPN*ATPTN | Bel300 | 0.5 | Be1600 | 4 | 4728.84 | 1822.76422 | 2.59 | 0.0098 | 0.05 | 1146.03 | 8311.65 |
| TRTPN*ATPTN | Bel300 | 0.5 | Be1900 | 0 | 299.01 | 1883.44422 | 0.16 | 0.8739 | 0.05 | -3403.08 | 4001.10 |
| TRTPN*ATPTN | Bel300 | 0.5 | Be1900 | 0.5 | -1135.66 | 1850.18422 | -0.61 | 0.5397 | 0.05 | -4772.37 | 2501.05 |
| TRTPN*ATPTN | Bel300 | 0.5 | Be1900 | 1 | 1683.81 | 1850.18422 | 0.91 | 0.3633 | 0.05 | -1952.89 | 5320.52 |
| TRTPN*ATPTN | Bel300 | 0.5 | Be1900 | 2 | 3441.57 | 1850.18422 | 1.86 | 0.0636 | 0.05 | -195.14 | 7078.28 |
| TRTPN*ATPTN | Bel300 | 0.5 | Be1900 | 3 | 4121.83 | 1850.18422 | 2.23 | 0.0264 | 0.05 | 485.12 | 7758.54 |
| TRTPN*ATPTN | Bel300 | 0.5 | Be1900 | 4 | 5170.32 | 1850.18422 | 2.79 | 0.0054 | 0.05 | 1533.61 | 8807.03 |
| TRTPN*ATPTN | Bel300 | 0.5 | 0xy30 | 0 | 1528.24 | 1922.13422 | 0.80 | 0.4270 | 0.05 | -2249.90 | 5306.39 |
| TRTPN*ATPTN | Bel300 | 0.5 | 0xy30 | 0.5 | 3800.39 | 1922.13422 | 1.98 | 0.0487 | 0.05 | 22.2455 | 7578.54 |
| TRTPN*ATPTN | Bel300 | 0.5 | 0xy30 | 1 | 5655.11 | 1883.53422 | 3.00 | 0.0028 | 0.05 | 1952.84 | 9357.38 |
| TRTPN*ATPTN | Bel300 | 0.5 | 0xy30 | 2 | 4799.96 | 1850.26422 | 2.59 | 0.0098 | 0.05 | 1163.09 | 8436.83 |
| TRTPN*ATPTN | Bel300 | 0.5 | 0xy30 | 3 | 3205.12 | 1850.26422 | 1.73 | 0.0840 | 0.05 | -431.74 | 6841.99 |
| TRTPN*ATPTN | Bel300 | 0.5 | 0xy30 | 4 | 2984.37 | 1850.26422 | 1.61 | 0.1075 | 0.05 | -652.50 | 6621.24 |
| TRTPN*ATPTN | Bel300 | 0.5 | Oxy60 | 0 | 2988.36 | 1886.80422 | 1.58 | 0.1140 | 0.05 | -720.34 | 6697.06 |
| TRTPN*ATPTN | Bel300 | 0.5 | Oxy60 | 0.5 | 5220.59 | 1886.80422 | 2.77 | 0.0059 | 0.05 | 1511.89 | 8929.29 |
| TRTPN*ATPTN | Bel300 | 0.5 | Oxy60 | 1 | 7312.12 | 1852.83422 | 3.95 | <.0001 | 0.05 | 3670.18 | 10954 |
| TRTPN*ATPTN | Bel300 | 0.5 | Oxy60 | 2 | 8304.67 | 1822.14422 | 4.56 | <.0001 | 0.05 | 4723.07 | 11886 |
| TRTPN*ATPTN | Bel300 | 0.5 | Oxy60 | 3 | 7637.85 | 1822.14422 | 4.19 | <.0001 | 0.05 | 4056.25 | 11219 |
| TRTPN*ATPTN | Bel300 | 0.5 | Oxy60 | 4 | 7518.71 | 1822.14422 | 4.13 | <.0001 | 0.05 | 3937.11 | 11100 |
| TRTPN*ATPTN | Bel300 | 0.5 | Plac | 0 | 3120.44 | 1821.91422 | 1.71 | 0.0875 | 0.05 | -460.71 | 6701.58 |
| TRTPN*ATPTN | Be1300 | 0.5 | Plac | 0.5 | 1594.81 | 1821.91422 | 0.88 | 0.3819 | 0.05 | -1986.33 | 5175.95 |
| TRTPN*ATPTN | Be1300 | 0.5 | Plac | 1 | 643.31 | 1821.91422 | 0.35 | 0.7242 | 0.05 | -2937.84 | 4224.45 |
| TRTPN*ATPTN | Bel300 | 0.5 | Plac | 2 | 4709.61 | 1821.91422 | 2.58 | 0.0101 | 0.05 | 1128.46 | 8290.75 |

Program: A Bio4.sas Created: 02APR2020 7:36 POSTLOCK 

# Appendix 16.1.9.2.4 Statistical Methods and Analysis Output Supporting Table 14.2.5 Supporting Table 14.2.4

# The Mixed Procedure

#### Parameter Code=MVMIPM

# Differences of Least Squares Means

| | Planned | Analysis | | Analvsis | or heade i | oquares means | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | | 4 | | Timepoint | | Standard | | | | | |
| Effect | (N) | (N) | (N) | (N) | Estimate | Error DFt | Value P | r > t 3 | Alpha | Lower | Upper |
| TRTPN*ATPT | , , | 0.5 | Plac | 3 | | 1821.91422 | 2.36 | 0.0188 | 0.05 | 714.40 | 7876.68 |
| TRTPN*ATPT1 | | 0.5 | Plac | 4 | | 1821.91422 | 1.71 | 0.0879 | | -464.84 | 6697.45 |
| TRTPN*ATPT1 | | 1 | Be1300 | 2 | | 1848.84422 | -0.08 | | | 3778.57 | 3489.59 |
| TRTPN*ATPTI | NBel300 | 1 | Be1300 | 3 | 4268.50 | 1848.84422 | 2.31 | 0.0214 | 0.05 | 634.42 | 7902.57 |
| TRTPN*ATPTI | NBel300 | 1 | Be1300 | 4 | 3713.32 | 1848.84422 | 2.01 | 0.0452 | 0.05 | 79.2444 | 7347.40 |
| TRTPN*ATPTI | NBel300 | 1 | Be1600 | 0 | 157.33 | 1852.53422 | 0.08 | 0.9324 | 0.05 - | 3484.00 | 3798.66 |
| TRTPN*ATPT | NBe1300 | 1 | Be1600 | 0.5 | -829.40 | 1852.53422 | -0.45 | 0.6546 | 0.05 - | 4470.73 | 2811.94 |
| TRTPN*ATPT | NBe1300 | 1 | Be1600 | 1 | 555.23 | 1822.76422 | 0.30 | 0.7608 | 0.05 - | 3027.58 | 4138.04 |
| TRTPN*ATPT | NBe1300 | 1 | Be1600 | 2 | 2160.46 | 1822.76422 | 1.19 | 0.2366 | 0.05 - | 1422.35 | 5743.27 |
| TRTPN*ATPT | NBe1300 | 1 | Be1600 | 3 | 3000.10 | 1822.76422 | 1.65 | 0.1005 | 0.05 | -582.71 | 6582.91 |
| TRTPN*ATPT | NBe1300 | 1 | Be1600 | 4 | 2816.66 | 1822.76422 | 1.55 | 0.1230 | 0.05 | -766.15 | 6399.47 |
| TRTPN*ATPT | NBe1300 | 1 | Be1900 | 0 | -1613.16 | 1883.44422 | -0.86 | 0.3922 | 0.05 - | 5315.25 | 2088.92 |
| TRTPN*ATPT | NBel300 | 1 | Be1900 | 0.5 | -3047.84 | 1850.18422 | -1.65 | 0.1002 | 0.05 - | 6684.54 | 588.87 |
| TRTPN*ATPT | NBel300 | 1 | Be1900 | 1 | -228.36 | 1850.18422 | -0.12 | 0.9018 | 0.05 - | 3865.07 | 3408.35 |
| TRTPN*ATPT | NBel300 | 1 | Be1900 | 2 | 1529.39 | 1850.18422 | 0.83 | 0.4089 | 0.05 - | 2107.32 | 5166.10 |
| TRTPN*ATPT | NBel300 | 1 | Be1900 | 3 | 2209.66 | 1850.18422 | 1.19 | 0.2330 | 0.05 - | 1427.05 | 5846.36 |
| TRTPN*ATPT | NBel300 | 1 | Be1900 | 4 | 3258.15 | 1850.18422 | 1.76 | 0.0790 | 0.05 | -378.56 | 6894.85 |
| TRTPN*ATPT | NBel300 | 1 | Oxy30 | 0 | -383.93 | 1922.13422 | -0.20 | 0.8418 | 0.05 - | 4162.08 | 3394.21 |
| TRTPN*ATPT | NBe1300 | 1 | Oxy30 | 0.5 | 1888.22 | 1922.13422 | 0.98 | 0.3265 | 0.05 - | 1889.93 | 5666.36 |
| TRTPN*ATPT | NBe1300 | 1 | Oxy30 | 1 | 3742.94 | 1883.53422 | 1.99 | 0.0475 | 0.05 | 40.6684 | 7445.20 |
| TRTPN*ATPT | NBe1300 | 1 | Oxy30 | 2 | 2887.79 | 1850.26422 | 1.56 | 0.1193 | 0.05 | -749.08 | 6524.65 |
| TRTPN*ATPT | NBe1300 | 1 | 0xy30 | 3 | 1292.95 | 1850.26422 | 0.70 | 0.4851 | 0.05 - | 2343.92 | 4929.82 |
| TRTPN*ATPT | NBe1300 | 1 | 0xy30 | 4 | 1072.20 | 1850.26422 | 0.58 | 0.5626 | 0.05 - | 2564.67 | 4709.06 |
| TRTPN*ATPT | NBe1300 | 1 | Oxy60 | 0 | 1076.18 | 1886.80422 | 0.57 | 0.5687 | 0.05 - | 2632.52 | 4784.88 |
| TRTPN*ATPTI | NBe1300 | 1 | Oxy60 | 0.5 | 3308.42 | 1886.80422 | 1.75 | 0.0803 | 0.05 | -400.29 | 7017.12 |

Program: A Bio4.sas Created: 02APR2020 7:36 POSTLOCK 

# Appendix 16.1.9.2.4 Statistical Methods and Analysis Output Supporting Table 14.2.5 Supporting Table 14.2.4

# The Mixed Procedure

#### Parameter Code=MVMIPM

# Differences of Least Squares Means

| | | | בב | TCTCIICCD V | or nease i | oquares means | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | Planned | Analysis | Planned | Analysis | | | | | | | |
| | Treatment | Timepoint | Treatment | Timepoint | | Standard | | | | | |
| Effect | (N) | (N) | (N) | (N) | Estimate | Error DF t | Value Pi | r > t . | Alpha | Lower | Upper |
| TRTPN*ATPTN | Bel300 | 1 | Oxy60 | 1 | 5399.94 | 1852.83422 | 2.91 | 0.0038 | 0.05 | 1758.01 | 9041.88 |
| TRTPN*ATPTN | Bel300 | 1 | Oxy60 | 2 | 6392.49 | 1822.14422 | 3.51 | 0.0005 | 0.05 | 2810.89 | 9974.09 |
| TRTPN*ATPTN | Bel300 | 1 | Oxy60 | 3 | 5725.68 | 1822.14422 | 3.14 | 0.0018 | 0.05 | 2144.08 | 9307.28 |
| TRTPN*ATPTN | Bel300 | 1 | Oxy60 | 4 | 5606.54 | 1822.14422 | 3.08 | 0.0022 | 0.05 | 2024.94 | 9188.14 |
| TRTPN*ATPTN | Bel300 | 1 | Plac | 0 | 1208.26 | 1821.91422 | 0.66 | 0.5076 | 0.05- | -2372.88 | 4789.40 |
| TRTPN*ATPTN | Bel300 | 1 | Plac | 0.5 | -317.37 | 1821.91422 | -0.17 | 0.8618 | 0.05- | -3898.51 | 3263.78 |
| TRTPN*ATPTN | Bel300 | 1 | Plac | 1 | -1268.87 | 1821.91422 | -0.70 | 0.4865 | 0.05- | -4850.01 | 2312.27 |
| TRTPN*ATPTN | Bel300 | 1 | Plac | 2 | 2797.43 | 1821.91422 | 1.54 | 0.1254 | 0.05 | -783.71 | 6378.57 |
| TRTPN*ATPTN | Bel300 | 1 | Plac | 3 | 2383.36 | 1821.91422 | 1.31 | 0.1915 | 0.05- | -1197.78 | 5964.50 |
| TRTPN*ATPTN | Bel300 | 1 | Plac | 4 | 1204.13 | 1821.91422 | 0.66 | 0.5090 | 0.05- | -2377.01 | 4785.27 |
| TRTPN*ATPTN | Bel300 | 2 | Be1300 | 3 | 4412.99 | 1848.84422 | 2.39 | 0.0174 | 0.05 | 778.91 | 8047.06 |
| TRTPN*ATPTN | Bel300 | 2 | Be1300 | 4 | 3857.81 | 1848.84422 | 2.09 | 0.0375 | 0.05 | 223.73 | 7491.89 |
| TRTPN*ATPTN | Bel300 | 2 | Be1600 | 0 | 301.82 | 1852.53422 | 0.16 | 0.8707 | 0.05- | -3339.51 | 3943.15 |
| TRTPN*ATPTN | Bel300 | 2 | Be1600 | 0.5 | -684.91 | 1852.53422 | -0.37 | 0.7118 | 0.05- | -4326.24 | 2956.43 |
| TRTPN*ATPTN | Bel300 | 2 | Be1600 | 1 | 699.72 | 1822.76422 | 0.38 | 0.7013 | 0.05- | -2883.09 | 4282.53 |
| TRTPN*ATPTN | Bel300 | 2 | Be1600 | 2 | 2304.95 | 1822.76422 | 1.26 | 0.2067 | 0.05- | -1277.86 | 5887.76 |
| TRTPN*ATPTN | Bel300 | 2 | Be1600 | 3 | 3144.59 | 1822.76422 | 1.73 | 0.0852 | 0.05 | -438.22 | 6727.40 |
| TRTPN*ATPTN | Bel300 | 2 | Be1600 | 4 | 2961.15 | 1822.76422 | 1.62 | 0.1050 | 0.05 | -621.66 | 6543.96 |
| TRTPN*ATPTN | Bel300 | 2 | Be1900 | 0 | -1468.68 | 1883.44422 | -0.78 | 0.4360 | 0.05- | -5170.76 | 2233.41 |
| TRTPN*ATPTN | Bel300 | 2 | Be1900 | 0.5 | -2903.35 | 1850.18422 | -1.57 | 0.1173 | 0.05- | -6540.05 | 733.36 |
| TRTPN*ATPTN | Bel300 | 2 | Be1900 | 1 | -83.8725 | 1850.18422 | -0.05 | 0.9639 | 0.05- | -3720.58 | 3552.84 |
| TRTPN*ATPTN | Bel300 | 2 | Be1900 | 2 | 1673.88 | 1850.18422 | 0.90 | 0.3661 | 0.05- | -1962.83 | 5310.59 |
| TRTPN*ATPTN | Bel300 | 2 | Be1900 | 3 | 2354.15 | 1850.18422 | 1.27 | 0.2039 | 0.05- | -1282.56 | 5990.85 |
| TRTPN*ATPTN | Bel300 | 2 | Be1900 | 4 | 3402.64 | 1850.18422 | 1.84 | 0.0666 | 0.05 | -234.07 | 7039.34 |
| TRTPN*ATPTN | Bel300 | 2 | 0xy30 | 0 | -239.44 | 1922.13422 | -0.12 | 0.9009 | 0.05- | -4017.59 | 3538.70 |

Program: A Bio4.sas Created: 02APR2020 7:36 POSTLOCK 

# Appendix 16.1.9.2.4 Statistical Methods and Analysis Output Supporting Table 14.2.5 Supporting Table 14.2.4

# The Mixed Procedure

#### Parameter Code=MVMIPM

# Differences of Least Squares Means

| | | | בב | TCTCIICCD V | or nease i | oquares means | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | Planned | Analysis | | Analysis | | | | | | | |
| | | - | Treatment | - | | Standard | | | | | |
| Effect | (N) | (N) | (N) | (N) | Estimate | Error DFt | | | - | Lower | Upper |
| TRTPN*ATPTN | Be1300 | 2 | 0xy30 | 0.5 | 2032.71 | 1922.13422 | 1.06 | 0.2909 | 0.05 - | 1745.44 | 5810.85 |
| TRTPN*ATPTN | Be1300 | 2 | 0xy30 | 1 | 3887.43 | 1883.53422 | 2.06 | 0.0396 | 0.05 | 185.16 | 7589.69 |
| TRTPN*ATPTN | Be1300 | 2 | 0xy30 | 2 | 3032.28 | 1850.26422 | 1.64 | 0.1020 | 0.05 - | -604.59 | 6669.14 |
| TRTPN*ATPTN | Be1300 | 2 | 0xy30 | 3 | 1437.44 | 1850.26422 | 0.78 | 0.4377 | 0.05 -2 | 2199.43 | 5074.31 |
| TRTPN*ATPTN | Be1300 | 2 | Oxy30 | 4 | 1216.68 | 1850.26422 | 0.66 | 0.5112 | 0.05 -2 | 2420.18 | 4853.55 |
| TRTPN*ATPTN | Bel300 | 2 | Oxy60 | 0 | 1220.67 | 1886.80422 | 0.65 | 0.5180 | 0.05 -2 | 2488.03 | 4929.37 |
| TRTPN*ATPTN | Be1300 | 2 | Oxy60 | 0.5 | 3452.91 | 1886.80422 | 1.83 | 0.0680 | 0.05 - | -255.80 | 7161.61 |
| TRTPN*ATPTN | Bel300 | 2 | Oxy60 | 1 | 5544.43 | 1852.83422 | 2.99 | 0.0029 | 0.05 | 1902.50 | 9186.37 |
| TRTPN*ATPTN | Be1300 | 2 | Oxy60 | 2 | 6536.98 | 1822.14422 | 3.59 | 0.0004 | 0.05 2 | 2955.38 | 10119 |
| TRTPN*ATPTN | Bel300 | 2 | Oxy60 | 3 | 5870.17 | 1822.14422 | 3.22 | 0.0014 | 0.05 2 | 2288.57 | 9451.77 |
| TRTPN*ATPTN | Bel300 | 2 | Oxy60 | 4 | 5751.03 | 1822.14422 | 3.16 | 0.0017 | 0.05 2 | 2169.43 | 9332.63 |
| TRTPN*ATPTN | Bel300 | 2 | Plac | 0 | 1352.75 | 1821.91422 | 0.74 | 0.4582 | 0.05 -2 | 2228.39 | 4933.89 |
| TRTPN*ATPTN | Bel300 | 2 | Plac | 0.5 | -172.88 | 1821.91422 | -0.09 | 0.9244 | 0.05 -3 | 3754.02 | 3408.27 |
| TRTPN*ATPTN | Bel300 | 2 | Plac | 1 | -1124.38 | 1821.91422 | -0.62 | 0.5375 | 0.05 - | 4705.52 | 2456.76 |
| TRTPN*ATPTN | Bel300 | 2 | Plac | 2 | 2941.92 | 1821.91422 | 1.61 | 0.1071 | 0.05 - | -639.22 | 6523.06 |
| TRTPN*ATPTN | Bel300 | 2 | Plac | 3 | 2527.85 | 1821.91422 | 1.39 | 0.1660 | 0.05 - | 1053.29 | 6108.99 |
| TRTPN*ATPTN | Bel300 | 2 | Plac | 4 | 1348.62 | 1821.91422 | 0.74 | 0.4596 | 0.05 -2 | 2232.52 | 4929.76 |
| TRTPN*ATPTN | Bel300 | 3 | Bel300 | 4 | -555.18 | 1848.84422 | -0.30 | 0.7641 | 0.05 - | 4189.25 | 3078.90 |
| TRTPN*ATPTN | Bel300 | 3 | Be1600 | 0 | -4111.17 | 1852.53422 | -2.22 | 0.0270 | 0.05 - | 7752.50 | -469.84 |
| TRTPN*ATPTN | Bel300 | 3 | Be1600 | 0.5 | -5097.89 | 1852.53422 | -2.75 | 0.0062 | 0.05 -8 | 3739.22- | -1456.56 |
| TRTPN*ATPTN | Bel300 | 3 | Be1600 | 1 | -3713.27 | 1822.76422 | -2.04 | 0.0423 | 0.05 - | 7296.08 | -130.46 |
| TRTPN*ATPTN | Bel300 | 3 | Be1600 | 2 | -2108.04 | 1822.76422 | -1.16 | 0.2481 | 0.05 - | 5690.85 | 1474.77 |
| TRTPN*ATPTN | Bel300 | 3 | Be1600 | 3 | -1268.39 | 1822.76422 | -0.70 | 0.4869 | 0.05 - | 4851.20 | 2314.42 |
| TRTPN*ATPTN | Bel300 | 3 | Be1600 | 4 | -1451.84 | 1822.76422 | -0.80 | 0.4262 | 0.05 - | 5034.65 | 2130.97 |
| TRTPN*ATPTN | Bel300 | 3 | Be1900 | 0 | -5881.66 | 1883.44422 | -3.12 | 0.0019 | 0.05 -9 | 9583.75- | -2179.57 |

Program: A Bio4.sas Created: 02APR2020 7:36 POSTLOCK 

# Appendix 16.1.9.2.4 Statistical Methods and Analysis Output Supporting Table 14.2.5 Supporting Table 14.2.4

# The Mixed Procedure

#### Parameter Code=MVMIPM

# Differences of Least Squares Means

| | Planned | Analysis | | Analvsis | or bease . | oquares neans | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | Treatment | _ | | :Timepoint | | Standard | | | | | |
| Effect | (N) | (N) | (N) | (N) | Estimate | Error DFt | Value Pa | r > t . | Alpha L | ower | Upper |
| TRTPN*ATPTI | N Bel300 | 3 | Be1900 | 0.5 | -7316.33 | 1850.18422 | -3.95 | <.0001 | 0.05 -1 | 0953 | -3679.63 |
| TRTPN*ATPTI | N Bel300 | 3 | Be1900 | 1 | -4496.86 | 1850.18422 | -2.43 | 0.0155 | 0.05-813 | 3.57 | -860.15 |
| TRTPN*ATPTI | N Bel300 | 3 | Be1900 | 2 | -2739.11 | 1850.18422 | -1.48 | 0.1395 | 0.05-637 | 5.81 | 897.60 |
| TRTPN*ATPT | N Bel300 | 3 | Be1900 | 3 | -2058.84 | 1850.18422 | -1.11 | 0.2664 | 0.05-569 | 5.55 | 1577.87 |
| TRTPN*ATPTI | N Bel300 | 3 | Be1900 | 4 | -1010.35 | 1850.18422 | -0.55 | 0.5853 | 0.05-464 | 7.06 | 2626.36 |
| TRTPN*ATPTI | N Bel300 | 3 | Oxy30 | 0 | -4652.43 | 1922.13422 | -2.42 | 0.0159 | 0.05-843 | 0.58 | -874.28 |
| TRTPN*ATPT | N Bel300 | 3 | Oxy30 | 0.5 | -2380.28 | 1922.13422 | -1.24 | 0.2163 | 0.05-615 | 8.43 | 1397.86 |
| TRTPN*ATPT | N Bel300 | 3 | Oxy30 | 1 | -525.56 | 1883.53422 | -0.28 | 0.7804 | 0.05-422 | 7.83 | 3176.71 |
| TRTPN*ATPT | NBel300 | 3 | Oxy30 | 2 | -1380.71 | 1850.26422 | -0.75 | 0.4559 | 0.05-501 | 7.58 | 2256.16 |
| TRTPN*ATPT | N Bel300 | 3 | Oxy30 | 3 | -2975.55 | 1850.26422 | -1.61 | 0.1085 | 0.05-661 | 2.42 | 661.32 |
| TRTPN*ATPT | N Bel300 | 3 | Oxy30 | 4 | -3196.30 | 1850.26422 | -1.73 | 0.0848 | 0.05-683 | 3.17 | 440.57 |
| TRTPN*ATPT | N Bel300 | 3 | Oxy60 | 0 | -3192.32 | 1886.80422 | -1.69 | 0.0914 | 0.05-690 | 1.02 | 516.39 |
| TRTPN*ATPT | NBel300 | 3 | Oxy60 | 0.5 | -960.08 | 1886.80422 | -0.51 | 0.6111 | 0.05-466 | 8.78 | 2748.62 |
| TRTPN*ATPT | NBel300 | 3 | Oxy60 | 1 | 1131.44 | 1852.83422 | 0.61 | 0.5418 | 0.05-251 | 0.49 | 4773.38 |
| TRTPN*ATPT | N Bel300 | 3 | Oxy60 | 2 | 2124.00 | 1822.14422 | 1.17 | 0.2444 | 0.05-145 | 7.60 | 5705.59 |
| TRTPN*ATPT | NBel300 | 3 | Oxy60 | 3 | 1457.18 | 1822.14422 | 0.80 | 0.4243 | 0.05-212 | 4.42 | 5038.78 |
| TRTPN*ATPT | NBel300 | 3 | Oxy60 | 4 | 1338.04 | 1822.14422 | 0.73 | 0.4632 | 0.05-224 | 3.56 | 4919.64 |
| TRTPN*ATPT | N Bel300 | 3 | Plac | 0 | -3060.24 | 1821.91422 | -1.68 | 0.0938 | 0.05-664 | 1.38 | 520.90 |
| TRTPN*ATPT | NBel300 | 3 | Plac | 0.5 | -4585.86 | 1821.91422 | -2.52 | 0.0122 | 0.05-816 | 7.01 | -1004.72 |
| TRTPN*ATPT | NBel300 | 3 | Plac | 1 | -5537.37 | 1821.91422 | -3.04 | 0.0025 | 0.05-911 | 8.51 | -1956.22 |
| TRTPN*ATPT | N Bel300 | 3 | Plac | 2 | -1471.07 | 1821.91422 | -0.81 | 0.4199 | 0.05-505 | 2.21 | 2110.08 |
| TRTPN*ATPT | NBel300 | 3 | Plac | 3 | -1885.14 | 1821.91422 | -1.03 | 0.3014 | 0.05-546 | 6.28 | 1696.01 |
| TRTPN*ATPT | N Bel300 | 3 | Plac | 4 | -3064.37 | 1821.91422 | -1.68 | 0.0933 | 0.05-664 | 5.51 | 516.77 |
| TRTPN*ATPT | N Bel300 | 4 | Be1600 | 0 | -3555.99 | 1852.53422 | -1.92 | 0.0556 | 0.05-719 | 7.32 | 85.3376 |
| TRTPN*ATPT | N Bel300 | 4 | Be1600 | 0.5 | -4542.71 | 1852.53422 | -2.45 | 0.0146 | 0.05-818 | 4.05 | -901.38 |

Program: A Bio4.sas Created: 02APR2020 7:36 POSTLOCK 

# Appendix 16.1.9.2.4 Statistical Methods and Analysis Output Supporting Table 14.2.5 Supporting Table 14.2.4

# The Mixed Procedure

#### Parameter Code=MVMIPM

# Differences of Least Squares Means

| | Planned | Analysis | Planned | Analysis | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| | Treatment | t Timepoint | t Treatmen | t Timepoint | | Standard | | | | |
| Effect | (N) | (N) | (N) | (N) | Estimate | Error DFt | Value P | r > t . | Alpha Lower | Upper |
| TRTPN*ATPT | N Bel300 | 4 | Be1600 | 1 | -3158.09 | 1822.76422 | -1.73 | 0.0839 | 0.05-6740.90 | 424.72 |
| TRTPN*ATPT | N Bel300 | 4 | Be1600 | 2 | -1552.86 | 1822.76422 | -0.85 | 0.3947 | 0.05-5135.67 | 2029.95 |
| TRTPN*ATPT | N Bel300 | 4 | Be1600 | 3 | -713.22 | 1822.76422 | -0.39 | 0.6958 | 0.05-4296.03 | 2869.59 |
| TRTPN*ATPT | N Bel300 | 4 | Be1600 | 4 | -896.66 | 1822.76422 | -0.49 | 0.6230 | 0.05-4479.47 | 2686.15 |
| TRTPN*ATPT | N Bel300 | 4 | Be1900 | 0 | -5326.48 | 1883.44422 | -2.83 | 0.0049 | 0.05-9028.57 | -1624.40 |
| TRTPN*ATPT | N Bel300 | 4 | Be1900 | 0.5 | -6761.16 | 1850.18422 | -3.65 | 0.0003 | 0.05 -10398 | -3124.45 |
| TRTPN*ATPT | N Bel300 | 4 | Be1900 | 1 | -3941.68 | 1850.18422 | -2.13 | 0.0337 | 0.05-7578.39 | -304.97 |
| TRTPN*ATPT | N Bel300 | 4 | Be1900 | 2 | -2183.93 | 1850.18422 | -1.18 | 0.2385 | 0.05-5820.64 | 1452.78 |
| TRTPN*ATPT | N Bel300 | 4 | Be1900 | 3 | -1503.66 | 1850.18422 | -0.81 | 0.4168 | 0.05-5140.37 | 2133.04 |
| TRTPN*ATPT | N Bel300 | 4 | Be1900 | 4 | -455.17 | 1850.18422 | -0.25 | 0.8058 | 0.05-4091.88 | 3181.53 |
| TRTPN*ATPT | N Bel300 | 4 | Oxy30 | 0 | -4097.25 | 1922.13422 | -2.13 | 0.0336 | 0.05-7875.40 | -319.11 |
| TRTPN*ATPT | N Bel300 | 4 | Oxy30 | 0.5 | -1825.10 | 1922.13422 | -0.95 | 0.3429 | 0.05-5603.25 | 1953.04 |
| TRTPN*ATPT | N Bel300 | 4 | Oxy30 | 1 | 29.6164 | 1883.53422 | 0.02 | 0.9875 | 0.05-3672.65 | 3731.88 |
| TRTPN*ATPT | N Bel300 | 4 | Oxy30 | 2 | -825.53 | 1850.26422 | -0.45 | 0.6557 | 0.05-4462.40 | 2811.33 |
| TRTPN*ATPT | N Bel300 | 4 | Oxy30 | 3 | -2420.37 | 1850.26422 | -1.31 | 0.1915 | 0.05-6057.24 | 1216.50 |
| TRTPN*ATPT | N Bel300 | 4 | Oxy30 | 4 | -2641.12 | 1850.26422 | -1.43 | 0.1542 | 0.05-6277.99 | 995.74 |
| TRTPN*ATPT | N Bel300 | 4 | Oxy60 | 0 | -2637.14 | 1886.80422 | -1.40 | 0.1629 | 0.05-6345.84 | 1071.56 |
| TRTPN*ATPT | N Bel300 | 4 | Oxy60 | 0.5 | -404.90 | 1886.80422 | -0.21 | 0.8302 | 0.05-4113.61 | 3303.80 |
| TRTPN*ATPT | N Bel300 | 4 | Oxy60 | 1 | 1686.62 | 1852.83422 | 0.91 | 0.3632 | 0.05-1955.31 | 5328.56 |
| TRTPN*ATPT | N Bel300 | 4 | Oxy60 | 2 | 2679.17 | 1822.14422 | 1.47 | 0.1422 | 0.05 -902.43 | 6260.77 |
| TRTPN*ATPT | N Bel300 | 4 | Oxy60 | 3 | 2012.36 | 1822.14422 | 1.10 | 0.2701 | 0.05-1569.24 | 5593.96 |
| TRTPN*ATPT | N Bel300 | 4 | Oxy60 | 4 | 1893.22 | 1822.14422 | 1.04 | 0.2994 | 0.05-1688.38 | 5474.82 |
| TRTPN*ATPT | N Bel300 | 4 | Plac | 0 | -2505.06 | 1821.91422 | -1.37 | 0.1699 | 0.05-6086.20 | 1076.08 |
| TRTPN*ATPT | N Bel300 | 4 | Plac | 0.5 | -4030.69 | 1821.91422 | -2.21 | 0.0275 | 0.05-7611.83 | -449.54 |
| TRTPN*ATPT | N Bel300 | 4 | Plac | 1 | -4982.19 | 1821.91422 | -2.73 | 0.0065 | 0.05-8563.33 | -1401.05 |

Program: A\_Bio4.sas Created: 02APR2020 7:36 POSTLOCK 

# Appendix 16.1.9.2.4 Statistical Methods and Analysis Output Supporting Table 14.2.5 Supporting Table 14.2.4

# The Mixed Procedure

#### Parameter Code=MVMIPM

# Differences of Least Squares Means

| | | | | | | . 1 | | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| | Planned | Analysis | Planned | Analysis | | | | | | |
| | Treatmen | t Timepoin | t Treatmen | t Timepoint | | Standard | | | | |
| Effect | (N) | (N) | (N) | (N) | Estimate | Error DFt | Value P | r > t | Alpha Lowe | r Upper |
| TRTPN*ATP1 | 'N Bel300 | 4 | Plac | 2 | -915.89 | 1821.91422 | -0.50 | 0.6154 | 0.05-4497.0 | 3 2665.25 |
| TRTPN*ATP1 | 'N Bel300 | 4 | Plac | 3 | -1329.96 | 1821.91422 | -0.73 | 0.4658 | 0.05-4911.1 | 2251.18 |
| TRTPN*ATP1 | 'N Bel300 | 4 | Plac | 4 | -2509.19 | 1821.91422 | -1.38 | 0.1692 | 0.05-6090.3 | 3 1071.95 |
| TRTPN*ATP1 | 'N Bel600 | 0 | Be1600 | 0.5 | -986.72 | 1848.84422 | -0.53 | 0.5938 | 0.05-4620.8 | 2647.35 |
| TRTPN*ATP1 | 'N Bel600 | 0 | Be1600 | 1 | 397.90 | 1820.87422 | 0.22 | 0.8271 | 0.05-3181.2 | 1 3977.02 |
| TRTPN*ATP1 | N Bel600 | 0 | Be1600 | 2 | 2003.13 | 1820.87422 | 1.10 | 0.2719 | 0.05-1575.9 | 8 5582.24 |
| TRTPN*ATP1 | 'N Bel600 | 0 | Be1600 | 3 | 2842.78 | 1820.87422 | 1.56 | 0.1192 | 0.05 -736.3 | 4 6421.89 |
| TRTPN*ATP1 | N Bel600 | 0 | Be1600 | 4 | 2659.33 | 1820.87422 | 1.46 | 0.1449 | 0.05 -919.7 | 8 6238.45 |
| TRTPN*ATP1 | N Bel600 | 0 | Be1900 | 0 | -1770.49 | 1886.03422 | -0.94 | 0.3484 | 0.05-5477.6 | 7 1936.69 |
| TRTPN*ATP1 | N Bel600 | 0 | Be1900 | 0.5 | -3205.16 | 1852.11422 | -1.73 | 0.0843 | 0.05-6845.6 | 7 435.35 |
| TRTPN*ATP1 | N Bel600 | 0 | Be1900 | 1 | -385.69 | 1852.11422 | -0.21 | 0.8351 | 0.05-4026.2 | 3254.82 |
| TRTPN*ATP1 | N Bel600 | 0 | Be1900 | 2 | 1372.07 | 1852.11422 | 0.74 | 0.4592 | 0.05-2268.4 | 4 5012.57 |
| TRTPN*ATP1 | N Bel600 | 0 | Be1900 | 3 | 2052.33 | 1852.11422 | 1.11 | 0.2684 | 0.05-1588.1 | 8 5692.84 |
| TRTPN*ATP1 | N Bel600 | 0 | Be1900 | 4 | 3100.82 | 1852.11422 | 1.67 | 0.0948 | 0.05 -539.6 | 9 6741.33 |
| TRTPN*ATP1 | N Bel600 | 0 | Oxy30 | 0 | -541.26 | 1925.09422 | -0.28 | 0.7787 | 0.05-4325.2 | 1 3242.69 |
| TRTPN*ATP1 | N Bel600 | 0 | Oxy30 | 0.5 | 1730.89 | 1925.09422 | 0.90 | 0.3691 | 0.05-2053.0 | 5514.84 |
| TRTPN*ATP1 | N Bel600 | 0 | Oxy30 | 1 | 3585.61 | 1886.28422 | 1.90 | 0.0580 | 0.05 -122.0 | 7 7293.29 |
| TRTPN*ATP1 | N Bel600 | 0 | Oxy30 | 2 | 2730.46 | 1852.82422 | 1.47 | 0.1413 | 0.05 -911.4 | 5 6372.37 |
| TRTPN*ATP1 | N Bel600 | 0 | Oxy30 | 3 | 1135.62 | 1852.82422 | 0.61 | 0.5403 | 0.05-2506.2 | 9 4777.53 |
| TRTPN*ATP1 | N Bel600 | 0 | Oxy30 | 4 | 914.87 | 1852.82422 | 0.49 | 0.6217 | 0.05-2727.0 | 4 4556.78 |
| TRTPN*ATP1 | N Bel600 | 0 | Oxy60 | 0 | 918.86 | 1886.96422 | 0.49 | 0.6265 | 0.05-2790.1 | 6 4627.87 |
| TRTPN*ATP1 | N Bel600 | 0 | Oxy60 | 0.5 | 3151.09 | 1886.96422 | 1.67 | 0.0957 | 0.05 -557.9 | 2 6860.11 |
| TRTPN*ATP1 | N Bel600 | 0 | Oxy60 | 1 | 5242.62 | 1853.41422 | 2.83 | 0.0049 | 0.05 1599.5 | 5 8885.68 |
| TRTPN*ATP1 | 'N Bel600 | 0 | Oxy60 | 2 | 6235.17 | 1822.19422 | 3.42 | 0.0007 | 0.05 2653.4 | 7 9816.86 |
| TRTPN*ATP1 | N Bel600 | 0 | Oxy60 | 3 | 5568.35 | 1822.19422 | 3.06 | 0.0024 | 0.05 1986.6 | 6 9150.05 |

Program: A Bio4.sas Created: 02APR2020 7:36 POSTLOCK 

Appendix 16.1.9.2.4
Statistical Methods and Analysis Output Supporting Table 14.2.5
Supporting Table 14.2.4

# The Mixed Procedure

#### Parameter Code=MVMIPM

# Differences of Least Squares Means

| | | | D11 | . ICICIICCO I | or nease i | squares means | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | Planned | Analysis | Planned | Analysis | | | | | | | |
| | Treatment | Timepoint | Treatment | Timepoint | | Standard | | | | | |
| Effect | (N) | (N) | (N) | (N) | Estimate | Error DF t | Value Pi | r > t . | Alpha | Lower | Upper |
| TRTPN*ATPTN | Be1600 | 0 | Oxy60 | 4 | 5449.21 | 1822.19422 | 2.99 | 0.0029 | 0.05 | 1867.52 | 9030.91 |
| TRTPN*ATPTN | Be1600 | 0 | Plac | 0 | 1050.93 | 1820.82422 | 0.58 | 0.5641 | 0.05 - | 2528.08 | 4629.94 |
| TRTPN*ATPTN | Bel600 | 0 | Plac | 0.5 | -474.69 | 1820.82422 | -0.26 | 0.7944 | 0.05 - | 4053.70 | 3104.32 |
| TRTPN*ATPTN | Be1600 | 0 | Plac | 1 | -1426.19 | 1820.82422 | -0.78 | 0.4339 | 0.05 - | 5005.20 | 2152.81 |
| TRTPN*ATPTN | Bel600 | 0 | Plac | 2 | 2640.11 | 1820.82422 | 1.45 | 0.1478 | 0.05 | -938.90 | 6219.11 |
| TRTPN*ATPTN | Bel600 | 0 | Plac | 3 | 2226.04 | 1820.82422 | 1.22 | 0.2222 | 0.05 - | 1352.97 | 5805.05 |
| TRTPN*ATPTN | Bel600 | 0 | Plac | 4 | 1046.80 | 1820.82422 | 0.57 | 0.5657 | 0.05 - | 2532.21 | 4625.81 |
| TRTPN*ATPTN | Bel600 | 0.5 | Be1600 | 1 | 1384.63 | 1820.87422 | 0.76 | 0.4474 | 0.05 - | 2194.49 | 4963.74 |
| TRTPN*ATPTN | Bel600 | 0.5 | Be1600 | 2 | 2989.85 | 1820.87422 | 1.64 | 0.1013 | 0.05 | -589.26 | 6568.97 |
| TRTPN*ATPTN | Bel600 | 0.5 | Be1600 | 3 | 3829.50 | 1820.87422 | 2.10 | 0.0360 | 0.05 | 250.38 | 7408.61 |
| TRTPN*ATPTN | Bel600 | 0.5 | Be1600 | 4 | 3646.05 | 1820.87422 | 2.00 | 0.0459 | 0.05 | 66.9402 | 7225.17 |
| TRTPN*ATPTN | Be1600 | 0.5 | Be1900 | 0 | -783.77 | 1886.03422 | -0.42 | 0.6779 | 0.05- | 4490.95 | 2923.41 |
| TRTPN*ATPTN | Bel600 | 0.5 | Be1900 | 0.5 | -2218.44 | 1852.11422 | -1.20 | 0.2317 | 0.05 - | 5858.95 | 1422.07 |
| TRTPN*ATPTN | Be1600 | 0.5 | Be1900 | 1 | 601.03 | 1852.11422 | 0.32 | 0.7457 | 0.05- | 3039.47 | 4241.54 |
| TRTPN*ATPTN | Be1600 | 0.5 | Be1900 | 2 | 2358.79 | 1852.11422 | 1.27 | 0.2035 | 0.05 - | 1281.72 | 5999.29 |
| TRTPN*ATPTN | Bel600 | 0.5 | Be1900 | 3 | 3039.05 | 1852.11422 | 1.64 | 0.1016 | 0.05 | -601.46 | 6679.56 |
| TRTPN*ATPTN | Be1600 | 0.5 | Be1900 | 4 | 4087.54 | 1852.11422 | 2.21 | 0.0279 | 0.05 | 447.03 | 7728.05 |
| TRTPN*ATPTN | Be1600 | 0.5 | 0xy30 | 0 | 445.46 | 1925.09422 | 0.23 | 0.8171 | 0.05 - | 3338.49 | 4229.41 |
| TRTPN*ATPTN | Bel600 | 0.5 | 0xy30 | 0.5 | 2717.61 | 1925.09422 | 1.41 | 0.1588 | 0.05 - | 1066.34 | 6501.56 |
| TRTPN*ATPTN | Be1600 | 0.5 | 0xy30 | 1 | 4572.33 | 1886.28422 | 2.42 | 0.0158 | 0.05 | 864.65 | 8280.01 |
| TRTPN*ATPTN | Be1600 | 0.5 | 0xy30 | 2 | 3717.18 | 1852.82422 | 2.01 | 0.0455 | 0.05 | 75.2728 | 7359.09 |
| TRTPN*ATPTN | Bel600 | 0.5 | Oxy30 | 3 | 2122.34 | 1852.82422 | 1.15 | 0.2527 | 0.05 - | 1519.57 | 5764.25 |
| TRTPN*ATPTN | Bel600 | 0.5 | 0xy30 | 4 | 1901.59 | 1852.82422 | 1.03 | 0.3053 | 0.05 - | 1740.32 | 5543.50 |
| TRTPN*ATPTN | Bel600 | 0.5 | Oxy60 | 0 | 1905.58 | 1886.96422 | 1.01 | 0.3131 | 0.05 - | 1803.44 | 5614.59 |
| TRTPN*ATPTN | Be1600 | 0.5 | Oxy60 | 0.5 | 4137.81 | 1886.96422 | 2.19 | 0.0289 | 0.05 | 428.80 | 7846.83 |

Program: A Bio4.sas Created: 02APR2020 7:36 POSTLOCK 

Appendix 16.1.9.2.4
Statistical Methods and Analysis Output Supporting Table 14.2.5
Supporting Table 14.2.4

# The Mixed Procedure

#### Parameter Code=MVMIPM

# Differences of Least Squares Means

| | D1 | | | | or heade i | oquares neans | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | Planned | Analysis | | Analysis | | 0+ | | | | | |
| D.C.C. | | - | | Timepoint | | Standard | 77. 1 . D | | | Ŧ | TT |
| Effect | (N) | (N) | (N) | (N) | Estimate | Error DFt | | | | Lower | Upper |
| TRTPN*ATPTN | | 0.5 | Oxy60 | 1 | | 1853.41422 | 3.36 | 0.0008 | | 2586.28 | 9872.40 |
| TRTPN*ATPTN | Bel600 | 0.5 | Oxy60 | 2 | | 1822.19422 | 3.96 | <.0001 | | 3640.19 | 10804 |
| TRTPN*ATPTN | Be1600 | 0.5 | Oxy60 | 3 | 6555.07 | 1822.19422 | 3.60 | 0.0004 | 0.05 | 2973.38 | 10137 |
| TRTPN*ATPTN | Bel600 | 0.5 | Oxy60 | 4 | 6435.93 | 1822.19422 | 3.53 | 0.0005 | 0.05 | 2854.24 | 10018 |
| TRTPN*ATPTN | Bel600 | 0.5 | Plac | 0 | 2037.66 | 1820.82422 | 1.12 | 0.2637 | 0.05- | -1541.35 | 5616.67 |
| TRTPN*ATPTN | Be1600 | 0.5 | Plac | 0.5 | 512.03 | 1820.82422 | 0.28 | 0.7787 | 0.05- | -3066.98 | 4091.04 |
| TRTPN*ATPTN | Be1600 | 0.5 | Plac | 1 | -439.47 | 1820.82422 | -0.24 | 0.8094 | 0.05- | -4018.48 | 3139.54 |
| TRTPN*ATPTN | Bel600 | 0.5 | Plac | 2 | 3626.83 | 1820.82422 | 1.99 | 0.0470 | 0.05 | 47.8170 | 7205.84 |
| TRTPN*ATPTN | Be1600 | 0.5 | Plac | 3 | 3212.76 | 1820.82422 | 1.76 | 0.0784 | 0.05 | -366.25 | 6791.77 |
| TRTPN*ATPTN | Bel600 | 0.5 | Plac | 4 | 2033.52 | 1820.82422 | 1.12 | 0.2647 | 0.05- | -1545.49 | 5612.53 |
| TRTPN*ATPTN | Bel600 | 1 | Be1600 | 2 | 1605.23 | 1790.13422 | 0.90 | 0.3704 | 0.05- | -1913.45 | 5123.90 |
| TRTPN*ATPTN | Bel600 | 1 | Be1600 | 3 | 2444.87 | 1790.13422 | 1.37 | 0.1727 | 0.05- | -1073.81 | 5963.55 |
| TRTPN*ATPTN | Be1600 | 1 | Be1600 | 4 | 2261.43 | 1790.13422 | 1.26 | 0.2072 | 0.05- | -1257.25 | 5780.11 |
| TRTPN*ATPTN | Bel600 | 1 | Be1900 | 0 | -2168.40 | 1856.55422 | -1.17 | 0.2435 | 0.05- | -5817.63 | 1480.84 |
| TRTPN*ATPTN | Bel600 | 1 | Be1900 | 0.5 | -3603.07 | 1822.36422 | -1.98 | 0.0487 | 0.05- | -7185.09 | -21.0431 |
| TRTPN*ATPTN | Bel600 | 1 | Be1900 | 1 | -783.59 | 1822.36422 | -0.43 | 0.6674 | 0.05- | -4365.62 | 2798.43 |
| TRTPN*ATPTN | Bel600 | 1 | Be1900 | 2 | 974.16 | 1822.36422 | 0.53 | 0.5932 | 0.05- | -2607.86 | 4556.18 |
| TRTPN*ATPTN | Bel600 | 1 | Be1900 | 3 | 1654.43 | 1822.36422 | 0.91 | 0.3645 | 0.05- | -1927.60 | 5236.45 |
| TRTPN*ATPTN | Bel600 | 1 | Be1900 | 4 | 2702.91 | 1822.36422 | 1.48 | 0.1388 | 0.05 | -879.11 | 6284.94 |
| TRTPN*ATPTN | Bel600 | 1 | 0xy30 | 0 | -939.16 | 1896.89422 | -0.50 | 0.6208 | 0.05- | -4667.68 | 2789.36 |
| TRTPN*ATPTN | Bel600 | 1 | Oxy30 | 0.5 | 1332.98 | 1896.89422 | 0.70 | 0.4826 | 0.05- | -2395.54 | 5061.51 |
| TRTPN*ATPTN | Bel600 | 1 | Oxy30 | 1 | 3187.71 | 1856.86422 | 1.72 | 0.0868 | 0.05 | -462.14 | 6837.55 |
| TRTPN*ATPTN | Bel600 | 1 | 0xy30 | 2 | 2332.55 | 1822.29422 | 1.28 | 0.2012 | 0.05- | -1249.33 | 5914.44 |
| TRTPN*ATPTN | Bel600 | 1 | Oxy30 | 3 | 737.72 | 1822.29422 | 0.40 | 0.6858 | 0.05- | -2844.17 | 4319.60 |
| TRTPN*ATPTN | Bel600 | 1 | Oxy30 | 4 | 516.96 | 1822.29422 | 0.28 | 0.7768 | 0.05- | -3064.92 | 4098.85 |

Program: A Bio4.sas Created: 02APR2020 7:36 POSTLOCK 

# Appendix 16.1.9.2.4 Statistical Methods and Analysis Output Supporting Table 14.2.5 Supporting Table 14.2.4

# The Mixed Procedure

#### Parameter Code=MVMIPM

# Differences of Least Squares Means

| | Planned | Analysis | | Analvsis | or bease . | oquares neams | | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| | Treatment | _ | | . Timepoint | | Standard | | | | |
| Effect | (N) | (N) | (N) | (N) | Estimate | Error DFt | Value P | r > t . | Alpha Lower | Upper |
| TRTPN*ATPT | N Bel600 | 1 | Oxy60 | 0 | 520.95 | 1857.43422 | 0.28 | 0.7793 | 0.05-3130.02 | 4171.93 |
| TRTPN*ATPT | N Bel600 | 1 | Oxy60 | 0.5 | 2753.19 | 1857.43422 | 1.48 | 0.1390 | 0.05 -897.79 | 6404.16 |
| TRTPN*ATPT | N Bel600 | 1 | Oxy60 | 1 | 4844.71 | 1822.82422 | 2.66 | 0.0082 | 0.05 1261.78 | 8427.64 |
| TRTPN*ATPTI | NBel600 | 1 | Oxy60 | 2 | 5837.26 | 1791.36422 | 3.26 | 0.0012 | 0.05 2316.16 | 9358.37 |
| TRTPN*ATPT | N Bel600 | 1 | Oxy60 | 3 | 5170.45 | 1791.36422 | 2.89 | 0.0041 | 0.05 1649.34 | 8691.55 |
| TRTPN*ATPT | N Bel600 | 1 | Oxy60 | 4 | 5051.31 | 1791.36422 | 2.82 | 0.0050 | 0.05 1530.20 | 8572.41 |
| TRTPN*ATPTI | NBel600 | 1 | Plac | 0 | 653.03 | 1790.78422 | 0.36 | 0.7155 | 0.05-2866.93 | 4172.99 |
| TRTPN*ATPTI | NBel600 | 1 | Plac | 0.5 | -872.60 | 1790.78422 | -0.49 | 0.6263 | 0.05-4392.55 | 2647.36 |
| TRTPN*ATPT | N Bel600 | 1 | Plac | 1 | -1824.10 | 1790.78422 | -1.02 | 0.3090 | 0.05-5344.06 | 1695.86 |
| TRTPN*ATPT | NBel600 | 1 | Plac | 2 | 2242.20 | 1790.78422 | 1.25 | 0.2112 | 0.05-1277.76 | 5762.16 |
| TRTPN*ATPT | NBel600 | 1 | Plac | 3 | 1828.13 | 1790.78422 | 1.02 | 0.3079 | 0.05-1691.83 | 5348.09 |
| TRTPN*ATPTI | NBel600 | 1 | Plac | 4 | 648.90 | 1790.78422 | 0.36 | 0.7173 | 0.05-2871.06 | 4168.85 |
| TRTPN*ATPT | N Bel600 | 2 | Be1600 | 3 | 839.65 | 1790.13422 | 0.47 | 0.6393 | 0.05-2679.03 | 4358.33 |
| TRTPN*ATPT | N Bel600 | 2 | Be1600 | 4 | 656.20 | 1790.13422 | 0.37 | 0.7141 | 0.05-2862.48 | 4174.88 |
| TRTPN*ATPT | NBel600 | 2 | Be1900 | 0 | -3773.62 | 1856.55422 | -2.03 | 0.0427 | 0.05-7422.86 | -124.39 |
| TRTPN*ATPT | N Bel600 | 2 | Be1900 | 0.5 | -5208.29 | 1822.36422 | -2.86 | 0.0045 | 0.05-8790.32 | -1626.27 |
| TRTPN*ATPT | NBel600 | 2 | Be1900 | 1 | -2388.82 | 1822.36422 | -1.31 | 0.1906 | 0.05-5970.84 | 1193.20 |
| TRTPN*ATPT | NBel600 | 2 | Be1900 | 2 | -631.06 | 1822.36422 | -0.35 | 0.7293 | 0.05-4213.09 | 2950.96 |
| TRTPN*ATPT | N Bel600 | 2 | Be1900 | 3 | 49.1998 | 1822.36422 | 0.03 | 0.9785 | 0.05-3532.82 | 3631.22 |
| TRTPN*ATPT | N Bel600 | 2 | Be1900 | 4 | 1097.69 | 1822.36422 | 0.60 | 0.5473 | 0.05-2484.33 | 4679.71 |
| TRTPN*ATPT | NBel600 | 2 | Oxy30 | 0 | -2544.39 | 1896.89422 | -1.34 | 0.1805 | 0.05-6272.91 | 1184.13 |
| TRTPN*ATPT | N Bel600 | 2 | Oxy30 | 0.5 | -272.24 | 1896.89422 | -0.14 | 0.8859 | 0.05-4000.76 | 3456.28 |
| TRTPN*ATPT | NBel600 | 2 | Oxy30 | 1 | 1582.48 | 1856.86422 | 0.85 | 0.3946 | 0.05-2067.37 | 5232.33 |
| TRTPN*ATPTI | NBel600 | 2 | Oxy30 | 2 | 727.33 | 1822.29422 | 0.40 | 0.6900 | 0.05-2854.56 | 4309.22 |
| TRTPN*ATPTI | NBel600 | 2 | Oxy30 | 3 | -867.51 | 1822.29422 | -0.48 | 0.6343 | 0.05-4449.40 | 2714.38 |

Program: A Bio4.sas Created: 02APR2020 7:36 POSTLOCK 

Appendix 16.1.9.2.4
Statistical Methods and Analysis Output Supporting Table 14.2.5
Supporting Table 14.2.4

# The Mixed Procedure

#### Parameter Code=MVMIPM

# Differences of Least Squares Means

| | | | | | or nease . | squares neams | | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| | Planned | Analysis | | Analysis | | | | | | |
| | Treatment | Timepoint | Treatment | Timepoint | | Standard | | | | |
| Effect | (N) | (N) | (N) | (N) | Estimate | Error DFt | | | - | Upper |
| TRTPN*ATPTN | Be1600 | 2 | 0xy30 | 4 | -1088.26 | 1822.29422 | -0.60 | 0.5507 | 0.05-4670.15 | 2493.62 |
| TRTPN*ATPTN | Be1600 | 2 | Oxy60 | 0 | -1084.27 | 1857.43422 | -0.58 | 0.5597 | 0.05-4735.25 | 2566.70 |
| TRTPN*ATPTN | Be1600 | 2 | Oxy60 | 0.5 | 1147.96 | 1857.43422 | 0.62 | 0.5369 | 0.05-2503.02 | 4798.94 |
| TRTPN*ATPTN | Be1600 | 2 | Oxy60 | 1 | 3239.49 | 1822.82422 | 1.78 | 0.0763 | 0.05 -343.45 | 6822.42 |
| TRTPN*ATPTN | Be1600 | 2 | Oxy60 | 2 | 4232.04 | 1791.36422 | 2.36 | 0.0186 | 0.05 710.93 | 7753.14 |
| TRTPN*ATPTN | Bel600 | 2 | Oxy60 | 3 | 3565.22 | 1791.36422 | 1.99 | 0.0472 | 0.05 44.1157 | 7086.33 |
| TRTPN*ATPTN | Be1600 | 2 | Oxy60 | 4 | 3446.08 | 1791.36422 | 1.92 | 0.0551 | 0.05-75.0234 | 6967.19 |
| TRTPN*ATPTN | Bel600 | 2 | Plac | 0 | -952.20 | 1790.78422 | -0.53 | 0.5952 | 0.05-4472.15 | 2567.76 |
| TRTPN*ATPTN | Be1600 | 2 | Plac | 0.5 | -2477.82 | 1790.78422 | -1.38 | 0.1672 | 0.05-5997.78 | 1042.13 |
| TRTPN*ATPTN | Bel600 | 2 | Plac | 1 | -3429.33 | 1790.78422 | -1.91 | 0.0562 | 0.05-6949.28 | 90.6325 |
| TRTPN*ATPTN | Bel600 | 2 | Plac | 2 | 636.97 | 1790.78422 | 0.36 | 0.7222 | 0.05-2882.98 | 4156.93 |
| TRTPN*ATPTN | Bel600 | 2 | Plac | 3 | 222.91 | 1790.78422 | 0.12 | 0.9010 | 0.05-3297.05 | 3742.86 |
| TRTPN*ATPTN | Bel600 | 2 | Plac | 4 | -956.33 | 1790.78422 | -0.53 | 0.5936 | 0.05-4476.29 | 2563.63 |
| TRTPN*ATPTN | Bel600 | 3 | Be1600 | 4 | -183.44 | 1790.13422 | -0.10 | 0.9184 | 0.05-3702.12 | 3335.23 |
| TRTPN*ATPTN | Bel600 | 3 | Be1900 | 0 | -4613.27 | 1856.55422 | -2.48 | 0.0133 | 0.05-8262.50 | -964.03 |
| TRTPN*ATPTN | Bel600 | 3 | Be1900 | 0.5 | -6047.94 | 1822.36422 | -3.32 | 0.0010 | 0.05-9629.96 | -2465.92 |
| TRTPN*ATPTN | Bel600 | 3 | Be1900 | 1 | -3228.47 | 1822.36422 | -1.77 | 0.0772 | 0.05-6810.49 | 353.56 |
| TRTPN*ATPTN | Bel600 | 3 | Be1900 | 2 | -1470.71 | 1822.36422 | -0.81 | 0.4201 | 0.05-5052.74 | 2111.31 |
| TRTPN*ATPTN | Bel600 | 3 | Be1900 | 3 | -790.45 | 1822.36422 | -0.43 | 0.6647 | 0.05-4372.47 | 2791.58 |
| TRTPN*ATPTN | Bel600 | 3 | Be1900 | 4 | 258.04 | 1822.36422 | 0.14 | 0.8875 | 0.05-3323.98 | 3840.07 |
| TRTPN*ATPTN | Bel600 | 3 | 0xy30 | 0 | -3384.04 | 1896.89422 | -1.78 | 0.0751 | 0.05-7112.56 | 344.48 |
| TRTPN*ATPTN | Bel600 | 3 | Oxy30 | 0.5 | -1111.89 | 1896.89422 | -0.59 | 0.5581 | 0.05-4840.41 | 2616.63 |
| TRTPN*ATPTN | Bel600 | 3 | 0xy30 | 1 | 742.83 | 1856.86422 | 0.40 | 0.6893 | 0.05-2907.01 | 4392.68 |
| TRTPN*ATPTN | Bel600 | 3 | Oxy30 | 2 | -112.32 | 1822.29422 | -0.06 | 0.9509 | 0.05-3694.20 | 3469.57 |
| TRTPN*ATPTN | Bel600 | 3 | 0xy30 | 3 | -1707.16 | 1822.29422 | -0.94 | 0.3494 | 0.05-5289.04 | 1874.73 |

Program: A Bio4.sas Created: 02APR2020 7:36 POSTLOCK 

# Appendix 16.1.9.2.4 Statistical Methods and Analysis Output Supporting Table 14.2.5 Supporting Table 14.2.4

# The Mixed Procedure

#### Parameter Code=MVMIPM

# Differences of Least Squares Means

| | | | | | or nease t | squares means | | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| | Planned | Analysis | | Analysis | | | | | | |
| | | - | Treatment | - | | Standard | | | | |
| Effect | (N) | (N) | (N) | (N) | Estimate | Error DF t | | | - | Upper |
| TRTPN*ATPTN | Be1600 | 3 | 0xy30 | 4 | -1927.91 | 1822.29422 | -1.06 | 0.2907 | 0.05-5509.80 | 1653.98 |
| TRTPN*ATPTN | Be1600 | 3 | Oxy60 | 0 | -1923.92 | 1857.43422 | -1.04 | 0.3009 | 0.05-5574.90 | 1727.05 |
| TRTPN*ATPTN | Be1600 | 3 | Oxy60 | 0.5 | 308.31 | 1857.43422 | 0.17 | 0.8682 | 0.05-3342.66 | 3959.29 |
| TRTPN*ATPTN | Be1600 | 3 | Oxy60 | 1 | 2399.84 | 1822.82422 | 1.32 | 0.1887 | 0.05-1183.09 | 5982.77 |
| TRTPN*ATPTN | Be1600 | 3 | Oxy60 | 2 | 3392.39 | 1791.36422 | 1.89 | 0.0589 | 0.05 -128.72 | 6913.49 |
| TRTPN*ATPTN | Bel600 | 3 | Oxy60 | 3 | 2725.57 | 1791.36422 | 1.52 | 0.1289 | 0.05 -795.53 | 6246.68 |
| TRTPN*ATPTN | Be1600 | 3 | Oxy60 | 4 | 2606.43 | 1791.36422 | 1.46 | 0.1464 | 0.05 -914.67 | 6127.54 |
| TRTPN*ATPTN | Bel600 | 3 | Plac | 0 | -1791.84 | 1790.78422 | -1.00 | 0.3176 | 0.05-5311.80 | 1728.11 |
| TRTPN*ATPTN | Be1600 | 3 | Plac | 0.5 | -3317.47 | 1790.78422 | -1.85 | 0.0646 | 0.05-6837.43 | 202.49 |
| TRTPN*ATPTN | Bel600 | 3 | Plac | 1 | -4268.97 | 1790.78422 | -2.38 | 0.0176 | 0.05-7788.93 | -749.01 |
| TRTPN*ATPTN | Bel600 | 3 | Plac | 2 | -202.67 | 1790.78422 | -0.11 | 0.9099 | 0.05-3722.63 | 3317.29 |
| TRTPN*ATPTN | Bel600 | 3 | Plac | 3 | -616.74 | 1790.78422 | -0.34 | 0.7307 | 0.05-4136.70 | 2903.22 |
| TRTPN*ATPTN | Bel600 | 3 | Plac | 4 | -1795.98 | 1790.78422 | -1.00 | 0.3165 | 0.05-5315.93 | 1723.98 |
| TRTPN*ATPTN | Bel600 | 4 | Be1900 | 0 | -4429.82 | 1856.55422 | -2.39 | 0.0175 | 0.05-8079.06 | -780.59 |
| TRTPN*ATPTN | Bel600 | 4 | Be1900 | 0.5 | -5864.50 | 1822.36422 | -3.22 | 0.0014 | 0.05-9446.52 | -2282.47 |
| TRTPN*ATPTN | Bel600 | 4 | Be1900 | 1 | -3045.02 | 1822.36422 | -1.67 | 0.0955 | 0.05-6627.05 | 537.00 |
| TRTPN*ATPTN | Bel600 | 4 | Be1900 | 2 | -1287.27 | 1822.36422 | -0.71 | 0.4803 | 0.05-4869.29 | 2294.76 |
| TRTPN*ATPTN | Bel600 | 4 | Be1900 | 3 | -607.00 | 1822.36422 | -0.33 | 0.7392 | 0.05-4189.03 | 2975.02 |
| TRTPN*ATPTN | Bel600 | 4 | Be1900 | 4 | 441.49 | 1822.36422 | 0.24 | 0.8087 | 0.05-3140.54 | 4023.51 |
| TRTPN*ATPTN | Bel600 | 4 | 0xy30 | 0 | -3200.59 | 1896.89422 | -1.69 | 0.0923 | 0.05-6929.11 | 527.93 |
| TRTPN*ATPTN | Bel600 | 4 | 0xy30 | 0.5 | -928.44 | 1896.89422 | -0.49 | 0.6248 | 0.05-4656.96 | 2800.08 |
| TRTPN*ATPTN | Bel600 | 4 | 0xy30 | 1 | 926.28 | 1856.86422 | 0.50 | 0.6182 | 0.05-2723.57 | 4576.12 |
| TRTPN*ATPTN | Bel600 | 4 | 0xy30 | 2 | 71.1266 | 1822.29422 | 0.04 | 0.9689 | 0.05-3510.76 | 3653.01 |
| TRTPN*ATPTN | Bel600 | 4 | 0xy30 | 3 | -1523.71 | 1822.29422 | -0.84 | 0.4035 | 0.05-5105.60 | 2058.17 |
| TRTPN*ATPTN | Bel600 | 4 | 0xy30 | 4 | -1744.46 | 1822.29422 | -0.96 | 0.3390 | 0.05-5326.35 | 1837.42 |

Program: A Bio4.sas Created: 02APR2020 7:36 POSTLOCK


Appendix 16.1.9.2.4
Statistical Methods and Analysis Output Supporting Table 14.2.5
Supporting Table 14.2.4

# The Mixed Procedure

#### Parameter Code=MVMIPM

# Differences of Least Squares Means

| | D1 1 | 3 | | | or bease i | oquares means | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | Planned | Analysis | | Analysis<br>Timepoint | | Standard | | | | | |
| Effect | | - | | - | | | 17-1 D. | | 7 7 1 | T | TT |
| | (N) | (N) | (N) | (N) | Estimate | Error DFt | | | | Lower | Upper |
| TRTPN*ATPT | | 4 | Oxy60 | 0 | | 1857.43422 | -0.94 | | 0.05-53 | | 1910.50 |
| TRTPN*ATPT | | 4 | Oxy60 | 0.5 | | 1857.43422 | 0.26 | 0.7913 | 0.05-31 | | 4142.73 |
| TRTPN*ATPT | N Bel600 | 4 | Oxy60 | 1 | 2583.28 | 1822.82422 | 1.42 | 0.1572 | 0.05 -9 | 999.65 | |
| TRTPN*ATPT | NBel600 | 4 | Oxy60 | 2 | 3575.83 | 1791.36422 | 2.00 | 0.0466 | 0.05 54 | 1.7283 | 7096.94 |
| TRTPN*ATPT | NBel600 | 4 | Oxy60 | 3 | 2909.02 | 1791.36422 | 1.62 | 0.1051 | 0.05 -6 | 512.09 | 6430.12 |
| TRTPN*ATPT | NBel600 | 4 | Oxy60 | 4 | 2789.88 | 1791.36422 | 1.56 | 0.1201 | 0.05 -7 | 731.23 | 6310.98 |
| TRTPN*ATPT | N Bel600 | 4 | Plac | 0 | -1608.40 | 1790.78422 | -0.90 | 0.3696 | 0.05-51 | L28.36 | 1911.56 |
| TRTPN*ATPT | NBel600 | 4 | Plac | 0.5 | -3134.03 | 1790.78422 | -1.75 | 0.0808 | 0.05-66 | 553.98 | 385.93 |
| TRTPN*ATPT | N Bel600 | 4 | Plac | 1 | -4085.53 | 1790.78422 | -2.28 | 0.0230 | 0.05-76 | 505.49 | -565.57 |
| TRTPN*ATPT | NBel600 | 4 | Plac | 2 | -19.2279 | 1790.78422 | -0.01 | 0.9914 | 0.05-35 | 539.19 | 3500.73 |
| TRTPN*ATPT | NBel600 | 4 | Plac | 3 | -433.30 | 1790.78422 | -0.24 | 0.8089 | 0.05-39 | 953.25 | 3086.66 |
| TRTPN*ATPT | NBel600 | 4 | Plac | 4 | -1612.53 | 1790.78422 | -0.90 | 0.3684 | 0.05-51 | 132.49 | 1907.43 |
| TRTPN*ATPT | N Bel900 | 0 | Be1900 | 0.5 | -1434.67 | 1882.76422 | -0.76 | 0.4465 | 0.05-51 | 135.43 | 2266.09 |
| TRTPN*ATPT | NBe1900 | 0 | Be1900 | 1 | 1384.80 | 1882.76422 | 0.74 | 0.4624 | 0.05-23 | 315.95 | 5085.56 |
| TRTPN*ATPT | N Bel900 | 0 | Be1900 | 2 | 3142.56 | 1882.76422 | 1.67 | 0.0958 | 0.05 -5 | 558.20 | 6843.31 |
| TRTPN*ATPT | N Bel900 | 0 | Be1900 | 3 | 3822.82 | 1882.76422 | 2.03 | 0.0429 | 0.05 1 | 122.06 | 7523.58 |
| TRTPN*ATPT | NBe1900 | 0 | Be1900 | 4 | 4871.31 | 1882.76422 | 2.59 | 0.0100 | 0.05 11 | 170.55 | 8572.07 |
| TRTPN*ATPT | NBe1900 | 0 | Oxy30 | 0 | 1229.23 | 1955.46422 | 0.63 | 0.5299 | 0.05-26 | 514.42 | 5072.88 |
| TRTPN*ATPT | NBe1900 | 0 | Oxy30 | 0.5 | 3501.38 | 1955.46422 | 1.79 | 0.0741 | 0.05 -3 | 342.27 | 7345.03 |
| TRTPN*ATPT | N Bel900 | 0 | Oxy30 | 1 | 5356.10 | 1917.18422 | 2.79 | 0.0054 | 0.05 15 | 587.70 | 9124.50 |
| TRTPN*ATPT | N Bel900 | 0 | Oxy30 | 2 | 4500.95 | 1884.18422 | 2.39 | 0.0173 | 0.05 | 797.40 | 8204.50 |
| TRTPN*ATPT | N Bel900 | 0 | Oxy30 | 3 | 2906.11 | 1884.18422 | 1.54 | 0.1237 | 0.05 -7 | 797.44 | 6609.66 |
| TRTPN*ATPT | N Bel900 | 0 | Oxy30 | 4 | 2685.36 | 1884.18422 | 1.43 | 0.1548 | 0.05-10 | 018.19 | 6388.91 |
| TRTPN*ATPT | N Bel900 | 0 | 0xy60 | 0 | 2689.35 | 1919.01422 | 1.40 | 0.1618 | 0.05-10 | 082.65 | 6461.35 |
| TRTPN*ATPT | N Bel900 | 0 | 0xy60 | 0.5 | 4921.58 | 1919.01422 | 2.56 | 0.0107 | 0.05 11 | L49.58 | 8693.58 |
| | | | - | | | | | | | | |

Program: A Bio4.sas Created: 02APR2020 7:36 POSTLOCK 

Appendix 16.1.9.2.4
Statistical Methods and Analysis Output Supporting Table 14.2.5
Supporting Table 14.2.4

# The Mixed Procedure

#### Parameter Code=MVMIPM

# Differences of Least Squares Means

| | Planned | Analysis | | Analysis | or heade . | oquares means | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | Treatment | | | t Timepoint | | Standard | | | | | |
| Effect | (N) | (N) | (N) | (N) | Estimate | Error DFt | Value P | r > t . | Alpha | Lower | Upper |
| TRTPN*ATPTI | N Bel900 | 0 | Oxy60 | 1 | 7013.11 | 1886.16422 | 3.72 | 0.0002 | 0.05 | 3305.67 | 10721 |
| TRTPN*ATPT | N Bel900 | 0 | Oxy60 | 2 | 8005.66 | 1855.83422 | 4.31 | <.0001 | 0.05 | 4357.83 | 11653 |
| TRTPN*ATPT | N Bel900 | 0 | Oxy60 | 3 | 7338.84 | 1855.83422 | 3.95 | <.0001 | 0.05 | 3691.02 | 10987 |
| TRTPN*ATPT | N Bel900 | 0 | Oxy60 | 4 | 7219.70 | 1855.83422 | 3.89 | 0.0001 | 0.05 | 3571.88 | 10868 |
| TRTPN*ATPT | N Bel900 | 0 | Plac | 0 | 2821.43 | 1856.35422 | 1.52 | 0.1293 | 0.05 | -827.42 | 6470.27 |
| TRTPN*ATPT | N Bel900 | 0 | Plac | 0.5 | 1295.80 | 1856.35422 | 0.70 | 0.4855 | 0.05 | -2353.04 | 4944.64 |
| TRTPN*ATPT | N Bel900 | 0 | Plac | 1 | 344.30 | 1856.35422 | 0.19 | 0.8529 | 0.05 | -3304.55 | 3993.14 |
| TRTPN*ATPT | N Bel900 | 0 | Plac | 2 | 4410.60 | 1856.35422 | 2.38 | 0.0179 | 0.05 | 761.75 | 8059.44 |
| TRTPN*ATPT | N Bel900 | 0 | Plac | 3 | 3996.53 | 1856.35422 | 2.15 | 0.0319 | 0.05 | 347.69 | 7645.37 |
| TRTPN*ATPT | N Bel900 | 0 | Plac | 4 | 2817.29 | 1856.35422 | 1.52 | 0.1299 | 0.05 | -831.55 | 6466.13 |
| TRTPN*ATPT | N Bel900 | 0.5 | Be1900 | 1 | 2819.47 | 1848.84422 | 1.52 | 0.1280 | 0.05 | -814.60 | 6453.55 |
| TRTPN*ATPT | N Bel900 | 0.5 | Be1900 | 2 | 4577.23 | 1848.84422 | 2.48 | 0.0137 | 0.05 | 943.15 | 8211.30 |
| TRTPN*ATPT | N Bel900 | 0.5 | Be1900 | 3 | 5257.49 | 1848.84422 | 2.84 | 0.0047 | 0.05 | 1623.42 | 8891.57 |
| TRTPN*ATPT | N Bel900 | 0.5 | Be1900 | 4 | 6305.98 | 1848.84422 | 3.41 | 0.0007 | 0.05 | 2671.91 | 9940.06 |
| TRTPN*ATPT | N Bel900 | 0.5 | Oxy30 | 0 | 2663.90 | 1922.09422 | 1.39 | 0.1665 | 0.05 | -1114.16 | 6441.96 |
| TRTPN*ATPT | N Bel900 | 0.5 | 0xy30 | 0.5 | 4936.05 | 1922.09422 | 2.57 | 0.0106 | 0.05 | 1157.99 | 8714.11 |
| TRTPN*ATPT | N Bel900 | 0.5 | Oxy30 | 1 | 6790.77 | 1883.48422 | 3.61 | 0.0003 | 0.05 | 3088.59 | 10493 |
| TRTPN*ATPT | N Bel900 | 0.5 | Oxy30 | 2 | 5935.62 | 1850.21422 | 3.21 | 0.0014 | 0.05 | 2298.84 | 9572.40 |
| TRTPN*ATPT | N Bel900 | 0.5 | Oxy30 | 3 | 4340.78 | 1850.21422 | 2.35 | 0.0194 | 0.05 | 704.00 | 7977.56 |
| TRTPN*ATPT | N Bel900 | 0.5 | Oxy30 | 4 | 4120.03 | 1850.21422 | 2.23 | 0.0265 | 0.05 | 483.25 | 7756.81 |
| TRTPN*ATPT | N Bel900 | 0.5 | Oxy60 | 0 | 4124.02 | 1886.21422 | 2.19 | 0.0293 | 0.05 | 416.48 | 7831.56 |
| TRTPN*ATPT | N Bel900 | 0.5 | Oxy60 | 0.5 | 6356.25 | 1886.21422 | 3.37 | 0.0008 | 0.05 | 2648.71 | 10064 |
| TRTPN*ATPT | N Bel900 | 0.5 | Oxy60 | 1 | 8447.78 | 1853.71422 | 4.56 | <.0001 | 0.05 | 4804.11 | 12091 |
| TRTPN*ATPT | N Bel900 | 0.5 | Oxy60 | 2 | 9440.33 | 1822.31422 | 5.18 | <.0001 | 0.05 | 5858.39 | 13022 |
| TRTPN*ATPT | N Bel900 | 0.5 | Oxy60 | 3 | 8773.51 | 1822.31422 | 4.81 | <.0001 | 0.05 | 5191.57 | 12355 |

Program: A Bio4.sas Created: 02APR2020 7:36 POSTLOCK 

# Appendix 16.1.9.2.4 Statistical Methods and Analysis Output Supporting Table 14.2.5 Supporting Table 14.2.4

# The Mixed Procedure

#### Parameter Code=MVMIPM

# Differences of Least Squares Means

| | D1 1 | | | | or bease i | oquares means | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | Planned | Analysis | | Analysis | | Standard | | | | | |
| Effect | (N) | (N) | (N) | Timepoint (N) | Estimate | Error DF t | 772 luo D | v > 1+1 | 7 l mh n | Lower | Ilnnor |
| TRTPN*ATPT | . , | ` , | ` , | | | 1822.31422 | 4.75 | <.0001 | | 5072.43 | Upper<br>12236 |
| | | 0.5 | Oxy60 | 4 | | | | | | | |
| TRTPN*ATPTI | | 0.5 | Plac | 0 | | 1822.11422 | 2.34 | 0.0200 | | 674.55 | 7837.64 |
| TRTPN*ATPTI | | 0.5 | Plac | 0.5 | | 1822.11422 | 1.50 | | | -851.07 | 6312.01 |
| TRTPN*ATPT | | 0.5 | Plac | 1 | | 1822.11422 | 0.98 | 0.3295 | | -1802.58 | 5360.51 |
| TRTPN*ATPT | | 0.5 | Plac | 2 | | 1822.11422 | 3.21 | 0.0014 | | 2263.72 | |
| TRTPN*ATPTI | | 0.5 | Plac | 3 | | 1822.11422 | 2.98 | | | 1849.65 | |
| TRTPN*ATPTI | 1Bel900 | 0.5 | Plac | 4 | 4251.96 | 1822.11422 | 2.33 | 0.0201 | 0.05 | 670.42 | 7833.51 |
| TRTPN*ATPT | 1Bel900 | 1 | Be1900 | 2 | 1757.75 | 1848.84422 | 0.95 | 0.3423 | 0.05 | -1876.32 | 5391.83 |
| TRTPN*ATPT | 1Bel900 | 1 | Be1900 | 3 | 2438.02 | 1848.84422 | 1.32 | 0.1880 | 0.05 | -1196.06 | 6072.09 |
| TRTPN*ATPTI | 1Bel900 | 1 | Be1900 | 4 | 3486.51 | 1848.84422 | 1.89 | 0.0600 | 0.05 | -147.57 | 7120.58 |
| TRTPN*ATPTI | NBe1900 | 1 | Oxy30 | 0 | -155.57 | 1922.09422 | -0.08 | 0.9355 | 0.05 | -3933.63 | 3622.49 |
| TRTPN*ATPT | NBe1900 | 1 | Oxy30 | 0.5 | 2116.58 | 1922.09422 | 1.10 | 0.2714 | 0.05 | -1661.48 | 5894.64 |
| TRTPN*ATPTI | NBel900 | 1 | Oxy30 | 1 | 3971.30 | 1883.48422 | 2.11 | 0.0356 | 0.05 | 269.12 | 7673.48 |
| TRTPN*ATPT | 1Bel900 | 1 | Oxy30 | 2 | 3116.15 | 1850.21422 | 1.68 | 0.0929 | 0.05 | -520.63 | 6752.93 |
| TRTPN*ATPT | 1Bel900 | 1 | 0xy30 | 3 | 1521.31 | 1850.21422 | 0.82 | 0.4114 | 0.05 | -2115.47 | 5158.09 |
| TRTPN*ATPT | 1Bel900 | 1 | Oxy30 | 4 | 1300.56 | 1850.21422 | 0.70 | 0.4825 | 0.05 | -2336.22 | 4937.34 |
| TRTPN*ATPTI | NBe1900 | 1 | Oxy60 | 0 | 1304.54 | 1886.21422 | 0.69 | 0.4896 | 0.05 | -2403.00 | 5012.08 |
| TRTPN*ATPT1 | NBel900 | 1 | Oxy60 | 0.5 | 3536.78 | 1886.21422 | 1.88 | 0.0615 | 0.05 | -170.76 | 7244.32 |
| TRTPN*ATPTI | NBe1900 | 1 | Oxy60 | 1 | 5628.30 | 1853.71422 | 3.04 | 0.0025 | 0.05 | 1984.64 | 9271.97 |
| TRTPN*ATPT | NBel900 | 1 | Oxy60 | 2 | 6620.86 | 1822.31422 | 3.63 | 0.0003 | 0.05 | 3038.91 | 10203 |
| TRTPN*ATPTI | JBel900 | 1 | Oxy60 | 3 | 5954.04 | 1822.31422 | 3.27 | 0.0012 | 0.05 | 2372.10 | |
| TRTPN*ATPT | JBe1900 | 1 | Oxy60 | 4 | | 1822.31422 | 3.20 | 0.0015 | | 2252.96 | 9416.84 |
| TRTPN*ATPT | | 1 | Plac | 0 | | 1822.11422 | 0.79 | 0.4309 | | | 5018.17 |
| TRTPN*ATPT | | 1 | Plac | 0.5 | | 1822.11 422 | -0.05 | 0.9611 | | -3670.55 | 3492.54 |
| TRTPN*ATPT | | 1 | Plac | 1 | | 1822.11422 | -0.57 | | | -4622.05 | |
| TIVILIN MILLI | v DCT 200 | _ | 1 1 4 0 | ± | 10.01.01 | 1022.11.422 | 0.57 | 0.5005 | 0.00 | 1022.00 | 2011.01 |

Program: A Bio4.sas Created: 02APR2020 7:36 POSTLOCK 

Appendix 16.1.9.2.4
Statistical Methods and Analysis Output Supporting Table 14.2.5
Supporting Table 14.2.4

# The Mixed Procedure

#### Parameter Code=MVMIPM

# Differences of Least Squares Means

| | Planned | Analysis | | Analvsis | or heade . | oquares neams | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | | _ | | Timepoint | | Standard | | | | | |
| Effect | (N) | (N) | (N) | (N) | Estimate | Error DFt | Value P | r > t | Alpha | Lower | Upper |
| TRTPN*ATPT | N Bel900 | 1 | Plac | 2 | 3025.79 | 1822.11422 | 1.66 | 0.0975 | 0.05 - | 555.75 | 6607.34 |
| TRTPN*ATPT | NBe1900 | 1 | Plac | 3 | 2611.72 | 1822.11422 | 1.43 | 0.1525 | 0.05 - | 969.82 | 6193.27 |
| TRTPN*ATPT | NBe1900 | 1 | Plac | 4 | 1432.49 | 1822.11422 | 0.79 | 0.4322 | 0.05-2 | 149.05 | 5014.03 |
| TRTPN*ATPTI | N Bel900 | 2 | Be1900 | 3 | 680.26 | 1848.84422 | 0.37 | 0.7131 | 0.05-2 | 953.81 | 4314.34 |
| TRTPN*ATPT | NBe1900 | 2 | Be1900 | 4 | 1728.75 | 1848.84422 | 0.94 | 0.3503 | 0.05-1 | 905.32 | 5362.83 |
| TRTPN*ATPT | NBe1900 | 2 | Oxy30 | 0 | -1913.32 | 1922.09422 | -1.00 | 0.3201 | 0.05-5 | 691.38 | 1864.73 |
| TRTPN*ATPTI | N Bel900 | 2 | Oxy30 | 0.5 | 358.82 | 1922.09422 | 0.19 | 0.8520 | 0.05 -3 | 419.24 | 4136.88 |
| TRTPN*ATPTI | N Bel900 | 2 | Oxy30 | 1 | 2213.54 | 1883.48422 | 1.18 | 0.2406 | 0.05-1 | 488.64 | 5915.72 |
| TRTPN*ATPT | N Bel900 | 2 | Oxy30 | 2 | 1358.39 | 1850.21422 | 0.73 | 0.4632 | 0.05 -2 | 278.39 | 4995.17 |
| TRTPN*ATPT | N Bel900 | 2 | Oxy30 | 3 | -236.44 | 1850.21422 | -0.13 | 0.8984 | 0.05 -3 | 873.23 | 3400.34 |
| TRTPN*ATPT | N Bel900 | 2 | Oxy30 | 4 | -457.20 | 1850.21422 | -0.25 | 0.8049 | 0.05-4 | 093.98 | 3179.58 |
| TRTPN*ATPTI | N Bel900 | 2 | Oxy60 | 0 | -453.21 | 1886.21422 | -0.24 | 0.8102 | 0.05-4 | 160.75 | 3254.33 |
| TRTPN*ATPT | NBe1900 | 2 | Oxy60 | 0.5 | 1779.02 | 1886.21422 | 0.94 | 0.3461 | 0.05-1 | 928.51 | 5486.56 |
| TRTPN*ATPT | NBe1900 | 2 | Oxy60 | 1 | 3870.55 | 1853.71422 | 2.09 | 0.0374 | 0.05 | 226.89 | 7514.21 |
| TRTPN*ATPT | N Bel900 | 2 | Oxy60 | 2 | 4863.10 | 1822.31422 | 2.67 | 0.0079 | 0.05 1 | 281.16 | 8445.04 |
| TRTPN*ATPT | N Bel900 | 2 | Oxy60 | 3 | 4196.29 | 1822.31422 | 2.30 | 0.0218 | 0.05 | 614.34 | 7778.23 |
| TRTPN*ATPT | N Bel900 | 2 | Oxy60 | 4 | 4077.15 | 1822.31422 | 2.24 | 0.0258 | 0.05 | 495.20 | 7659.09 |
| TRTPN*ATPTI | N Bel900 | 2 | Plac | 0 | -321.13 | 1822.11422 | -0.18 | 0.8602 | 0.05 -3 | 902.68 | 3260.41 |
| TRTPN*ATPT | NBe1900 | 2 | Plac | 0.5 | -1846.76 | 1822.11422 | -1.01 | 0.3114 | 0.05-5 | 428.30 | 1734.79 |
| TRTPN*ATPT | NBe1900 | 2 | Plac | 1 | -2798.26 | 1822.11422 | -1.54 | 0.1254 | 0.05-6 | 379.80 | 783.28 |
| TRTPN*ATPTI | N Bel900 | 2 | Plac | 2 | 1268.04 | 1822.11422 | 0.70 | 0.4869 | 0.05 -2 | 313.50 | 4849.58 |
| TRTPN*ATPT | NBe1900 | 2 | Plac | 3 | 853.97 | 1822.11422 | 0.47 | 0.6395 | 0.05 -2 | 727.57 | 4435.51 |
| TRTPN*ATPTI | N Bel900 | 2 | Plac | 4 | -325.26 | 1822.11422 | -0.18 | 0.8584 | 0.05 -3 | 906.81 | 3256.28 |
| TRTPN*ATPTI | N Bel900 | 3 | Be1900 | 4 | 1048.49 | 1848.84422 | 0.57 | 0.5709 | 0.05 -2 | 585.59 | 4682.56 |
| TRTPN*ATPTI | N Bel900 | 3 | Oxy30 | 0 | -2593.59 | 1922.09422 | -1.35 | 0.1779 | 0.05-6 | 371.65 | 1184.47 |

Program: A\_Bio4.sas Created: 02APR2020 7:36 POSTLOCK 

# Appendix 16.1.9.2.4 Statistical Methods and Analysis Output Supporting Table 14.2.5 Supporting Table 14.2.4

# The Mixed Procedure

#### Parameter Code=MVMIPM

# Differences of Least Squares Means

| | Planned | Analysis | | Analvsis | or bease . | squares means | | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| | Treatment | 4 | | t Timepoint | | Standard | | | | |
| Effect | (N) | (N) | (N) | (N) | Estimate | Error DFt | Value P | r > t | Alpha Lower | Upper |
| TRTPN*ATPT | N Bel900 | 3 | Oxy30 | 0.5 | -321.44 | 1922.09422 | -0.17 | 0.8673 | 0.05-4099.50 | 3456.62 |
| TRTPN*ATPT | N Bel900 | 3 | Oxy30 | 1 | 1533.28 | 1883.48422 | 0.81 | 0.4161 | 0.05-2168.90 | 5235.46 |
| TRTPN*ATPT | N Bel900 | 3 | Oxy30 | 2 | 678.13 | 1850.21422 | 0.37 | 0.7142 | 0.05-2958.65 | 4314.91 |
| TRTPN*ATPT | N Bel900 | 3 | Oxy30 | 3 | -916.71 | 1850.21422 | -0.50 | 0.6205 | 0.05-4553.49 | 2720.07 |
| TRTPN*ATPT | N Bel900 | 3 | Oxy30 | 4 | -1137.46 | 1850.21422 | -0.61 | 0.5390 | 0.05-4774.24 | 2499.32 |
| TRTPN*ATPT | N Bel900 | 3 | Oxy60 | 0 | -1133.47 | 1886.21422 | -0.60 | 0.5482 | 0.05-4841.01 | 2574.06 |
| TRTPN*ATPT | N Bel900 | 3 | Oxy60 | 0.5 | 1098.76 | 1886.21422 | 0.58 | 0.5605 | 0.05-2608.78 | 4806.30 |
| TRTPN*ATPT | N Bel900 | 3 | Oxy60 | 1 | 3190.29 | 1853.71422 | 1.72 | 0.0860 | 0.05 -453.38 | 6833.95 |
| TRTPN*ATPT | N Bel900 | 3 | Oxy60 | 2 | 4182.84 | 1822.31422 | 2.30 | 0.0222 | 0.05 600.89 | 7764.78 |
| TRTPN*ATPT | N Bel900 | 3 | Oxy60 | 3 | 3516.02 | 1822.31422 | 1.93 | 0.0543 | 0.05-65.9217 | 7097.96 |
| TRTPN*ATPT | N Bel900 | 3 | Oxy60 | 4 | 3396.88 | 1822.31422 | 1.86 | 0.0630 | 0.05 -185.06 | 6978.83 |
| TRTPN*ATPT | N Bel900 | 3 | Plac | 0 | -1001.40 | 1822.11422 | -0.55 | 0.5829 | 0.05-4582.94 | 2580.15 |
| TRTPN*ATPT | N Bel900 | 3 | Plac | 0.5 | -2527.02 | 1822.11422 | -1.39 | 0.1662 | 0.05-6108.57 | 1054.52 |
| TRTPN*ATPT | N Bel900 | 3 | Plac | 1 | -3478.52 | 1822.11422 | -1.91 | 0.0569 | 0.05-7060.07 | 103.02 |
| TRTPN*ATPT | N Bel900 | 3 | Plac | 2 | 587.78 | 1822.11422 | 0.32 | 0.7472 | 0.05-2993.77 | 4169.32 |
| TRTPN*ATPT | N Bel900 | 3 | Plac | 3 | 173.71 | 1822.11422 | 0.10 | 0.9241 | 0.05-3407.84 | 3755.25 |
| TRTPN*ATPT | N Bel900 | 3 | Plac | 4 | | 1822.11422 | -0.55 | 0.5813 | 0.05-4587.07 | |
| TRTPN*ATPT | N Bel900 | 4 | 0xy30 | 0 | -3642.08 | 1922.09422 | -1.89 | 0.0588 | 0.05-7420.14 | 135.98 |
| TRTPN*ATPT | N Bel900 | 4 | 0xy30 | 0.5 | -1369.93 | 1922.09422 | -0.71 | 0.4764 | 0.05-5147.99 | 2408.13 |
| TRTPN*ATPT | N Bel900 | 4 | 0xy30 | 1 | 484.79 | 1883.48422 | 0.26 | 0.7970 | 0.05-3217.39 | 4186.97 |
| TRTPN*ATPT | N Bel900 | 4 | Oxy30 | 2 | -370.36 | 1850.21422 | -0.20 | 0.8414 | 0.05-4007.14 | 3266.42 |
| TRTPN*ATPT | N Bel900 | 4 | 0xy30 | 3 | -1965.20 | 1850.21422 | -1.06 | 0.2888 | 0.05-5601.98 | 1671.58 |
| TRTPN*ATPT | N Bel900 | 4 | 0xy30 | 4 | -2185.95 | 1850.21422 | -1.18 | 0.2381 | | |
| TRTPN*ATPT | N Bel900 | 4 | Oxy60 | 0 | -2181.96 | 1886.21422 | -1.16 | 0.2480 | 0.05-5889.50 | 1525.58 |
| TRTPN*ATPT | N Bel900 | 4 | Oxy60 | 0.5 | 50.2714 | 1886.21422 | 0.03 | 0.9787 | 0.05-3657.27 | 3757.81 |

Program: A Bio4.sas Created: 02APR2020 7:36 POSTLOCK 

# Appendix 16.1.9.2.4 Statistical Methods and Analysis Output Supporting Table 14.2.5 Supporting Table 14.2.4

# The Mixed Procedure

#### Parameter Code=MVMIPM

# Differences of Least Squares Means

| | _, , | | | | or heade i | oquares means | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | Planned | Analysis | | Analysis | | Q. 1 1 | | | | | |
| | | - | Treatment | - | | Standard | _ | | | | |
| Effect | (N) | (N) | (N) | (N) | Estimate | Error DFt | | | | Lower | Upper |
| TRTPN*ATPTN | Be1900 | 4 | Oxy60 | 1 | 2141.80 | 1853.71422 | 1.16 | 0.2486 | 0.05-15 | 01.87 | 5785.46 |
| TRTPN*ATPTN | Be1900 | 4 | Oxy60 | 2 | 3134.35 | 1822.31422 | 1.72 | 0.0862 | 0.05 -4 | 47.60 | 6716.29 |
| TRTPN*ATPTN | Be1900 | 4 | Oxy60 | 3 | 2467.53 | 1822.31422 | 1.35 | 0.1764 | 0.05-11 | 14.41 | 6049.48 |
| TRTPN*ATPTN | Be1900 | 4 | Oxy60 | 4 | 2348.39 | 1822.31422 | 1.29 | 0.1982 | 0.05-123 | 33.55 | 5930.34 |
| TRTPN*ATPTN | Be1900 | 4 | Plac | 0 | -2049.89 | 1822.11422 | -1.13 | 0.2612 | 0.05-563 | 31.43 | 1531.66 |
| TRTPN*ATPTN | Be1900 | 4 | Plac | 0.5 | -3575.51 | 1822.11422 | -1.96 | 0.0504 | 0.05-71 | 57.06 | 6.0322 |
| TRTPN*ATPTN | Be1900 | 4 | Plac | 1 | -4527.01 | 1822.11422 | -2.48 | 0.0134 | 0.05-81 | 08.56 | -945.47 |
| TRTPN*ATPTN | Be1900 | 4 | Plac | 2 | -460.71 | 1822.11422 | -0.25 | 0.8005 | 0.05-40 | 42.26 | 3120.83 |
| TRTPN*ATPTN | Be1900 | 4 | Plac | 3 | -874.78 | 1822.11422 | -0.48 | 0.6314 | 0.05-44 | 56.33 | 2706.76 |
| TRTPN*ATPTN | Be1900 | 4 | Plac | 4 | -2054.02 | 1822.11422 | -1.13 | 0.2603 | 0.05-563 | 35.56 | 1527.53 |
| TRTPN*ATPTN | Oxy30 | 0 | 0xy30 | 0.5 | 2272.15 | 1985.97422 | 1.14 | 0.2532 | 0.05-163 | 31.47 | 6175.77 |
| TRTPN*ATPTN | Oxy30 | 0 | 0xy30 | 1 | 4126.87 | 1951.67422 | 2.11 | 0.0351 | 0.05 2 | 90.66 | 7963.08 |
| TRTPN*ATPTN | Oxy30 | 0 | 0xy30 | 2 | 3271.72 | 1922.33422 | 1.70 | 0.0895 | 0.05 -50 | 06.82 | 7050.26 |
| TRTPN*ATPTN | Oxy30 | 0 | 0xy30 | 3 | 1676.88 | 1922.33422 | 0.87 | 0.3835 | 0.05-21 | 01.66 | 5455.42 |
| TRTPN*ATPTN | Oxy30 | 0 | 0xy30 | 4 | 1456.13 | 1922.33422 | 0.76 | 0.4492 | 0.05-23 | 22.41 | 5234.66 |
| TRTPN*ATPTN | Oxy30 | 0 | Oxy60 | 0 | 1460.11 | 1958.61422 | 0.75 | 0.4564 | 0.05-23 | 39.73 | 5309.95 |
| TRTPN*ATPTN | Oxy30 | 0 | Oxy60 | 0.5 | 3692.35 | 1958.61422 | 1.89 | 0.0601 | 0.05 -1 | 57.49 | 7542.19 |
| TRTPN*ATPTN | Oxy30 | 0 | Oxy60 | 1 | 5783.87 | 1927.80422 | 3.00 | 0.0029 | 0.05 19 | 94.59 | 9573.16 |
| TRTPN*ATPTN | Oxy30 | 0 | Oxy60 | 2 | 6776.43 | 1896.92422 | 3.57 | 0.0004 | 0.05 30 | 47.84 | 10505 |
| TRTPN*ATPTN | Oxy30 | 0 | Oxy60 | 3 | 6109.61 | 1896.92422 | 3.22 | 0.0014 | 0.05 23 | 31.03 | 9838.19 |
| TRTPN*ATPTN | Oxy30 | 0 | Oxy60 | 4 | 5990.47 | 1896.92422 | 3.16 | 0.0017 | 0.05 22 | 61.89 | 9719.05 |
| TRTPN*ATPTN | Oxy30 | 0 | Plac | 0 | 1592.19 | 1895.07422 | 0.84 | 0.4013 | 0.05-21 | 32.76 | 5317.15 |
| TRTPN*ATPTN | Oxy30 | 0 | Plac | 0.5 | 66.5664 | 1895.07422 | 0.04 | 0.9720 | 0.05-36 | 58.39 | 3791.52 |
| TRTPN*ATPTN | Oxy30 | 0 | Plac | 1 | -884.94 | 1895.07422 | -0.47 | 0.6408 | 0.05-46 | 09.89 | 2840.02 |
| TRTPN*ATPTN | Oxy30 | 0 | Plac | 2 | 3181.36 | 1895.07422 | 1.68 | 0.0939 | 0.05 -5 | 43.59 | 6906.32 |

Program: A\_Bio4.sas Created: 02APR2020 7:36 POSTLOCK

# Appendix 16.1.9.2.4 Statistical Methods and Analysis Output Supporting Table 14.2.5 Supporting Table 14.2.4

# The Mixed Procedure

#### Parameter Code=MVMIPM

# Differences of Least Squares Means

| | Planned | Analysis | | Analysis | or hease . | oquares neams | | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| | Treatment | 4 | | t Timepoint | | Standard | | | | |
| Effect | (N) | (N) | (N) | (N) | Estimate | Error DFt | Value P | r > t | Alpha Lower | Upper |
| TRTPN*ATPT | M Oxy30 | 0 | Plac | 3 | 2767.29 | 1895.07422 | 1.46 | 0.1450 | 0.05 -957.66 | 6492.25 |
| TRTPN*ATPT | NOxy30 | 0 | Plac | 4 | 1588.06 | 1895.07422 | 0.84 | 0.4025 | 0.05-2136.89 | 5313.01 |
| TRTPN*ATPT | NOxy30 | 0.5 | Oxy30 | 1 | 1854.72 | 1951.67422 | 0.95 | 0.3425 | 0.05-1981.49 | 5690.93 |
| TRTPN*ATPT | NOxy30 | 0.5 | Oxy30 | 2 | 999.57 | 1922.33422 | 0.52 | 0.6034 | 0.05-2778.97 | 4778.11 |
| TRTPN*ATPT | NOxy30 | 0.5 | Oxy30 | 3 | -595.27 | 1922.33422 | -0.31 | 0.7570 | 0.05-4373.81 | 3183.27 |
| TRTPN*ATPT | NOxy30 | 0.5 | Oxy30 | 4 | -816.02 | 1922.33422 | -0.42 | 0.6714 | 0.05-4594.56 | 2962.52 |
| TRTPN*ATPT | 4 | 0.5 | Oxy60 | 0 | -812.03 | 1958.61422 | -0.41 | 0.6786 | 0.05-4661.87 | 3037.81 |
| TRTPN*ATPT | NOxy30 | 0.5 | Oxy60 | 0.5 | 1420.20 | 1958.61422 | 0.73 | 0.4688 | 0.05-2429.64 | 5270.04 |
| TRTPN*ATPT | NOxy30 | 0.5 | Oxy60 | 1 | 3511.73 | 1927.80422 | 1.82 | 0.0692 | 0.05 -277.56 | 7301.02 |
| TRTPN*ATPT | NOxy30 | 0.5 | Oxy60 | 2 | 4504.28 | 1896.92422 | 2.37 | 0.0180 | 0.05 775.69 | 8232.86 |
| TRTPN*ATPT | NOxy30 | 0.5 | Oxy60 | 3 | 3837.46 | 1896.92422 | 2.02 | 0.0437 | 0.05 108.88 | 7566.04 |
| TRTPN*ATPT | NOxy30 | 0.5 | Oxy60 | 4 | 3718.32 | 1896.92422 | 1.96 | 0.0506 | 0.05-10.2601 | 7446.91 |
| TRTPN*ATPT | NOxy30 | 0.5 | Plac | 0 | -679.96 | 1895.07422 | -0.36 | 0.7199 | 0.05-4404.91 | 3045.00 |
| TRTPN*ATPT | NOxy30 | 0.5 | Plac | 0.5 | -2205.58 | 1895.07422 | -1.16 | 0.2451 | 0.05-5930.54 | 1519.37 |
| TRTPN*ATPT | NOxy30 | 0.5 | Plac | 1 | -3157.08 | 1895.07422 | -1.67 | 0.0965 | 0.05-6882.04 | 567.87 |
| TRTPN*ATPT | NOxy30 | 0.5 | Plac | 2 | 909.22 | 1895.07422 | 0.48 | 0.6316 | 0.05-2815.74 | 4634.17 |
| TRTPN*ATPT | NOxy30 | 0.5 | Plac | 3 | 495.15 | 1895.07422 | 0.26 | 0.7940 | 0.05-3229.81 | 4220.10 |
| TRTPN*ATPT | NOxy30 | 0.5 | Plac | 4 | -684.09 | 1895.07422 | -0.36 | 0.7183 | 0.05-4409.04 | 3040.87 |
| TRTPN*ATPT | NOxy30 | 1 | Oxy30 | 2 | -855.15 | 1882.89422 | -0.45 | 0.6499 | 0.05-4556.16 | 2845.86 |
| TRTPN*ATPT | NOxy30 | 1 | Oxy30 | 3 | -2449.99 | 1882.89422 | -1.30 | 0.1939 | 0.05-6150.99 | 1251.02 |
| TRTPN*ATPT | NOxy30 | 1 | Oxy30 | 4 | -2670.74 | 1882.89422 | -1.42 | 0.1568 | 0.05-6371.75 | 1030.26 |
| TRTPN*ATPT | NOxy30 | 1 | Oxy60 | 0 | -2666.75 | 1920.15422 | -1.39 | 0.1656 | 0.05-6441.00 | 1107.49 |
| TRTPN*ATPTI | NOxy30 | 1 | Oxy60 | 0.5 | -434.52 | 1920.15422 | -0.23 | 0.8211 | 0.05-4208.76 | 3339.72 |
| TRTPN*ATPTI | NOxy30 | 1 | Oxy60 | 1 | 1657.01 | 1888.02422 | 0.88 | 0.3806 | 0.05-2054.09 | 5368.10 |
| TRTPN*ATPTI | NOxy30 | 1 | Oxy60 | 2 | 2649.56 | 1856.88422 | 1.43 | 0.1544 | 0.05-1000.32 | 6299.43 |

Program: A Bio4.sas Created: 02APR2020 7:36 POSTLOCK 

# Appendix 16.1.9.2.4 Statistical Methods and Analysis Output Supporting Table 14.2.5 Supporting Table 14.2.4

# The Mixed Procedure

#### Parameter Code=MVMIPM

# Differences of Least Squares Means

| | Planned | Analysis | | Analysis | or bease . | oquares neans | | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| | Treatment | _ | | t Timepoint | | Standard | | | | |
| Effect | (N) | (N) | (N) | (N) | Estimate | Error DFt | Value P | r > t | Alpha Lower | Upper |
| TRTPN*ATPT | 10xy30 | 1 | Oxy60 | 3 | 1982.74 | 1856.88422 | 1.07 | 0.2862 | 0.05-1667.14 | 5632.62 |
| TRTPN*ATPT | N 0xy30 | 1 | Oxy60 | 4 | 1863.60 | 1856.88422 | 1.00 | 0.3161 | 0.05-1786.27 | 5513.48 |
| TRTPN*ATPT | N 0xy30 | 1 | Plac | 0 | -2534.68 | 1855.92422 | -1.37 | 0.1728 | 0.05-6182.68 | 1113.32 |
| TRTPN*ATPTI | N 0xy30 | 1 | Plac | 0.5 | -4060.30 | 1855.92422 | -2.19 | 0.0292 | 0.05-7708.30 | -412.30 |
| TRTPN*ATPTI | N 0xy30 | 1 | Plac | 1 | -5011.80 | 1855.92422 | -2.70 | 0.0072 | 0.05-8659.81 | -1363.80 |
| TRTPN*ATPTI | N 0xy30 | 1 | Plac | 2 | -945.50 | 1855.92422 | -0.51 | 0.6107 | 0.05-4593.51 | 2702.50 |
| TRTPN*ATPTI | N 0xy30 | 1 | Plac | 3 | -1359.57 | 1855.92422 | -0.73 | 0.4642 | 0.05-5007.57 | 2288.43 |
| TRTPN*ATPTI | N 0xy30 | 1 | Plac | 4 | -2538.81 | 1855.92422 | -1.37 | 0.1721 | 0.05-6186.81 | 1109.19 |
| TRTPN*ATPT | 0 EyxO | 2 | Oxy30 | 3 | -1594.84 | 1848.84422 | -0.86 | 0.3888 | 0.05-5228.91 | 2039.24 |
| TRTPN*ATPTI | 0 EyxO V | 2 | Oxy30 | 4 | -1815.59 | 1848.84422 | -0.98 | 0.3267 | 0.05-5449.67 | 1818.48 |
| TRTPN*ATPTI | 0 EyxO V | 2 | Oxy60 | 0 | -1811.60 | 1886.98422 | -0.96 | 0.3376 | 0.05-5520.66 | 1897.45 |
| TRTPN*ATPTI | 4 | 2 | Oxy60 | 0.5 | 420.63 | 1886.98422 | 0.22 | 0.8237 | 0.05-3288.43 | 4129.69 |
| TRTPN*ATPT | 0 EyxO | 2 | Oxy60 | 1 | 2512.16 | 1853.66422 | 1.36 | 0.1761 | 0.05-1131.39 | 6155.71 |
| TRTPN*ATPT | 0 EyxO | 2 | Oxy60 | 2 | 3504.71 | 1822.29422 | 1.92 | 0.0551 | 0.05-77.1821 | 7086.60 |
| TRTPN*ATPT | 0 EyxO | 2 | Oxy60 | 3 | 2837.89 | 1822.29422 | 1.56 | 0.1201 | 0.05 -744.00 | 6419.78 |
| TRTPN*ATPT | 0 EyxO | 2 | Oxy60 | 4 | 2718.75 | 1822.29422 | 1.49 | 0.1365 | 0.05 -863.14 | 6300.64 |
| TRTPN*ATPT | 0 EyxO | 2 | Plac | 0 | -1679.53 | 1822.16422 | -0.92 | 0.3572 | 0.05-5261.16 | 1902.11 |
| TRTPN*ATPTI | 0 EyxO V | 2 | Plac | 0.5 | -3205.15 | 1822.16422 | -1.76 | 0.0793 | 0.05-6786.79 | 376.49 |
| TRTPN*ATPT | 0 EyxO | 2 | Plac | 1 | -4156.65 | 1822.16422 | -2.28 | 0.0230 | 0.05-7738.29 | -575.02 |
| TRTPN*ATPT | 0 EyxO | 2 | Plac | 2 | -90.3546 | 1822.16422 | -0.05 | 0.9605 | 0.05-3671.99 | 3491.28 |
| TRTPN*ATPTI | 0 EyxO V | 2 | Plac | 3 | -504.42 | 1822.16422 | -0.28 | 0.7820 | 0.05-4086.06 | 3077.21 |
| TRTPN*ATPT | 0 EyxO | 2 | Plac | 4 | -1683.66 | 1822.16422 | -0.92 | 0.3560 | 0.05-5265.30 | 1897.98 |
| TRTPN*ATPT | 0 EyxO | 3 | Oxy30 | 4 | -220.75 | 1848.84422 | -0.12 | 0.9050 | 0.05-3854.83 | 3413.32 |
| TRTPN*ATPTI | NOxy30 | 3 | Oxy60 | 0 | -216.77 | 1886.98422 | -0.11 | 0.9086 | 0.05-3925.82 | 3492.29 |
| TRTPN*ATPTI | 0 EyxO | 3 | Oxy60 | 0.5 | 2015.47 | 1886.98422 | 1.07 | 0.2861 | 0.05-1693.59 | 5724.53 |

Program: A Bio4.sas Created: 02APR2020 7:36 POSTLOCK 

# Appendix 16.1.9.2.4 Statistical Methods and Analysis Output Supporting Table 14.2.5 Supporting Table 14.2.4

# The Mixed Procedure

#### Parameter Code=MVMIPM

# Differences of Least Squares Means

| | | | | | or heade . | oquares means | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | Planned | Analysis | | Analysis | | Q1 1 1 | | | | | |
| T. C. C | | - | Treatment | - | | Standard | | | | _ | |
| Effect | (N) | (N) | (N) | (N) | Estimate | Error DF t | | | | Lower | Upper |
| TRTPN*ATPTN | - | 3 | Oxy60 | 1 | | 1853.66422 | 2.22 | 0.0273 | | 463.44 | 7750.55 |
| TRTPN*ATPTN | Oxy30 | 3 | Oxy60 | 2 | 5099.55 | 1822.29422 | 2.80 | 0.0054 | 0.05 | 1517.66 | 8681.43 |
| TRTPN*ATPTN | Oxy30 | 3 | Oxy60 | 3 | 4432.73 | 1822.29422 | 2.43 | 0.0154 | 0.05 | 850.84 | 8014.62 |
| TRTPN*ATPTN | Oxy30 | 3 | Oxy60 | 4 | 4313.59 | 1822.29422 | 2.37 | 0.0184 | 0.05 | 731.70 | 7895.48 |
| TRTPN*ATPTN | Oxy30 | 3 | Plac | 0 | -84.6873 | 1822.16422 | -0.05 | 0.9630 | 0.05- | -3666.33 | 3496.95 |
| TRTPN*ATPTN | Oxy30 | 3 | Plac | 0.5 | -1610.31 | 1822.16422 | -0.88 | 0.3773 | 0.05- | -5191.95 | 1971.32 |
| TRTPN*ATPTN | Oxy30 | 3 | Plac | 1 | -2561.82 | 1822.16422 | -1.41 | 0.1605 | 0.05- | -6143.45 | 1019.82 |
| TRTPN*ATPTN | Oxy30 | 3 | Plac | 2 | 1504.48 | 1822.16422 | 0.83 | 0.4095 | 0.05- | -2077.15 | 5086.12 |
| TRTPN*ATPTN | Oxy30 | 3 | Plac | 3 | 1090.41 | 1822.16422 | 0.60 | 0.5499 | 0.05- | -2491.22 | 4672.05 |
| TRTPN*ATPTN | Oxy30 | 3 | Plac | 4 | -88.8197 | 1822.16422 | -0.05 | 0.9611 | 0.05- | -3670.46 | 3492.82 |
| TRTPN*ATPTN | Oxy30 | 4 | Oxy60 | 0 | 3.9867 | 1886.98422 | 0.00 | 0.9983 | 0.05- | -3705.07 | 3713.04 |
| TRTPN*ATPTN | Oxy30 | 4 | Oxy60 | 0.5 | 2236.22 | 1886.98422 | 1.19 | 0.2367 | 0.05- | -1472.83 | 5945.28 |
| TRTPN*ATPTN | Oxy30 | 4 | Oxy60 | 1 | 4327.75 | 1853.66422 | 2.33 | 0.0200 | 0.05 | 684.20 | 7971.30 |
| TRTPN*ATPTN | Oxy30 | 4 | Oxy60 | 2 | 5320.30 | 1822.29422 | 2.92 | 0.0037 | 0.05 | 1738.41 | 8902.19 |
| TRTPN*ATPTN | Oxy30 | 4 | Oxy60 | 3 | 4653.48 | 1822.29422 | 2.55 | 0.0110 | 0.05 | 1071.59 | 8235.37 |
| TRTPN*ATPTN | Oxy30 | 4 | Oxy60 | 4 | 4534.34 | 1822.29422 | 2.49 | 0.0132 | 0.05 | 952.45 | 8116.23 |
| TRTPN*ATPTN | Oxy30 | 4 | Plac | 0 | 136.07 | 1822.16422 | 0.07 | 0.9405 | 0.05- | -3445.57 | 3717.70 |
| TRTPN*ATPTN | Oxy30 | 4 | Plac | 0.5 | -1389.56 | 1822.16422 | -0.76 | 0.4461 | 0.05- | -4971.20 | 2192.08 |
| TRTPN*ATPTN | Oxy30 | 4 | Plac | 1 | -2341.06 | 1822.16422 | -1.28 | 0.1996 | 0.05- | -5922.70 | 1240.57 |
| TRTPN*ATPTN | Oxy30 | 4 | Plac | 2 | 1725.24 | 1822.16422 | 0.95 | 0.3443 | 0.05- | -1856.40 | 5306.87 |
| TRTPN*ATPTN | Oxy30 | 4 | Plac | 3 | 1311.17 | 1822.16422 | 0.72 | 0.4722 | 0.05- | -2270.47 | 4892.81 |
| TRTPN*ATPTN | Oxy30 | 4 | Plac | 4 | 131.93 | 1822.16422 | 0.07 | 0.9423 | 0.05- | -3449.71 | 3713.57 |
| TRTPN*ATPTN | Oxy60 | 0 | Oxy60 | 0.5 | 2232.24 | 1913.73422 | 1.17 | 0.2441 | 0.05- | -1529.39 | 5993.86 |
| TRTPN*ATPTN | Oxy60 | 0 | Oxy60 | 1 | 4323.76 | 1885.44422 | 2.29 | 0.0223 | 0.05 | 617.73 | 8029.79 |
| TRTPN*ATPTN | Oxy60 | 0 | Oxy60 | 2 | 5316.31 | 1855.33422 | 2.87 | 0.0044 | 0.05 | 1669.47 | 8963.15 |

Program: A Bio4.sas Created: 02APR2020 7:36 POSTLOCK 

Appendix 16.1.9.2.4
Statistical Methods and Analysis Output Supporting Table 14.2.5
Supporting Table 14.2.4

# The Mixed Procedure

#### Parameter Code=MVMIPM

# Differences of Least Squares Means

| Planned | Analysis | Planned | Analysis | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| Treatmen | t Timepoint | t Treatmen | t Timepoint | | Standard | | | | | |
| (N) | (N) | (N) | (N) | Estimate | Error DFt | Value P | r > t | Alpha | Lower | Upper |
| N Оху60 | 0 | Oxy60 | 3 | 4649.50 | 1855.33422 | 2.51 | 0.0126 | 0.05 | 1002.66 | 8296.33 |
| N Оху60 | 0 | Oxy60 | 4 | 4530.36 | 1855.33422 | 2.44 | 0.0150 | 0.05 | 883.52 | 8177.20 |
| NOxy60 | 0 | Plac | 0 | 132.08 | 1856.77422 | 0.07 | 0.9433 | 0.05 | -3517.59 | 3781.75 |
| N Оху60 | 0 | Plac | 0.5 | -1393.55 | 1856.77422 | -0.75 | 0.4534 | 0.05 | -5043.22 | 2256.12 |
| NOxy60 | 0 | Plac | 1 | -2345.05 | 1856.77422 | -1.26 | 0.2073 | 0.05 | -5994.72 | 1304.62 |
| и Охуб0 | 0 | Plac | 2 | 1721.25 | 1856.77422 | 0.93 | 0.3544 | 0.05 | -1928.42 | 5370.92 |
| N Оху60 | 0 | Plac | 3 | 1307.18 | 1856.77422 | 0.70 | 0.4818 | 0.05 | -2342.49 | 4956.85 |
| NOxy60 | 0 | Plac | 4 | 127.95 | 1856.77422 | 0.07 | 0.9451 | 0.05 | -3521.72 | 3777.62 |
| N Оху60 | 0.5 | Oxy60 | 1 | 2091.53 | 1885.44422 | 1.11 | 0.2679 | 0.05 | -1614.50 | 5797.55 |
| N Оху60 | 0.5 | Oxy60 | 2 | 3084.08 | 1855.33422 | 1.66 | 0.0972 | 0.05 | -562.76 | 6730.91 |
| N Оху60 | 0.5 | Oxy60 | 3 | 2417.26 | 1855.33422 | 1.30 | 0.1933 | 0.05 | -1229.58 | 6064.10 |
| NOxy60 | 0.5 | Oxy60 | 4 | 2298.12 | 1855.33422 | 1.24 | 0.2162 | 0.05 | -1348.72 | 5944.96 |
| N Оху60 | 0.5 | Plac | 0 | -2100.16 | 1856.77422 | -1.13 | 0.2587 | 0.05 | -5749.83 | 1549.51 |
| N Оху60 | 0.5 | Plac | 0.5 | -3625.78 | 1856.77422 | -1.95 | 0.0515 | 0.05 | -7275.45 | 23.8874 |
| NOxy60 | 0.5 | Plac | 1 | -4577.29 | 1856.77422 | -2.47 | 0.0141 | 0.05 | -8226.96 | -927.62 |
| NOxy60 | 0.5 | Plac | 2 | -510.99 | 1856.77422 | -0.28 | 0.7833 | 0.05 | -4160.66 | 3138.68 |
| N Оху60 | 0.5 | Plac | 3 | -925.05 | 1856.77422 | -0.50 | 0.6186 | 0.05 | -4574.72 | 2724.62 |
| NOxy60 | 0.5 | Plac | 4 | -2104.29 | 1856.77422 | -1.13 | 0.2577 | 0.05 | -5753.96 | 1545.38 |
| N Оху60 | 1 | Oxy60 | 2 | 992.55 | 1820.88422 | 0.55 | 0.5860 | 0.05 | -2586.57 | 4571.67 |
| NOxy60 | 1 | Oxy60 | 3 | 325.74 | 1820.88422 | 0.18 | 0.8581 | 0.05 | -3253.39 | 3904.86 |
| и Охуб0 | 1 | Oxy60 | 4 | 206.60 | 1820.88422 | 0.11 | 0.9097 | 0.05 | -3372.52 | 3785.72 |
| NOxy60 | 1 | Plac | 0 | -4191.68 | 1822.94422 | -2.30 | 0.0220 | 0.05 | -7774.85 | -608.51 |
| NOxy60 | 1 | Plac | 0.5 | -5717.31 | 1822.94422 | -3.14 | 0.0018 | 0.05 | -9300.48 | -2134.14 |
| N Oxy60 | 1 | Plac | 1 | -6668.81 | 1822.94422 | -3.66 | 0.0003 | 0.05 | -10252 | -3085.64 |
| и Охуб0 | 1 | Plac | 2 | -2602.51 | 1822.94422 | -1.43 | 0.1541 | 0.05 | -6185.68 | 980.66 |
| | Treatmen | Treatment Timepoint (N) (N) N Oxy60 0 N Oxy60 0 N Oxy60 0 N Oxy60 0 N Oxy60 0 N Oxy60 0 N Oxy60 0 N Oxy60 0.5 N Oxy60 1 N Oxy60 1 N Oxy60 1 N Oxy60 1 N Oxy60 1 | Treatment Timepoint Treatment (N) (N) (N) (N) N Oxy60 0 Oxy60 N Oxy60 0 Plac N Oxy60 0.5 Oxy60 N Oxy60 0.5 Oxy60 N Oxy60 0.5 Oxy60 N Oxy60 0.5 Plac N Oxy60 1 Oxy60 N Oxy60 1 Oxy60 N Oxy60 1 Oxy60 N Oxy60 1 Oxy60 N Oxy60 1 Plac N Oxy60 1 Plac | Treatment Timepoint Treatment Timepoint (N) (N) (N) (N) N Oxy60 0 Oxy60 3 N Oxy60 0 Oxy60 4 N Oxy60 0 Plac 0.5 N Oxy60 0 Plac 1 N Oxy60 0 Plac 1 N Oxy60 0 Plac 2 N Oxy60 0 Plac 3 N Oxy60 0 Plac 3 N Oxy60 0 Plac 4 N Oxy60 0.5 Oxy60 1 N Oxy60 0.5 Oxy60 2 N Oxy60 0.5 Oxy60 3 N Oxy60 0.5 Plac 0 N Oxy60 0.5 Plac 0 N Oxy60 0.5 Plac 1 N Oxy60 0.5 Plac 3 N Oxy60 0.5 Plac 1 N Oxy60 0.5 Plac 3 N Oxy60 0.5 Plac 3 N Oxy60 0.5 Plac 4 N Oxy60 0.5 Plac 3 N Oxy60 0.5 Plac 3 N Oxy60 0.5 Plac 4 N Oxy60 0.5 Plac 4 N Oxy60 0.5 Plac 4 N Oxy60 1 Oxy60 3 N Oxy60 1 Oxy60 4 N Oxy60 1 Oxy60 4 N Oxy60 1 Oxy60 4 N Oxy60 1 Plac 0 N Oxy60 1 Plac 0.5 N Oxy60 1 Plac 0.5 | Treatment Timepoint Treatment Timepoint (N) (N) (N) (N) Estimate N Oxy60 0 Oxy60 3 4649.50 N Oxy60 0 Oxy60 4 4530.36 N Oxy60 0 Plac 0 132.08 N Oxy60 0 Plac 0.5 -1393.55 N Oxy60 0 Plac 1 -2345.05 N Oxy60 0 Plac 2 1721.25 N Oxy60 0 Plac 3 1307.18 N Oxy60 0 Plac 3 1307.18 N Oxy60 0 Plac 4 127.95 N Oxy60 0.5 Oxy60 1 2091.53 N Oxy60 0.5 Oxy60 2 3084.08 N Oxy60 0.5 Oxy60 3 2417.26 N Oxy60 0.5 Oxy60 4 2298.12 N Oxy60 0.5 Plac 0 -2100.16 N Oxy60 0.5 Plac 0 -2100.16 N Oxy60 0.5 Plac 1 -4577.29 N Oxy60 0.5 Plac 2 -510.99 N Oxy60 0.5 Plac 4 -2204.29 N Oxy60 0.5 Plac 3 -925.05 N Oxy60 0.5 Plac 4 -2104.29 N Oxy60 0.5 Plac 4 -2104.29 N Oxy60 0.5 Plac 4 -2104.29 N Oxy60 0.5 Plac 4 -2104.29 N Oxy60 1 Oxy60 3 325.74 N Oxy60 1 Oxy60 4 206.60 N Oxy60 1 Plac 0 -4191.68 N Oxy60 1 Plac 0 -5717.31 N Oxy60 1 Plac 0 -5717.31 N Oxy60 1 Plac 0 -5717.31 | Treatment Timepoint Treatment Timepoint (N) (N) (N) (N) Estimate Error DFt Noxy60 0 Oxy60 3 4649.50 1855.33 422 Noxy60 0 Oxy60 4 4530.36 1855.33 422 Noxy60 0 Plac 0 132.08 1856.77 422 Noxy60 0 Plac 0.5 -1393.55 1856.77 422 Noxy60 0 Plac 1 -2345.05 1856.77 422 Noxy60 0 Plac 2 1721.25 1856.77 422 Noxy60 0 Plac 3 1307.18 1856.77 422 Noxy60 0 Plac 3 1307.18 1856.77 422 Noxy60 0 Plac 4 127.95 1856.77 422 Noxy60 0.5 Oxy60 1 2091.53 1885.44 422 Noxy60 0.5 Oxy60 2 3084.08 1855.33 422 Noxy60 0.5 Oxy60 3 2417.26 1855.33 422 Noxy60 0.5 Oxy60 4 2298.12 1855.33 422 Noxy60 0.5 Plac 0 -2100.16 1856.77 422 Noxy60 0.5 Plac 0 -510.99 1856.77 422 Noxy60 0.5 Plac 1 -4577.29 1856.77 422 Noxy60 0.5 Plac 1 -4577.29 1856.77 422 Noxy60 0.5 Plac 2 -510.99 1856.77 422 Noxy60 0.5 Plac 3 -925.05 1856.77 422 Noxy60 0.5 Plac 3 -925.05 1856.77 422 Noxy60 0.5 Plac 4 -2104.29 1856.77 422 Noxy60 0.5 Plac 3 -925.05 1856.77 422 Noxy60 0.5 Plac 4 -2104.29 1856.77 422 Noxy60 0.5 Plac 3 -925.05 1856.77 422 Noxy60 1 Oxy60 4 206.60 1820.88 422 Noxy60 1 Oxy60 4 206.60 1820.88 422 Noxy60 1 Plac 0 -4191.68 1822.94 422 Noxy60 1 Plac 0 -4191.68 1822.94 422 Noxy60 1 Plac 0 -5717.31 1822.94 422 Noxy60 1 Plac 0 -5717.31 1822.94 422 Noxy60 1 Plac 1 -6668.81 1822.94 422 | Treatment Timepoint Treatment Timepoint (N) (N) (N) (N) Estimate Error DFt Value P NOxy60 0 Oxy60 3 4649.50 1855.33 422 2.51 NOxy60 0 Oxy60 4 4530.36 1855.33 422 2.44 NOxy60 0 Plac 0 132.08 1856.77 422 0.07 NOxy60 0 Plac 1 -2345.05 1856.77 422 -0.75 NOxy60 0 Plac 1 -2345.05 1856.77 422 -1.26 NOxy60 0 Plac 2 1721.25 1856.77 422 0.93 NOxy60 0 Plac 3 1307.18 1856.77 422 0.70 NOxy60 0 Plac 3 1307.18 1856.77 422 0.70 NOxy60 0 Plac 4 127.95 1856.77 422 0.70 NOxy60 0 Plac 4 127.95 1856.77 422 1.11 NOxy60 0.5 Oxy60 1 2091.53 1885.44 422 1.11 NOxy60 0.5 Oxy60 2 3084.08 1855.33 422 1.66 NOxy60 0.5 Oxy60 3 2417.26 1855.33 422 1.24 NOxy60 0.5 Oxy60 4 2298.12 1855.33 422 1.24 NOxy60 0.5 Plac 0 -2100.16 1856.77 422 -1.13 NOxy60 0.5 Plac 0 -2100.16 1856.77 422 -1.95 NOxy60 0.5 Plac 1 -4577.29 1856.77 422 -2.47 NOxy60 0.5 Plac 1 -4577.29 1856.77 422 -0.28 NOxy60 0.5 Plac 3 -925.05 1856.77 422 -0.28 NOxy60 0.5 Plac 4 -2104.29 1856.77 422 -0.50 NOxy60 0.5 Plac 3 -925.05 1856.77 422 -0.50 NOxy60 0.5 Plac 4 -2104.29 1856.77 422 -1.13 NOxy60 0.5 Plac 3 -925.05 1856.77 422 -0.50 NOxy60 0.5 Plac 4 -2104.29 1856.77 422 -0.50 NOxy60 1 Oxy60 3 325.74 1820.88 422 0.55 NOxy60 1 Oxy60 3 325.74 1820.88 422 0.55 NOxy60 1 Oxy60 4 206.60 1820.88 422 0.55 NOxy60 1 Oxy60 3 325.74 1820.88 422 0.55 NOxy60 1 Oxy60 4 206.60 1820.88 422 0.55 NOxy60 1 Plac 0 -4191.68 1822.94 422 -2.30 NOxy60 1 Plac 0 -5717.31 1822.94 422 -3.14 NOxy60 1 Plac 0 -5717.31 1822.94 422 -3.16 | Treatment Timepoint Treatment Timepoint (N) (N) (N) (N) (S) Estimate Error DFt Value Pr > t Noxy60 | Treatment Timepoint Treatment Timepoint (N) (N) (N) (N) (Signature) Noxy60 0 0xy60 3 4649.50 1855.33 422 2.51 0.0126 0.05 Noxy60 0 0xy60 4 4530.36 1855.33 422 2.44 0.0150 0.05 Noxy60 0 Plac 0 132.08 1856.77 422 0.07 0.9433 0.05 Noxy60 0 Plac 0.5 -1393.55 1856.77 422 -0.75 0.4534 0.05 Noxy60 0 Plac 1 -2345.05 1856.77 422 -1.26 0.2073 0.05 Noxy60 0 Plac 2 1721.25 1856.77 422 0.93 0.3544 0.05 Noxy60 0 Plac 3 1307.18 1856.77 422 0.70 0.4818 0.05 Noxy60 0 Plac 4 127.95 1856.77 422 0.07 0.9451 0.05 Noxy60 0.5 0xy60 1 2091.53 1885.43 422 1.11 0.2679 0.05 Noxy60 0.5 0xy60 2 3084.08 1855.33 422 1.66 0.0972 0.05 Noxy60 0.5 0xy60 3 2417.26 1855.33 422 1.66 0.0972 0.05 Noxy60 0.5 Plac 0 -2100.16 1856.77 422 -1.13 0.2587 0.05 Noxy60 0.5 Plac 1 -4577.29 1856.77 422 -1.95 0.0515 0.05 Noxy60 0.5 Plac 2 -510.99 1856.77 422 -0.28 0.7833 0.05 Noxy60 0.5 Plac 2 -510.99 1856.77 422 -0.50 0.6186 0.05 Noxy60 0.5 Plac 3 -925.05 1856.77 422 -0.50 0.6186 0.05 Noxy60 0.5 Plac 3 -925.05 1856.77 422 -0.50 0.6186 0.05 Noxy60 0.5 Plac 3 -925.05 1856.77 422 -0.28 0.7833 0.05 Noxy60 0.5 Plac 4 -2104.29 1856.77 422 -0.28 0.7833 0.05 Noxy60 0.5 Plac 3 -925.05 1856.77 422 -0.28 0.7833 0.05 Noxy60 0.5 Plac 3 -925.05 1856.77 422 -0.50 0.6186 0.05 Noxy60 0.5 Plac 4 -2104.29 1856.77 422 -0.28 0.7833 0.05 Noxy60 0.5 Plac 3 -925.05 1856.77 422 -0.28 0.7833 0.05 Noxy60 0.5 Plac 4 -2104.29 1856.77 422 -0.28 0.7833 0.05 Noxy60 0.5 Plac 3 -925.05 1856.77 422 -0.28 0.7833 0.05 Noxy60 1 0xy60 3 325.74 1820.88 422 0.11 0.9097 0.05 Noxy60 1 0xy60 3 325.74 1820.88 422 0.11 0.9097 0.05 Noxy60 1 Plac 0 -4191.68 1822.94 422 -3.14 0.0018 0.05 Noxy60 1 Plac 0 -4191.68 1822.94 422 -3.16 0.0003 0.05 | Treatment Timepoint Treatment Timepoint (N) (N) (N) (N) (N) (Estimate Error DFt Value Pr > t Alpha Lower N0xy60 0 0 0xy60 3 4649.50 1855.33422 2.51 0.0126 0.05 1002.66 N0xy60 0 0xy60 4 4530.36 1855.33422 2.44 0.0150 0.05 883.52 N0xy60 0 Plac 0 132.08 1856.77422 0.07 0.9433 0.05-3517.59 N0xy60 0 Plac 0.5 -1393.55 1856.77422 -0.75 0.4534 0.05-5043.22 N0xy60 0 Plac 1 -2345.05 1856.77422 -1.26 0.2073 0.05-5994.72 N0xy60 0 Plac 2 1721.25 1856.77422 0.93 0.3544 0.05-5994.72 N0xy60 0 Plac 3 1307.18 1856.77422 0.93 0.3544 0.05-5994.72 N0xy60 0 Plac 3 1307.18 1856.77422 0.93 0.3544 0.05-5994.72 N0xy60 0 Plac 4 127.95 1856.77422 0.070 0.4818 0.05-2342.49 N0xy60 0.5 0xy60 1 2091.53 1885.44422 1.11 0.2679 0.05-1614.50 N0xy60 0.5 0xy60 1 2091.53 1885.44422 1.11 0.2679 0.05-1614.50 N0xy60 0.5 0xy60 3 2417.26 1855.33422 1.66 0.0972 0.05 -5527.6 N0xy60 0.5 0xy60 3 2417.26 1855.33422 1.60 0.0972 0.05 -5282.76 N0xy60 0.5 0xy60 4 2298.12 1855.33422 1.30 0.1933 0.05-1229.58 N0xy60 0.5 Plac 0 -2100.16 1856.77422 -1.13 0.2587 0.05-5749.83 N0xy60 0.5 Plac 0 -2100.16 1856.77422 -1.13 0.2587 0.05-5749.83 N0xy60 0.5 Plac 1 -4577.29 1856.77422 -1.95 0.0515 0.05-7275.45 N0xy60 0.5 Plac 1 -4577.29 1856.77422 -0.28 0.7833 0.05-4160.66 N0xy60 0.5 Plac 2 -510.99 1856.77422 -0.28 0.7833 0.05-4160.66 N0xy60 0.5 Plac 3 -925.05 1856.77422 -0.50 0.6186 0.05-4574.72 N0xy60 0.5 Plac 4 -2104.29 1856.77422 -0.50 0.6186 0.05-4574.72 N0xy60 0.5 Plac 4 -2104.29 1856.77422 -0.50 0.6186 0.05-4574.72 N0xy60 1 0xy60 4 206.60 1820.88422 0.15 0.55-5753.96 N0xy60 1 0xy60 4 206.60 1820.88422 0.15 0.5970 0.05-5753.96 N0xy60 1 0xy60 4 206.60 1820.88422 0.16 0.9970 0.05-5735.39 N0xy60 1 0xy60 4 206.60 1820.88422 0.11 0.9097 0.05-5735.39 N0xy60 1 0xy60 4 206.60 1820.88422 0.11 0.9097 0.05-7774.85 N0xy60 1 Plac 0 -4191.68 1822.94422 -2.30 0.0020 0.05-7774.85 N0xy60 1 Plac 0 -4191.68 1822.94422 -3.14 0.0018 0.05-9300.48 N0xy60 1 Plac 0 -4191.68 1822.94422 -3.16 0.0008 0.05-9300.48 N0xy60 1 Plac 0 -4191.68 1822.94422 -3.16 0.0008 0.05-9300.48 N0xy60 1 Plac 0 -4191.68 |

Program: A\_Bio4.sas Created: 02APR2020 7:36 POSTLOCK

# Appendix 16.1.9.2.4 Statistical Methods and Analysis Output Supporting Table 14.2.5 Supporting Table 14.2.4

# The Mixed Procedure

#### Parameter Code=MVMIPM

# Differences of Least Squares Means

| | D1 1 | 7 1 | | | or heade i | oquares neans | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | Planned | Analysis | | Analysis<br>Timepoint | | Standard | | | | | |
| Effect | (N) | (N) | (N) | (N) | Estimate | Error DF t | 7/2 ] 110 P: | ^ \ I+I | Λlnha | Lower | Upper |
| | ` ' | 1 | . , | 3 | | 1822.94422 | -1.65 | | | -6599.75 | 566.59 |
| TRTPN*ATPT | 4 | _ | Plac | - | | | | | | | |
| TRTPN*ATPT | 4 | 1 | Plac | 4 | | 1822.94422 | -2.30 | | | | -612.64 |
| TRTPN*ATPT | 4 | 2 | Oxy60 | 3 | | 1790.13422 | -0.37 | | | | 2851.86 |
| TRTPN*ATPT | 4 | 2 | Oxy60 | 4 | | 1790.13422 | -0.44 | | | | 2732.72 |
| TRTPN*ATPT | N 0xy60 | 2 | Plac | 0 | -5184.23 | 1791.43422 | -2.89 | 0.0040 | 0.05- | -8705.46 | -1663.00 |
| TRTPN*ATPT | NOxy60 | 2 | Plac | 0.5 | -6709.86 | 1791.43422 | -3.75 | 0.0002 | 0.05 | -10231 | -3188.63 |
| TRTPN*ATPT | NOxy60 | 2 | Plac | 1 | -7661.36 | 1791.43422 | -4.28 | <.0001 | 0.05 | -11183 | -4140.13 |
| TRTPN*ATPT | NOxy60 | 2 | Plac | 2 | -3595.06 | 1791.43422 | -2.01 | 0.0454 | 0.05- | -7116.29 | -73.8314 |
| TRTPN*ATPT | NOxy60 | 2 | Plac | 3 | -4009.13 | 1791.43422 | -2.24 | 0.0257 | 0.05- | -7530.36 | -487.90 |
| TRTPN*ATPT | NOxy60 | 2 | Plac | 4 | -5188.37 | 1791.43422 | -2.90 | 0.0040 | 0.05- | -8709.60 | -1667.13 |
| TRTPN*ATPT | NOxy60 | 3 | Oxy60 | 4 | -119.14 | 1790.13422 | -0.07 | 0.9470 | 0.05- | -3637.82 | 3399.54 |
| TRTPN*ATPT | NOxy60 | 3 | Plac | 0 | -4517.42 | 1791.43422 | -2.52 | 0.0120 | 0.05- | -8038.65 | -996.19 |
| TRTPN*ATPT | NOxy60 | 3 | Plac | 0.5 | -6043.04 | 1791.43422 | -3.37 | 0.0008 | 0.05- | -9564.27 | -2521.81 |
| TRTPN*ATPT | NOxy60 | 3 | Plac | 1 | -6994.55 | 1791.43422 | -3.90 | 0.0001 | 0.05 | -10516 | -3473.32 |
| TRTPN*ATPT | NOxy60 | 3 | Plac | 2 | -2928.25 | 1791.43422 | -1.63 | 0.1029 | 0.05- | -6449.48 | 592.98 |
| TRTPN*ATPT | NOxy60 | 3 | Plac | 3 | -3342.32 | 1791.43422 | -1.87 | 0.0628 | 0.05- | -6863.55 | 178.91 |
| TRTPN*ATPT | NOxy60 | 3 | Plac | 4 | -4521.55 | 1791.43422 | -2.52 | 0.0120 | 0.05- | -8042.78 | -1000.32 |
| TRTPN*ATPT | NOxy60 | 4 | Plac | 0 | -4398.28 | 1791.43422 | -2.46 | 0.0145 | 0.05- | -7919.51 | -877.05 |
| TRTPN*ATPT | NOxy60 | 4 | Plac | 0.5 | -5923.90 | 1791.43422 | -3.31 | 0.0010 | 0.05- | -9445.13 | -2402.67 |
| TRTPN*ATPT | NOxy60 | 4 | Plac | 1 | -6875.41 | 1791.43422 | -3.84 | 0.0001 | 0.05 | -10397 | -3354.18 |
| TRTPN*ATPT | NOxy60 | 4 | Plac | 2 | -2809.11 | 1791.43422 | -1.57 | 0.1176 | 0.05- | -6330.34 | 712.12 |
| TRTPN*ATPT | NOxy60 | 4 | Plac | 3 | -3223.18 | 1791.43422 | -1.80 | 0.0727 | 0.05- | -6744.41 | 298.05 |
| TRTPN*ATPT | NOxy60 | 4 | Plac | 4 | -4402.41 | 1791.43422 | -2.46 | 0.0144 | 0.05- | -7923.64 | -881.18 |
| TRTPN*ATPT | N Plac | 0 | Plac | 0.5 | -1525.63 | 1790.13422 | -0.85 | 0.3946 | 0.05- | -5044.30 | 1993.05 |
| TRTPN*ATPT | N Plac | 0 | Plac | 1 | -2477.13 | 1790.13422 | -1.38 | 0.1672 | 0.05- | -5995.81 | 1041.55 |

Program: A Bio4.sas Created: 02APR2020 7:36 POSTLOCK 

# Appendix 16.1.9.2.4 Statistical Methods and Analysis Output Supporting Table 14.2.5 Supporting Table 14.2.4

# The Mixed Procedure

#### Parameter Code=MVMIPM

# Differences of Least Squares Means

| | Planned | Analysis | Planned | Analysis | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| | Treatment | Timepoint | Treatment | Timepoint | | Standard | | | | |
| Effect | (N) | (N) | (N) | (N) | Estimate | Error DFt | Value Pr | > t . | Alpha Lower | Upper |
| TRTPN*ATPTN | Plac | 0 | Plac | 2 | 1589.17 | 1790.13422 | 0.89 | 0.3752 | 0.05-1929.51 | 5107.85 |
| TRTPN*ATPTN | Plac | 0 | Plac | 3 | 1175.10 | 1790.13422 | 0.66 | 0.5119 | 0.05-2343.58 | 4693.78 |
| TRTPN*ATPTN | Plac | 0 | Plac | 4 | -4.1324 | 1790.13422 | -0.00 | 0.9982 | 0.05-3522.81 | 3514.55 |
| TRTPN*ATPTN | Plac | 0.5 | Plac | 1 | -951.50 | 1790.13422 | -0.53 | 0.5953 | 0.05-4470.18 | 2567.18 |
| TRTPN*ATPTN | Plac | 0.5 | Plac | 2 | 3114.80 | 1790.13422 | 1.74 | 0.0826 | 0.05 -403.88 | 6633.48 |
| TRTPN*ATPTN | Plac | 0.5 | Plac | 3 | 2700.73 | 1790.13422 | 1.51 | 0.1321 | 0.05 -817.95 | 6219.41 |
| TRTPN*ATPTN | Plac | 0.5 | Plac | 4 | 1521.49 | 1790.13422 | 0.85 | 0.3958 | 0.05-1997.18 | 5040.17 |
| TRTPN*ATPTN | Plac | 1 | Plac | 2 | 4066.30 | 1790.13422 | 2.27 | 0.0236 | 0.05 547.62 | 7584.98 |
| TRTPN*ATPTN | Plac | 1 | Plac | 3 | 3652.23 | 1790.13422 | 2.04 | 0.0420 | 0.05 133.55 | 7170.91 |
| TRTPN*ATPTN | Plac | 1 | Plac | 4 | 2473.00 | 1790.13422 | 1.38 | 0.1679 | 0.05-1045.68 | 5991.68 |
| TRTPN*ATPTN | Plac | 2 | Plac | 3 | -414.07 | 1790.13422 | -0.23 | 0.8172 | 0.05-3932.75 | 3104.61 |
| TRTPN*ATPTN | Plac | 2 | Plac | 4 | -1593.30 | 1790.13422 | -0.89 | 0.3739 | 0.05-5111.98 | 1925.38 |
| TRTPN*ATPTN | Plac | 3 | Plac | 4 | -1179.23 | 1790.13422 | -0.66 | 0.5104 | 0.05-4697.91 | 2339.44 |

# Tests of Effect Slices Analysis

# Timepoint Num Den

| Effect | (N) | DF | DF F | Value P | r > | F |
|-----------|--------|-----|------|---------|-----|----|
| TRTPN*ATP | TN 0 | 5 - | 422 | 0.610 | .69 | 06 |
| TRTPN*ATP | TN 0.5 | 5 - | 422 | 3.110 | .00 | 90 |
| TRTPN*ATP | TN 1 | 5 - | 422 | 3.970 | .00 | 16 |
| TRTPN*ATP | TN 2 | 5 - | 422 | 2.840 | .01 | 55 |
| TRTPN*ATP | TN 3 | 5 - | 422 | 1.550 | .17 | 19 |
| TRTPN*ATP | TN 4 | 5 - | 422 | 1.750 | .12 | 15 |

Program: A\_Bio4.sas Created: 02APR2020 7:36 POSTLOCK

Appendix 16.1.9.2.4
Statistical Methods and Analysis Output Supporting Table 14.2.5
Supporting Table 14.2.4

The Mixed Procedure

Parameter Code=MVMIPM

Program: A\_Bio4.sas Created: 02APR2020 7:36 POSTLOCK 